## **CLINICAL STUDY REPORT**

EFFICACY AND SAFETY STUDY OF F373280 FOR MAINTENANCE OF SINUS RHYTHM AFTER ELECTRICAL CARDIOVERSION IN PATIENTS WITH PERSISTENT ATRIAL FIBRILLATION AND CHRONIC HEART FAILURE

## 16. APPENDICES

## 16.1. STUDY INFORMATION

## 16.1.1. Protocol and protocol amendments

Final version 1/1185

## Study F323280 CA 2 01

## 16.1. STUDY INFORMATION

16.1.1. Protocol and protocol amendments

Final version 2/1185

- 16.1.1.1. Protocol and appendices (version 1: 09 November 2012)
- 16.1.1.2. Protocol and appendices (version 2: 15 January 2013)
- 16.1.1.3. Protocol amendment n° PA01 local (Italy) and substantial dated on 01 March 2013 linked to Protocol and appendices (version3: 01 March 2013)
- 16.1.1.4. Protocol amendment n°PA02 General and non-substantial dated on 28 March 2013 linked to Protocol and appendices (version 4: 28 March 2013)
- 16.1.1.5. Protocol amendment n°PA03 General and substantial dated on 23 October 2013 linked to Protocol and appendices (version 5: 23 October 2013)
- 16.1.1.6. Protocol and appendices (version 6: 02 December 2013)
- 16.1.1.7. Protocol amendment n°PA04 General and non-substantial dated on 03

  June 2014 linked to Protocol and appendices (version 7: 03 June 2014)
- 16.1.1.8 Protocol amendment n°PA05 General and substantial dated on 22 October 2014 linked to Protocol and appendices (version 8: 22 October 2014)
- 16.1.1.9 Protocol amendment n°PA06 General and non-substantial dated on 06

  June 2016
- 16.1.1.10 Protocol amendment n°PA07 General and substantial dated on 28 September 2016 linked to Protocol and appendices (version 9: 28 September 2016)
- 16.1.1.11 Protocol amendment n° PA07 Local (Italy) and non-substantial dated on 06 December 2016 linked to Protocol and appendices (version 9: 06 December 2016)

Final version 3/1185

16.1.1.1. Protocol and appendices (version 1: 09 November 2012)

Final version 4/1185

F 373280 CA 2 01

Final version 5/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

## CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

**Sponsor's Representative:** Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 63 48 Fax:+33 5 34 50 65 92

E-mail:marlene.guiraud@pierre-fabre.com

Pr Savina NODARI Section of Cardiology

**Department of Experimental and Applied Sciences** 

**University of Brescia BRESCIA, ITALY** 

Phone: +39 030 3996 587 - Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>

## Version 1-09 NOV 2012

**Study Coordinating Investigator** 

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 6/1185

## **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

## **Clinical Study Manager (Monitor)**

Marlène GUIRAUD, Pharm D Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 63 48 Fax: +33 5 34 50 65 92

E-mail: marlene.guiraud@pierre-

fabre.com

#### **Head of Therapeutic Area**

Alain DELARUE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1

Phone: +33 5 34 50 61 88 Fax: +33 5 34 50 65 92

E-mail: alain.delarue@pierre-

fabre.com

## **Clinical Development Physician**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 65 92 E-mail: richard.roche@pierre-

fabre.com

Final version 7/1185

## CONTRACT RESEARCH ORGANISATIONS

## For Feasibility, Monitoring and Regulatory issues:

Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

## For Centralised Randomisation and Electronic Case Report Form

#### **S-Clinica**

6, Chaussée de Boondael B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

## For Centralised Reading of Holder ECG and TTEM and equipment supply:

## **Biomedical System**

1945 Chaussée de Wavre B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

## For intra erythrocyte DHA dosage

## **Agrocampus Ouest**

Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

Final version 8/1185

## Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 1 – 09 NOV 2012

Sponsor's Representative:

**Head of Therapeutic Area:** 

Alain DELARUE, MD

Date:

Signature:

12 November 2012 <

16 November 2012 Sorrue

**Study Coordinating Investigator:** 

Savina NODARI, MD

Date:

Signature:

## Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

## **Protocol Version 1 – 09 NOV 2012**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 10/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

Protocol Version1 – 09 NOV 2012

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 09 November 2012 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

## Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * To be adapted | |
|-----------------|------|
| | Data |

| Date: | Signature |
|-------|-----------|

Final version 11/1185

## TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| <b>1.</b> ] | INTRODUCTION AND STUDY RATIONALE | 21 |
|-------------------|----------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 21 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 23 |
| 1.2.1. | Chemical and pharmaceutical characteristics | 24 |
| 1.2.1. | | |
| 1.2.1.2 | σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ | |
| 1.2.2.<br>1.2.2.1 | | |
| 1.2.2.2 | | |
| 1.2.2.3 | | |
| 1.2.2.4 | C 1 | |
| 1.2.3. | Clinical data | 26 |
| 1.3. | STUDY RATIONALE | 29 |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 29 |
| 2. | STUDY OBJECTIVES | 32 |
| 2.1. | PRIMARY OBJECTIVE | 32 |
| 2.2. | SECONDARY OBJECTIVES | 32 |
| <b>3.</b> ] | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 32 |
| 4. | STUDY DESIGN | 34 |
| 4.1. | OVERALL DESCRIPTION | 34 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | $\mathcal{F}$ | |
| 4.2.3. | | |
| 4.2.4. | 1 | |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 38 |
| 5.3. | NUMBER OF PATIENTS | 39 |
| 5.4. | RECRUITMENT MODALITIES | 40 |
| 5.5. | PATIENTS IDENTIFICATION | 40 |
| 5.6. | WITHDRAWAL CRITERIA | 40 |
| 5.7. | REPLACEMENT OF PATIENTS | 41 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 41 |
| 5.9. | STUDY CARD | 41 |

| 6. S | TUDY TREATMENT | 42 |
|---|---|---|
| 5.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 42 |
| 5.2. | PACKAGING AND LABELLING | |
| 5.2.1. | Packaging | |
| 5.2.2. | Labelling | |
| 5.3. | DISTRIBUTION TO CENTRE AND STORAGE | |
| 5.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | |
| 5.5. | DRUG ADMINISTRATION | |
| 5.5.1. | Duration of Treatment | |
| 5.5.2. | Dose Schedule | |
| 5.5.3. | Route and Conditions of Administration. | |
| 5.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 46 |
| 5.7. | RECALL OF INVESTIGATIONAL PRODUCTS | 47 |
| 7. ( | CONCOMITANT TREATMENTS | 47 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 48 |
| 7.2. | PROHIBITED TREATMENTS | 48 |
| 7.3. | AUTHORISED TREATMENTS | |
| 8. E | EVALUATION CRITERIA | 49 |
| 8.1. | PRIMARY EFFICACY CRITERION: | 49 |
| 3.1.1. | Time to the first Atrial Fibrillation Recurrence | 49 |
| 8.1.1.1 | | |
| 3.1.1.2 | | |
| 8.1.1.3<br>8.1.2. | | |
| 3.1.2.<br>3.1.2.1 | Secondary Efficacy Criteria | 30 |
| 3.1.4.1 | visit) | 50 |
| 8.1.2.2 | · | |
| | visit) | |
| 8.1.2.3 | 1 | |
| 3.1.2.4 | | |
| 8.1.2.5 | | 53 |
| 3.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA | 53 |
| 3.2.1. | Definition | |
| 3.2.1. | Blood samples | |
| 3.2.2.1 | • | |
| 3.2.2.2 | | |
| 8.2.3. | DHA concentration measurement | 54 |
| 3.3. | SAFETY ASSESSMENT | 55 |

| 3.3.1. Adverse Events | 55 |
|----------------------------------------------------------------|----|
| 8.3.2. Laboratory Investigations | 55 |
| 8.3.2.1. Schedule | 55 |
| 8.3.2.2. Technical Procedures and Parameters | 55 |
| 8.3.3. Global Physical Examination | 56 |
| 8.3.4. Vital Signs | 56 |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.3.7. Concomitant Treatments | |
| 8.4. COMPLIANCE | 58 |
| 9. STUDY PROCEDURES | 59 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 65 |
| 10.1. ADVERSE EVENTS | 65 |
| 10.1.1. Definition of Adverse Events | 65 |
| 10.1.2. Grading of Adverse Events | |
| 10.1.3. Reporting of Adverse Events | 66 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 66 |
| 10.2.1. Definition | 66 |
| 10.2.2. Reporting of SAE | 67 |
| 10.2.3. Follow-up of SAE | |
| 10.2.4. SAE Occurring After the Study | 67 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 68 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 68 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | 69 |
| 11. DATA COLLECTION AND STUDY MONITORING | 69 |
| 11.1. DATA COLLECTION | 69 |
| 11.1.1. Case Report Form | 69 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | 70 |
| 11.2.1. Monitoring visits | 70 |
| 11.2.1.1. Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | 71 |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | 72 |
| 12 DATA MANACEMENT | 72 |

| 12.1. DATA ENTRY | 73 |
|---|---|
| 12.2. DATA CLEANING | 73 |
| 12.3. DATA CODING | 73 |
| 12.4. DATA STORAGE | 73 |
| 12.5. DATABASE LOCK | 74 |
| 13. STATISTICAL ANALYSIS | 74 |
| 13.1. GENERAL CONSIDERATIONS | 74 |
| 13.2. SAMPLE SIZE | 74 |
| 13.3. PROTOCOL DEVIATIONS | 75 |
| 13.4. DATA SETS ANALYSED | |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 76 |
| 13.7. EFFICACY ANALYSIS | 77 |
| 13.7.1. Primary Criterion | 77 |
| 13.7.1.1. Primary Analysis | 77 |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2. Secondary Criteria | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | 78 |
| 13.8.1. Adverse Events | 78 |
| 13.8.2. Clinical Laboratory Evaluation | 80 |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | |
| 13.8.4.2. Body weight | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | |
| 14. GENERAL ETHICAL CONSIDERATIONS | |
| 14.1. ETHICAL CONDITIONS | |
| 14.2 ETHICS COMMITTEE AND LEGAL REQUIREMENTS | |

| 14.3. | PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 84 |
|---|---|---|
| 14.4. | PERSONAL DATA PROTECTION | 85 |
| 14.5. | INSURANCE POLICY | 85 |
| 15. | ADMINISTRATIVE PROCEDURES | 86 |
| 15.1. | PROTOCOL AMENDMENT | 86 |
| 15.2. | SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 86 |
| 15.3. | END OF THE STUDY | 87 |
| 15.3. | J | |
| 15.3. | | |
| 15.3. | | |
| | 2.2. Early Study Termination Decided by the Competent Authorities | |
| 15.4. | | |
| 15.5. | INSPECTION | |
| 15.6. | CONFIDENTIALITY | 88 |
| 15.7. | CLINICAL STUDY REPORT | 88 |
| 15.8. | STUDY RESULTS COMMUNICATION | 89 |
| 15.9. | STUDY RESULTS PUBLICATION | 89 |
| 16. | REFERENCES | 91 |
| 17. | APPENDICES | 94 |
| 17.1. | DECLARATION OF HELSINKI | 95 |
| 17.2. | SAE REPORT FORM | 99 |
| 17.3. | PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 102 |

## **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of Atrial Fibrillation (AF) induced by burst pacing.[1] Moreover, the effectiveness of PUFA (PolyUnsaturated Fatty Acid) has been proven in the following conditions: - prevention of Atrial Fibrillation recurrence in patients with persistent Atrial Fibrillation, in co-administration with amiodarone (add on therapy) [2] - Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – April 2014 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>Salety and tolerability of F3/3280</li> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 (anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> <li>Treatment duration: 24 weeks</li> </ul> |
| Study Schedule | 9 visits will be scheduled: - V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit) - V2/D1: Inclusion visit (start of treatment) - V3/W4 (D28 -2/+7 days): cardioversion visit (Outpatient or hospitalization according to |

Final version 17/1185

| | clinical practice of the centre) (installation of the Holter device) |
|---|---|
| | - V4/W5 (D35± 2 days): follow-up visit (removing of the Holter device and installation of |
| | the TTEM) |
| | - V5/W8 (D56± 7 days): follow-up visit |
| | - V6/W12 (D84 $\pm$ 7 days): follow-up visit |
| | - $V7/W16$ (D112 ± 7 days): follow-up visit |
| | - V8/W20 (D140 ± 7 days): follow-up visit |
| | - V9/W24 (D168 $\pm$ 7 days): final study visit |
| Number of Patients: | 76 x 2 patients |

#### **Diagnosis and Criteria for Inclusion:**

#### **Inclusion Criteria:**

Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive),
- 2. Patients with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) ) at selection and at inclusion
- On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$ ) at selection and at inclusion
- 9. Patients treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:
  - use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment
  - documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion

#### Ethical /legal considerations:

- 12. Having signed his/her written informed consent,
- 13. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 1 year
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6
- Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- Severe chronic kidney disease (creatinine 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection</li>
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (K>5.5 mEq/L or K  $\leq$  3.5 mEq/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

Final version 18/1185

| | <ul> <li>Criteria related to treatments:</li> <li>11. Previously ineffective pharmacological or electrical cardioversion</li> <li>12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers</li> <li>13. Previous treatment with oral amiodarone within 12 months prior to inclusion</li> <li>14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion</li> <li>15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months</li> <li>16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months</li> <li>17. Dietary supplement with ω3 or ω6 according to investigator's judgement</li> <li>18. Having undergone any form of ablation therapy for AF</li> <li>19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel</li> </ul> |
|---|---|
| | <ul> <li>Other criteria:</li> <li>20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion</li> <li>21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection</li> <li>22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints</li> <li>23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator</li> <li>24. Patient having forfeited his / her freedom by administrative or legal award or being</li> </ul> |
| Exclusion criteria before V3: | under guardianship Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV) ECV will be performed in patients without dyskalemia If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: Dose: | F373280 Soft Capsules Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules Placebo will be administered in the same conditions as the tested product. |
| Mode of Administration: | Oral, one capsule each evening with dinner |
| Evaluation Criteria: | <ul> <li>Efficacy evaluation variables:</li> <li>Primary evaluation variable:</li> <li>Time to first Atrial Fibrillation recurrence defined by the first episode of Atrial Fibrillation lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit)</li> <li>Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24.</li> <li>For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).</li> <li>Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM.</li> <li>All ECG traces will be evaluated by a Central Reading Laboratory.</li> <li>Secondary evaluation variables:</li> <li>During the 7-day continuous ECG monitoring,</li> <li>Numbers of AF episodes</li> </ul> |

Final version 19/1185

Duration of AF episodes

#### Clinical parameters:

During the whole study:

- Number of recurrence of symptomatic AF episodes
- EHRA score
- Hospitalization for cardiovascular events
- Hospitalization for thromboembolic stroke
- All cause of hospitalization

#### Cardioversion:

- Assessment of spontaneous cardioversion
- Assessment of successful cardioversion
- Number of patients needing an other cardioversion after the initial ECV

#### Other:

- Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m², Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))
- Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).

#### Safety criteria:

- Adverse events (observed and / or spontaneously reported)
- Vital signs (Blood pressure (supine and standing), heart rate
- Physical examination (body weight),
- **Standard 12-lead ECG**: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized).
- Haematology: haematocrit, haemoglobin, RBC, WBC, differential count, platelets
- **Biochemistry:** sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)
- **Coagulation parameters:** Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR *(local laboratory)*, Prothrombine Time *(PT)*

#### **Statistical Methods:**

#### Sample Size:

Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary to achieve, using a log-rank test of survival curves, a difference between groups of 20%.

#### **Primary Efficacy Analysis**

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### Secondary Analyses

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

#### Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment)

Final version 20/1185

## STUDY FLOW-CHART

Final version 21/1185

| F373280 CA 201 | V1 | V2 | <b>V</b> 3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 +/-2 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(116+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | х | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic characteristics | х | | | | | | | | |
| Medico-surgical history | х | | | | | | | | |
| Concomitant disease | х | | | | | | | | |
| Concomitant treatment | х | х | x | × | х | х | х | х | х |
| Habits | х | | | | | | | | |
| Global physical examination (body weight) | х | х | x | | х | х | х | х | х |
| Echocardiography | х | х | | x | | х | | | х |
| Eligibility criteria check | х | х | | | | | | | |
| Blood pressure, heart rate | х | х | x | × | х | х | х | x | х |
| 12-Lead ECG Recording | х | х | x | | х | х | х | х | х |
| INR | - | | (2) | | х | х | х | х | х |
| аРТТ, ТСТ | × | x | × | | x | x | x | x | х |
| Biochemistry | × | | | | | | | | x |
| Hematology | × | | | | | | | | x |
| Urinary pregnancy test | | x | | | | | | | x |
| Red Blood Cell concentrations of DHA | | x | × | | | x | | | x |
| Treatment allocation | | x | | | | x | | | |
| IVRS | х | х | | | х | х | | | |
| ECV (3) | | | × | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | × | х | x | х | х | х | x | х |
| Holter ECG | (4) | | - | (5) | | | | | |
| TTEM (6) | _ | | t or hospitalization a | | | | | | <del></del> |

Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)

Final version 22/1185

<sup>(2)</sup> In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF (4) 24-hour Holter ECG

<sup>(5) 7-</sup>day Holter ECG

<sup>1-</sup>vay rioline ECG (6) TTEM everyday from week 6 to week 8. Then every 2 days from week 9 to week 24. In case of AF symptoms. In case of AF recurrence for at least 10 minutes and the patient does not stop the study treatment then TTEM every 4 weeks

## LIST OF ABBREVIATIONS

aPTT Activated partial thromboplastin time

AE : Adverse event

AERP Atrial effective refractory period

AF : Atrial fibrillation
ALA Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK Anti vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP Blood pressure
BSA : Body Surface Area

CEP Protocol evaluation committee

CHF : Congestive heart failure

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT Cardiac resynchronization therapy

"Clinically Significant Change", i.e., Predefined potentially clinically

CSC : significant change leading to a potentially clinically significant value (vital

signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO –TE Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA European heart rhythm association

EPA Eicosapentaenoic acid eCRF Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

Final version 23/1185

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL High density lipoprotein

HF Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR International normalized ratio
IRPF: Institut de Recherche Pierre Fabre
IVRS Interactive voice response system

LAA Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL Low density lipoprotein LOQ : Limit of quantification

LVEF Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR Mineralocorticoid receptor
MR perfusion Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change

(lab or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

POC Proof of concept

PUFA : PolyUnsaturated fatty acid

PK : Pharmacokinetics

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE
 Serious adverse event
 SBP
 Systolic blood pressure
 SD
 Standard deviation
 T<sub>1/2</sub>
 Terminal half-life

To : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT Thrombin clotting time

TEAEs Treatment emergent adverse events
TTEM TransTelephonic ECG monitoring

VTP : Ventricular tachypacing

Final version 24/1185

WBC White blood cells

WHO-DRUG: World health organization drug reference list

## 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of atrial fibrillation (AF) in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the PUFAs (Polyunsaturated Fatty Acids) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are ALA, EPA and DHA. First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or atrial fibrillation.

Final version 25/1185

The potential anti-arrythmic effects of a PUFA was previously developed in atrial fibrillation: nicotinyl ester of DHA (pro-drug based on DHA delivery) were assessed in a two-week ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of atrial fibrillation (AF) induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll assessed n-3 Polyunsaturated Fatty Acids in the prevention of atrial fibrillation recurrences after electrical cardioversion. All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct electrical cardioversion (ECV) 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95%] confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent atrial fibrillation on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion [2]. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFA on top of traditional treatment (amiodarone, beta blockers, reninangiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than placebo group at one month (3.3% vs 10%; p=0.043), at 3 months (10% vs 25%; p=0.004) and at 6 months (13.3% vs 40%; p<0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effect of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of

Final version 26/1185

functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with a chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for HF were 6% in the n-3 PUFAs and 30% in the placebo group (p < 0.0002).

Moertl and coll **[4]** performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (P = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, P = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent atrial fibrillation and heart failure in the maintenance of sinus rhythm after electrical cardioversion.

## 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA (docosahexaenoic acid) is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of atrial fibrillation.

F373280 is a prodrug of DHA.

Final version 27/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

## 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

## 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

Trimethylpentane: Slightly soluble

Final version 28/1185

#### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period (AERP) were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased AERP (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, P<0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the ECG intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing (VTP)-induced congestive heart failure (CHF) provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses CHF-induced AF-promotion and fibrosis in the VTP canine model. Nicotinyl ester of DHA was tested in this model, at 1g/day and 5g/day, during 4 weeks, to prevent CHF-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in atrial fibrillation duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus  $637 \pm 196$  sec, n=5 in the presence of 1g/kg/d Nicotinyl ester of DHA and  $79 \pm 51$  sec, n=5, in the presence of 5g/kg/d Nicotinyl ester of DHA The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280

Final version 29/1185

similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the

compound may exert a similar protective effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 gm/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 30/1185

6 consecutive single ascending doses were tested (0.5g, 1g, 2g, 4g, 8g and 16g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 4 were observed in the placebo group (palpitation, dizziness in standing position, 2 symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events were reported in the groups of F373280 at the dosages of 0.5g, 1g, 2g, 4g and 8g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5g to 16 g in 36 young male healthy subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirm that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding PK parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16g with no departure from proportionality (baseline corrected parameters).

Final version 31/1185

#### Part B: Multiple dose

Three consecutive repeated ascending doses (1, 2 and 4g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280 5/9 TEAE were classified according the SOC in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAE have already been reported with Poly Unsaturated Fatty Acids and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 32/1185

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of atrial fibrillation (AF) induced by burst pacing [1].

Moreover, the effectiveness of PUFA has been proven in the following conditions:

- Prevention of atrial fibrillation recurrence in patients with persistent atrial fibrillation in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

#### 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor®, [9]:

Final version 33/1185

- The frequencies of adverse reactions are ranked according to the following: common (> 1/100, < 1/10); uncommon (>1/1000 < 1/100); rare (>1/10000, < 1/1000); very rare ( < 1/10000), not known (cannot be estimated from the available data).
  - The reported adverse events are:
- Infection and infestations

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

• Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

• Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

Final version 34/1185

#### • Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1g and 4g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in Atrial Fibrillation studies [2, 8]. The range of PUFAs doses tested was between 2g to 3g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in heart failure patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1g to 5g (1g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Final version 35/1185

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

#### 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct electrical cardioversion
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

Final version 36/1185
After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of atrial fibrillation and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (AVK), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication,
- Anticoagulation with anti-vitamin K for at least 3 weeks before ECV,
- ECV in patients with stabilized INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

Final version 37/1185

- Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent atrial fibrillation and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35  $\pm$  2D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit

Final version 38/1185

- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent atrial fibrillation and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent atrial fibrillation with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters,
  morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- early persistent atrial fibrillation history (less than one year) with a duration of a the current episode between 7 days to 6 months
- a moderately abnormal moderately systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- A Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or

Final version 39/1185

unstable ischemic coronaropathy (assessed by coronarography or cardiac stress test or effort test within 6 months before selection).

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on anti-arrhythmics on atrial fibrillation (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be developed as a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, anti-arhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent atrial fibrillation and requiring an electrical cardioversion will be included in order to assess the time to first documented recurrence of atrial fibrillation since cardioversion.

To confirm the persistent nature of atrial fibrillation, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before electrical cardioversion. According to guidelines for the management of atrial fibrillation [6], anti-vitamin K should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation, of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodary study [2], the duration of pre-treatment with PUFA before cardioversion appears to be a contributing factor in

Final version 40/1185

success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of atrial fibrillation recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of atrial fibrillation recurrence occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using a more easy to carry and easy to use device, a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

#### 4.2.3. Choice of the Dose

According to a previous study in patients with atrial fibrillation [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of atrial fibrillation after cardioversion. Moreover, PUFAs at dosage of 1g and 2g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95mg/mL and 60 to 90mg/mL, respectively) (phase I study of F373280 and Salm and coll study) [16]. With regard to the rythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA.Therefore, a dose of 1 g daily of F373280 is considered to be appropriate to be tested in this POC study.

Final version 41/1185

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive),
- 2. Patient with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:
  - use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
  - documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion

## Ethical /legal considerations:

- 12. Having signed his/her written informed consent,
- 13. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation),

## 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

1. History of first documented episode of persistent AF more than 1 year,

Final version 42/1185

- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be check in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (K > 5.5 mEq/L or K < 3.5 mEq/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship.

#### **5.3. NUMBER OF PATIENTS**

76 x 2 patients (taking into account 15 % of non evaluable patients).

Final version 43/1185

#### 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO,...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENTS IDENTIFICATION

The patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

#### 5.6. WITHDRAWAL CRITERIA

The reasons for a patient's premature withdrawal from the study may be the following:

- The patient's decision. A patient who wishes to withdraw from the study for any reason may do so at any time but must inform the investigator. In all cases, the Investigator should attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form
  - obtain the reason(s) for withdrawal and report it/them in the case report form
  - evaluate the patient's clinical condition
  - if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- The Investigator's decision in the patient's interest. Particularly, if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.

Final version 44/1185

- An erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion / non inclusion criteria will immediately be withdrawn and an appropriate treatment will be instored by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with anti-vitamin K for at least 3 weeks before ECV,
- Patients who will not stabilize INR between 2 and 3 on at least 3 consecutive weekly tests
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 week for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV (i.e. unsuccessful ECV) will be considered to have finished follow-up.
- An occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and uncomfortable clinical symptoms.

#### 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit, a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator

Final version 45/1185

and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83.

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.

# 6.1. SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT

F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

Final version 46/1185

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number,
- c) packaging batch number,
- d) the treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
  - "for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose".

On the treatment unit, another label will be affixed with the mention of the investigator name and patient number (completed by the investigator).

In addition, on each case, will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

Final version 47/1185

## 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person.

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

Final version 48/1185

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion Visit and another one at Visit 6.

For each patient, the treatment number given at Visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Calls the vocal server
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the vocal server.
- The IVRS/IWRS company:
  - Confirms this information by fax/email to the Investigator
  - Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 5, the Investigator will contact again the IVRS/IWRS to obtain for visit 6 the treatment number for the last 12-week period of treatment according to the same process as described above.

Final version 49/1185

#### 6.5. DRUG ADMINISTRATION

## **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure will be 24 weeks, with F373280 or placebo.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

## 6.6. ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT

The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

Final version 50/1185

## 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator, in collaboration with the Sponsor representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF, according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (Selection Visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on e-CRF. All treatments should be evaluated by the investigator at selection and their prolongation during the study or their stop should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

Final version 51/1185

#### 7.1. ANTI-VITAMIN K TREATMENT

Anti-vitamin K should be given for at least 3 weeks before ECV and continued for the whole study duration. The anti-vitamin K used will be left to the decision of the each investigator according to his/her local practice.

## 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
    - Class IA: Disopyramide, Procainamide, Quinidine
    - Class IB: Lidocaine, Mexiletine
    - Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Any Polyunsaturated Fatty Acid (PUFA)
- Any anticoagulant treatment other than antivitamin K: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

#### 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the case report form. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

Final version 52/1185

## 8. EVALUATION CRITERIA

## **8.1. PRIMARY EFFICACY CRITERION:**

## **8.1.1.** Time to the first Atrial Fibrillation Recurrence

## 8.1.1.1. Definition

Time to first Atrial Fibrillation recurrence is defined by the first episode of Atrial Fibrillation (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of electrical cardioversion visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

#### 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM)

• Trans Telephonic ECG Monitoring (TTEM):

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 to visit 6. Then, every two days from visit 6 to visit 9.

Moreover, during this TTEM period, if patient experiences AF symptoms, it should be documented using the TTEM.

Final version 53/1185

In case of AF recurrence, and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at the investigator's judgement, he/she could be maintained in the study with the treatment, in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

## 8.1.2. Secondary Efficacy Criteria

# 8.1.2.1. Numbers of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

## 8.1.2.1.1. *Definition*

Number of Atrial Fibrillation episodes will consist in the assessment of episodes of AF with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

## 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the study visit 4.

#### 8.1.2.1.3. Evaluation Methods

## • 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

Final version 54/1185

# 8.1.2.2. Duration of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

## 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episodes.

## 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the follow up study visit (visit 4).

#### 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

## 8.1.2.3. Clinical parameters evaluation

## 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition:

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

Final version 55/1185

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month); intermediate (1/month to almost daily); and frequent at least daily.

#### 8.1.2.3.1.2. Schedule

This evaluation will be performed in case of symptoms evocative of arrhythmia.

## 8.1.2.3.1.3. Evaluation Methods

This evaluation will be collected by Central Reading Laboratory during all the study period.

## 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of number of AF recurrence associated with a symptom (Palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG in atrial fibrillation.

## 8.1.2.3.3. Number and duration of hospitalization

- Number and duration of hospitalization for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
  - Hospitalization for myocardial infarction
  - All cause of hospitalization
- Number and duration of hospitalization for thromboembolic stroke

## 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

Final version 56/1185

## 8.1.2.5. Evolution of echocardiographic parameters

## 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), Left atrial area (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m<sup>2</sup>, Left ventricular end diastolic diameter (mm) Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL),

## 8.1.2.5.2. Schedule

The measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

The measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

## 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, for volume measurements, the recommended method is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

## 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

## 8.2.1. Definition

Because of the limited accessibility of human tissues for biopsy, red blood cell DHA contents is a marker for tissue DHA concentration [13], [14].

Final version 57/1185

## 8.2.2. Blood samples

## 8.2.2.1. Collection schedule

Blood samples will be collected for determination of red blood cells (RBC) concentrations of DHA.

Blood samples will be performed as follows:

• Visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the electronic Case Report Forms (e-CRFs).

## 8.2.2.2. Technical handling

Two blood samples will be collected containing EDTA. They will be gently shaken and centrifuged at 3000g for 15 min at room temperature, within 30 minutes after collection. Plasma and white blood cells will be discarded. Red blood cells will be stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C) within 3 weeks following collection. Analysis will be performed within 2 weeks following reception at the Analytical centre.

#### **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol, after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will

Final version 58/1185

be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells

(expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk

for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end

of the study, and will be provided only at the end of the study (after database lock), in a separate

file.

8.3. SAFETY ASSESSMENT

8.3.1. Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the

occurrence of adverse events (AEs) since the last visit will be based on the patient's spontaneous

reporting, the investigator's non-leading questioning and his/her clinical evaluation. All AEs will

be reported on the e-CRF (see section 10).

8.3.2. Laboratory Investigations

8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of

treatment) or End of Treatment visit.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The volume of blood samples complete haematology, biochemistry should not exceed 30 mL.

8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells

(WBC) count, WBC differential counts (% and absolute), platelets.

<u>Chemistry</u>: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate

Final version 59/1185

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning, in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula

Cockeroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L],

in women:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patients' interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

## 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

## 8.3.4.1. Schedule

Vital signs will be measured at each visit.

Final version 60/1185

#### 8.3.4.2. Technical Procedure and Parameters

Systolic (SBP) and diastolic (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation, after at least 5 minutes in supine position and after 2 minutes in standing position by counting the beats for at least 30 seconds.

Bodyweight will be measured in patient in underwear and with the same balance at each visit.

## 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An electrocardiogram will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

## 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram (ECG):

The global interpretation from manual reading (normality, clinical relevance) and heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

#### • 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent atrial fibrillation.

## 8.3.6. Coagulation parameters

The assessment of coagulation will be evaluated by the following parameters:

Final version 61/1185

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV,
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV,
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by anti-vitamin K should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial can be found in section 7.

## 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back any remaining soft capsules, blister, case (used or unused) at the following visit.

At each visit, the Investigator will record the number of supplied and remaining Soft Capsules in the e-CRF.

Final version 62/1185

## 9. STUDY PROCEDURES

## Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If he/she accepts to participate in the study, he/she will sign the informed consent and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and Atrial Fibrillation characteristics
- Echocardiography using a two-dimensional echocardiography.
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

Final version 63/1185

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory (CRL). The CRL will send his/her assessment regarding the confirmation of persistent atrial fibrillation within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will contact the IVRS/IWRS system to confirm the patient selection and order the treatment delivery and organise the appointment for the next visit.

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

Final version 64/1185

Visit 2 - Inclusion Visit (Day 1)

If the patient's behaviour during the selection period and/or the result of complementary

examinations particularly the confirmation of the presence of persistent atrial fibrillation by the

CRL during this period, the INR and laboratory tests, are compatible with the inclusion criteria,

the patient will be assessed for the following:

Adverse events

• Concomitant treatments (authorised, disallowed)

• Laboratory examination: red blood cell concentrations of DHA and coagulation parameters

Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin

Clotting Time (TCT)

Global Physical examination/bodyweight

Vital signs

• Echocardiography using a two-dimensional echocardiography.

• 12-lead ECG

• Urine pregnancy test for women of child bearing potential.

If the results of the above assessments are compatible with the inclusion criteria, the patient will

be included and allocated a treatment number using the IVRS/IWRS system.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to

paragraph 8.3.6), in order to ensure that the INR is stable, between 2 to 3 before electrical

cardioversion.

At the end of the visit, the Investigator will organise the appointment for the next visit and give

the treatment to be taken during the next 4-week period.

Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Patient will be assessed for the following criteria:

Final version 65/1185

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Red Blood Cell concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO -TE (transesophageal echocardiograph) performed in the same day (before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

Final version 66/1185

## Visit 4 (Week 5: D35 $\pm$ 2 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of Adverse Events
- Concomitant treatments (authorised, disallowed)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device (Trans Telephonic ECG Monitoring) for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG

Final version 67/1185

• The cardiac monitoring will be continued using a TTEM device (Trans Telephonic ECG Monitoring). The device will be given to the patient who will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week treatment period.

#### In addition:

- at visit 5, the investigator will contact the IVRS/IWRS to obtain another treatment unit to be dispensed at visit 6 for the last 12-week period.
- at visit 6, an echocardiography will be performed and, the red blood cell concentration of DHA will be measured.

## End-of-Study Visit - Visit 9 (Week 24: D168 $\pm$ 7 days)

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential

Final version 68/1185

• Echocardiography using a two-dimensional echocardiography

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused soft capsules.

## 10. ADVERSE EVENTS: DEFINITION AND REPORTING

## 10.1. ADVERSE EVENTS

## 10.1.1. Definition of Adverse Events

An adverse event is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

This includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values, which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified

## 10.1.2. Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity.

Final version 69/1185

## **10.1.3.** Reporting of Adverse Events

The records of adverse events in the electronic Case Report Form (e-CRF) describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

## 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A serious adverse event (SAE) includes, but is not necessarily restricted to any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect.

Other events such as cancer, and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough, or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

- \* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:
  - planned (as per protocol) medical/surgical procedure,
  - preparation for routine health assessment/procedure (e.g. routine colonoscopy),
  - planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required),
  - administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

Final version 70/1185

will not be reported as a SAE.

10.2.2. Reporting of SAE

All serious adverse events, according to the above-mentioned definitions and regardless of

treatment or relationship to study drug, must be recorded by the Investigator as soon as he/she is

informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the

"Notification of serious adverse event" form ("first notification") (see appendix 17.2) with all the

available information about the event, to the Sponsor's representative:

Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE.

Centre de R&D Pierre Fabre – BP 13562

3 Avenue Hubert Curien

31035 TOULOUSE Cedex 1

Phone: +33 5 35 50 63 48

Fax: +33 5 34 50 65 92

Email: marlene.guiraud@pierre-fabre.com

In case of non-inclusion the reporting period ends when the non-inclusion is documented.

10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious

adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out

examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be

notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for

the patient which may be related to the study treatment in the Investigator's opinion.

Final version 71/1185

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage, and associated adverse event if any, are reported only on the Adverse Event page of the CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must be also transmitted to the sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug(s) should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is discontinued from the study.

The investigators must report to the sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The investigator must immediately notify the sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Women who become pregnant after exposure to the study drug must be followed by the investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the sponsor (baby's healthy status).

Final version 72/1185
# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

## 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An electronic Case Report Forms (e-CRF) will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files and which will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants who will use this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation.

Final version 73/1185

At the end of the study, a CD-ROM containing the pdf version of all e-CRF (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

#### 11.2. STUDY MONITORING

## 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

## 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

Final version 74/1185

## 11.2.1.2. Initiation Visit

Before the start of the study at all investigation sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
  - has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

## 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

• Verify that the e-CRFs CD-ROM with pdf files are correctly stored

Final version 75/1185

- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes,
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

## 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of measures of primary end point, the safety data and to recommend to the Sponsor whether to continue, modify, or to stop the study.

The IDMC operating procedures will be described in an independent document.

## 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

Final version 76/1185

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on a e-CRF.

The e-CRF used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate coding.

## 12.4. DATA STORAGE

The computer data files, as well as their modifications, will be archived by the subcontractor and kept available upon request of the Sponsor.

Final version 77/1185

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e.: data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

## 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by Pierre Fabre Biométrie (PFB) or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan (SAP) approved by the Validation Committee.

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

## 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 evaluable patients per group is required to achieve, using a log-rang test of survival curves with a 80 % power and a 5 % two-sided significance level.

Final version 78/1185

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

## 13.4. DATA SETS ANALYSED

The following 2 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses.

Final version 79/1185

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

## **13.5.1. Dropouts**

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

## 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

## 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

## 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- <u>Quantitative parameters</u> will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

Final version 80/1185

## 13.7. EFFICACY ANALYSIS

## 13.7.1. Primary Criterion

## 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

## 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

## 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

## 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

## 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

## 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

Final version 81/1185

## 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

## 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

#### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patients will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

Final version 82/1185

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event.
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAE
- With at least three TEAE
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.
- Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:
- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Final version 83/1185

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

"The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TE AE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (for all patient).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

Serious adverse events will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

## 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all blood laboratory parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate. Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower

Final version 84/1185

and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

Clinically noteworthy abnormal laboratory values (CNALV) (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

## 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

Final version 85/1185

## 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

## 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and heart rate in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

## 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

Final version 86/1185

## **13.8.6.** Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

## 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" (ATC) classification on the safety set.

## 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated \_actual \_consumption}{Theoretical \ consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) – number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days).

## 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

Final version 87/1185

## 14. GENERAL ETHICAL CONSIDERATIONS

## 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

## 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

Final version 88/1185

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study.

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

## 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

Final version 89/1185

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament, are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

## 15. ADMINISTRATIVE PROCEDURES

## 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

## 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF, drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not

Final version 90/1185

- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents
- Authorises direct access to source documents for monitoring, audits and inspections
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

## 15.3. END OF THE STUDY

## 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

## 15.3.2. Early Study Termination

## 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

## 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if it considers that the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

Final version 91/1185

#### **15.4.** AUDIT

The Sponsor is responsible for making sure that both his representatives (Study Manager, CRA, ...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

#### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed to in writing with the Study Manager, the investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

## 15.7. CLINICAL STUDY REPORT

Data analysis, and clinical study report writing are under the Sponsor's responsibility.

Upon completion of the data analysis, a final report, including a review of the objectives and methods, a presentation and discussion of the results are drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

Final version 92/1185

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

#### 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

## 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

Final version 93/1185

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 94/1185

## 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version October 2012
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 95/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

[14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83 : 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 96/1185

## [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

## [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

## [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

## [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

## [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 97/1185

## 17. APPENDICES

Final version 98/1185

#### 17.1. DECLARATION OF HELSINKI

## WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 99/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 100/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 101/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

## C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 102/1185

## 17.2. SAE REPORT FORM

Final version 103/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE PRODUCT SAFETY DEPARTMENT |
|---|
| TO BE TRANSMITTED TO THE MONITOR BY FAX WITHIN 24H: M. GUIRAUDFax n° +33 5 34 50 65 92 |
| Transmission date |
| SAE N° FIRST NOTIFICATION FOLLOW-UP |
| > SUBJECT CHARACTERISTICS |
| Surname Birth date Birth date |
| Gender1=M, 2=F Heightcm Weight kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date |
| Seriousness onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| Date of first study treatment administration (ddmmyyyy) |
| Date of last study treatment administration before the occurence of SAE (ddmmyyyy) |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |
| 1 |

Final version 104/1185

| INN or trade name | Daily dose | Start date (ddmmyy) | Ongoing at occurence of the event | Stop date (ddmmyy) | Route of admin. | Indication |
|---|---|---|---|---|---|---|
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAK | EN FOLLOWI | NG THE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage mod | ification, specify | / : | Modi | fication Date : | / | / |
| ☐ Temporarily | ☐ Temporarily discontinued Readministration date :// | | | | | |
| ☐ Withdrawn | | End date :// | | | | |
| ☐ Not applicab | ole | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription | of corrective or | symptomatic treatme | ents (specify names and | d dosages): | | |
| ☐ Discontinuation of concomitant treatments (specify names): | | | | | | |
| | | | • | | | |
| ☐ Others, spec | 11y : | | | | | |
| > OUTCOME | | | | | | |
| | ☐ Not recovered/Not resolved ☐ Recovering/Resolving ☐ Recovered/Resolved | | | | | |
| ☐ Recovered/Res | ☐ Recovered/Resolved with sequelae ☐ Fatal ☐ Unknown | | | | | |
| In case of de | ath, has an autop | sy been conducted? | ☐ Yes ☐ No | | | |
| | CAUSALITY A | ASSESSMENT (inve | estigator's assessmen | t to be done as soor | as possible) | |
| ➤ INVESTIGATOR | | | | | | |
| | | • | | | | |
| ➤ INVESTIGATOR □ Not Suspected comments: | □ Sus | • | Insufficient data | | | |

Final version 105/1185

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| TO THE TOTAL | Protein | g/1 | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/l | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pH | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 106/1185

<sup>(

)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

## **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | <ul> <li>Decrease of at least 2g/dl and value &lt; 10 g/dl whatever the baseline value</li> <li>If missing baseline: value &lt;10g/dl</li> </ul> |
| NEUTROPHILS WBC (if missing value for neutrophils) | | • < 1 500/mm $^3$ whatever the baseline value • < 3 000/mm $^3$ whatever the baseline value |
| SERUM CREATININE | | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N: <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline: <ul> <li>TB &gt; 1.5 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>TB &gt; 2 N</li> </ul> </li> </ul> |

## N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 107/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | HR ≥ 110 bpm and increase ≥ 10 bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Chan<br>Post-baseline Vo | ge from Baseline<br>alue | to the Maximum | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>aseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | A11 | A11 | A11 | All |
| ≥ 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the for each parame | | aseline Value | |
|---|---|---|---|---|---|---|
| | SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| | < 120 | < 80 | ≤50 | ≤90 | ≤ 50 | ≤50 |
| | [120;140] | [80;90[ | <i>[50 ;75]</i> | [90 ;120] | [50;80[ | [50;75] |
| | [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| | ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3BI 2 90 01 DBI 2 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq 20$ mmHg or DBP Decrease $\geq 10$ mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 108/1185
16.1.1.2. Protocol and appendices (version 2: 15 January 2013)

Final version 109/1185

F 373280 CA 2 01

Final version 110/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

## CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

**Sponsor's Representative:** Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 63 48 Fax:+33 5 34 50 65 92

E-mail:marlene.guiraud@pierre-fabre.com

Pr Savina NODARI Section of Cardiology

**Department of Experimental and Applied Sciences** 

**University of Brescia BRESCIA, ITALY** 

Phone: +39 030 3996 587 - Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>

#### Version 2-15 JAN 2013

**Study Coordinating Investigator** 

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 111/1185

## **SPONSOR PERSONNEL**

## PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

## **Clinical Study Manager (Monitor)**

Marlène GUIRAUD, Pharm D Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Fax: +33 5 34 50 65 92

Phone: +33 5 34 50 63 48

E-mail: marlene.guiraud@pierre-

fabre.com

## **Head of Therapeutic Area**

Alain DELARUE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1

Phone: + 33 5 34 50 61 88 Fax: +33 5 34 50 65 92

E-mail: alain.delarue@pierre-

fabre.com

## **Clinical Development Physician**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3. Avenue Hubert Curien 31035 TOULOUSE Cedex 1

Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 65 92 E-mail: richard.roche@pierre-

fabre.com

Final version 112/1185

## CONTRACT RESEARCH ORGANISATIONS

## For Feasibility, Monitoring and Regulatory issues:

Pharmaceutical Service Network (PSN)

Rufino Gonzalez 28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

## For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6, Chaussée de Boondael B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

## For Centralised Reading of Holder ECG and TTEM and equipment supply:

## **Biomedical System**

1945 Chaussée de Wavre B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

## For intra erythrocyte DHA dosage

## **Agrocampus Ouest**

Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

Final version 113/1185

# Protocol F 373280 CA 2 01

## APPROVAL FORM

Protocol Version 2 – 15 JAN 2013

| Sponsor's Representative: | | £3.* |
|---|---|---|
| Head of Therapeutic Area: Alain DELARUE, MD | Date: | Signature: |
| | 18 January 20-13 | HOLL |
| I con from that my orogonal sugnature was dated in 18 January | 2013. | er 2013 |
| Study Coordinating Investigator: Savina NODARI, MD | Date: | Signature: |
| Savina ito prasty itali | 29/02/2013 | Some hode |

## Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

## **Protocol Version 2 – 15 JAN 2013**

| Country: | | |
|------------------------------------|-------|------------|
| Country Coordinating Investigator: | | |
| "Name" | Date: | Signature: |

Final version 115/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

**Protocol Version 2 – 15 JAN 2013** 

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 15 January 2013 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * To be adapted |
|-----------------|
|-----------------|

| Date: | Signature: |
|-------|------------|

Final version 116/1185

# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| <b>1.</b> ] | INTRODUCTION AND STUDY RATIONALE | 21 |
|-------------------|----------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 21 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 23 |
| 1.2.1. | Chemical and pharmaceutical characteristics | 24 |
| 1.2.1. | | |
| 1.2.1.2 | σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ σ | |
| 1.2.2.<br>1.2.2.1 | | |
| 1.2.2.2 | | |
| 1.2.2.3 | | |
| 1.2.2.4 | C 1 | |
| 1.2.3. | Clinical data | 26 |
| 1.3. | STUDY RATIONALE | 29 |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 29 |
| 2. | STUDY OBJECTIVES | 32 |
| 2.1. | PRIMARY OBJECTIVE | 32 |
| 2.2. | SECONDARY OBJECTIVES | 32 |
| <b>3.</b> ] | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 32 |
| 4. | STUDY DESIGN | 34 |
| 4.1. | OVERALL DESCRIPTION | 34 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | $\mathcal{F}$ | |
| 4.2.3. | | |
| 4.2.4. | 1 | |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 38 |
| 5.3. | NUMBER OF PATIENTS | 39 |
| 5.4. | RECRUITMENT MODALITIES | 40 |
| 5.5. | PATIENTS IDENTIFICATION | 40 |
| 5.6. | WITHDRAWAL CRITERIA | 40 |
| 5.7. | REPLACEMENT OF PATIENTS | 41 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 41 |
| 5.9. | STUDY CARD | 41 |

| 6. | STUDY TREATMENT | 42 |
|---|---|---|
| 6.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 42 |
| 6.2. | PACKAGING AND LABELLING | |
| 6.2.1. | Packaging | |
| 6.2.2. | Labelling | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | |
| 6.5. | DRUG ADMINISTRATION | |
| 6.5.1. | Duration of Treatment | |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration. | 46 |
| 6.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 46 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| 7. | CONCOMITANT TREATMENTS | 47 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 48 |
| 7.2. | PROHIBITED TREATMENTS | 48 |
| 7.3. | AUTHORISED TREATMENTS | |
| <b>8.</b> ] | EVALUATION CRITERIA | 49 |
| 8.1. | PRIMARY EFFICACY CRITERION: | 49 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence | 49 |
| 8.1.1. | | |
| 8.1.1.2<br>8.1.1.3 | | |
| 8.1.1.3<br>8.1.2. | B. Evaluation MethodsSecondary Efficacy Criteria | |
| 8.1.2.1 | | 50 |
| | visit) | 50 |
| 8.1.2.2 | | |
| 012 | visit) | |
| 8.1.2.3<br>8.1.2.4 | 1 | |
| 8.1.2.5 | | |
| 8.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF | |
| o. <b></b> | DHA | 53 |
| 8.2.1. | Definition | 53 |
| 8.2.2. | Blood samples | |
| 8.2.2. | | |
| 8.2.2.2<br>8.2.3. | 2. Technical handling | |
| 8.2.3.<br>8.3. | SAFETY ASSESSMENT | 55 |
| ()). | DATEL ADDEDONIONI | |

| 8.3.1. Adverse Events | 55 |
|-----------------------------------------------------------------|----|
| 8.3.2. Laboratory Investigations | 55 |
| 8.3.2.1. Schedule | 55 |
| 8.3.2.2. Technical Procedures and Parameters | 55 |
| 8.3.3. Global Physical Examination | 56 |
| 8.3.4. Vital Signs | 56 |
| 8.3.4.1. Schedule | |
| 3.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.3.7. Concomitant Treatments | |
| 8.4. COMPLIANCE | 58 |
| 9. STUDY PROCEDURES | 59 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 64 |
| 10.1. ADVERSE EVENTS | 64 |
| 10.1.1. Definition of Adverse Events | 64 |
| 10.1.2. Grading of Adverse Events | |
| 10.1.3. Reporting of Adverse Events | 65 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 65 |
| 10.2.1. Definition | 65 |
| 10.2.2. Reporting of SAE | 66 |
| 10.2.3. Follow-up of SAE | 67 |
| 10.2.4. SAE Occurring After the Study | 67 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 67 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 67 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES. | |
| 11. DATA COLLECTION AND STUDY MONITORING | 68 |
| 11.1. DATA COLLECTION | 68 |
| 11.1.1. Case Report Form | 68 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | 70 |
| 11.2.1. Monitoring visits | 70 |
| 11.2.1.1. Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | 71 |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | 71 |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | 72 |
| 12 DATA MANACEMENT | 72 |

| 12.1. DATA ENTRY | 72 |
|---|---|
| 12.2. DATA CLEANING | 72 |
| 12.3. DATA CODING | 73 |
| 12.4. DATA STORAGE | 73 |
| 12.5. DATABASE LOCK | 73 |
| 13. STATISTICAL ANALYSIS | 73 |
| 13.1. GENERAL CONSIDERATIONS | 74 |
| 13.2. SAMPLE SIZE | 74 |
| 13.3. PROTOCOL DEVIATIONS | 74 |
| 13.4. DATA SETS ANALYSED | |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 76 |
| 13.7. EFFICACY ANALYSIS | 76 |
| 13.7.1. Primary Criterion | 76 |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | 76 |
| 13.7.2. Secondary Criteria | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | 81 |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 83 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 83 |
| 14.1. ETHICAL CONDITIONS | 83 |
| 14.2 ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 83 |

| 14.3. | PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 84 |
|---|---|---|
| 14.4. | PERSONAL DATA PROTECTION | 85 |
| 14.5. | INSURANCE POLICY | 85 |
| 15. | ADMINISTRATIVE PROCEDURES | 85 |
| 15.1. | PROTOCOL AMENDMENT | 85 |
| 15.2. | SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 86 |
| 15.3. | END OF THE STUDY | 86 |
| 15.3. | J | |
| 15.3. | | |
| | 2.1. Early Study Termination Decided by the Sponsor | |
| | 2.2. Early Study Termination Decided by the Competent Authorities | |
| 15.4. | AUDIT | 87 |
| 15.5. | INSPECTION | 88 |
| 15.6. | CONFIDENTIALITY | 88 |
| 15.7. | CLINICAL STUDY REPORT | 88 |
| 15.8. | STUDY RESULTS COMMUNICATION | 88 |
| 15.9. | STUDY RESULTS PUBLICATION | 88 |
| 16. | REFERENCES | 90 |
| <b>17.</b> | APPENDICES | 93 |
| 17.1. | DECLARATION OF HELSINKI | 94 |
| 17.2. | SAE REPORT FORM | 98 |
| 17.3. | PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 101 |

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of Atrial Fibrillation (AF) induced by burst pacing.[1] Moreover, the effectiveness of PUFA (PolyUnsaturated Fatty Acid) has been proven in the following conditions: — prevention of Atrial Fibrillation recurrence in patients with persistent Atrial Fibrillation, in co-administration with amiodarone (add on therapy) [2] — Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – April 2014 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 (anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> <li>Treatment duration: 24 weeks</li> </ul> |
| Study Schedule | <ul> <li>9 visits will be scheduled:</li> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (Outpatient or hospitalization according to</li> </ul> |

Final version 122/1185

| | <ul> <li>clinical practice of the centre) (installation of the Holter device)</li> <li>V4/ W5 (D35± 2 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V5/ W8 (D56± 7 days): follow-up visit</li> <li>V6/ W12 (D84± 7 days): follow-up visit</li> </ul> |
|---|---|
| | - V6/ W12 (D64 ± 7 days): follow-up visit - V7/ W16 (D112 ± 7 days): follow-up visit - V8/ W20 (D140 ± 7 days): follow-up visit - V9/ W24 (D168 ± 7 days): final study visit |
| Number of Patients: | 76 x 2 patients |

#### Diagnosis and Criteria for Inclusion:

#### **Inclusion Criteria:**

Demographic Characteristics and Other Baseline Characteristics:

- Men or women aged more than 18 years (inclusive),
- Patients with persistent AF between 7 days and 6 months duration for whom electrical 2. cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- History of ischemic or non ischemic heart failure
- NYHA class I or II chronic heart failure at selection and at inclusion
- Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) ) at selection and at inclusion
- On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- Left atrial area  $\leq 40 \text{ cm}^2$ ) at selection and at inclusion
- 9. Patients treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:
  - use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment
  - documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion

#### Ethical /legal considerations:

- 12. Having signed his/her written informed consent,
- 13. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

## Non-Inclusion Criteria:

Criteria related to pathologies:

- History of first documented episode of persistent AF more than 1 year
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
- NYHA class III or IV heart failure at selection or at inclusion
- Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- Bradycardia (HR ≤ 50 bpm)
- Hyperkalemia or hypokalemia (K>5.5 mEq/L or K  $\leq$  3.5 mEq/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

Final version 123/1185

| | <ul> <li>Criteria related to treatments:</li> <li>11. Previously ineffective pharmacological or electrical cardioversion</li> <li>12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers</li> <li>13. Previous treatment with oral amiodarone within 12 months prior to inclusion</li> <li>14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion</li> <li>15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months</li> <li>16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months</li> <li>17. Dietary supplement with ω3 or ω6 according to investigator's judgement</li> <li>18. Having undergone any form of ablation therapy for AF</li> <li>19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel</li> </ul> |
|---|---|
| | <ul> <li>Other criteria:</li> <li>20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion</li> <li>21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection</li> <li>22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints</li> <li>23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator</li> <li>24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship</li> <li>25. Breastfeeding female patient</li> </ul> |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV) ECV will be performed in patients without dyskalemia If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280<br>Soft Capsules |
| Dose: | Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules Placebo will be administered in the same conditions as the tested product. |
| Mode of Administration: | Oral, one capsule each evening with dinner |
| Evaluation Criteria: | <ul> <li>Efficacy evaluation variables:</li> <li>Primary evaluation variable:</li> <li>Time to first Atrial Fibrillation recurrence defined by the first episode of Atrial Fibrillation lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit) Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24.</li> <li>For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).</li> <li>Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM.</li> <li>All ECG traces will be evaluated by a Central Reading Laboratory.</li> </ul> |
| | December of the tention of the tenti |

Final version 124/1185

During the 7-day continuous ECG monitoring,

- Numbers of AF episodes
- Duration of AF episodes

## Clinical parameters:

During the whole study:

- Number of recurrence of symptomatic AF episodes
- EHRA score
- Hospitalization for cardiovascular events
- Hospitalization for thromboembolic stroke
- All cause of hospitalization

#### Cardioversion:

- Assessment of spontaneous cardioversion
- Assessment of successful cardioversion
- Number of patients needing an other cardioversion after the initial ECV

#### Other:

- Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m², Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))
- Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).

#### Safety criteria:

- Adverse events (observed and / or spontaneously reported)
- Vital signs (Blood pressure (supine and standing), heart rate
- Physical examination (body weight),
- Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized).
- Haematology: haematocrit, haemoglobin, RBC, WBC, differential count, platelets
- **Biochemistry:** sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (*local laboratory*)
- Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR (local laboratory), Prothrombine Time (PT)

#### **Statistical Methods:**

## Sample Size:

Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%.

## **Primary Efficacy Analysis**

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### Secondary Analyses

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

## Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment)

Final version 125/1185

## STUDY FLOW-CHART

Final version 126/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 +/-2 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | х | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic characteristics | х | | | | | | | | |
| Medico-surgical history | х | | | | | | | | |
| Concomitant disease | х | | | | | | | | |
| Concomitant treatment | х | х | х | х | х | х | х | x | х |
| Habits | х | | | | | | | | |
| Global physical examination (body weight) | х | х | х | | х | х | х | х | х |
| Echocardiography | х | х | | х | | х | | | х |
| Eligibility criteria check | х | х | | | | | | | |
| Blood pressure, heart rate | х | х | х | х | х | х | х | х | х |
| 12-Lead ECG Recording | х | х | х | | х | х | х | х | х |
| INR | <b>—</b> | | (2) | | х | х | х | х | х |
| аРТТ, ТСТ | х | х | х | | х | х | х | x | х |
| Biochemistry | х | | | | | | | | x |
| Hematology | х | | X | | | X | | | х |
| Urinary pregnancy test | | х | | | | | | | x |
| Red Blood Cell concentrations of DHA | | х | х | | | х | | | x |
| Treatment allocation | | х | | | | х | | | |
| IVRS | х | х | | | х | х | | | |
| ECV (3) | | | х | | | | | | |
| Drug administration | | <b>—</b> | | | | | | | <b></b> |
| Adverse events recording | | х | х | х | х | х | х | x | x |
| Holter ECG | (4) | | <b>←</b> | (5) | | | | 4 | |
| TTEM (6) | | | | | | | 24 ( | | $\rightarrow$ |

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)

Final version 127/1185

<sup>(2)</sup> In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(5) 7-</sup>day Holter ECG

<sup>&</sup>quot;O'TTEM everyday from week 6 to week 8. Then every 2 days from week 9 to week 24. In case of AF symptoms. In case of AF recurrence for at least 10 minutes and the patient does not stop the study treatment then TTEM every 4 weeks

## LIST OF ABBREVIATIONS

aPTT Activated partial thromboplastin time

AE : Adverse event

AERP Atrial effective refractory period

AF : Atrial fibrillation
ALA Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK Anti vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP Blood pressure
BSA : Body Surface Area

CEP Protocol evaluation committee

CHF : Congestive heart failure

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO –TE Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA European heart rhythm association

EPA Eicosapentaenoic acid eCRF Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

Final version 128/1185

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL High density lipoprotein

HF Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR International normalized ratio
IRPF: Institut de Recherche Pierre Fabre
IVRS Interactive voice response system

LAA Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL Low density lipoprotein LOQ : Limit of quantification

LVEF Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR Mineralocorticoid receptor
MR perfusion Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie
POC Proof of concept

PUFA : PolyUnsaturated fatty acid

PK : Pharmacokinetics

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT Thrombin clotting time

TEAEs Treatment emergent adverse events
TTEM TransTelephonic ECG monitoring

VTP : Ventricular tachypacing

WBC White blood cells

WHO-DRUG: World health organization drug reference list

Final version 129/1185

## 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of atrial fibrillation (AF) in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the PUFAs (Polyunsaturated Fatty Acids) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are ALA, EPA and DHA. First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or atrial fibrillation.

The potential anti-arrythmic effects of a PUFA was previously developed in atrial fibrillation: nicotinyl ester of DHA (pro-drug based on DHA delivery) were assessed in a two-week

Final version 130/1185

ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of atrial fibrillation (AF) induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll assessed n-3 Polyunsaturated Fatty Acids in the prevention of atrial fibrillation recurrences after electrical cardioversion. All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct electrical cardioversion (ECV) 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95%] confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent atrial fibrillation on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion [2]. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFA on top of traditional treatment (amiodarone, beta blockers, reninangiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than placebo group at one month (3.3% vs 10%; p=0.043), at 3 months (10% vs 25%; p=0.004) and at 6 months (13.3% vs 40%; p<0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effect of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Final version 131/1185

Nodari and coll [3] performed a trial in patients with a chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (P = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, P = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent atrial fibrillation and heart failure in the maintenance of sinus rhythm after electrical cardioversion.

#### 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA (docosahexaenoic acid) is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of atrial fibrillation.

F373280 is a prodrug of DHA.

Final version 132/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

## 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

## 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

Trimethylpentane: Slightly soluble

Final version 133/1185

## 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an  $IC_{50}$  value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period (AERP) were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased AERP (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, P<0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the ECG intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing (VTP)-induced congestive heart failure (CHF) provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses CHF-induced AF-promotion and fibrosis in the VTP canine model. Nicotinyl ester of DHA was tested in this model, at 1g/day and 5g/day, during 4 weeks, to prevent CHF-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in atrial fibrillation duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus  $637 \pm 196$  sec, n=5 in the presence of 1g/kg/d Nicotinyl ester of DHA and  $79 \pm 51$  sec, n=5, in the presence of 5g/kg/d Nicotinyl ester of DHA The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280

Final version 134/1185

similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the

compound may exert a similar protective effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 gm/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 135/1185

6 consecutive single ascending doses were tested (0.5g, 1g, 2g, 4g, 8g and 16g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 4 were observed in the placebo group (palpitation, dizziness in standing position, 2 symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events were reported in the groups of F373280 at the dosages of 0.5g, 1g, 2g, 4g and 8g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5g to 16 g in 36 young male healthy subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirm that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding PK parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16g with no departure from proportionality (baseline corrected parameters).

Final version 136/1185

## Part B: Multiple dose

Three consecutive repeated ascending doses (1, 2 and 4g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280 5/9 TEAE were classified according the SOC in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAE have already been reported with Poly Unsaturated Fatty Acids and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 137/1185

### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of atrial fibrillation (AF) induced by burst pacing [1].

Moreover, the effectiveness of PUFA has been proven in the following conditions:

- Prevention of atrial fibrillation recurrence in patients with persistent atrial fibrillation in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor®, [9]:

Final version 138/1185

- The frequencies of adverse reactions are ranked according to the following: common (> 1/100, < 1/10); uncommon (>1/1000 < 1/100); rare (>1/10000, < 1/1000); very rare ( < 1/10000), not known (cannot be estimated from the available data).
  - The reported adverse events are:
- Infection and infestations

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

• Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

Final version 139/1185

## • Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1g and 4g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in Atrial Fibrillation studies [2, 8]. The range of PUFAs doses tested was between 2g to 3g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in heart failure patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1g to 5g (1g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Final version 140/1185

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct electrical cardioversion
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

Final version 141/1185

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of atrial fibrillation and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (AVK), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication,
- Anticoagulation with anti-vitamin K for at least 3 weeks before ECV,
- ECV in patients with stabilized INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

Final version 142/1185

- Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent atrial fibrillation and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35  $\pm$  2D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit

Final version 143/1185

- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent atrial fibrillation and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent atrial fibrillation with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters,
   morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- early persistent atrial fibrillation history (less than one year) with a duration of a the current episode between 7 days to 6 months
- a moderately abnormal moderately systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- A Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or

Final version 144/1185
unstable ischemic coronaropathy (assessed by coronarography or cardiac stress test or effort test within 6 months before selection).

# 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on anti-arrhythmics on atrial fibrillation (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be developed as a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, anti-arhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent atrial fibrillation and requiring an electrical cardioversion will be included in order to assess the time to first documented recurrence of atrial fibrillation since cardioversion.

To confirm the persistent nature of atrial fibrillation, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before electrical cardioversion. According to guidelines for the management of atrial fibrillation [6], anti-vitamin K should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation, of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodary study [2], the duration of pre-treatment with PUFA before cardioversion appears to be a contributing factor in

Final version 145/1185

success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of atrial fibrillation recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of atrial fibrillation recurrence occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using a more easy to carry and easy to use device, a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

#### 4.2.3. Choice of the Dose

According to a previous study in patients with atrial fibrillation [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of atrial fibrillation after cardioversion. Moreover, PUFAs at dosage of 1g and 2g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95mg/mL and 60 to 90mg/mL, respectively) (phase I study of F373280 and Salm and coll study) [16]. With regard to the rythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a dose of 1 g daily of F373280 is considered to be appropriate to be tested in this POC study.

Final version 146/1185

# 4.2.4. Choice of the Sample Size

See chapter 13.

# 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive),
- 2. Patient with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:
  - use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
  - documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion

#### Ethical /legal considerations:

- 12. Having signed his/her written informed consent,
- 13. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation),

# 5.2. NON INCLUSION CRITERIA

# Criteria related to pathologies:

1. History of first documented episode of persistent AF more than 1 year,

Final version 147/1185

- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be check in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (K > 5.5 mEg/L or K < 3.5 mEg/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection.
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship.
- 25. Breastfeeding female patient.

#### 5.3. NUMBER OF PATIENTS

76 x 2 patients (taking into account 15 % of non evaluable patients).

Final version 148/1185

#### 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO,...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENTS IDENTIFICATION

The patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

#### 5.6. WITHDRAWAL CRITERIA

The reasons for a patient's premature withdrawal from the study may be the following:

- The patient's decision. A patient who wishes to withdraw from the study for any reason may do so at any time but must inform the investigator. In all cases, the Investigator should attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form
  - obtain the reason(s) for withdrawal and report it/them in the case report form
  - evaluate the patient's clinical condition
  - if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- The Investigator's decision in the patient's interest. Particularly, if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.

Final version 149/1185

- An erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion / non inclusion criteria will immediately be withdrawn and an appropriate treatment will be instored by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with anti-vitamin K for at least 3 weeks before ECV,
- Patients who will not stabilize INR between 2 and 3 on at least 3 consecutive weekly tests
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 week for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV (i.e. unsuccessful ECV) will be considered to have finished follow-up.
- An occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and uncomfortable clinical symptoms.

#### 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

# 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

# 5.9. STUDY CARD

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit, a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator

Final version 150/1185

and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83.

# 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

#### 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

# 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

Final version 151/1185

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

# 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number,
- c) packaging batch number,
- d) the treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
  - "for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose".

On the treatment unit, another label will be affixed with the mention of the investigator name and patient number (completed by the investigator).

In addition, on each case, will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

Final version 152/1185

#### 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person.

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

Final version 153/1185

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion Visit and another one at Visit 6.

For each patient, the treatment number given at Visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Calls the vocal server
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the vocal server.
- The IVRS/IWRS company:
  - Confirms this information by fax/email to the Investigator
  - Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 5, the Investigator will contact again the IVRS/IWRS to obtain for visit 6 the treatment number for the last 12-week period of treatment according to the same process as described above.

Final version 154/1185

#### 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure will be 24 weeks, with F373280 or placebo.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

#### 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

# 6.6. ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT

The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

Final version 155/1185

# 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator, in collaboration with the Sponsor representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF, according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (Selection Visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on e-CRF. All treatments should be evaluated by the investigator at selection and their prolongation during the study or their stop should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

Final version 156/1185

### 7.1. ANTI-VITAMIN K TREATMENT

Anti-vitamin K should be given for at least 3 weeks before ECV and continued for the whole study duration. The anti-vitamin K used will be left to the decision of the each investigator according to his/her local practice.

# 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
    - Class IA: Disopyramide, Procainamide, Quinidine
    - Class IB: Lidocaine, Mexiletine
    - Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Any Polyunsaturated Fatty Acid (PUFA)
- Any anticoagulant treatment other than antivitamin K: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

#### 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the case report form. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

Final version 157/1185

# 8. EVALUATION CRITERIA

#### **8.1. PRIMARY EFFICACY CRITERION:**

#### **8.1.1.** Time to the first Atrial Fibrillation Recurrence

# 8.1.1.1. Definition

Time to first Atrial Fibrillation recurrence is defined by the first episode of Atrial Fibrillation (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of electrical cardioversion visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

#### 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM)

• Trans Telephonic ECG Monitoring (TTEM):

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 to visit 6. Then, every two days from visit 6 to visit 9.

Moreover, during this TTEM period, if patient experiences AF symptoms, it should be documented using the TTEM.

Final version 158/1185

In case of AF recurrence, and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at the investigator's judgement, he/she could be maintained in the study with the treatment, in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

# 8.1.2. Secondary Efficacy Criteria

# 8.1.2.1. Numbers of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

# 8.1.2.1.1. *Definition*

Number of Atrial Fibrillation episodes will consist in the assessment of episodes of AF with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

#### 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the study visit 4.

#### 8.1.2.1.3. Evaluation Methods

#### • 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

Final version 159/1185

# 8.1.2.2. Duration of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

# 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episodes.

# 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the follow up study visit (visit 4).

#### 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

# 8.1.2.3. Clinical parameters evaluation

# 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition:

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

Final version 160/1185

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month); intermediate (1/month to almost daily); and frequent at least daily.

#### 8.1.2.3.1.2. Schedule

This evaluation will be performed in case of symptoms evocative of arrhythmia.

## 8.1.2.3.1.3. Evaluation Methods

This evaluation will be collected by Central Reading Laboratory during all the study period.

# 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of number of AF recurrence associated with a symptom (Palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG in atrial fibrillation.

# 8.1.2.3.3. Number and duration of hospitalization

- Number and duration of hospitalization for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
  - Hospitalization for myocardial infarction
  - All cause of hospitalization
- Number and duration of hospitalization for thromboembolic stroke

#### 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

Final version 161/1185

# 8.1.2.5. Evolution of echocardiographic parameters

## 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), Left atrial area (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m<sup>2</sup>, Left ventricular end diastolic diameter (mm) Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL),

#### 8.1.2.5.2. Schedule

The measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

The measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, for volume measurements, the recommended method is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.1. Definition

Because of the limited accessibility of human tissues for biopsy, red blood cell DHA contents is a marker for tissue DHA concentration [13], [14].

Final version 162/1185

# 8.2.2. Blood samples

#### 8.2.2.1. Collection schedule

Blood samples will be collected for determination of red blood cells (RBC) concentrations of DHA.

Blood samples will be performed as follows:

• Visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the electronic Case Report Forms (e-CRFs).

# 8.2.2.2. Technical handling

Two blood samples will be collected containing EDTA. They will be gently shaken and centrifuged at 3000g for 15 min at room temperature, within 30 minutes after collection. Plasma and white blood cells will be discarded. Red blood cells will be stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C) within 3 weeks following collection. Analysis will be performed within 2 weeks following reception at the Analytical centre.

#### **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol, after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will

Final version 163/1185

be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells

(expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk

for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end

of the study, and will be provided only at the end of the study (after database lock), in a separate

file.

8.3. SAFETY ASSESSMENT

**8.3.1.** Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the

occurrence of adverse events (AEs) since the last visit will be based on the patient's spontaneous

reporting, the investigator's non-leading questioning and his/her clinical evaluation. All AEs will

be reported on the e-CRF (see section 10).

8.3.2. Laboratory Investigations

8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of

treatment) or End of Treatment visit.

At visit 3 and 6, only an haematology examination will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The volume of blood samples complete haematology, biochemistry should not exceed 30 mL.

8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells

(WBC) count, WBC differential counts (% and absolute), reticulocytes,

platelets.

Final version 164/1185

Chemistry:

sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning, in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L],

in women:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patients' interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

# 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

Final version 165/1185

#### 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic (SBP) and diastolic (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation, after at least 5 minutes in supine position and after 2 minutes in standing position by counting the beats for at least 30 seconds.

Bodyweight will be measured in patient in underwear and with the same balance at each visit.

# 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An electrocardiogram will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

## 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram (ECG):

The global interpretation from manual reading (normality, clinical relevance) and heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

#### • 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent atrial fibrillation.

Final version 166/1185

# **8.3.6.** Coagulation parameters

The assessment of coagulation will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV,
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV,
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by anti-vitamin K should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial can be found in section 7.

#### 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back any remaining soft capsules, blister, case (used or unused) at the following visit.

At each visit, the Investigator will record the number of supplied and remaining Soft Capsules in the e-CRF.

Final version 167/1185

# 9. STUDY PROCEDURES

## Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If he/she accepts to participate in the study, he/she will sign the informed consent and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and Atrial Fibrillation characteristics
- Echocardiography using a two-dimensional echocardiography.
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

Final version 168/1185

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory (CRL). The CRL will send his/her assessment regarding the confirmation of persistent atrial fibrillation within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will contact the IVRS/IWRS system to confirm the patient selection and order the treatment delivery and organise the appointment for the next visit.

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

### Visit 2 - Inclusion Visit (Day 1)

If the patient's behaviour during the selection period and/or the result of complementary examinations particularly the confirmation of the presence of persistent atrial fibrillation by the CRL during this period, the INR and laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography.

Final version 169/1185

- 12-lead ECG
- Urine pregnancy test for women of child bearing potential.

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and allocated a treatment number using the IVRS/IWRS system.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.3.6), in order to ensure that the INR is stable, between 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

#### Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, Red Blood Cell concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (transesophageal echocardiograph) performed in the same day (before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be

Final version 170/1185

induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

#### Visit 4 (Week 5: D35 $\pm$ 2 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of Adverse Events
- Concomitant treatments (authorised, disallowed)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device (Trans Telephonic ECG Monitoring) for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

Final version 171/1185

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$ 

7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

Adverse events

• Concomitant treatments (authorised, disallowed)

• Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin

Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of

anticoagulation after ECV, the monitoring of INR, aPTT and TCT should be stopped.

Global Physical examination/bodyweight

• Vital signs

12-lead ECG

• The cardiac monitoring will be continued using a TTEM device (Trans Telephonic ECG

Monitoring). The device will be given to the patient who will be requested to performed daily

transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in

case of AF symptoms additional transmission may be performed.

The Investigator will collect all the cases, blisters and any unused soft capsules and count the

unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give

the treatment to be taken during the next 4-week treatment period.

In addition:

- at visit 5, the investigator will contact the IVRS/IWRS to obtain another treatment unit to be

dispensed at visit 6 for the last 12-week period.

- at visit 6, an echocardiography will be performed, an haematology examination will be done and

the red blood cell concentration of DHA will be measured.

End-of-Study Visit - Visit 9 (Week 24: D168  $\pm$  7 days)

Final version 172/1185

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused soft capsules.

# 10. ADVERSE EVENTS: DEFINITION AND REPORTING

## 10.1. ADVERSE EVENTS

### 10.1.1. Definition of Adverse Events

An adverse event is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

This includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values, which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as

Final version 173/1185

those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

# **10.1.2.** Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity.

# **10.1.3.** Reporting of Adverse Events

The records of adverse events in the electronic Case Report Form (e-CRF) describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A serious adverse event (SAE) includes, but is not necessarily restricted to any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect.

Final version 174/1185

Other events such as cancer, and any additional adverse experience or abnormal laboratory values

occurring during the study period, defined by the protocol as serious or which the Investigator

considers significant enough, or that suggest a significant hazard, contra-indications, side effect or

precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the

SAE notification form (see section 10.4).

\* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:

- planned (as per protocol) medical/surgical procedure,

- preparation for routine health assessment/procedure (e.g. routine colonoscopy),

- planned medical/surgical admission (planned prior to entry into study trial, appropriate

documentation required),

- administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver

respite, family circumstances)

will not be reported as a SAE.

10.2.2. Reporting of SAE

All serious adverse events, according to the above-mentioned definitions and regardless of

treatment or relationship to study drug, must be recorded by the Investigator as soon as he/she is

informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the

"Notification of serious adverse event" form ("first notification") (see appendix 17.2) with all the

available information about the event, to the Sponsor's representative:

Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE,

Centre de R&D Pierre Fabre – BP 13562

3 Avenue Hubert Curien

31035 TOULOUSE Cedex 1

Phone: +33 5 35 50 63 48

Fax: + 33 5 34 50 65 92

Email: marlene.guiraud@pierre-fabre.com

Final version 175/1185

In case of non-inclusion the reporting period ends when the non-inclusion is documented.

## 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

# 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage, and associated adverse event if any, are reported only on the Adverse Event page of the CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must be also transmitted to the sponsor.

#### 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and be withdrawn immediately from the study.

Final version 176/1185

If pregnancy is suspected while the patient is receiving study treatment, the study drug(s) should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is discontinued from the study.

The investigators must report to the sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The investigator must immediately notify the sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Women who become pregnant after exposure to the study drug must be followed by the investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

# 11.1.1. Case Report Form

An electronic Case Report Forms (e-CRF) will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files and which will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and include a traceability system for data corrections and deletions (audit trail).

Final version 177/1185

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants who will use this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation.

At the end of the study, a CD-ROM containing the pdf version of all e-CRF (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

Final version 178/1185

#### 11.2. STUDY MONITORING

# 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

## 11.2.1.2. Initiation Visit

Before the start of the study at all investigation sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
  - has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

Final version 179/1185

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

# 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes,
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

Final version 180/1185
#### 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of measures of primary end point, the safety data and to recommend to the Sponsor whether to continue, modify, or to stop the study.

The IDMC operating procedures will be described in an independent document.

# 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on a e-CRF.

The e-CRF used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

Final version 181/1185

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate coding.

#### 12.4. DATA STORAGE

The computer data files, as well as their modifications, will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e.: data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

# 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by Pierre Fabre Biométrie (PFB) or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan (SAP) approved by the Validation Committee.

Final version 182/1185

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 evaluable patients per group is required, using a log-rang test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

Final version 183/1185

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

#### 13.4. DATA SETS ANALYSED

The following 2 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

# **13.5.1.** Dropouts

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

# 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

#### 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

Final version 184/1185

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- Quantitative parameters will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

### 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

Final version 185/1185

# 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

# 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

### 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

### 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

#### 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

Final version 186/1185

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patients will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAE

Final version 187/1185

- With at least three TEAE
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.
- Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:
- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

"The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TE AE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (<u>for all patient</u>).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

Serious adverse events will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time

Final version 188/1185

of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

### 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

Final version 189/1185

Clinically noteworthy abnormal laboratory values (CNALV) (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and heart rate in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

Final version 190/1185

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

#### 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

#### 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" (ATC) classification on the safety set.

Final version 191/1185

#### 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated \_actual \_consumption}{Theoretical \_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) – number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days).

#### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

# 14. GENERAL ETHICAL CONSIDERATIONS

# 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

#### 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

Final version 192/1185

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study.

Final version 193/1185

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament, are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

#### 15. ADMINISTRATIVE PROCEDURES

#### 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Final version 194/1185

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

# 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF, drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not
- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents
- Authorises direct access to source documents for monitoring, audits and inspections
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

#### 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

Final version 195/1185

# 15.3.2. Early Study Termination

# 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if it considers that the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both his representatives (Study Manager, CRA, ...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

Final version 196/1185

#### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed to in writing with the Study Manager, the investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

#### 15.7. CLINICAL STUDY REPORT

Data analysis, and clinical study report writing are under the Sponsor's responsibility.

Upon completion of the data analysis, a final report, including a review of the objectives and methods, a presentation and discussion of the results are drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

#### 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

Final version 197/1185

To allow use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 198/1185

#### 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version January 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 199/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

[14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 200/1185

# [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

# [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

### [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

### [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

#### [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 201/1185

# 17. APPENDICES

Final version 202/1185

#### 17.1. DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 203/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 204/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 205/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 206/1185

# 17.2. SAE REPORT FORM

Final version 207/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE PRODUCT SAFETY DEPARTMENT |
|---|
| TO BE TRANSMITTED TO THE MONITOR BY FAX WITHIN 24H: M. GUIRAUDFax n° +33 5 34 50 65 92 |
| Transmission date |
| SAE N° FIRST NOTIFICATION FOLLOW-UP |
| > SUBJECT CHARACTERISTICS |
| Surname Birth date Birth date |
| Gender1=M, 2=F Heightcm Weight kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date |
| Seriousness onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| Date of first study treatment administration (ddmmyyyy) |
| Date of last study treatment administration before the occurence of SAE (ddmmyyyy) |
| • Was the blind broken? |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 208/1185

| INN or trade name | Daily dose | Start date (ddmmyy) | Ongoing at occurence of the event | Stop date (ddmmyy) | Route of admin. | Indication |
|---|---|---|---|---|---|---|
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAK | EN FOLLOWI | NG THE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage mod | lification, specify | / : | Modi | fication Date : | / | / |
| ☐ Temporarily | discontinued | | Readministr | ration date : | / | / |
| ☐ Withdrawn | | | | End date : | / | / |
| ☐ Not applicat | ole | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription | of corrective or | symptomatic treatme | ents (specify names and | d dosages): | | |
| ☐ Discontinua | tion of concomit | ant treatments (specif | fy names): | | | |
| | | | • | | | |
| ☐ Others, spec | 11y : | | | | | |
| > OUTCOME | | | | | | |
| ☐ Not recovered/ | | ☐ Recovering | - | Recovered/Resolve | ed | |
| ☐ Recovered/Res | solved with seque | elae 🗖 Fatal | <b>-</b> 1 | Unknown | | |
| T C 1 | ath, has an autop | sy been conducted? | ☐ Yes ☐ No | | | |
| In case of de | | | | | | |
| | CAUSALITY A | ASSESSMENT (inve | estigator's assessment | t to be done as soor | as possible) | |
| > INVESTIGATOR | | • | | t to be done as soon | as possible) | |
| In case of de ➤ INVESTIGATOR □ Not Suspected comments: | □ Sus | • | estigator's assessment Insufficient data | t to be done as soon | as possible) | |

Final version 209/1185

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| TO THE TOTAL | Protein | g/1 | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/l | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pH | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 210/1185

<sup>(¤)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

# **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| HAEMOGLOBIN | | <ul> <li>Decrease of at least 2g/dl and value &lt; 10 g/dl whatever the baseline value</li> <li>If missing baseline: value &lt;10g/dl</li> </ul> |
| NEUTROPHILS | | • < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing value for neutrophils) | | • < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM CREATININE | | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N: <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline:</li> <li>TB &gt; 1.5 N</li> <li>If abnormal baseline:</li> <li>TB &gt; 2 N</li> </ul> |

#### N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 211/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \leq 50$ mmHg and decrease $\geq 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>paseline Value | to the | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | Classes for the for each parame | Minimum Post-bo<br>ter | aseline Value | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤50 | ≤90 | ≤ 50 | ≤50 |
| [120;140[ | [80;90[ | ]50 ;75[ | [90 ;120[ | [50;80[ | ]50 ;75[ |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3BI 2 90 01 DBI 2 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq$ 20 mmHg or DBP Decrease $\geq$ 10 mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 212/1185

16.1.1.3. Protocol amendment n° PA01 Local (Italy) and substantial dated on 01 March 2013 linked to Protocol and appendices (version3: 01 March 2013)

Final version 213/1185

CLINICAL STUDY PROTOCOL AMENDMENT n° PA01 – Version 1 Local (Italy) - Substantial

Final version 214/1185

Pierre Fabre Médicament

Represented by: Institut de Recherche Pierre Fabre

45, Place Abel Gance F-92100 Boulogne

#### CLINICAL STUDY PROTOCOL AMENDMENT nº PA01 – Version 1

# **Local (Italy) - Substantial**

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

**Pierre Fabre Study Code:** F373280 CA 2 01

**EudraCT Number:** 2012-003487-48

**Sponsor's Representative:** Marlène GUIRAUD

**Coordinating Investigator:** Pr Savina NODARI

**Date of amendment PA01:** 1st March 2013

Final version 215/1185



Protocol: F373280 CA 2 01

#### Confidential

# Clinical Study Protocol Amendment n° PA01 – Version 1

# **Local (Italy) - Substantial SIGNATURE FORM**

| Sponsor's representative: | | |
|----------------------------------|------------|------------|
| · Head of Therapeutic Area | Date: | Signature: |
| Alain DELARUE, MD | 08-03-2013 | Ajohe |
| | | Ci. |
| Study Coordinating Investigator: | Date: | Signature: |
| Pr Savina NODARI | | |

Clinical study protocol amendment no PA 01 - Version 1 (Local/substantial)

Date: 01MAR13

# Clinical Study Protocol Amendment n° PA 01 – Version 1

Local (Italy) - Substantial

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

| Country Coordinating Investigator: | Date: | Signature: |
|------------------------------------|-------|------------|
| Pr Savina NODARI | | |

Final version 217/1185

# Clinical Study Protocol Amendment n° PA 01 – Version 1

Local (Italy) - Substantial

# INVESTIGATOR SIGNATURE FORM

| By my signature below, I, Dr | , hereby confirm that I have read, taken | l |
|---|---|---|
| note of (and will apply) the modifications brough | nt by the protocol amendment n° PA 01, dated $\_/\_/$ | |
| and I will conduct the trial according to these ne | ew modalities. | |
| Date: | Signature: | |

Final version 218/1185

# HISTORY OF PROTOCOL VERSIONS

| PROTOCOL VERSIONS | | MODIFICATIONS | COMMENTS |
|---|---|---|---|
| Version 1 | 09/11/2012 | Initial version | Version 1 submitted in<br>Italy (to Central Ethics<br>Committee) |
| Version 2 | 15/01/2013 | Following French CA request (ANSM): - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 | Version 2 not submitted<br>to CEC in Italy –<br>The version 3 will be<br>directly submitted |

Final version 219/1185

#### 1. AMENDMENT RATIONALE

This substantial local amendment follows the submission of the study protocol and Informed Consent Form (ICF) to the Central Ethics Committee (CEC) and Competent Authority (CA) in Italy.

According to the CEC and CA requirements and, in order to harmonise the protocol and the ICF, the following changes have been done to the study protocol:

- adjustment of the selection criteria n°10 related to the contraception method
- addition of a letter that is given by the patient to his/her general practitioner (GP)
- precision that the sponsor can not collect a copy of the Informed Consent Form
- precision that the patient card is in Italian language only (without any English mention)

In addition, the modification performed in the protocol version 2, on French Medicinal Agency have been included:

- Addition of a non-inclusion criteria related to breast-feeding female patient
- Addition of haematology dosage at visit 3 and 6

Final version 220/1185

# 2. CHANGES DESCRIPTION

| PREVIOUS<br>VERSION | MODIFIED VERSION |
|---------------------|------------------|

Final version 221/1185

# STUDY SYNOPSIS AND 5.1 INCLUSION CRITERIA

Demographic Characteristics and Other Baseline

*Characteristics:* 10. For female

10. For female patient of child-bearing potential:

use of an effective of method contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or

documented as

#### STUDY SYNOPSIS AND 5.1 INCLUSION CRITERIA

Demographic Characteristics and Other Baseline Characteristics:

10. For female patient of child-bearing potential:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- **use of double barrier contraception method** (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion

#### 12. For male with a childbearing potential partner:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- **use of double barrier contraception method** (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study.

Final version 222/1185

| 11. For female patient of child-bearing potential: negative urine pregnancy test at | surgical<br>ly<br>sterilize<br>d | |
|---|---|---|
| inclusion | patient of child-<br>bearing potential<br>negative uring<br>pregnancy test a | l-<br>l:<br>e |

Final version 223/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| STUDY SYNOPSIS AND 5.2 NON INCLUSION CRITERIA | STUDY SYNOPSIS AND 5.2 NON INCLUSION CRITERIA |
| Others criteria: | Others criteria: |
| 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion, 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection, 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints, 23. Patient family member or work associate (secretary, nurse, technician) of the Investigator, 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship, | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion, 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection, 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints, 23. Patient family member or work associate (secretary, nurse, technician) of the Investigator, 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship, 25. Breastfeeding female patient. |

Final version 224/1185

#### PREVIOUS VERSION

#### **MODIFIED VERSION**

#### 5.9 STUDY CARD

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit, a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83.

# 5.9 STUDY CARD AND LETTER FOR GENERAL PRACTITIONERS (GP)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. **This card will be in Italian without any English mention.**
- a letter to be given to his/her general practitioner. This letter intends to inform the GP (and any other doctors who take care of the patient) that the patient participate to this clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

Final version 225/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 8.3 SAFETY ASSESSMENT 8.3.2 Laboratory Investigations | 8.3 SAFETY ASSESSMENT 8.3.2 Laboratory Investigations |
| 8.3.2.1 Schedule | 8.3.2.1 Schedule |
| Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit. | Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit. |
| Furthermore the kaliemia will be checked before electrical cardioversion at visit 3. | At visit 3 and 6, only an haematology examination will be performed. |
| | Furthermore the kaliemia will be checked before electrical cardioversion at visit 3. |
| 8.3.2.2. Technical Procedures and Parameters | 8.3.2.2. Technical Procedures and Parameters |
| The following tests will be performed: | The following tests will be performed: |
| Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells (WBC) count, WBC differential counts (% and absolute), platelets. | Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells (WBC) count, WBC differential counts (% and absolute), reticulocytes, platelets. |

Final version 226/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 9. STUDY PROCEDURES | 9. STUDY PROCEDURES |
| Visit 3 (Week 4: D28 -2/+7 days) cardioversion | Visit 3 (Week 4: D28 -2/+7 days) cardioversion |
| Patient will be assessed for the following criteria: | Patient will be assessed for the following criteria: |
| Laboratory examination: Red Blood Cell concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT) | Red Blood Cell concentrations of DHA, |
| Visit 5 (Week 8: D56 ± 7 days) – Visit 6 (Week 12: D84 ± 7 days) - Visit 7 (Week 16: D112 ± 7 days) - Visit 8 (Week 20: D140 ± 7 days) | Visit 5 (Week 8: D56 ± 7 days) – Visit 6 (Week 12: D84 ± 7 days) - Visit 7 (Week 16: D112 ± 7 days) - Visit 8 (Week 20: D140 ± 7 days) |
| Patient will be assessed for the following criteria: | Patient will be assessed for the following criteria: |
| - at visit 6, an echocardiography will be performed and the red blood cell concentration of DHA will be measured. | - at visit 6, an echocardiography will be performed, an haematology examination will be done and the red blood cell concentration of DHA will be measured. |

Final version 227/1185

#### PREVIOUS VERSION

#### **MODIFIED VERSION**

#### 11.2. STUDY MONITORING

#### 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes,
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2. STUDY MONITORING

#### 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirement),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

Final version 228/1185

#### PREVIOUS VERSION

#### **MODIFIED VERSION**

#### 13.8 SAFETY ANALYSIS

#### 13.8.2 Clinical Laboratory Evaluation

For all blood laboratory parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

#### 13.8 SAFETY ANALYSIS

#### 13.8.2 Clinical Laboratory Evaluation

For all **biochemistry** parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

Final version 229/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 14.3 PATIENT'S INFORMATION<br>LEAFLET AND INFORMED<br>CONSENT FORM | 14.3 PATIENT'S INFORMATION<br>LEAFLET AND INFORMED<br>CONSENT FORM |
| The information and consent document are made in | The information and consent document are made in |
| triplicate: the original copy is kept by the | triplicate: the original copy is kept by the |
| Investigator, one copy is given to the patient and the | Investigator, one copy is given to the patient and the |
| last copy is kept by the Clinical Quality Assurance | last copy is kept by the Clinical Quality Assurance |
| Unit of the Sponsor in a sealed envelope at the end | Unit of the Sponsor in a sealed envelope at the end |
| of study. | of study (except in case of specific country |
| | requirement). |

Final version 230/1185

F 373280 CA 2 01

Final version 231/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

#### CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

**Sponsor's Representative:** Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 63 48 Fax:+33 5 34 50 65 92

E-mail:marlene.guiraud@pierre-fabre.com

Pr Savina NODARI Section of Cardiology

**Department of Experimental and Applied Sciences** 

**University of Brescia BRESCIA, ITALY** 

Phone: +39 030 3996 587 - Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>

#### Version 3-01 MAR 2013

**Study Coordinating Investigator** 

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 232/1185

#### **SPONSOR PERSONNEL**

#### PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

### **Clinical Study Manager (Monitor)**

Marlène GUIRAUD, Pharm D Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1

#### **Head of Therapeutic Area**

Alain DELARUE, MD Institut de Recherche Pierre Fabre

Centre de R&D Pierre Fabre BP 13 562

3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1

#### **Clinical Development Physician**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3. Avenue Hubert Curien

31035 TOULOUSE Cedex 1

Phone: +33 5 34 50 63 48 Fax: +33 5 34 50 65 92

E-mail: marlene.guiraud@pierre-

fabre.com

Fax: +33 5 34 50 65 92 E-mail: alain.delarue@pierre-

Phone: + 33 5 34 50 61 88

fabre.com

Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 65 92

E-mail: richard.roche@pierre-

fabre.com

Final version 233/1185

#### CONTRACT RESEARCH ORGANISATIONS

#### For Feasibility, Monitoring and Regulatory issues:

Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

#### For Centralised Randomisation and Electronic Case Report Form

#### **S-Clinica**

6, Chaussée de Boondael B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

# For Centralised Reading of Holder ECG and TTEM and equipment supply:

#### **Biomedical System**

1945 Chaussée de Wavre B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage

#### **Agrocampus Ouest**

Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

Final version 234/1185

# Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 3 – 01 MAR 2013

| Sponsor' | S | Re | presenta | tive: |
|----------|---|----|----------|-------|

<u>Head of Therapeutic Area:</u> Alain DELARUE, MD

Date:

Signature:

05-03-2013

**Study Coordinating Investigator:** 

Savina NODARI, MD

Date:

Signature:

#### Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

#### **Protocol Version 3 – 01 MAR 2013**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 236/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

**Protocol Version 3 – 01 MAR 2013** 

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 1<sup>st</sup> March 2013 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * To t | be adaj | pted | |
|--------|---------|------|---|
| | | | _ |

| Date: | Signature: |
|-------|------------|

Final version 237/1185

# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|-------------|----------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 24 |
| 1.2.1. | Chemical and pharmaceutical characteristics | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1. | 5 | |
| 1.2.2. | | |
| 1.2.2. | $\mathcal{E}$ 1 | |
| 1.2.2. | | |
| 1.2.2. | OF I | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 33 |
| 2.1. | PRIMARY OBJECTIVE | 33 |
| 2.2. | SECONDARY OBJECTIVES | 33 |
| <b>3.</b> ] | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 35 |
| 4.1. | OVERALL DESCRIPTION | 35 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 36 |
| 4.2.1. | Choice of the Study Population | 36 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 39 |
| <b>5.</b> | STUDY POPULATION | 39 |
| 5.1. | INCLUSION CRITERIA | 39 |
| 5.2. | NON INCLUSION CRITERIA | 40 |
| 5.3. | NUMBER OF PATIENTS | 41 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENTS IDENTIFICATION | 41 |
| 5.6. | WITHDRAWAL CRITERIA | 41 |
| 5.7. | REPLACEMENT OF PATIENTS | 42 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 43 |
| 5.9. | STUDY CARD | 43 |

| 6. S | TUDY TREATMENT | 43 |
|---|---|---|
| 5.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 43 |
| 5.2. | PACKAGING AND LABELLING | |
| 5.2.1. | Packaging | |
| 5.2.2. | Labelling | |
| 5.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 5.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 5.5. | DRUG ADMINISTRATION | |
| 5.5.1. | Duration of Treatment | |
| 5.5.2. | Dose Schedule | |
| 5.5.3. | Route and Conditions of Administration. | 47 |
| 5.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 47 |
| 5.7. | RECALL OF INVESTIGATIONAL PRODUCTS | 48 |
| 7. ( | CONCOMITANT TREATMENTS | 48 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | 49 |
| 7.3. | AUTHORISED TREATMENTS | 49 |
| 8. E | EVALUATION CRITERIA | 50 |
| 8.1. | PRIMARY EFFICACY CRITERION: | 50 |
| 3.1.1. | Time to the first Atrial Fibrillation Recurrence | 50 |
| 8.1.1.1 | | |
| 8.1.1.2 | | |
| 8.1.1.3<br>8.1.2. | Evaluation Methods Secondary Efficacy Criteria | |
| 3.1.2.<br>3.1.2.1 | · | 31 |
| J.1. <b>2</b> .1 | visit) | 51 |
| 8.1.2.2 | · · | |
| | visit) | |
| 3.1.2.3 | 1 | |
| 8.1.2.4<br>8.1.2.5 | | |
| 3.1.2. <i>3</i><br>3.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF | 94 |
| 5.2. | DHA | 54 |
| 3.2.1. | Definition | |
| 3.2.2. | Blood samples | |
| 8.2.2.1 | . Collection schedule | |
| 8.2.2.2 | $\mathcal{C}$ | |
| 3.2.3. | DHA concentration measurement | |
| 3.3. | SAFETY ASSESSMENT | 56 |

| 8.3.1. Adverse Events | 56 |
|----------------------------------------------------------------|----|
| 8.3.2. Laboratory Investigations | 56 |
| 8.3.2.1. Schedule | |
| 8.3.2.2. Technical Procedures and Parameters | 56 |
| 8.3.3. Global Physical Examination | 57 |
| 8.3.4. Vital Signs | |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.4. COMPLIANCE | |
| 9. STUDY PROCEDURES | 60 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 65 |
| 10.1. ADVERSE EVENTS | 65 |
| 10.1.1. Definition of Adverse Events | 65 |
| 10.1.2. Grading of Adverse Events | |
| 10.1.3. Reporting of Adverse Events | 66 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 66 |
| 10.2.1. Definition | 66 |
| 10.2.2. Reporting of SAE | 67 |
| 10.2.3. Follow-up of SAE | |
| 10.2.4. SAE Occurring After the Study | |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 68 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 68 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | 69 |
| 11. DATA COLLECTION AND STUDY MONITORING | 69 |
| 11.1. DATA COLLECTION | 69 |
| 11.1.1. Case Report Form | 69 |
| 11.1.2. Source Documents | 70 |
| 11.2. STUDY MONITORING | 71 |
| 11.2.1. Monitoring visits | |
| 11.2.1.1. Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | 73 |
| 12. DATA MANAGEMENT | 73 |

| 12.1. DATA ENTRY | 73 |
|---|---|
| 12.2. DATA CLEANING | 73 |
| 12.3. DATA CODING | 74 |
| 12.4. DATA STORAGE | 74 |
| 12.5. DATABASE LOCK | 74 |
| 13. STATISTICAL ANALYSIS | 74 |
| 13.1. GENERAL CONSIDERATIONS | 75 |
| 13.2. SAMPLE SIZE | 75 |
| 13.4. DATA SETS ANALYSED | 76 |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | 76 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 77 |
| 13.7. EFFICACY ANALYSIS | 77 |
| 13.7.1. Primary Criterion | 77 |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | 77 |
| 13.7.2. Secondary Criteria | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | |
| 14. GENERAL ETHICAL CONSIDERATIONS | |
| 14.1. ETHICAL CONDITIONS | |
| 14.2 ETHICS COMMITTEE AND LEGAL REQUIREMENTS | |

| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 85 |
|---|---|
| 14.4. PERSONAL DATA PROTECTION | 86 |
| 14.5. INSURANCE POLICY | 86 |
| 15. ADMINISTRATIVE PROCEDURES | 86 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 87 |
| 15.3. END OF THE STUDY | 87 |
| 15.3.1. Definition of the End of Study | |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | 88 |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | |
| 15.4. AUDIT | 88 |
| 15.5. INSPECTION | |
| 15.6. CONFIDENTIALITY | |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 89 |
| 15.9. STUDY RESULTS PUBLICATION | 89 |
| 16. REFERENCES | 91 |
| 17. APPENDICES | 94 |
| 17.1. DECLARATION OF HELSINKI | 95 |
| 17.2. SAE REPORT FORM | 99 |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 102 |

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| <b>Study Centres:</b> | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of Atrial Fibrillation (AF) induced by burst pacing.[1] Moreover, the effectiveness of PUFA (PolyUnsaturated Fatty Acid) has been proven in the following conditions: — prevention of Atrial Fibrillation recurrence in patients with persistent Atrial Fibrillation, in co-administration with amiodarone (add on therapy) [2] — Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – April 2014 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 (anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> </ul> |
| Study Schedule | <ul> <li>Treatment duration: 24 weeks</li> <li>9 visits will be scheduled:</li> <li>V1/ W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/ D1: Inclusion visit (start of treatment)</li> <li>V3/ W4 (D28 -2/+7 days): cardioversion visit (Outpatient or hospitalization according to</li> </ul> |

Final version 243/1185

| | clinical practice of the centre) (installation of the Holter device) - V4/ W5 (D35± 2 days): follow-up visit (removing of the Holter device and installation of the TTEM) |
|---|---|
| | - V5/ W8 (D56± 7 days): follow-up visit<br>- V6/ W12 (D84 ± 7 days): follow-up visit<br>- V7/ W16 (D112 ± 7 days): follow-up visit<br>- V8/ W20 (D140 ± 7 days): follow-up visit<br>- V9/ W24 (D168 ± 7 days): final study visit |
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | <ol> <li>Demographic Characteristics and Other Baseline Characteristics:</li> <li>Men or women aged more than 18 years (inclusive),</li> <li>Patients with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.</li> <li>History of first documented persistent AF less than 1 year</li> <li>History of ischemic or non ischemic heart failure</li> <li>NYHA class I or II chronic heart failure at selection and at inclusion</li> <li>Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) ) at selection and at inclusion</li> <li>On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers</li> <li>Left atrial area ≤ 40 cm² ) at selection and at inclusion</li> <li>Patients treated or having to be treated by anti-vitamin K</li> </ol> |
| | <ul> <li>in all the countries except Italy: <ul> <li>use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment</li> <li>documented as surgically sterilized</li> </ul> </li> <li>in Italy only: <ul> <li>absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or</li> <li>use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of</li> </ul> </li> </ul> |

- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study.

#### Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

. History of first documented episode of persistent AF more than 1 year

Final version 244/1185

| | More than two successful cardioversions (electrical or pharmacological) in the last 6 months |
|---|---|
| | Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV) |
| | 4. NYHA class III or IV heart failure at selection or at inclusion |
| | 5. Thyroid disease uncontrolled by treatment: TSH $\pm$ T4L $\pm$ T3L to be checked in case of |
| | treatment for thyroid disease |
| | 6. Myocardial infarction or unstable angina or presence of unstable ischemic |
| | coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice |
| | stress test, nuclear or MR perfusion evaluation methods) within 6 months before |
| | selection |
| | 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration |
| | rate < 30 mL/min) at selection |
| | 8. Bradycardia (HR ≤ 50 bpm) |
| | 9. Hyperkalemia or hypokalemia (K>5.5 mEq/L or K < 3.5 mEq/L) at selection |
| | 10. Cardiac surgery within 3 months before selection or planned during the study duration |
| | Criteria related to treatments: |
| | 11. Previously ineffective pharmacological or electrical cardioversion |
| | 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), |
| | except stable dose of digoxin, betablockers, calcium-blockers |
| | 13. Previous treatment with oral amiodarone within 12 months prior to inclusion |
| | 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion |
| | 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT |
| | implantation within the last 6 months |
| | 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months |
| | 17. Dietary supplement with ω3 or ω6 according to investigator's judgement |
| | 18. Having undergone any form of ablation therapy for AF |
| | 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor |
| | such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel |
| | of Frasugrei |
| | Other criteria: |
| | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the |
| | investigator's opinion |
| | 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a |
| | trial at the time of selection |
| | 22. Patient linguistically or mentally unable to understand the nature, objectives and |
| | possible consequences of the trial, or refusing to patient himself/herself to its constraints |
| | 23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator |
| | 24. Patient having forfeited his / her freedom by administrative or legal award or being |
| | under guardianship |
| | 25. Breastfeeding female patient |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly |
| | tests performed before ECV will be excluded from the study, unless the presence of atrial |
| | thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the some day (before ECV) |
| | in the same day (before ECV) ECV will be performed in patients without dyskalemia |
| | If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) |
| | could be postponed by 7 days. |
| Test Product: | F373280 |
| 1 cot 1 toutet. | Soft Capsules |
| Dose: | Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules |
| _ ~ ~ | Placebo will be administered in the same conditions as the tested product. |

Final version 245/1185

| Mode of Administration: | Oral, one capsule each evening with dinner |
|---|---|
| Evaluation Criteria: | Efficacy evaluation variables: |
| | <ul> <li>Primary evaluation variable:</li> <li>Time to first Atrial Fibrillation recurrence defined by the first episode of Atrial Fibrillation lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit) Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24.</li> <li>For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).</li> <li>Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM.</li> <li>All ECG traces will be evaluated by a Central Reading Laboratory.</li> </ul> |
| | Secondary evaluation variables: During the 7-day continuous ECG monitoring, Numbers of AF episodes Duration of AF episodes |
| | Clinical parameters: During the whole study: Number of recurrence of symptomatic AF episodes EHRA score Hospitalization for cardiovascular events Hospitalization for thromboembolic stroke All cause of hospitalization |
| | <ul> <li>Cardioversion: <ul> <li>Assessment of spontaneous cardioversion</li> <li>Assessment of successful cardioversion</li> <li>Number of patients needing an other cardioversion after the initial ECV</li> </ul> </li> </ul> |
| | <ul> <li>Other: <ul> <li>Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m², Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))</li> <li>Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).</li> </ul> </li> </ul> |
| | <ul> <li>Safety criteria:</li> <li>Adverse events (observed and / or spontaneously reported)</li> <li>Vital signs (Blood pressure (supine and standing), heart rate</li> <li>Physical examination (body weight),</li> <li>Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized).</li> <li>Haematology: haematocrit, haemoglobin, RBC, WBC, differential count, platelets</li> <li>Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)</li> <li>Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR (local laboratory), Prothrombine Time (PT)</li> </ul> |
| Statistical Methods: | Sample Size: Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. |

Final version 246/1185

#### **Primary Efficacy Analysis**

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### **Secondary Analyses**

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

#### Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment)

Final version 247/1185

# STUDY FLOW-CHART

Final version 248/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 +/-2 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | x | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic characteristics | х | | | | | | | | |
| Medico-surgical history | х | | | | | | | | |
| Concomitant disease | х | | | | | | | | |
| Concomitant treatment | х | х | х | х | х | х | х | x | x |
| Habits | х | | | | | | | | |
| Global physical examination (body weight) | х | х | х | | х | х | х | х | х |
| Echocardiography | х | x | | х | | х | | | x |
| Eligibility criteria check | х | x | | | | | | | |
| Blood pressure, heart rate | х | х | х | х | х | х | х | x | x |
| 12-Lead ECG Recording | х | x | х | | х | х | х | x | x |
| INR | <b>─</b> | | (2) | | х | х | х | x | х |
| аРТТ, ТСТ | х | х | х | | х | х | х | x | x |
| Biochemistry | х | | | | | | | | x |
| Hematology | х | | X | | | X | | | x |
| Urinary pregnancy test | | x | | | | | | | x |
| Red Blood Cell concentrations of DHA | | x | х | | | х | | | x |
| Treatment allocation | | x | | | | х | | | |
| IVRS | х | x | | | х | х | | | |
| ECV (3) | | | х | | | | | | |
| Drug administration | | 1 | | | | | | | <b>—</b> |
| Adverse events recording | | х | х | х | х | х | х | x | x |
| Holter ECG | (4) | | <b>—</b> | (5) | | | | 4 | |
| TTEM (6) | | | | | | | | 4 | Ť |

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)

Final version 249/1185

<sup>(2)</sup> In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(5) 7-</sup>day Holter ECG

<sup>&</sup>quot;O'TTEM everyday from week 6 to week 8. Then every 2 days from week 9 to week 24. In case of AF symptoms. In case of AF recurrence for at least 10 minutes and the patient does not stop the study treatment then TTEM every 4 weeks

#### LIST OF ABBREVIATIONS

aPTT Activated partial thromboplastin time

AE : Adverse event

AERP Atrial effective refractory period

AF : Atrial fibrillation
ALA Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK Anti vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP Blood pressure
BSA : Body Surface Area

CEP Protocol evaluation committee

CHF : Congestive heart failure

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO –TE Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA European heart rhythm association

EPA Eicosapentaenoic acid eCRF Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

Final version 250/1185

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL High density lipoprotein

HF Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS Interactive voice response system

LAA Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL Low density lipoprotein LOQ : Limit of quantification

LVEF Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR Mineralocorticoid receptor
MR perfusion Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie
POC Proof of concept

PUFA : PolyUnsaturated fatty acid

PK : Pharmacokinetics

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT Thrombin clotting time

TEAEs Treatment emergent adverse events
TTEM TransTelephonic ECG monitoring

VTP : Ventricular tachypacing

WBC White blood cells

WHO-DRUG: World health organization drug reference list

Final version 251/1185

#### 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of atrial fibrillation (AF) in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the PUFAs (Polyunsaturated Fatty Acids) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are ALA, EPA and DHA. First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or atrial fibrillation.

The potential anti-arrythmic effects of a PUFA was previously developed in atrial fibrillation: nicotinyl ester of DHA (pro-drug based on DHA delivery) were assessed in a two-week

Final version 252/1185
ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of atrial fibrillation (AF) induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll assessed n-3 Polyunsaturated Fatty Acids in the prevention of atrial fibrillation recurrences after electrical cardioversion. All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct electrical cardioversion (ECV) 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95%] confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent atrial fibrillation on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion [2]. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFA on top of traditional treatment (amiodarone, beta blockers, reninangiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than placebo group at one month (3.3% vs 10%; p=0.043), at 3 months (10% vs 25%; p=0.004) and at 6 months (13.3% vs 40%; p<0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effect of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Final version 253/1185

Nodari and coll [3] performed a trial in patients with a chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (P = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, P = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent atrial fibrillation and heart failure in the maintenance of sinus rhythm after electrical cardioversion.

#### 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA (docosahexaenoic acid) is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of atrial fibrillation.

F373280 is a prodrug of DHA.

Final version 254/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

# 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

# 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

Trimethylpentane: Slightly soluble

Final version 255/1185

#### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

# 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period (AERP) were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased AERP (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, P<0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the ECG intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing (VTP)-induced congestive heart failure (CHF) provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses CHF-induced AF-promotion and fibrosis in the VTP canine model. Nicotinyl ester of DHA was tested in this model, at 1g/day and 5g/day, during 4 weeks, to prevent CHF-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in atrial fibrillation duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus  $637 \pm 196$  sec, n=5 in the presence of 1g/kg/d Nicotinyl ester of DHA and  $79 \pm 51$  sec, n=5, in the presence of 5g/kg/d Nicotinyl ester of DHA The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280

Final version 256/1185

similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the

compound may exert a similar protective effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 gm/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 257/1185

6 consecutive single ascending doses were tested (0.5g, 1g, 2g, 4g, 8g and 16g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 4 were observed in the placebo group (palpitation, dizziness in standing position, 2 symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events were reported in the groups of F373280 at the dosages of 0.5g, 1g, 2g, 4g and 8g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5g to 16 g in 36 young male healthy subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirm that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding PK parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16g with no departure from proportionality (baseline corrected parameters).

Final version 258/1185

## Part B: Multiple dose

Three consecutive repeated ascending doses (1, 2 and 4g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280 5/9 TEAE were classified according the SOC in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAE have already been reported with Poly Unsaturated Fatty Acids and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 259/1185

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of atrial fibrillation (AF) induced by burst pacing [1].

Moreover, the effectiveness of PUFA has been proven in the following conditions:

- Prevention of atrial fibrillation recurrence in patients with persistent atrial fibrillation in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor®, [9]:

Final version 260/1185

- The frequencies of adverse reactions are ranked according to the following: common (> 1/100, < 1/10); uncommon (>1/1000 < 1/100); rare (>1/10000, < 1/1000); very rare ( < 1/10000), not known (cannot be estimated from the available data).
  - The reported adverse events are:
- Infection and infestations

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

General disorders and administration site conditions:

Rare: malaise sensation

Final version 261/1185

## • Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1g and 4g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in Atrial Fibrillation studies [2, 8]. The range of PUFAs doses tested was between 2g to 3g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in heart failure patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1g to 5g (1g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Final version 262/1185

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct electrical cardioversion
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

Final version 263/1185

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of atrial fibrillation and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (AVK), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication,
- Anticoagulation with anti-vitamin K for at least 3 weeks before ECV,
- ECV in patients with stabilized INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

Final version 264/1185

- Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent atrial fibrillation and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35  $\pm$  2D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit

Final version 265/1185

- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent atrial fibrillation and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent atrial fibrillation with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters,
  morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- early persistent atrial fibrillation history (less than one year) with a duration of a the current episode between 7 days to 6 months
- a moderately abnormal moderately systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- A Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or

Final version 266/1185

unstable ischemic coronaropathy (assessed by coronarography or cardiac stress test or effort test within 6 months before selection).

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on anti-arrhythmics on atrial fibrillation (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be developed as a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, anti-arhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent atrial fibrillation and requiring an electrical cardioversion will be included in order to assess the time to first documented recurrence of atrial fibrillation since cardioversion.

To confirm the persistent nature of atrial fibrillation, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before electrical cardioversion. According to guidelines for the management of atrial fibrillation [6], anti-vitamin K should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation, of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodary study [2], the duration of pre-treatment with PUFA before cardioversion appears to be a contributing factor in

Final version 267/1185

success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of atrial fibrillation recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of atrial fibrillation recurrence occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using a more easy to carry and easy to use device, a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

#### 4.2.3. Choice of the Dose

According to a previous study in patients with atrial fibrillation [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of atrial fibrillation after cardioversion. Moreover, PUFAs at dosage of 1g and 2g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95mg/mL and 60 to 90mg/mL, respectively) (phase I study of F373280 and Salm and coll study) [16]. With regard to the rythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a dose of 1 g daily of F373280 is considered to be appropriate to be tested in this POC study.

Final version 268/1185

# 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive),
- 2. Patient with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

## • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- documented as surgically sterilized

## • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or

Final version 269/1185

- use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study.

## Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation),

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 1 year,
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be check in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (K > 5.5 mEq/L or K < 3.5 mEq/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,

Final version 270/1185

- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship,
- 25. Breastfeeding female patient.

#### **5.3. NUMBER OF PATIENTS**

76 x 2 patients (taking into account 15 % of non evaluable patients).

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO,...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENTS IDENTIFICATION

The patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

The reasons for a patient's premature withdrawal from the study may be the following:

- The patient's decision. A patient who wishes to withdraw from the study for any reason may do so at any time but must inform the investigator. In all cases, the Investigator should attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form

Final version 271/1185

- obtain the reason(s) for withdrawal and report it/them in the case report form
- evaluate the patient's clinical condition
- if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- The Investigator's decision in the patient's interest. Particularly, if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.
- An erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion / non inclusion criteria will immediately be withdrawn and an appropriate treatment will be instored by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with anti-vitamin K for at least 3 weeks before ECV,
- Patients who will not stabilize INR between 2 and 3 on at least 3 consecutive weekly tests
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 week for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV (i.e. unsuccessful ECV) will be considered to have finished follow-up.
- An occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and uncomfortable clinical symptoms.

#### 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

Final version 272/1185

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.
- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

Final version 273/1185

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

#### 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number,
- c) packaging batch number,
- d) the treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units

Final version 274/1185

- i) direction for use
- k) legal statements:
  - "for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose".

On the treatment unit, another label will be affixed with the mention of the investigator name and patient number (completed by the investigator).

In addition, on each case, will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

## 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person.

Final version 275/1185

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

## 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion Visit and another one at Visit 6.

For each patient, the treatment number given at Visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Calls the vocal server
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the vocal server.
- The IVRS/IWRS company:
  - Confirms this information by fax/email to the Investigator

Final version 276/1185

- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 5, the Investigator will contact again the IVRS/IWRS to obtain for visit 6 the treatment number for the last 12-week period of treatment according to the same process as described above.

#### 6.5. DRUG ADMINISTRATION

## **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure will be 24 weeks, with F373280 or placebo.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made

Final version 277/1185

available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

## 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator, in collaboration with the Sponsor representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF, according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (Selection Visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on e-CRF. All treatments should be evaluated by the investigator at selection and their prolongation during the study or their stop should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

Final version 278/1185

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

## 7.1. ANTI-VITAMIN K TREATMENT

Anti-vitamin K should be given for at least 3 weeks before ECV and continued for the whole study duration. The anti-vitamin K used will be left to the decision of the each investigator according to his/her local practice.

## 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
    - Class IA: Disopyramide, Procainamide, Quinidine
    - Class IB: Lidocaine, Mexiletine
    - Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Any Polyunsaturated Fatty Acid (PUFA)
- Any anticoagulant treatment other than antivitamin K: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

Final version 279/1185

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the case report form. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

## 8. EVALUATION CRITERIA

## **8.1. PRIMARY EFFICACY CRITERION:**

## **8.1.1.** Time to the first Atrial Fibrillation Recurrence

# 8.1.1.1. Definition

Time to first Atrial Fibrillation recurrence is defined by the first episode of Atrial Fibrillation (symptomatic or not) lasting for at least 10 minutes.

## 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of electrical cardioversion visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM)

• Trans Telephonic ECG Monitoring (TTEM):

Final version 280/1185

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 to visit 6. Then, every two days from visit 6 to visit 9.

Moreover, during this TTEM period, if patient experiences AF symptoms, it should be documented using the TTEM.

In case of AF recurrence, and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at the investigator's judgement, he/she could be maintained in the study with the treatment, in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

## 8.1.2. Secondary Efficacy Criteria

# 8.1.2.1. Numbers of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

## 8.1.2.1.1. *Definition*

Number of Atrial Fibrillation episodes will consist in the assessment of episodes of AF with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

## 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the study visit 4.

#### 8.1.2.1.3. Evaluation Methods

• 7-day holter monitor:

Final version 281/1185

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

# 8.1.2.2. Duration of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

## 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episodes.

#### 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the follow up study visit (visit 4).

#### 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

# 8.1.2.3. Clinical parameters evaluation

## 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition:

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

Final version 282/1185

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month); intermediate (1/month to almost daily); and frequent at least daily.

#### 8.1.2.3.1.2. Schedule

This evaluation will be performed in case of symptoms evocative of arrhythmia.

#### 8.1.2.3.1.3. Evaluation Methods

This evaluation will be collected by Central Reading Laboratory during all the study period.

## 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of number of AF recurrence associated with a symptom (Palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG in atrial fibrillation.

## 8.1.2.3.3. Number and duration of hospitalization

- Number and duration of hospitalization for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
  - Hospitalization for myocardial infarction
  - All cause of hospitalization
- Number and duration of hospitalization for thromboembolic stroke

#### 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

Final version 283/1185

## 8.1.2.5. Evolution of echocardiographic parameters

## 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), Left atrial area (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m<sup>2</sup>, Left ventricular end diastolic diameter (mm) Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL),

## 8.1.2.5.2. Schedule

The measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

The measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

## 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, for volume measurements, the recommended method is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

## 8.2.1. Definition

Because of the limited accessibility of human tissues for biopsy, red blood cell DHA contents is a marker for tissue DHA concentration [13], [14].

Final version 284/1185

## 8.2.2. Blood samples

## 8.2.2.1. Collection schedule

Blood samples will be collected for determination of red blood cells (RBC) concentrations of DHA.

Blood samples will be performed as follows:

• Visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the electronic Case Report Forms (e-CRFs).

## 8.2.2.2. Technical handling

Two blood samples will be collected containing EDTA. They will be gently shaken and centrifuged at 3000g for 15 min at room temperature, within 30 minutes after collection. Plasma and white blood cells will be discarded. Red blood cells will be stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C) within 3 weeks following collection. Analysis will be performed within 2 weeks following reception at the Analytical centre.

#### **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol, after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will

Final version 285/1185

be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells

(expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk

for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end

of the study, and will be provided only at the end of the study (after database lock), in a separate

file.

8.3. SAFETY ASSESSMENT

**8.3.1.** Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the

occurrence of adverse events (AEs) since the last visit will be based on the patient's spontaneous

reporting, the investigator's non-leading questioning and his/her clinical evaluation. All AEs will

be reported on the e-CRF (see section 10).

8.3.2. Laboratory Investigations

8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of

treatment) or End of Treatment visit.

At visit 3 and 6, only an haematology examination will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The volume of blood samples complete haematology, biochemistry should not exceed 30 mL.

8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells

(WBC) count, WBC differential counts (% and absolute), reticulocytes,

platelets.

Final version 286/1185

Chemistry:

sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning, in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L],

in women:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patients' interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

Final version 287/1185

#### 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic (SBP) and diastolic (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation, after at least 5 minutes in supine position and after 2 minutes in standing position by counting the beats for at least 30 seconds.

Bodyweight will be measured in patient in underwear and with the same balance at each visit.

# 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An electrocardiogram will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

## 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram (ECG):

The global interpretation from manual reading (normality, clinical relevance) and heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

#### • 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent atrial fibrillation.

Final version 288/1185
# **8.3.6.** Coagulation parameters

The assessment of coagulation will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV,
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV,
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by anti-vitamin K should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

## **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial can be found in section 7.

## 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back any remaining soft capsules, blister, case (used or unused) at the following visit.

At each visit, the Investigator will record the number of supplied and remaining Soft Capsules in the e-CRF.

Final version 289/1185

# 9. STUDY PROCEDURES

# Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If he/she accepts to participate in the study, he/she will sign the informed consent and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and Atrial Fibrillation characteristics
- Echocardiography using a two-dimensional echocardiography.
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

Final version 290/1185

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory (CRL). The CRL will send his/her assessment regarding the confirmation of persistent atrial fibrillation within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will contact the IVRS/IWRS system to confirm the patient selection and order the treatment delivery and organise the appointment for the next visit.

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

# **Visit 2 - Inclusion Visit (Day 1)**

If the patient's behaviour during the selection period and/or the result of complementary examinations particularly the confirmation of the presence of persistent atrial fibrillation by the CRL during this period, the INR and laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography.

Final version 291/1185

- 12-lead ECG
- Urine pregnancy test for women of child bearing potential.

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and allocated a treatment number using the IVRS/IWRS system.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.3.6), in order to ensure that the INR is stable, between 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

## Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, Red Blood Cell concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (transesophageal echocardiograph) performed in the same day (before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be

Final version 292/1185

induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

## Visit 4 (Week 5: D35 $\pm$ 2 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of Adverse Events
- Concomitant treatments (authorised, disallowed)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device (Trans Telephonic ECG Monitoring) for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

Final version 293/1185

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$ 

7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

Adverse events

• Concomitant treatments (authorised, disallowed)

Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin

Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of

anticoagulation after ECV, the monitoring of INR, aPTT and TCT should be stopped.

Global Physical examination/bodyweight

Vital signs

• 12-lead ECG

• The cardiac monitoring will be continued using a TTEM device (Trans Telephonic ECG

Monitoring). The device will be given to the patient who will be requested to performed daily

transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in

case of AF symptoms additional transmission may be performed.

The Investigator will collect all the cases, blisters and any unused soft capsules and count the

unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give

the treatment to be taken during the next 4-week treatment period.

In addition:

- at visit 5, the investigator will contact the IVRS/IWRS to obtain another treatment unit to be

dispensed at visit 6 for the last 12-week period.

- at visit 6, an echocardiography will be performed, an haematology examination will be done and

the red blood cell concentration of DHA will be measured.

End-of-Study Visit - Visit 9 (Week 24: D168  $\pm$  7 days)

Final version 294/1185

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused soft capsules.

# 10. ADVERSE EVENTS: DEFINITION AND REPORTING

## 10.1. ADVERSE EVENTS

## 10.1.1. Definition of Adverse Events

An adverse event is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

This includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values, which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as

Final version 295/1185

those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

# **10.1.2.** Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity.

# 10.1.3. Reporting of Adverse Events

The records of adverse events in the electronic Case Report Form (e-CRF) describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

## 10.2.1. Definition

A serious adverse event (SAE) includes, but is not necessarily restricted to any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect.

Final version 296/1185

Other events such as cancer, and any additional adverse experience or abnormal laboratory values

occurring during the study period, defined by the protocol as serious or which the Investigator

considers significant enough, or that suggest a significant hazard, contra-indications, side effect or

precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the

SAE notification form (see section 10.4).

\* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:

- planned (as per protocol) medical/surgical procedure,

- preparation for routine health assessment/procedure (e.g. routine colonoscopy),

- planned medical/surgical admission (planned prior to entry into study trial, appropriate

documentation required),

- administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver

respite, family circumstances)

will not be reported as a SAE.

10.2.2. Reporting of SAE

All serious adverse events, according to the above-mentioned definitions and regardless of

treatment or relationship to study drug, must be recorded by the Investigator as soon as he/she is

informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the

"Notification of serious adverse event" form ("first notification") (see appendix 17.2) with all the

available information about the event, to the Sponsor's representative:

Marlène GUIRAUD, Pharm D

INSTITUT DE RECHERCHE PIERRE FABRE,

Centre de R&D Pierre Fabre – BP 13562

3 Avenue Hubert Curien

31035 TOULOUSE Cedex 1

Phone: +33 5 35 50 63 48

Fax: + 33 5 34 50 65 92

Email: marlene.guiraud@pierre-fabre.com

Final version 297/1185

In case of non-inclusion the reporting period ends when the non-inclusion is documented.

## 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

# 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

## 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage, and associated adverse event if any, are reported only on the Adverse Event page of the CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must be also transmitted to the sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and be withdrawn immediately from the study.

Final version 298/1185

If pregnancy is suspected while the patient is receiving study treatment, the study drug(s) should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is discontinued from the study.

The investigators must report to the sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The investigator must immediately notify the sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Women who become pregnant after exposure to the study drug must be followed by the investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

## 11.1. DATA COLLECTION

# 11.1.1. Case Report Form

An electronic Case Report Forms (e-CRF) will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files and which will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and include a traceability system for data corrections and deletions (audit trail).

Final version 299/1185

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants who will use this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation.

At the end of the study, a CD-ROM containing the pdf version of all e-CRF (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

Final version 300/1185

## 11.2. STUDY MONITORING

# 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

## 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

# 11.2.1.2. Initiation Visit

Before the start of the study at all investigation sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
  - has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

Final version 301/1185

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

# 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

## 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

Final version 302/1185

## 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of measures of primary end point, the safety data and to recommend to the Sponsor whether to continue, modify, or to stop the study.

The IDMC operating procedures will be described in an independent document.

# 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

## 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on a e-CRF.

The e-CRF used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

## 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

Final version 303/1185

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

## 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate coding.

## 12.4. DATA STORAGE

The computer data files, as well as their modifications, will be archived by the subcontractor and kept available upon request of the Sponsor.

## 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e.: data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

# 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by Pierre Fabre Biométrie (PFB) or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan (SAP) approved by the Validation Committee.

Final version 304/1185

## 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

## 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 evaluable patients per group is required, using a log-rang test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

## 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

Final version 305/1185

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

## 13.4. DATA SETS ANALYSED

The following 2 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses.

## 13.5. HANDLING OF DROPOUTS AND MISSING DATA

# **13.5.1.** Dropouts

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

# 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

## 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

Final version 306/1185

## 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- Quantitative parameters will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

## 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

## 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

Final version 307/1185

# 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

# 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

# 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

# 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

## 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

Final version 308/1185

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

## 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

## 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patients will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAE

Final version 309/1185

- With at least three TEAE
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.
- Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:
- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

"The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TE AE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (<u>for all patient</u>).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

Serious adverse events will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time

Final version 310/1185

of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

## 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

Final version 311/1185

Clinically noteworthy abnormal laboratory values (CNALV) (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and heart rate in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

Final version 312/1185

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

## 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

## 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

## 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" (ATC) classification on the safety set.

Final version 313/1185

## 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) – number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days).

## 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

## 14. GENERAL ETHICAL CONSIDERATIONS

# 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

## 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

Final version 314/1185

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Final version 315/1185

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

## 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

## 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament, are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

## 15. ADMINISTRATIVE PROCEDURES

## 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Final version 316/1185

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

# 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF, drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not
- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents
- Authorises direct access to source documents for monitoring, audits and inspections
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

## 15.3. END OF THE STUDY

## 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

Final version 317/1185

# 15.3.2. Early Study Termination

# 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if it considers that the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

## **15.4. AUDIT**

The Sponsor is responsible for making sure that both his representatives (Study Manager, CRA, ...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

Final version 318/1185

## 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

## 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed to in writing with the Study Manager, the investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

## 15.7. CLINICAL STUDY REPORT

Data analysis, and clinical study report writing are under the Sponsor's responsibility.

Upon completion of the data analysis, a final report, including a review of the objectives and methods, a presentation and discussion of the results are drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

## 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

Final version 319/1185

To allow use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 320/1185

## 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version January 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 321/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

[14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 322/1185

# [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

# [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

## [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

## [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

## [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 323/1185

# 17. APPENDICES

Final version 324/1185
#### 17.1. DECLARATION OF HELSINKI

## WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 325/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 326/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 327/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 328/1185

## 17.2. SAE REPORT FORM

Final version 329/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE PRODUCT SAFETY DEPARTMENT |
|---|
| TO BE TRANSMITTED TO THE MONITOR BY FAX WITHIN 24H: M. GUIRAUDFax n° +33 5 34 50 65 92 |
| Transmission date |
| SAE N° FIRST NOTIFICATION FOLLOW-UP |
| > SUBJECT CHARACTERISTICS |
| Surname Birth date Birth date |
| Gender1=M, 2=F Heightcm Weight kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date |
| Seriousness onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| Date of first study treatment administration (ddmmyyyy) |
| Date of last study treatment administration before the occurence of SAE (ddmmyyyy) |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 330/1185

| Transmission date | | | (ddmmyyyy) | Country: | ••••• | |
|---|---|---|---|---|---|---|
| SAE N° | | FIRST NOTIFICATION FOLLOW-UP | | | | |
| > CONCOMITANT MEDICATION SINCE TRIAL INITIATION and UP UNTIL THE OCCURRENCE OF THE SAE (EXCEPT THE TREATMENTS GIVEN FOR THE SAE) | | | | | | |
| INN or trade name | Daily dose | Start date (ddmmyy) | Ongoing at occurence of the event | Stop date (ddmmyy) | Route of admin. | Indication |
| | | // | | // | | |
| | | / | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAK | EN FOLLOWIN | NG THE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage mod | ification, specify | | Modi | fication Date : | / | / |
| ☐ Temporarily | discontinued | | Readministr | ration date: | / | / |
| ☐ Withdrawn | | | | End date: | / | / |
| ☐ Not applicab | ole | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription | of corrective or s | symptomatic treatment | s (specify names and | d dosages): | | |
| ☐ Discontinuat | tion of concomita | ant treatments (specify | names): | | | |
| ☐ Others, spec | ify · | | | | | |
| <b>a</b> others, spec | | | | | | |
| > OUTCOME | | | | | | |
| □ Not recovered/ | | ☐ Recovering/I | • | Recovered/Resolve | ed | |
| ☐ Recovered/Resolved with sequelae ☐ Fatal ☐ Unknown | | | | | | |
| In case of de | ath, has an autop | sy been conducted? | ☐ Yes ☐ No | | | |
| > INVESTIGATOR | CAUSALITY A | SSESSMENT (invest | tigator's assessment | t to be done as soor | ı as possible) | |
| □ Not Suspected □ Suspected □ Insufficient data | | | | | | |
| comments : | | | | | | |
| Enc | close in the notific | ation the results of carr | ied out examinations, | reports of hospitalisa | ation, etc | |

Final version 331/1185

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|----------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| 1,61141101,112 | Protein | g/1 | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pН | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/1 | | N x (30/95) |

N = upper limit of normal range

Final version 332/1185

<sup>(

)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

#### **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| HAEMOGLOBIN | | Decrease of at least 2g/dl and value < 10 g/dl whatever the baseline value If missing baseline : value <10g/dl |
| NEUTRO | PHILS | $\bullet$ < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N: <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline:</li> <li>TB &gt; 1.5 N</li> <li>If abnormal baseline:</li> <li>TB &gt; 2 N</li> </ul> |

#### N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 333/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg}$ and increase $\ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>baseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the for each parame | Minimum Post-bo<br>ter | aseline Value |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤ <i>50</i> | ≤90 | ≤ 50 | ≤50 |
| [120;140] | [80;90[ | <i>[50 ;75]</i> | [90 ;120] | [50;80[ | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3B1 ≥ 90 01 DB1 ≥ 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq 20$ mmHg or DBP Decrease $\geq 10$ mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 334/1185

16.1.1.4. Protocol amendment n° PA02 General and non-substantial dated on 28 March 2013 linked to Protocol and appendices (version 4: 28 March 2013)

Final version 335/1185

CLINICAL STUDY PROTOCOL AMENDMENT n° PA02 – Version 1 General – Non Substantial

Final version 336/1185

Pierre Fabre Médicament

Represented by : Institut de Recherche Pierre Fabre

45, Place Abel Gance F-92100 Boulogne

#### CLINICAL STUDY PROTOCOL AMENDMENT nº PA02 – Version 1

#### General - Non Substantial

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

**Pierre Fabre Study Code:** F373280 CA 2 01

**EudraCT Number:** 2012-003487-48

**Sponsor's Representative:** Gaëlle ALCARAZ

**Coordinating Investigator:** Pr Savina NODARI

**Date of amendment PA02:** 28 March 2013

Final version 337/1185



Protocol: F373280 CA 2 01


# Clinical Study Protocol Amendment n° PA02 - Version 1

# General – Non Substantial SIGNATURE FORM

| 67 | i | 4 42 |
|---------|---|-----------------|
| Sponsor | 8 | representative: |

Medical Director

Richard ROCHE, MD

Date: 14/05/13 Signature:

Study Coordinating Investigator:

Pr Savina NODARI

Date:

Signature:

Clinical study protocol amendment no PA 02 – Version 1 (General/Non Date: 28MAR13 substantial)


# Clinical Study Protocol Amendment n° PA 02 – Version 1

General – Non substantial

## COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

| <b>Country Coordinating Investigator:</b> | Date: | Signature: |
|-------------------------------------------|-------|------------|

Final version 339/1185

# Clinical Study Protocol Amendment n° PA 02 – Version 1

General – Non Substantial

## INVESTIGATOR SIGNATURE FORM

| By my signature below, I, Dr | , hereby confirm that I have read, taken |
|---|---|
| note of (and will apply) the modifications brough | ht by the protocol amendment n° PA 02, dated 28 MAR |
| 2013 and I will conduct the trial according to the | ese new modalities. |
| Date: | Signature: |

Final version 340/1185

## HISTORY OF PROTOCOL VERSIONS

| PROTOCOL VERSIONS | DATE | MODIFICATIONS | COMMENTS |
|---|---|---|---|
| Version 1 | 09/11/2012 | Initial version | General |
| Version 2<br>(General) | 15/01/2013 | Following French CA request (ANSM): - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 | General |
| Version 3<br>(Local Italy) | 01/03/2013 | Following to the <b>Italian</b> Central Ethics Committee and Competent Authority requirements and, in order to harmonise the protocol and the Informed Consent Form, the following changes have been done to the study protocol: - adjustment of the selection criteria n°10 related to the contraception method - addition of a letter that is given by the patient to his/her general practitioner (GP) - precision that the sponsor can not collect a copy of the Informed Consent Form - precision that the patient card is in Italian language only (without any English mention) | Local Italy |

Final version 341/1185

| N° | DATES | TYPE | APPLICATION<br>AREA | MODIFICATIONS | _ | FOCOL<br>SIONS |
|---|---|---|---|---|---|---|
| NA | | NA | General | | Version 1 | 09/11/2012 |
| NA | | NA | General | Following French CA request (ANSM): - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 | Version 2 | 15/01/2013 |
| PA01 | 01.03.2013 | Substantial | Local (Italy) | Following to the <b>Italian</b> Central Ethics Committee and Competent Authority requirements and, in order to harmonise the protocol and the Informed Consent Form, the following changes have been done to the study protocol: - Integration of the modification included in the protocol version 2 - Harmonisation of the protocol and the Informed Consent Form: * adjustment of the selection criteria n°10 related to the contraception method * addition of a letter that is given by the patient to his/her general practitioner (GP) * precision that the sponsor can not collect a copy of the Informed Consent Form * precision that the patient card is in Italian language only (without any English mention) | Version 3 | 01/03/2013 |

Final version 342/1185

#### 1. AMENDMENT RATIONALE

The clinical study protocol is updated with the following changes:

- change of Sponsor's Representative (Clinical Study Manager),
- modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed,
- precision on the function and address of the International Study Coordinator Pr Nodari,
- add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study),
- adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage",
- precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee),
- correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized).
- addition of the changes included in the local italian substantial protocol amendment (i.e : contraception method, letter to General Practionner, patient card in Italian and no collection of the consent form by the sponsor in Italy).

Final version 343/1185

## 2. CHANGES DESCRIPTION

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| Sponsor's Representative:<br>Marlène GUIRAUD, Pharm D | Sponsor's Representative:<br>Gaëlle ALCARAZ |
| INSTITUT DE RECHERCHE PIERRE FABRE -<br>Centre de R&D Pierre Fabre - BP 13562<br>3 avenue Hubert Curien<br>31035 TOULOUSE Cédex 1<br>Phone: +33 5 34 50 63 48 | INSTITUT DE RECHERCHE PIERRE FABRE -<br>Centre de R&D Pierre Fabre - BP 13562<br>3 avenue Hubert Curien<br>31035 TOULOUSE Cédex 1<br>Phone: +33 5 34 50 62 16 |
| Fax:+33 5 34 50 65 92<br>E-mail:marlene.guiraud@pierre-fabre.com | Fax:+33 5 34 50 XX XX (TBC)<br>E-mail:gaelle.alcaraz@pierre-fabre.com |
| Study Coordinating Investigator: | Study Coordinating Investigator: |
| Pr Savina NODARI Section of Cardiology Department of Experimental and Applied Sciences University of Brescia BRESCIA, ITALY Phone: +39 030 3996 587 - Fax: +39 030 3700 359 E-mail: savinanodari@gmail.com | Pr Savina NODARI – Associate Professor of Cardiology Department of Clinical and Surgical Specialities, Radiological Science and Public Health Section of Cardiovascular Diseases University Medical School and Spedali Civili Hospital of Brescia c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY Phone: +39 030 3996 587 - +39 030 393849 |
| | Fax:+39 030 3700359 E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a> ; <a href="mailto:nodari@med.unibs.it">nodari@med.unibs.it</a> |

Final version 344/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| CONTRACT RESEARCH ORGANISATIONS For intra erythrocyte DHA dosage: Agrocampus Ouest Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 | CONTRACT RESEARCH ORGANISATIONS For intra erythrocyte DHA dosage: Agrocampus Ouest Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 |
| 35042 RENNES Cedex - FRANCE Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr | 35042 RENNES Cedex - FRANCE Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr |
| | For transportation of blood sample to the Analytical centre (Agrocampus) and material supply: Theradis Pharma 41, chemin des Presses 06800 CAGNES-SUR-MER – France Phone: +33 (0)4 97 02 07 07 Fax: +33 (0)4 97 10 08 78 E-mail: chantal.raffy@theradis.pharma.com |
| | For refund of patients expenses linked to the patients expenses linked to the study: CLINACT 6-10 rue TROYON 92310 SEVRES – FRANCE Phone: +33 1 46 90 27 27 Fax: +33 1 46 23 01 56 Email: sebastien.beaumont@clinact.com |

Final version 345/1185

| PREVIOUS<br>VERSION | MODIFIED VERSION |
|---|---|
| STUDY | STUDY SYNOPSIS AND 5.1 INCLUSION CRITERIA |
| SYNOPSIS | Demographic Characteristics and Other Baseline Characteristics: |
| AND 5.1 | 10. For female patient of child-bearing potential: |
| INCLUSION | • in all the countries except Italy: |
| CRITERIA | - use of an effective method of contraception (hormonal contraception or intra-uterine |
| Demographic<br>Characteristics | device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to |
| and Other | 1 month after the last dose of the study treatment or |
| Baseline | - documented as surgically sterilized |
| Characteristics: | |
| 10. For female patient of child-bearing potential: | <ul> <li>in Italy only:</li> <li>absolute abstention from sexual intercourse during the whole duration of the study</li> </ul> |
| use of an effective method of contraception (hormonal contraception or intrauterine | <ul> <li>and for a month after the end of the study or</li> <li>use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or</li> <li>documented as surgically sterilized</li> </ul> |
| device) assessed by the investigator, for at least 2 months before | <ul> <li>11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion</li> <li>12. For male with a childbearing potential partner (In Italy only):</li> <li>absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or</li> </ul> |
| the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or - documented as surgica lly | - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study. |

Final version 346/1185

| steriliz<br>ed |
|----------------------------------|
| 11. For female patient of child- |
| bearing potential: |
| negative urine pregnancy test at |
| inclusion |

Final version 347/1185

#### PREVIOUS VERSION

#### **MODIFIED VERSION**

# STUDY SYNOPSIS, SECTION 3. Ethical CONSIDERATIONS RELATING TO THE STUDY and section 9. Study procedures:

STUDY SYNOPSIS, SECTION 3. Ethical CONSIDERATIONS RELATING TO THE STUDY and section 9. Study procedures:

Patients not stabilized for INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (transesophageal echocardiograph) performed in the same day (before ECV)

#### **5.9 Study CARD**

# 5.9 Study CARD and LETTER FOR GENERAL PRACTITIONERS (GP)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit, a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83.

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian without any English mention.
- a letter to be given to his/her general practitioner. This letter intends to inform the GP (and any other doctors who take care of the patient) that the patient participates to this clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

Final version 348/1185

#### **PREVIOUS VERSION**

#### **MODIFIED VERSION**

# 8.1. PRIMARY EFFICACY CRITERION:

#### 8.1.1.3. Evaluation Methods

• Trans Telephonic ECG Monitoring (TTEM):

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 to visit 6. Then, every two days from visit 6 to visit 9.

#### 8.2 BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.2.2 Technical handling

Two blood samples will be collected containing EDTA. They will be gently shaken and centrifuged at 3000g for 15 min at room temperature, within 30 minutes after collection. Plasma and white blood cells will be discarded. Red blood cells will be stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C) within 3 weeks following collection. Analysis will be performed within 2 weeks following reception at the Analytical centre.

# 8.1. PRIMARY EFFICACY CRITERION:

#### 8.1.1.3. Evaluation Methods

• Trans Telephonic ECG Monitoring (TTEM):

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 (week 6) to visit 5 (week 8). Then, every two days from visit 5 (week 8) to visit 9 (week 24 – End of study).

#### 8.2 BIOMARKER ASSESSMENT: RED BLOOD CELLCONCENTRATIONS OF DHA

#### 8.2.2.2 Technical handling

Two blood samples will be collected containing EDTA. They will be gently shaken, stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical centre.

Final version 349/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 8.3 SAFETY ASSESSMENT | 8.3 SAFETY ASSESSMENT |
| 8.3.2 Laboratory Investigations | 8.3.2 Laboratory Investigations |
| Laboratory investigations will be performed at | Laboratory investigations will be performed at |
| visit 1 (before treatment) and visit 9 (end of | visit 1 (before treatment) and visit 9 (end of |
| treatment) or End of Treatment visit. | treatment) or End of Treatment visit. |
| At visit 3 and 6, only an haematology examination will be performed. | At visit 3 and 6, only a standard haematologic dosage will be performed. |
| 10.2 Reporting of SAE | 10.2 Reporting of SAE |
| Marlène GUIRAUD, Pharm D | Gaëlle ALCARAZ |
| INSTITUT DE RECHERCHE PIERRE FABRE, Centre de R&D Pierre Fabre – BP 13562 3 Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 35 50 63 48 Fax: +33 5 34 50 65 92 Email: marlene.guiraud@pierre-fabre.com | INSTITUT DE RECHERCHE PIERRE FABRE, Centre de R&D Pierre Fabre – BP 13562 3 Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 35 50 62 16 Fax: +33 5 34 50 65 92 Email: gaelle.alcaraz@pierre-fabre.com |

Final version 350/1185

#### PREVIOUS VERSION MODIFIED VERSION 11.2. STUDY MONITORING 11.2. STUDY MONITORING 11.2.1.4. Closing Visit 11.2.1.4. Closing Visit At the end of the study, a final visit will be carried At the end of the study, a final visit will be carried out by the CRA to: out by the CRA to: • Verify that the e-CRFs CD-ROM with pdf files Verify that the e-CRFs CD-ROM with pdf files are correctly stored are correctly stored Control the accountability of intact and used Control the accountability of intact and used treatment units and return them to the Clinical treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction Pharmacy Department of the IRPF for destruction Obtain the last data clarifications and/or Obtain the last data clarifications and/or solutions if any solutions if any Collect the patient's consent forms in sealed Collect the patient's consent forms in sealed envelopes, envelopes (except in case of specific country requirement), Make an on-site review of all study Make on-site review study of documentation and complete it if necessary documentation and complete it if necessary And finally, remind the Investigator of his And finally, remind the Investigator of his regulatory obligations, study document archiving regulatory obligations, study document archiving process and duration. process and duration.

Final version 351/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 14.3 PATIENT'S INFORMATION<br>LEAFLET AND INFORMED<br>CONSENT FORM | 14.3 PATIENT'S INFORMATION<br>LEAFLET AND INFORMED<br>CONSENT FORM |
| The information and consent document are made in | The information and consent document are made in |
| triplicate: the original copy is kept by the | triplicate: the original copy is kept by the |
| Investigator, one copy is given to the patient and the | Investigator, one copy is given to the patient and the |
| last copy is kept by the Clinical Quality Assurance | last copy is kept by the Clinical Quality Assurance |
| Unit of the Sponsor in a sealed envelope at the end | Unit of the Sponsor in a sealed envelope at the end |
| of study. | of study (except in case of specific country |
| | requirement). |

Final version 352/1185

F 373280 CA 2 01

Final version 353/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

#### CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE - Centre de

R&D Pierre Fabre - BP 13562 3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 65 92

E-mail:gaelle.alcaraz@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI –

**Associate Professor of Cardiology** 

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>; nodari@med.unibs.it

#### Version 4-28 MAR 2013

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 354/1185

#### **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

#### **Clinical Study Manager (Monitor)**

Gaëlle ALCARAZ

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 62 16 Fax: +33 5 34 50 65 92

E-mail: gaelle.alcaraz@pierre-

fabre.com

#### **Medical Director**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 65 92

E-mail: richard.roche@pierre-

fabre.com

Final version 355/1185

#### CONTRACT RESEARCH ORGANISATIONS

#### For Feasibility, Monitoring and Regulatory issues:

#### Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

#### For Centralised Randomisation and Electronic Case Report Form

#### **S-Clinica**

6, Chaussée de Boondael B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

#### For Centralised Reading of Holder ECG and TTEM and equipment supply:

### **Biomedical System**

1945 Chaussée de Wavre B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage:

#### **Agrocampus Ouest**

Laboratoire de Biochimie 65 rue de Saint Brieuc – CS 84215 35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

#### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER - France

Phone: +33 (0)4 97 02 07 07 Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 356/1185

## **CONTRACT RESEARCH ORGANISATIONS**

## For refund of patients expenses linked to the study (in France):

**CLINACT** 

6-10 rue TROYON 92310 SEVRES – FRANCE Phone: +33 1 46 90 27 27

Fax: +33 1 46 23 01 56

Email: sebastien.beaumont@clinact.com

Final version 357/1185

# Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 4 - 28 MAR 2013

| Sponsor's | Repr | esentative: |
|-----------|------|-------------|
|-----------|------|-------------|

Medical Director: Richard ROCHE, MD Date: 14/08/18 Signature:

Study Coordinating Investigator: Savina NODARI, MD

20/05/13 Some

Signature

#### Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

#### **Protocol Version 4 – 28 MAR 2013**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 359/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

Protocol Version 4 – 28 MAR 2013

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 28 March 2013 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| " <u> </u> | 0 | be | adapted |
|------------|---|----|---------|
|------------|---|----|---------|

| Date: | Signature: |
|-------|------------|

Final version 360/1185
# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 23 |
|------------------|----------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 23 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | |
| 1.2.1. | Chemical and pharmaceutical characteristics | 26 |
| 1.2.1. | | |
| 1.2.1. | 5 | |
| 1.2.2. | | |
| 1.2.2. | 6 - 7 | |
| 1.2.2.<br>1.2.2. | | |
| 1.2.2. | | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 31 |
| 2. | STUDY OBJECTIVES | 34 |
| 2.1. | PRIMARY OBJECTIVE | 34 |
| 2.2. | SECONDARY OBJECTIVES | 34 |
| 3. | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 34 |
| 4. | STUDY DESIGN | 36 |
| 4.1. | OVERALL DESCRIPTION | 36 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 37 |
| 4.2.1. | . Choice of the Study Population | 37 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 40 |
| <b>5.</b> | STUDY POPULATION | 40 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 41 |
| 5.3. | NUMBER OF PATIENTS | 42 |
| 5.4. | RECRUITMENT MODALITIES | 42 |
| 5.5. | PATIENTS IDENTIFICATION | 42 |
| 5.6. | WITHDRAWAL CRITERIA | 42 |
| 5.7. | REPLACEMENT OF PATIENTS | 43 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 44 |
| 5.9. | STUDY CARD | 44 |

| 6. | STUDY TREATMENT | 44 |
|---|---|---|
| 6.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 11 |
| 6.2. | PACKAGING AND LABELLING | |
| 6.2.1. | | |
| 6.2.1.<br>6.2.2. | | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | |
| 6.5. | DRUG ADMINISTRATION | |
| 6.5.1. | | |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration | 48 |
| 6.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 49 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| 7. | CONCOMITANT TREATMENTS | 49 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 50 |
| 7.2. | PROHIBITED TREATMENTS | 50 |
| 7.3. | AUTHORISED TREATMENTS | 51 |
| 8. | EVALUATION CRITERIA | 51 |
| 8.1. | PRIMARY EFFICACY CRITERION: | 51 |
| 8.1.1. | | |
| 8.1.1. | | |
| 8.1.1.<br>8.1.1. | | |
| 8.1.1.<br>8.1.2. | | |
| 8.1.2. | 1. Numbers of Atrial Fibrillation episodes in the first week following visit 3 (ECV | |
| | visit) | 52 |
| 8.1.2. | | 52 |
| 8.1.2. | visit) | |
| 8.1.2. | | |
| 8.1.2. | 5. Evolution of echocardiographic parameters | 55 |
| 8.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF | |
| | DHA | |
| 8.2.1. | | |
| 8.2.2. | 1 | |
| 8.2.2.<br>8.2.2. | | |
| 8.2.3. | $\boldsymbol{\mathcal{E}}$ | |
| 8.3. | SAFETY ASSESSMENT | 57 |

| 3.3.1. Adverse Events | 57 |
|----------------------------------------------------------------|----|
| 8.3.2. Laboratory Investigations | 57 |
| 8.3.2.1. Schedule | 57 |
| 8.3.2.2. Technical Procedures and Parameters | 57 |
| 8.3.3. Global Physical Examination | 58 |
| 8.3.4. Vital Signs | 58 |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.3.7. Concomitant Treatments | |
| 8.4. COMPLIANCE | 60 |
| 9. STUDY PROCEDURES | 61 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 66 |
| 10.1. ADVERSE EVENTS | 66 |
| 10.1.1. Definition of Adverse Events | 66 |
| 10.1.2. Grading of Adverse Events | |
| 10.1.3. Reporting of Adverse Events | 67 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 67 |
| 10.2.1. Definition | 67 |
| 10.2.2. Reporting of SAE | 68 |
| 10.2.3. Follow-up of SAE | 69 |
| 10.2.4. SAE Occurring After the Study | 69 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 69 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 69 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | |
| 11. DATA COLLECTION AND STUDY MONITORING | 70 |
| 11.1. DATA COLLECTION | 70 |
| 11.1.1. Case Report Form | 70 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | 72 |
| 11.2.1. Monitoring visits | 72 |
| 11.2.1.1. Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | 73 |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | 73 |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | 74 |
| 12 DATA MANACEMENT | 74 |

| 12.1. DATA ENTRY | 74 |
|---|---|
| 12.2. DATA CLEANING | 74 |
| 12.3. DATA CODING | 75 |
| 12.4. DATA STORAGE | 75 |
| 12.5. DATABASE LOCK | 75 |
| 13. STATISTICAL ANALYSIS | 75 |
| 13.1. GENERAL CONSIDERATIONS | 76 |
| 13.2. SAMPLE SIZE | 76 |
| 13.3. PROTOCOL DEVIATIONS | 76 |
| 13.4. DATA SETS ANALYSED | |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | 77 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 78 |
| 13.7. EFFICACY ANALYSIS | 78 |
| 13.7.1. Primary Criterion | 78 |
| 13.7.1.1. Primary Analysis | 78 |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2. Secondary Criteria | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | 80 |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 85 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 85 |
| 14.1. ETHICAL CONDITIONS | 85 |
| 14.2 ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 85 |

| 14.3. | PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 86 |
|---|---|---|
| 14.4. | PERSONAL DATA PROTECTION | 87 |
| 14.5. | INSURANCE POLICY | 87 |
| 15. | ADMINISTRATIVE PROCEDURES | 87 |
| 15.1. | PROTOCOL AMENDMENT | 87 |
| 15.2. | SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 88 |
| 15.3. | END OF THE STUDY | 88 |
| 15.3. | J | |
| 15.3. | | |
| 15.3. | | |
| 15.3. | | |
| 15.4. | | |
| 15.5. | INSPECTION | |
| 15.6. | CONFIDENTIALITY | 90 |
| 15.7. | CLINICAL STUDY REPORT | 90 |
| 15.8. | STUDY RESULTS COMMUNICATION | 90 |
| 15.9. | STUDY RESULTS PUBLICATION | 90 |
| 16. | REFERENCES | 92 |
| <b>17.</b> | APPENDICES | 95 |
| 17.1. | DECLARATION OF HELSINKI | 96 |
| 17.2. | SAE REPORT FORM | 100 |
| 17.3. | PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 103 |

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | International, multicentric, randomised, double-blind, placebo controlled study Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of Atrial Fibrillation (AF) induced by burst pacing.[1] Moreover, the effectiveness of PUFA (PolyUnsaturated Fatty Acid) has been proven in the following conditions: - prevention of Atrial Fibrillation recurrence in patients with persistent Atrial Fibrillation, in co-administration with amiodarone (add on therapy) [2] - Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – April 2014 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 (anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> <li>Treatment duration: 24 weeks</li> </ul> |
| Study Schedule | 9 visits will be scheduled: - V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit) - V2/D1: Inclusion visit (start of treatment) - V3/W4 (D28 -2/+7 days): cardioversion visit (Outpatient or hospitalization according to |

Final version 366/1185

| | <ul> <li>clinical practice of the centre) (installation of the Holter device)</li> <li>V4/ W5 (D35± 2 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V5/ W8 (D56± 7 days): follow-up visit</li> <li>V6/ W12 (D84 ± 7 days): follow-up visit</li> <li>V7/ W16 (D112 ± 7 days): follow-up visit</li> <li>V8/ W20 (D140 ± 7 days): follow-up visit</li> <li>V9/ W24 (D168 ± 7 days): final study visit</li> </ul> |
|---|---|
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | Inclusion Criteria: |
| | Demographic Characteristics and Other Baseline Characteristics: |
| | <ol> <li>Men or women aged more than 18 years (inclusive),</li> <li>Patients with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.</li> <li>History of first documented persistent AF less than 1 year</li> <li>History of ischemic or non ischemic heart failure</li> <li>NYHA class I or II chronic heart failure at selection and at inclusion</li> <li>Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) ) at selection and at inclusion</li> <li>On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers</li> <li>Left atrial area ≤ 40 cm² ) at selection and at inclusion</li> <li>Patients treated or having to be treated by anti-vitamin K</li> <li>For female patient of child-bearing potential: <ul> <li>in all the countries except Italy:</li> <li>use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the</li> </ul> </li> </ol> |
| | selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment - documented as surgically sterilized in Italy only: - absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or |

- and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study.

## Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

History of first documented episode of persistent AF more than 1 year

Final version 367/1185

| | , |
|---|---|
| | More than two successful cardioversions (electrical or pharmacological) in the last 6 months |
| | 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV) |
| | 4. NYHA class III or IV heart failure at selection or at inclusion |
| | 5. Thyroid disease uncontrolled by treatment: TSH $\pm$ T4L $\pm$ T3L to be checked in case of |
| | treatment for thyroid disease 6. Myocardial infarction or unstable angina or presence of unstable ischemic |
| | coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice |
| | stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection |
| | 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection |
| | 8. Bradycardia (HR ≤ 50 bpm) |
| | <ul> <li>Hyperkalemia or hypokalemia (K&gt;5.5 mEq/L or K &lt; 3.5 mEq/L) at selection</li> <li>Cardiac surgery within 3 months before selection or planned during the study duration</li> </ul> |
| | Criteria related to treatments: |
| | 11. Previously ineffective pharmacological or electrical cardioversion |
| | 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers |
| | 13. Previous treatment with oral amiodarone within 12 months prior to inclusion |
| | 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion |
| | 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months |
| | 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months |
| | 17. Dietary supplement with ω3 or ω6 according to investigator's judgement |
| | 18. Having undergone any form of ablation therapy for AF |
| | <ol> <li>Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor<br/>such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel<br/>or Prasugrel</li> </ol> |
| | Other criteria: |
| | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion |
| | 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a |
| | trial at the time of selection 22. Patient linguistically or mentally unable to understand the nature, objectives and |
| | possible consequences of the trial, or refusing to patient himself/herself to its constraints 23. Patient family member or work associate (secretary, nurse, technician,) of the |
| | Investigator 24. Patient having forfeited his / her freedom by administrative or legal award or being |
| | under guardianship |
| | 25. Breastfeeding female patient |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive |
| | weekly tests performed before ECV will be excluded from the study, unless the presence of |
| | atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) |
| | performed in the same day (before ECV) ECV will be performed in patients without dyskalemia |
| | If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) |
| | could be postponed by 7 days. |
| Test Product: | F373280 |
| Dose: | Soft Capsules<br>Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| Duration of Treatment: | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules |
| | Placebo will be administered in the same conditions as the tested product. |

Final version 368/1185

| Mode of Administration: | Oral, one capsule each evening with dinner |
|---|---|
| Evaluation Criteria: | Efficacy evaluation variables: |
| | Primary evaluation variable: Time to first Atrial Fibrillation recurrence defined by the first episode of Atrial Fibrillation lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit) Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24. For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5). Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM. All ECG traces will be evaluated by a Central Reading Laboratory. |
| | Secondary evaluation variables: During the 7-day continuous ECG monitoring, Numbers of AF episodes Duration of AF episodes |
| | Clinical parameters: During the whole study: Number of recurrence of symptomatic AF episodes EHRA score Hospitalization for cardiovascular events Hospitalization for thromboembolic stroke All cause of hospitalization |
| | <ul> <li>Cardioversion: <ul> <li>Assessment of spontaneous cardioversion</li> <li>Assessment of successful cardioversion</li> <li>Number of patients needing an other cardioversion after the initial ECV</li> </ul> </li> </ul> |
| | Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m², Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL)) • Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized). |
| | <ul> <li>Safety criteria:</li> <li>Adverse events (observed and / or spontaneously reported)</li> <li>Vital signs (Blood pressure (supine and standing), heart rate</li> <li>Physical examination (body weight),</li> <li>Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized).</li> <li>Haematology: haematocrit, haemoglobin, RBC, WBC, differential count, platelets</li> <li>Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)</li> <li>Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR (local laboratory), Prothrombine Time (PT)</li> </ul> |
| Statistical Methods: | Sample Size: Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. |

Final version 369/1185

## **Primary Efficacy Analysis**

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### **Secondary Analyses**

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

## Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment)

Final version 370/1185

# STUDY FLOW-CHART

Final version 371/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 +/-2 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | х | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic characteristics | х | | | | | | | | |
| Medico-surgical history | х | | | | | | | | |
| Concomitant disease | х | | | | | | | | |
| Concomitant treatment | х | х | х | х | х | х | х | х | х |
| Habits | х | | | | | | | | |
| Global physical examination (body weight) | х | х | х | | х | х | х | х | х |
| Echocardiography | х | x | | х | | х | | | x |
| Eligibility criteria check | х | х | | | | | | | |
| Blood pressure, heart rate | х | х | х | х | х | х | х | x | x |
| 12-Lead ECG Recording | х | x | х | | х | х | х | х | x |
| INR | <b>→</b> | | (2) | | х | х | х | х | x |
| аРТТ, ТСТ | х | х | х | | х | х | х | х | x |
| Biochemistry | х | | | | | | | | x |
| Hematology | х | | х | | | х | | | х |
| Urinary pregnancy test | | x | | | | | | | x |
| Red Blood Cell concentrations of DHA | | x | х | | | х | | | x |
| Treatment allocation | | х | | | | х | | | |
| IVRS | х | x | | | х | х | | | |
| ECV (3) | | | х | | | | | | |
| Drug administration | | <b>+</b> | | | | | | | <b>—</b> |
| Adverse events recording | | х | x | x | x | х | х | х | x |
| Holter ECG | (4) | | - | (5) | | | | 4 | |
| TTEM (6) | | | | | | | | 4 | <b>→</b> |

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)

Final version 372/1185

<sup>(2)</sup> In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(5) 7-</sup>day Holter ECG

<sup>&</sup>quot;O'TTEM everyday from week 6 to week 8. Then every 2 days from week 9 to week 24. In case of AF symptoms. In case of AF recurrence for at least 10 minutes and the patient does not stop the study treatment then TTEM every 4 weeks

## LIST OF ABBREVIATIONS

aPTT Activated partial thromboplastin time

AE : Adverse event

AERP Atrial effective refractory period

AF : Atrial fibrillation
ALA Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK Anti vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP Blood pressure
BSA : Body Surface Area

CEP Protocol evaluation committee

CHF : Congestive heart failure

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO –TE Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA European heart rhythm association

EPA Eicosapentaenoic acid eCRF Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

Final version 373/1185

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL High density lipoprotein

HF Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS Interactive voice response system

LAA Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL Low density lipoprotein LOQ : Limit of quantification

LVEF Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR Mineralocorticoid receptor
MR perfusion Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie
POC Proof of concept

PUFA : PolyUnsaturated fatty acid

PK : Pharmacokinetics

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT Thrombin clotting time

TEAEs Treatment emergent adverse events
TTEM TransTelephonic ECG monitoring

VTP : Ventricular tachypacing

WBC White blood cells

WHO-DRUG: World health organization drug reference list

Final version 374/1185

## 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of atrial fibrillation (AF) in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the PUFAs (Polyunsaturated Fatty Acids) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are ALA, EPA and DHA. First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or atrial fibrillation.

The potential anti-arrythmic effects of a PUFA was previously developed in atrial fibrillation: nicotinyl ester of DHA (pro-drug based on DHA delivery) were assessed in a two-week

Final version 375/1185

ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of atrial fibrillation (AF) induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll assessed n-3 Polyunsaturated Fatty Acids in the prevention of atrial fibrillation recurrences after electrical cardioversion. All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct electrical cardioversion (ECV) 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95%] confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent atrial fibrillation on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion [2]. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFA on top of traditional treatment (amiodarone, beta blockers, reninangiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than placebo group at one month (3.3% vs 10%; p=0.043), at 3 months (10% vs 25%; p=0.004) and at 6 months (13.3% vs 40%; p<0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effect of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Final version 376/1185

Nodari and coll [3] performed a trial in patients with a chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (P = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, P = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent atrial fibrillation and heart failure in the maintenance of sinus rhythm after electrical cardioversion.

#### 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA (docosahexaenoic acid) is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of atrial fibrillation.

F373280 is a prodrug of DHA.

Final version 377/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

## 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

## 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

Final version 378/1185

#### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period (AERP) were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased AERP (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, P<0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the ECG intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing (VTP)-induced congestive heart failure (CHF) provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses CHF-induced AF-promotion and fibrosis in the VTP canine model. Nicotinyl ester of DHA was tested in this model, at 1g/day and 5g/day, during 4 weeks, to prevent CHF-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in atrial fibrillation duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus  $637 \pm 196$  sec, n=5 in the presence of 1g/kg/d Nicotinyl ester of DHA and  $79 \pm 51$  sec, n=5, in the presence of 5g/kg/d Nicotinyl ester of DHA The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280

Final version 379/1185

similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the

compound may exert a similar protective effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 gm/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 380/1185

6 consecutive single ascending doses were tested (0.5g, 1g, 2g, 4g, 8g and 16g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 4 were observed in the placebo group (palpitation, dizziness in standing position, 2 symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events were reported in the groups of F373280 at the dosages of 0.5g, 1g, 2g, 4g and 8g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5g to 16 g in 36 young male healthy subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirm that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding PK parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16g with no departure from proportionality (baseline corrected parameters).

Final version 381/1185

## Part B: Multiple dose

Three consecutive repeated ascending doses (1, 2 and 4g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280 5/9 TEAE were classified according the SOC in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAE have already been reported with Poly Unsaturated Fatty Acids and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 382/1185

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of atrial fibrillation (AF) induced by burst pacing [1].

Moreover, the effectiveness of PUFA has been proven in the following conditions:

- Prevention of atrial fibrillation recurrence in patients with persistent atrial fibrillation in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor®, [9]:

Final version 383/1185

- The frequencies of adverse reactions are ranked according to the following: common (> 1/100, < 1/10); uncommon (>1/1000 < 1/100); rare (>1/10000, < 1/1000); very rare ( < 1/10000), not known (cannot be estimated from the available data).
  - The reported adverse events are:
- Infection and infestations

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

• Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

• Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

Final version 384/1185

## • Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1g and 4g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in Atrial Fibrillation studies [2, 8]. The range of PUFAs doses tested was between 2g to 3g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in heart failure patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1g to 5g (1g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Final version 385/1185

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct electrical cardioversion
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

Final version 386/1185

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of atrial fibrillation and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (AVK), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication,
- Anticoagulation with anti-vitamin K for at least 3 weeks before ECV,
- ECV in patients with stabilized INR (i.e. values between 2 and 3) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

Final version 387/1185

- Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent atrial fibrillation and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35  $\pm$  2D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit

Final version 388/1185

- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent atrial fibrillation and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent atrial fibrillation with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters,
   morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- early persistent atrial fibrillation history (less than one year) with a duration of a the current episode between 7 days to 6 months
- a moderately abnormal moderately systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- A Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent atrial fibrillation associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or

Final version 389/1185

unstable ischemic coronaropathy (assessed by coronarography or cardiac stress test or effort test within 6 months before selection).

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on anti-arrhythmics on atrial fibrillation (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be developed as a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, anti-arhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent atrial fibrillation and requiring an electrical cardioversion will be included in order to assess the time to first documented recurrence of atrial fibrillation since cardioversion.

To confirm the persistent nature of atrial fibrillation, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before electrical cardioversion. According to guidelines for the management of atrial fibrillation [6], anti-vitamin K should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation, of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodary study [2], the duration of pre-treatment with PUFA before cardioversion appears to be a contributing factor in

Final version 390/1185

success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of atrial fibrillation recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of atrial fibrillation recurrence occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using a more easy to carry and easy to use device, a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

## 4.2.3. Choice of the Dose

According to a previous study in patients with atrial fibrillation [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of atrial fibrillation after cardioversion. Moreover, PUFAs at dosage of 1g and 2g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95mg/mL and 60 to 90mg/mL, respectively) (phase I study of F373280 and Salm and coll study) [16]. With regard to the rythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a dose of 1 g daily of F373280 is considered to be appropriate to be tested in this POC study.

Final version 391/1185

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive),
- 2. Patient with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted.
- 3. History of first documented persistent AF less than 1 year
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

## • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator, for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- documented as surgically sterilized

#### • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):

Final version 392/1185

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or

## Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation),

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 1 year,
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be check in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercice stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (K > 5.5 mEq/L or K < 3.5 mEq/L) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,

Final version 393/1185

- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship,
- 25. Breastfeeding female patient.

#### 5.3. NUMBER OF PATIENTS

76 x 2 patients (taking into account 15 % of non evaluable patients).

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO,...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENTS IDENTIFICATION

The patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

The reasons for a patient's premature withdrawal from the study may be the following:

- The patient's decision. A patient who wishes to withdraw from the study for any reason may do so at any time but must inform the investigator. In all cases, the Investigator should attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form

Final version 394/1185

- obtain the reason(s) for withdrawal and report it/them in the case report form
- evaluate the patient's clinical condition
- if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- The Investigator's decision in the patient's interest. Particularly, if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.
- An erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion / non inclusion criteria will immediately be withdrawn and an appropriate treatment will be instored by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with anti-vitamin K for at least 3 weeks before ECV,
- Patients who will not stabilize INR between 2 and 3 on at least 3 consecutive weekly tests
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 week for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV (i.e. unsuccessful ECV) will be considered to have finished follow-up.
- An occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and uncomfortable clinical symptoms.

#### 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

Final version 395/1185

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit,

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.

- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

• F373280

Final version 396/1185
Formulation of F373280, 1g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

#### 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

# 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1g F373280 soft capsules or placebo soft capsules each.

# 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number,
- c) packaging batch number,
- d) the treatment number
- e) storage conditions

Final version 397/1185

- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
  - "for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose".

On the treatment unit, another label will be affixed with the mention of the investigator name and patient number (completed by the investigator).

In addition, on each case, will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

#### 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

• Details of storage conditions that should be respected

Final version 398/1185

• And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person.

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion Visit and another one at Visit 6.

For each patient, the treatment number given at Visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Calls the vocal server
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the vocal server.

Final version 399/1185

- The IVRS/IWRS company:
  - Confirms this information by fax/email to the Investigator
  - Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 5, the Investigator will contact again the IVRS/IWRS to obtain for visit 6 the treatment number for the last 12-week period of treatment according to the same process as described above.

#### 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure will be 24 weeks, with F373280 or placebo.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

#### 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

Final version 400/1185


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

#### 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator, in collaboration with the Sponsor representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF, according to the Sponsor's procedures.

### 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (Selection Visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted

Final version 401/1185

on e-CRF. All treatments should be evaluated by the investigator at selection and their prolongation during the study or their stop should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

#### 7.1. ANTI-VITAMIN K TREATMENT

Anti-vitamin K should be given for at least 3 weeks before ECV and continued for the whole study duration. The anti-vitamin K used will be left to the decision of the each investigator according to his/her local practice.

# 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
    - Class IA: Disopyramide, Procainamide, Quinidine
    - Class IB: Lidocaine, Mexiletine
    - Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Any Polyunsaturated Fatty Acid (PUFA)
- Any anticoagulant treatment other than antivitamin K: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

Final version 402/1185

#### 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the case report form. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

# 8. EVALUATION CRITERIA

### **8.1. PRIMARY EFFICACY CRITERION:**

#### **8.1.1.** Time to the first Atrial Fibrillation Recurrence

# 8.1.1.1. **Definition**

Time to first Atrial Fibrillation recurrence is defined by the first episode of Atrial Fibrillation (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of electrical cardioversion visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

# 8.1.1.3. Evaluation Methods

# • 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM)

Final version 403/1185

# • Trans Telephonic ECG Monitoring (TTEM):

Thus, the follow up will be documented using the TTEM: daily transmission from visit 4 (week 6) to visit 5 (week 8). Then, every two days from visit 5 (week 8) to visit 9 (week 24 – End of study).

Moreover, during this TTEM period, if patient experiences AF symptoms, it should be documented using the TTEM.

In case of AF recurrence, and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at the investigator's judgement, he/she could be maintained in the study with the treatment, in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

# 8.1.2. Secondary Efficacy Criteria

# 8.1.2.1. Numbers of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

# 8.1.2.1.1. *Definition*

Number of Atrial Fibrillation episodes will consist in the assessment of episodes of AF with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

#### 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the study visit 4.

Final version 404/1185

#### 8.1.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

# 8.1.2.2. Duration of Atrial Fibrillation episodes in the first week following visit 3 (ECV visit)

# 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episodes.

#### 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful electrical cardioversion visit (visit 3) to the follow up study visit (visit 4).

#### 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

# 8.1.2.3. Clinical parameters evaluation

#### 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition:

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected

Final version 405/1185

- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month); intermediate (1/month to almost daily); and frequent at least daily.

#### 8.1.2.3.1.2. Schedule

This evaluation will be performed in case of symptoms evocative of arrhythmia.

#### 8.1.2.3.1.3. Evaluation Methods

This evaluation will be collected by Central Reading Laboratory during all the study period.

# 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of number of AF recurrence associated with a symptom (Palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG in atrial fibrillation.

# 8.1.2.3.3. Number and duration of hospitalization

- Number and duration of hospitalization for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
  - Hospitalization for myocardial infarction
  - All cause of hospitalization
- Number and duration of hospitalization for thromboembolic stroke

#### 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)

Final version 406/1185

• Number of patients needing another cardioversion after initial ECV

# 8.1.2.5. Evolution of echocardiographic parameters

# 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), Left atrial area (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m<sup>2</sup>, Left ventricular end diastolic diameter (mm) Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL),

#### 8.1.2.5.2. Schedule

The measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

The measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, for volume measurements, the recommended method is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.1. Definition

Because of the limited accessibility of human tissues for biopsy, red blood cell DHA contents is a marker for tissue DHA concentration [13], [14].

Final version 407/1185

# 8.2.2. Blood samples

#### 8.2.2.1. Collection schedule

Blood samples will be collected for determination of red blood cells (RBC) concentrations of DHA.

Blood samples will be performed as follows:

• Visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the electronic Case Report Forms (e-CRFs).

# 8.2.2.2. Technical handling

Two blood samples (4ml) will be collected in tubes containing EDTA. They will be gently shaken, stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical centre.

#### 8.2.3. DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol, after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells

Final version 408/1185

(expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk

for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end

of the study, and will be provided only at the end of the study (after database lock), in a separate

file.

8.3. SAFETY ASSESSMENT

8.3.1. Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the

occurrence of adverse events (AEs) since the last visit will be based on the patient's spontaneous

reporting, the investigator's non-leading questioning and his/her clinical evaluation. All AEs will

be reported on the e-CRF (see section 10).

8.3.2. Laboratory Investigations

8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of

treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The volume of blood samples complete haematology, biochemistry should not exceed 30 mL.

8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: Hematocrit, haemoglobin, Red blood cells (RBC) count, white blood cells

(WBC) count, WBC differential counts (% and absolute), reticulocytes,

platelets.

Final version 409/1185

Chemistry:

sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning, in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR  $(mL/min) = [(140-age)] \times weight / 7.2 \times serum creatinine in mg/L],$ 

in women:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as  $\mu$ mol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patients' interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

# 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

Final version 410/1185

#### 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic (SBP) and diastolic (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation, after at least 5 minutes in supine position and after 2 minutes in standing position by counting the beats for at least 30 seconds.

Bodyweight will be measured in patient in underwear and with the same balance at each visit.

# 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. *Schedule*

An electrocardiogram will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

## 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram (ECG):

The global interpretation from manual reading (normality, clinical relevance) and heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

#### • 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent atrial fibrillation.

Final version 411/1185

# **8.3.6.** Coagulation parameters

The assessment of coagulation will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV,
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV,
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by anti-vitamin K should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial can be found in section 7.

#### 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back any remaining soft capsules, blister, case (used or unused) at the following visit.

At each visit, the Investigator will record the number of supplied and remaining Soft Capsules in the e-CRF.

Final version 412/1185

# 9. STUDY PROCEDURES

## Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If he/she accepts to participate in the study, he/she will sign the informed consent and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and Atrial Fibrillation characteristics
- Echocardiography using a two-dimensional echocardiography.
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

Final version 413/1185

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory (CRL). The CRL will send his/her assessment regarding the confirmation of persistent atrial fibrillation within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (anti-vitamin K) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will contact the IVRS/IWRS system to confirm the patient selection and order the treatment delivery and organise the appointment for the next visit.

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

### Visit 2 - Inclusion Visit (Day 1)

If the patient's behaviour during the selection period and/or the result of complementary examinations particularly the confirmation of the presence of persistent atrial fibrillation by the CRL during this period, the INR and laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography.

Final version 414/1185

- 12-lead ECG
- Urine pregnancy test for women of child bearing potential.

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and allocated a treatment number using the IVRS/IWRS system.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.3.6), in order to ensure that the INR is stable, between 2 to 3 before electrical cardioversion.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

## Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, Red Blood Cell concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (transesophageal echocardiograph) performed in the same day (before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be

Final version 415/1185

induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

#### Visit 4 (Week 5: D35 $\pm$ 2 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of Adverse Events
- Concomitant treatments (authorised, disallowed)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device (Trans Telephonic ECG Monitoring) for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

Final version 416/1185

Visit 5 (Week 8: D56 ± 7 days) – Visit 6 (Week 12: D84 ± 7 days) - Visit 7 (Week 16: D112 ± 7 days) - Visit 8 (Week 20: D140 ± 7 days)

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- The cardiac monitoring will be continued using a TTEM device (Trans Telephonic ECG Monitoring). The device will be given to the patient who will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms additional transmission may be performed.

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week treatment period.

#### In addition:

- at visit 5, the investigator will contact the IVRS/IWRS to obtain another treatment unit to be dispensed at visit 6 for the last 12-week period.
- at visit 6, an echocardiography will be performed, an haematology examination will be done and the red blood cell concentration of DHA will be measured.

Final version 417/1185

## End-of-Study Visit - Visit 9 (Week 24: D168 ± 7 days)

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all the cases, blisters and any unused soft capsules and count the unused soft capsules.

# 10. ADVERSE EVENTS: DEFINITION AND REPORTING

#### 10.1. ADVERSE EVENTS

#### 10.1.1. Definition of Adverse Events

An adverse event is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

This includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values, which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as

Final version 418/1185

those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

# 10.1.2. Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity.

# **10.1.3.** Reporting of Adverse Events

The records of adverse events in the electronic Case Report Form (e-CRF) describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A serious adverse event (SAE) includes, but is not necessarily restricted to any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect.

Final version 419/1185

Other events such as cancer, and any additional adverse experience or abnormal laboratory values

occurring during the study period, defined by the protocol as serious or which the Investigator

considers significant enough, or that suggest a significant hazard, contra-indications, side effect or

precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the

SAE notification form (see section 10.4).

\* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:

planned (as per protocol) medical/surgical procedure,

- preparation for routine health assessment/procedure (e.g. routine colonoscopy),

- planned medical/surgical admission (planned prior to entry into study trial, appropriate

documentation required),

- administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver

respite, family circumstances)

will not be reported as a SAE.

10.2.2. Reporting of SAE

All serious adverse events, according to the above-mentioned definitions and regardless of

treatment or relationship to study drug, must be recorded by the Investigator as soon as he/she is

informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the

"Notification of serious adverse event" form ("first notification") (see appendix 17.2) with all the

available information about the event, to the Sponsor's representative:

Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE,

Centre de R&D Pierre Fabre – BP 13562

3 Avenue Hubert Curien

31035 TOULOUSE Cedex 1

Phone: +33 5 35 50 62 16

Fax: + 33 5 34 50 65 92

Email: gaelle.alcaraz@pierre-fabre.com

Final version 420/1185 In case of non-inclusion the reporting period ends when the non-inclusion is documented.

## 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

# 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage, and associated adverse event if any, are reported only on the Adverse Event page of the CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must be also transmitted to the sponsor.

#### 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and be withdrawn immediately from the study.

Final version 421/1185

If pregnancy is suspected while the patient is receiving study treatment, the study drug(s) should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is discontinued from the study.

The investigators must report to the sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The investigator must immediately notify the sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Women who become pregnant after exposure to the study drug must be followed by the investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

# 11.1.1. Case Report Form

An electronic Case Report Forms (e-CRF) will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files and which will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and include a traceability system for data corrections and deletions (audit trail).

Final version 422/1185

Prior to the start of the study, the Investigator will complete a "*Delegation of significant study-related duties*" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants who will use this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation.

At the end of the study, a CD-ROM containing the pdf version of all e-CRF (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

Final version 423/1185

## 11.2. STUDY MONITORING

# 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

## 11.2.1.2. Initiation Visit

Before the start of the study at all investigation sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
  - has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

Final version 424/1185

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

# 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

Final version 425/1185

#### 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of measures of primary end point, the safety data and to recommend to the Sponsor whether to continue, modify, or to stop the study.

The IDMC operating procedures will be described in an independent document.

# 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on a e-CRF.

The e-CRF used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

Final version 426/1185

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate coding.

#### 12.4. DATA STORAGE

The computer data files, as well as their modifications, will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e.: data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

# 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by Pierre Fabre Biométrie (PFB) or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan (SAP) approved by the Validation Committee.

Final version 427/1185

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 evaluable patients per group is required, using a log-rang test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

Final version 428/1185

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

#### 13.4. DATA SETS ANALYSED

The following 2 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

# **13.5.1.** Dropouts

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

# 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

#### 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

Final version 429/1185

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- Quantitative parameters will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

## 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

Final version 430/1185

# 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

# 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

# 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

## 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

# 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

Final version 431/1185

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

#### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patients will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAE

Final version 432/1185
- With at least three TEAE
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.
- Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:
- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

"The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TE AE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (<u>for all patient</u>).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

Serious adverse events will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time

Final version 433/1185

of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

# 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be identified differently. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of PSC range and CNALV range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

Final version 434/1185

Clinically noteworthy abnormal laboratory values (CNALV) (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and heart rate in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

Final version 435/1185

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

# 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

# 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by the rapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" (ATC) classification on the safety set.

Final version 436/1185

## 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) – number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days).

# 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

# 14. GENERAL ETHICAL CONSIDERATIONS

# 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

# 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

Final version 437/1185

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Final version 438/1185

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament, are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

# 15. ADMINISTRATIVE PROCEDURES

# 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Final version 439/1185

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

# 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF, drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not
- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents
- Authorises direct access to source documents for monitoring, audits and inspections
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

### 15.3. END OF THE STUDY

# 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

Final version 440/1185

# 15.3.2. Early Study Termination

# 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if it considers that the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both his representatives (Study Manager, CRA, ...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

Final version 441/1185

### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

# 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed to in writing with the Study Manager, the investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

# 15.7. CLINICAL STUDY REPORT

Data analysis, and clinical study report writing are under the Sponsor's responsibility.

Upon completion of the data analysis, a final report, including a review of the objectives and methods, a presentation and discussion of the results are drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

#### 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

Final version 442/1185

To allow use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 443/1185

# 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version January 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 444/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

# [14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 445/1185

# [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

# [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

# [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

# [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

# [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 446/1185

# 17. APPENDICES

Final version 447/1185

#### 17.1. DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 448/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 449/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 450/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 451/1185

# 17.2. SAE REPORT FORM

Final version 452/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE PRODUCT SAFETY DEPARTMENT |
|---|
| TO BE TRANSMITTED TO THE MONITOR BY FAX WITHIN 24H: G. ALCARAZFax n° +33 5 34 50 65 92 |
| Transmission date |
| SAE N° FIRST NOTIFICATION FOLLOW-UP |
| > SUBJECT CHARACTERISTICS |
| Surname Birth date Birth date |
| Gender1=M, 2=F Heightcm Weight kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date |
| Seriousness onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| Summary description (it enmed eduse, significant instory, progression of event, available according results, etc) |
| (*) Franch and braid limit and the district and a should be described by |
| (*) Except hospitalisations with durations and goals planned in the protocol > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| <ul> <li>□ During the selection or run-in period</li> <li>□ During the administration phase of the study treatment</li> <li>□ After the administration phase of the study treatment</li> </ul> |
| Date of first study treatment administration (ddmmyyyy) |
| Date of last study treatment administration before the occurrence of SAE (ddmmyyyy) |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 453/1185

| Transmission date | | | (ddmmyyyy) | Country: | | ••••• |
|---|---|---|---|---|---|---|
| SAE N° | FIRST NOTIFICATION ☐ FOLLOW-UP ☐ | | | | | |
| > CONCOMITANT MEDICATION SINCE TRIAL INITIATION and UP UNTIL THE OCCURRENCE OF THE SAE (EXCEPT THE TREATMENTS GIVEN FOR THE SAE) | | | | | | |
| INN or trade name | Daily dose | Start date (ddmmyy) | Ongoing at occurence of the event | Stop date (ddmmyy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAK | EN FOLLOWIN | NG THE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage mod | ification, specify | ······ | Modi | fication Date : | /_ | / |
| ☐ Temporarily | discontinued | | Readministr | ration date: | / | / |
| ☐ Withdrawn | | | | End date : | / | / |
| ☐ Not applicab | le | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription | of corrective or s | symptomatic treatmen | ts (specify names and | d dosages): | | |
| ☐ Discontinuat | tion of concomita | ant treatments (specify | names) : | | | |
| Others spec | :c | | | | | |
| ☐ Others, spec | iiy : | | | | | |
| <b>&gt;</b> OUTCOME | | | | | | |
| □ Not recovered/ | | ☐ Recovering/ | - | Recovered/Resolve | ed | |
| ☐ Recovered/Resolved with sequelae ☐ Fatal ☐ Unknown | | | | | | |
| In case of death, has an autopsy been conducted? $\square$ Yes $\square$ No | | | | | | |
| > INVESTIGATOR CAUSALITY ASSESSMENT (investigator's assessment to be done as soon as possible) | | | | | | |
| □ Not Suspected □ Suspected □ Insufficient data | | | | | | |
| comments : | | | | | | |
| Eng | close in the notific | ation the results of carr | ried out examinations | renorts of hospitalisa | ition, etc | |

Final version 454/1185

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| NOTATIONAL | Protein | g/l | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pH | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/I | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 455/1185

<sup>(

)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

# **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | Decrease of at least 2g/dl and value < 10 g/dl whatever the baseline value If missing baseline : value <10g/dl |
| NEUTRO | PHILS | $\bullet$ < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC<br>(if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline: <ul> <li>TB &gt; 1.5 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>TB &gt; 2 N</li> </ul> </li> </ul> |

# N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 456/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>oaseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the for each parame | Minimum Post-bo<br>ter | aseline Value |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤ <i>50</i> | ≤90 | ≤ 50 | ≤50 |
| [120;140] | [80;90[ | <i>[50 ;75]</i> | [90 ;120] | [50;80[ | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) SBP < 140 and DBP < 90 | Pressure (mmHg) SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100<br>or DBP [90;100[ and SBP < 160 | $SBP \le 90 \text{ or } DBP \le 50$ |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq 20$ mmHg or DBP Decrease $\geq 10$ mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 457/1185

16.1.1.5. Protocol amendment n° PA03
General and substantial dated on 23 October
2013 linked to Protocol and appendices
(version 5: 23 October 2013)

Final version 458/1185

CLINICAL STUDY PROTOCOL AMENDMENT n° PA03 Version 1 (General – Substantial)

Final version 459/1185

Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne, France

#### CLINICAL STUDY PROTOCOL AMENDMENT n° PA03 Version 1

(General – Substantial)

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Pierre Fabre Study Code: F373280 CA 2 01

**EudraCT Number or equivalent:** 2012-003487-48

Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE - Centre de R&D Pierre

**Sponsor's Representative:**Fabre - BP 13562
3 avenue Hubert Curien

31035 TOULOUSE Cedex 1

Pr Savina NODARI

Department of Clinical and Surgical Specialities, Radiological

Science and Public Health

Section of Cardiovascular Diseases

Study Coordinating Investigator: University Medical School and Spedali Civili Hospital of Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

**Date of amendment PA03:** 23 October 2013

Final version 460/1185




Study code: F373280 CA 2 01

# APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Clinical Study Protocol Amendment no PA03 Version 1

(General - Substantial)

Dated:23/10/2013

| Sponsor's representative(s) Medical Director | Dr Richard ROCHE | Date: 291121313 | Signature: | //e} |
|---|---|---|---|---|
| · Clinical Study Manager : | Gaëlle ALCARAZ | Date: 23 OCT 233 | Signature: | |
| Study Coordinating Investigate | or:<br>Pr Savina NODARI | Date: | Signature: | Shadd |




Study code: F373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Clinical Study Protocol Amendment no PA03 Version 1

(General – Substantial) Dated: 23/10/2013

Country Coordinating Investigator: SAVINA NODAN Date: 13/01/2014 Signature: Some Wall

# **INVESTIGATOR SIGNATURE FORM**

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

# Clinical Study Protocol Amendment nº PA03 Version 1

(General – Substantial)

Dated: 23/10/2013

| By my signature below, I, Dr | , hereby confirm that I have read, taken |
|---|---|
| | ght by the protocol amendment n° PA03 and I will |
| conduct the trial according to these new modalities | <b>5.</b> |
| Date: | Signature: |

Final version 463/1185

# HISTORY OF AMENDMENTS

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| NA | NA | General | NA | Following French CA request (ANSM) and leading to protocol version 2: - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 |
| PA01 | Substantial | Local (Italy) | 01.03.2013 | Corresponding to Protocol Version 3: - Integration of the modification included in the protocol version 2 - Harmonisation of the protocol and the Informed Consent Form: * adjustment of the selection criteria n°10 related to the contraception method * addition of a letter that is given by the patient to his/her general practitioner (GP) * precision that the sponsor can not collect a copy of the Informed Consent Form * precision that the patient card is in Italian language only (without any English mention) |
| PA02 | Non<br>Substantial | General | 28.03.2013 | Corresponding to Protocol Version 4: - change of Sponsor's Representative (Clinical Study Manager), - modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed, - precision on the function and address of the International Study Coordinator Pr Nodari, - add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study), - adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage", - precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee), - correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized) addition of the changes included in the local italian substantial protocol amendment (i.e: contraception method, letter to General Practionner, patient card in Italian and no collection of the consent form by the sponsor in Italy). |

Final version 464/1185

#### 1. AMENDMENT RATIONALE

This amendment relates to an adjustment of some criteria in order to improve the feasibility of the study and to minor changes as typographical errors or style. Finally a change affects the recipient of the SAEs reports.

The clinical study protocol is updated with the following changes:

- Due to a recruitment rate significantly lower than expected the planned end of study is postponed to January 2015.
- The authorized history of the first documented persistent atrial fibrillation passes from less than 1 year to less than 3 years. This modification will expand our target population without changing the characteristics of the selected patients by enabling the management of patients who experienced a longer period without relapse.
- At selection a hyperkalemia or a hypokalemia will be better defined by the standards of the local laboratories.
- Regarding previous treatments by amiodarone the non inclusion criteria of the protocol are adapted as follow:
  - Previous treatment with oral amiodarone within 4 months prior to inclusion
  - Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion.
  - Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion

Despite the long half life of amiodarone, these time limits relating to its non-use before inclusion allow to ensure the absence of amiodarone at sufficient levels to interfere with the assessment of the product.

- For male with a child-bearing potential partner (in Italy only):

  Taking into account the duration of spermatogenesis the absolute abstention from sexual intercourse or the use of double barrier contraception method are extended to 3 months after the end of the study.
- Ranolazine is an antiangina treatment with antiarrhythmic properties. This treatment is added to the prohibited treatments in order to exclude a potential association between the study product and a treatment having an antiarrhythmic effect.
- Updated Serious Adverse Events (SAEs) form. Main change is the SAE sending: SAEs have to be reported to the Corporate Vigilance Department, and not anymore to the clinical study manager. Also SAEs can be sent by e-mail and by fax.
- Addition of Alpha Bioresearch as CRO involved for Feasibility, Monitoring and Regulatory issues in Spain.
- Some minor typographic errors are corrected in the protocol.

Final version 465/1185

# 2. CHANGES DESCRIPTION

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| Sponsor's Representative: | Sponsor's Representative: |
| Gaëlle ALCARAZ INSTITUT DE RECHERCHE PIERRE FABRE - Centre de R&D Pierre Fabre - BP 13562 3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 65 92 E-mail:gaelle.alcaraz@pierre-fabre.com | Gaëlle ALCARAZ INSTITUT DE RECHERCHE PIERRE FABRE - Centre de R&D Pierre Fabre - BP 13562 3 avenue Hubert Curien 31035 TOULOUSE Cédex 1 Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 69 69 E-mail:gaelle.alcaraz@pierre-fabre.com |
| <b>Medical Director:</b> | Medical Director: |
| Richard ROCHE, MD | Richard ROCHE, MD |
| Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 65 92 E-mail: richard.roche@pierre-fabre.com | Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1 Phone: +33 5 34 50 69 69 E-mail: richard.roche@pierre-fabre.com |
| CONTRACT RESEARCH | CONTRACT RESEARCH |
| ORGANISATIONS | ORGANISATIONS |
| For Feasibility, Monitoring and Regulatory issues: Pharmaceutical Service Network (PSN) Rufino Gonzalez 28 037 Madrid - SPAIN Phone: +34 91 375 6930 - Fax: +34 91 375 6931 E-mail: www.psnglobal.org | For Feasibility, Monitoring and Regulatory issues: Pharmaceutical Service Network (PSN) Rufino Gonzalez 28 037 Madrid - SPAIN Phone: +34 91 375 6930 - Fax: +34 91 375 6931 E-mail: www.psnglobal.org For Feasibility, Monitoring and Regulatory issues (in Spain): Alpha Bioresearch Paseo de la Castellana, 163 - 2° Izquierda 28 046 Madrid - SPAIN Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com |
| SYNOPSIS | SYNOPSIS |
| Planned Study Period: | Planned Study Period: |
| January 2013 – April 2014 | January 2013 – <b>January 2015</b> |
| Diagnosis and Criteria for Inclusion: | Diagnosis and Criteria for Inclusion: |
| Inclusion Criteria: 2. Patients with persistent AF between 7 days and 6 months duration for whom electrical cardioversion is | Inclusion Criteria: 2. Patients with <b>current episode</b> of persistent AF between 7 days and 6 months duration for whom electrical |

Final version 466/1185

warranted.

- History of first documented persistent AF less than 1 year.
- 12. For male with a child-bearing potential partner (In Italy only):
- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study

#### Non-Inclusion Criteria:

Criteria related to pathologies:

 History of first documented episode of persistent AF more than 1 year

[...]

Hyperkalemia or hypokalemia (K>5.5 mEq/L or K < 3.5 mEq/L) at selection</li>

Criteria related to treatments:

ſ...

- Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion

## **Evaluation Criteria:**

Efficacy evaluation variables:

Other:

Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))

#### Safety criteria:

Haematology: haematocrit, haemoglobin, RBC, WBC, differential count, platelets

#### STUDY FLOW-CHART

Please see flow-chart of previous version in appendix 1.

cardioversion is warranted

- 3. History of first documented persistent AF less than 3 years
- 12. For male with a child-bearing potential partner (In Italy only):
- absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
- use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study

Non-Inclusion Criteria:

Criteria related to pathologies:

 History of first documented episode of persistent AF more than 3 years

[...]

9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection

Criteria related to treatments:

[...]

12. Concomitant treatment with **ranolazine or** any antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calciumblockers

#### 13. Oral amiodarone:

13a Previous treatment with oral amiodarone within 4 months prior to inclusion

13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion

14. Previous treatment with intravenous amiodarone within **4 weeks** prior to inclusion

# **Evaluation Criteria:**

Efficacy evaluation variables:

Other:

• Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA (mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))

Safety criteria:

 Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, differential count, reticulocytes, platelets

### STUDY FLOW-CHART

Please see flow-chart of modified version in appendix 2.

Final version 467/1185

# 1. INTRODUCTION AND STUDY RATIONALE

### 1.2. Information on the test product

#### 1.2.3. Clinical data

#### Part A: Single dose

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 4 were observed in the placebo group (palpitation, dizziness in standing position, 2 symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position).

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

During the study, in case of AF recurrence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure

#### 4. STUDY DESIGN

### 4.1. Overall description

 Visit 4 (V4): W5 (D35 ± 2D): follow-up visit (removing of Holter ECG device and installation of the TTEM)

#### 4.2. Discussion of the study design

### 4.2.1. Choice of the study population

The study aim is to investigate the product effect in patients with:

Persistent AF history (less than one year) with a duration of the current episode from 7 days to 6 months

[...]

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or unstable ischemic coronaropathy (assessed by coronarography or cardiac stress test or effort test within 6 months before selection).

#### 5. STUDY POPULATION

# 5.1.Inclusion criteria

# 1. INTRODUCTION AND STUDY RATIONALE

#### 1.2. Information on the test product

#### 1.2.3. Clinical data

### Part A: Single dose

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, **3 TEAs** were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotensions without loss of consciousness) and 4 in the group of F373280 at the dosage of 16g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position).

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

During the study, in case of AF recurrence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical **symptoms for instance**, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure

# 4. STUDY DESIGN

### 4.1. Overall description

 Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)

#### 4.2. Discussion of the study design

# 4.2.1. Choice of the study population

The study aim is to investigate the product effect in patients with:

Persistent AF history (less than **three** years) with a duration of the current episode from 7 days to 6 months

[...]

For the successful rate of electrical cardioversion, patients should have a stable medical treatment of heart failure and should not have myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

#### 5. STUDY POPULATION

#### 5.1.Inclusion criteria

Final version 468/1185
Demographic Characteristics and Other Baseline Characteristics:

- 1. [...]
- Patient with persistent AF between 7 days and 6 months duration for whomelectrical cardioversion is warranted
- 3. History of first documented persistent AF less than 1 year

[...]

- 12 For male with a child-bearing potential partner (In Italy only):
- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or

-use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to a month after the end of the study

#### 5.2. Non Inclusion criteria

Criteria related to pathologies:

1. History of first documented episode of persistent AF more than 1 year,

[...]

Hyperkalemia or hypokalemia (K > 5.5 mEq/L or K < 3.5 mEq/L) at selection</li>

Criteria related to treatments:

- Concomitant treatment with any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers
- 13. Previous treatment with oral amiodarone within 12 months prior to inclusion
- 14. Previous treatment with intravenous amiodarone within 6 months prior to inclusion

### 5.6. Withdrawal criteria

- Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV (i.e. unsuccessful ECV) will be considered to have finished follow-up.
- An occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and uncomfortable clinical symptoms.

Demographic Characteristics and Other Baseline Characteristics:

- 1. [...]
- 2. Patient with **current episode of** persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted
- 3. History of first documented persistent AF less than 3 years

[...]

- 12.For male with a child-bearing potential partner (In Italy only):
- absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
- -use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study

#### 5.2. Non Inclusion criteria

Criteria related to pathologies:

1. History of first documented episode of persistent AF more than 3 years,

[...]

9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection

Criteria related to treatments:

 Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calciumblockers

#### 13. Oral amiodarone:

13a Previous treatment with oral amiodarone within 4 months prior to inclusion

13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion

14. Previous treatment with intravenous amiodarone within **4 weeks** prior to inclusion

#### 5.6. Withdrawal criteria

- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early relapse within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance.

Final version 469/1185

## 6. STUDY TREATMENT

#### 6.3. Distribution to centre and storage

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's file.

## 6.4. Allocation of treatments and dispensation to patient

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Calls the vocal server
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the vocal server.

[...]

At visit 5, the Investigator will contact again the IVRS/IWRS to obtain for visit 6 the treatment number for the last 12-week period of treatment according to the same process as described above.

#### 6. STUDY TREATMENT

#### 6.3. Distribution to centre and storage

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file.

# 6.4. Allocation of treatments and dispensation to patient

Practically, once the patient's eligibility is confirmed, at selection visit:

- The Investigator:
  - Contacts the IVRS/IWRS
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

[...]

At visit 6, the Investigator will contact again the IVRS/IWRS to **obtain** the treatment number for the last 12-week period of treatment according to the same process as described above.

#### 7. CONCOMITANT TREATMENTS

#### 7.2. Prohibited treatments

 $[\ldots]$ 

#### 7. CONCOMITANT TREATMENTS

#### 7.2. Prohibited treatments

[...]

- Ranolazine

#### 8. EVALUATION CRITERIA

#### 8.1.2.5. Evolution of echocardiographic parameters

8.1.2.5.1. Definition

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%),Left ventricular volume (mL), Left ventricular volume/BSA(mL/m², Left ventricular end diastolic diameter (mm) Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL),

#### 8. EVALUATION CRITERIA

#### 8.1.2.5. Evolution of echocardiographic parameters

8.1.2.5.1. Definition

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), LVEF (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA (mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL).

## 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week -4 to Week -1)

• The patient will enter the selection period in which anticoagulant (anti-vitamin K) will be adjusted to achieve an

## 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week -4 to Week -1)

• The patient will enter the selection period in which anticoagulant (AVK) will be adjusted to achieve an

Final version 470/1185

International Normalized Ratio (INR) of 2 to 3 before electrical cardioversion.

International Normalized Ratio of 2 to 3 before ECV.

Visit 4 (Week 5: D35  $\pm$  2 days)

Visit 4 (Week 5: D35 -2/+7 days)

Body weight (body weight measured at V3 to be used)

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

In addition:

- at visit 5, the investigator will contact the IVRS/IWRS to obtain another treatment unit to be dispensed at visit 6 for the last 12-week period.

- at visit 6, an echocardiography will be performed, an haematology examination will be done and the red blood cell concentration of DHA will be measured.

In addition:

- at visit 6:

- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

#### 10.2.2. Reporting of SAE

All serious adverse events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") (see appendix 17.2) with all the available information about the event, to the Sponsor's representative:

Gaëlle ALCARAZ INSTITUT DE RECHERCHE PIERRE FABRE, Centre de R&D Pierre Fabre – BP 13562 3 Avenue Hubert Curien

31035 TOULOUSE Cedex 1 Phone: +33 5 35 50 62 16 Fax: +33 5 34 50 65 92

Email: gaelle.alcaraz@pierre-fabre.com

In case of non-inclusion the reporting period ends when the non-inclusion is documented.

#### 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

#### HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:
+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

### 13. STATISTICAL ANALYSIS

#### 13.4. Data sets analysed

The following 2 data sets will be analysed (as defined by the Validation Committee): [...]

• The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy

#### 13. STATISTICAL ANALYSIS

## 13.4. Data sets analysed

The following 3 data sets will be analysed (as defined by the Validation Committee): [...]

• The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy

Final version 471/1185

criteria available and without any major protocol deviation or other source of bias for primary criteria analyses.

criteria available and without any major protocol deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

## 16. REFERENCES

### 16. REFERENCES

[1] F373280 INVESTIGATOR'S BROCHURE, version January 2013

[1] F373280 INVESTIGATOR'S BROCHURE, version **October** 2013

Final version 472/1185

## **APPENDIX 1**

## STUDY FLOW-CHART FROM PROTOCOL VERSION 4

Final version 473/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 +/-2 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | х | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic characteristics | х | | | | | | | | |
| Medico-surgical history | х | | | | | | | | |
| Concomitant disease | х | | | | | | | | |
| Concomitant treatment | х | х | х | х | х | х | х | x | х |
| Habits | х | | | | | | | | |
| Global physical examination (body weight) | х | x | х | | x | х | х | x | х |
| Echocardiography | х | х | | х | | х | | | х |
| Eligibility criteria check | х | х | | | | | | | |
| Blood pressure, heart rate | х | х | х | х | х | х | х | x | х |
| 12-Lead ECG Recording | х | х | х | | х | х | х | x | х |
| INR | <b>─</b> | | (2) | | х | х | х | x | х |
| аРТТ, ТСТ | х | x | х | | x | x | х | x | х |
| Biochemistry | х | | | | | | | | х |
| Hematology | х | | X | | | x | | | х |
| Urinary pregnancy test | | х | | | | | | | х |
| Red Blood Cell concentrations of DHA | | х | х | | | х | | | х |
| Treatment allocation | | х | | | | х | | | |
| IVRS | х | х | | | х | х | | | |
| ECV (3) | | | х | | | | | | |
| Drug administration | | <b>+</b> | | | | | | | <b>→</b> |
| Adverse events recording | | х | х | х | х | х | х | x | х |
| Holter ECG | (4) | | - | (5) | | | | 4 | |
| TTEM (6) | | | t or hospitalization a | | | | | 4 | $\rightarrow$ |

Final version 474/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(5) 7-</sup>day Holter ECG

<sup>10</sup> TTEM everyday from week 6 to week 8. Then every 2 days from week 9 to week 24. In case of AF symptoms. In case of AF recurrence for at least 10 minutes and the patient does not stop the study treatment then TTEM every 4 weeks

## **APPENDIX 2**

STUDY FLOW-CHART FROM PROTOCOL VERSION 5 (modified version)

Final version 475/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | X | X | Х | X | Х | Х | Х | Х | X |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | X | X | X | | x | Х | x | x | X |
| Echocardiography | Х | X | | X | | Х | | | X |
| Eligibility criteria check | X | X | | | | | | | |
| Blood pressure, heart rate | X | X | X | X | x | Х | x | x | X |
| 12-Lead ECG Recording | X | X | X | | Х | Х | Х | Х | X |
| INR | <b>+</b> | | (2) | | Х | Х | Х | Х | X |
| aPTT, TCT | X | X | Х | | Х | Х | Х | Х | X |
| Biochemistry | Х | | | | | | | | Х |
| Hematology | Х | | Х | | | Х | | | Х |
| Urinary pregnancy test | | X | | | | | | | X |
| Red Blood Cell concentrations of DHA | | X | X | | | Х | | | X |
| Treatment allocation | | X | | | | Х | | | |
| IVRS/IWRS | X | X | | | | Χ | | | |
| ECV (3) | | | x | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | x | х | x | Х | Х | Х | Х | Х |
| Holter ECG | <b>←</b> (4) | | <b>+</b> | (5) | | | | | |
| TTEM (6) | | | | + | | | | | |

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)

Final version 476/1185

<sup>(2)</sup> In case of AVK introduction: INR 2 to 3 times a week, then weekly untill the ECV, then every 4 weeks after ECV.

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) TTEM: everyday from week 6 to week 8;. then every 2 days from week 9 to week 24; at any time in case of AF symptoms.

In case of AF recurrence for at least 10 minutes and if the patient does not stop the study treatment then TTEM once a week

F 373280 CA 2 01

Final version 477/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

## CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE - Centre de

R&D Pierre Fabre - BP 13562 3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 69 69

E-mail:gaelle.alcaraz@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

**Associate Professor of Cardiology** 

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>; nodari@med.unibs.it

#### **Version 5 –23OCT2013**

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 478/1185

## **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

## **Clinical Study Manager (Monitor)**

Gaëlle ALCARAZ

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 62 16 Fax: +33 5 34 50 69 69

E-mail: gaelle.alcaraz@pierre-

fabre.com

## **Medical Director**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 69 69

E-mail: richard.roche@pierre-

fabre.com

Final version 479/1185

## CONTRACT RESEARCH ORGANISATIONS

## For Feasibility, Monitoring and Regulatory issues:

## Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

## For Feasibility, Monitoring and Regulatory issues (in Spain):

## Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

## For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6, Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

## For Centralised Reading of Holder ECG and TTEM and equipment supply:

## **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage:

## Agrocampus Ouest

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

#### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER – FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 480/1185

## For refund of patients expenses linked to the study (in France):

**CLINACT** 

6-10 rue TROYON 92310 SEVRES – FRANCE

Phone: +33 1 46 90 27 27 - Fax: +33 1 46 23 01 56

Email: sebastien.beaumont@clinact.com

Final version 481/1185

# Protocol F 373280 CA 2 01 APPROVAL FORM

## Protocol Version 5 - 23 OCT 2013

Sponsor's Representative:

Medical Director: Richard ROCHE, MD Date: L9/10/2013 Signature:

Study Coordinating Investigator:

Savina NODARI, MD

Date:

Signature:

30/20/2013

## Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

## **Protocol Version 5 – 23 OCT 2013**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 483/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

**Protocol Version 5 – 23 OCT 2013** 

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 23 October 2013 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

\* To be adapted

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| 1000 | adapted |
|------|---------|

| Date: | Signature |
|-------|-----------|
|-------|-----------|

Final version 484/1185

## TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|-------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 24 |
| 1.2.1. | Chemical and pharmaceutical characteristics. | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1.2 | 7 | |
| 1.2.2. | | |
| 1.2.2. | $\mathcal{C}$ | |
| 1.2.2.3 | | |
| 1.2.2.4 | C, 1 | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 33 |
| 2.1. | PRIMARY OBJECTIVE | 33 |
| 2.2. | SECONDARY OBJECTIVES | |
| <b>3.</b> 1 | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 35 |
| 4.1. | OVERALL DESCRIPTION | 35 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | 38 |
| 5.2. | NON INCLUSION CRITERIA | 39 |
| 5.3. | NUMBER OF PATIENTS | 40 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 41 |
| 5.6. | WITHDRAWAL CRITERIA | 41 |
| 5.7. | REPLACEMENT OF PATIENTS | 42 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 42 |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | 42 |

| 6. | STUDY TREATMENT | 43 |
|---|---|---|
| 5.2. | PACKAGING AND LABELLING | 43 |
| 5.2.1. | Packaging | 44 |
| 5.2.2. | | |
| 5.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 5.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 5.5. | DRUG ADMINISTRATION | 47 |
| 5.5.1. | Duration of Treatment | 47 |
| 5.5.2. | | |
| 5.5.3. | Route and Conditions of Administration | 47 |
| 5.7. | RECALL OF INVESTIGATIONAL PRODUCTS | 48 |
| 7. | CONCOMITANT TREATMENTS | 48 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | 49 |
| 7.3. | AUTHORISED TREATMENTS | |
| 8. | EVALUATION CRITERIA | |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | | |
| 3.1.1. | | |
| 3.1.1. | | |
| 8.1.1. | | |
| 8.1.2. | | |
| 8.1.2.<br>8.1.2. | | |
| 3.1.2.<br>3.1.2. | | |
| 3.1.2.<br>3.1.2. | | |
| 8.1.2. | | |
| 3.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF | |
| | DHA | 54 |
| 3.2.1. | Definition | 54 |
| 8.2.2. | 1 | |
| 3.2.2. | | |
| 3.2.2. | $oldsymbol{arepsilon}$ | |
| 3.2.3. | | |
| 3.3. | SAFETY ASSESSMENT | |
| 3.3.1. | | |
| 3.3.2. | Laboratory Investigations | 56 |

| 8.3.2.1. Schedule | 56 |
|----------------------------------------------------------------|----------|
| 8.3.2.2. Technical Procedures and Parameters | 56 |
| 8.3.3. Global Physical Examination | 57 |
| 8.3.4. Vital Signs | 57 |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.3.7. Concomitant Treatments | |
| 8.4. COMPLIANCE | 59 |
| 9. STUDY PROCEDURES | 59 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 65 |
| 10.1. ADVERSE EVENTS | 65 |
| 10.1.1. Definition of Adverse Events | 65 |
| 10.1.2. Grading of Adverse Events | 66 |
| 10.1.3. Reporting of Adverse Events | 66 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 66 |
| 10.2.1. Definition | 66 |
| 10.2.2. Reporting of SAE | |
| 10.2.3. Follow-up of SAE | 67 |
| 10.2.4. SAE Occurring After the Study | 68 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 68 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 68 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | |
| 11. DATA COLLECTION AND STUDY MONITORING | 69 |
| 11.1. DATA COLLECTION | 69 |
| 11.1.1 Casa Panort Form | 60 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | |
| 11.2.1. Monitoring visits | |
| 11.2.1.1 Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | |
| 12. DATA MANAGEMENT | 73 |
| 12.1. DATA ENTRY | |
| 12.2 DATA CLEANING | 73<br>73 |

| 12.3. DATA CODING | 73 |
|---|---|
| 12.4. DATA STORAGE | 74 |
| 12.5. DATABASE LOCK | 74 |
| 13. STATISTICAL ANALYSIS | 74 |
| 13.1. GENERAL CONSIDERATIONS | 74 |
| 13.2. SAMPLE SIZE | 75 |
| 13.4. DATA SETS ANALYSED | 75 |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | 76 |
| 13.5.1. Dropouts | 76 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 13.7. EFFICACY ANALYSIS | 77 |
| 13.7.1. Primary Criterion | |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | |
| 14. GENERAL ETHICAL CONSIDERATIONS | 84 |
| 14.1. ETHICAL CONDITIONS | |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 85 |
| 14.4. PERSONAL DATA PROTECTION | 85 |

| 14.5. | INSURANCE POLICY | 86 |
|---|---|---|
| 15. | ADMINISTRATIVE PROCEDURES | 86 |
| 15.2. | SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 86 |
| 15.3. | END OF THE STUDY | 87 |
| 15.3. | 1. Definition of the End of Study | 87 |
| 15.3.2 | | |
| | 2.1. Early Study Termination Decided by the Sponsor | |
| 15.3.2 | 2.2. Early Study Termination Decided by the Competent Authorities | 88 |
| 15.4. | AUDIT | 88 |
| 15.5. | INSPECTION | 88 |
| 15.6. | CONFIDENTIALITY | 88 |
| 15.7. | CLINICAL STUDY REPORT | 89 |
| 15.8. | STUDY RESULTS COMMUNICATION | 89 |
| 15.9. | STUDY RESULTS PUBLICATION | 89 |
| 16. | REFERENCES | 91 |
| 17. | APPENDICES | 94 |
| 17.1. | DECLARATION OF HELSINKI | 95 |
| 17.2. | SAE REPORT FORM | 99 |
| 17.3. | PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY | |
| | CLINICALLY SIGNIFICANT CHANGES AND VALUES | 103 |

## **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | International, multicentric, randomised, double-blind, placebo controlled study Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing.[1] Moreover, the effectiveness of PolyUnsaturated Fatty Acid (PUFA) has been proven in the following conditions: — prevention of AF recurrence in patients with persistent AF, in co-administration with amiodarone (add on therapy) [2] — Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in |
| Planned Study Period: | patients with persistent atrial fibrillation and chronic heart failure. January 2013 – January 2015 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>Salety and tolerability of F373280</li> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> <li>Treatment duration: 24 weeks</li> </ul> |
| Study Schedule | 9 visits will be scheduled: - V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit) - V2/D1: Inclusion visit (start of treatment) - V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to |

Final version 490/1185

| | clinical practice of the centre) (installation of the Holter device) |
|---|---|
| | - V4/W5 (D35± 2 days): follow-up visit (removing of the Holter device and installation of |
| | the TTEM) |
| | - V5/W8 (D56± 7 days): follow-up visit |
| | - V6/W12 (D84 ± 7 days): follow-up visit |
| | - V7/W16 (D112 $\pm$ 7 days): follow-up visit |
| | - V8/W20 (D140 $\pm$ 7 days): follow-up visit |
| | - V9/W24 (D168 $\pm$ 7 days): final study visit |
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | Inclusion Criteria: |

Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted
- 3. History of first documented persistent AF less than 3 years.
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patients treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

#### • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment
- documented as surgically sterilized

#### • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 3 years
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6

Final version 491/1185

| | <ol> <li>months</li> <li>Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)</li> <li>NYHA class III or IV heart failure at selection or at inclusion</li> <li>Thyroid disease uncontrolled by treatment: TSH ± T4L ± T3L to be checked in case of treatment for thyroid disease</li> <li>Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress tests (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection</li> <li>Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate &lt; 30 mL/min) at selection</li> <li>Bradycardia (HR ≤ 50 bpm)</li> <li>Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection</li> <li>Cardiac surgery within 3 months before selection or planned during the study duration</li> <li>Criteria related to treatments:</li> <li>Previously ineffective pharmacological or electrical cardioversion</li> <li>Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers</li> <li>Oral amiodarone: <ul> <li>13a Previous treatment with oral amiodarone within 4 months prior to inclusion</li> <li>13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion</li> </ul> </li> <li>Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion</li> <li>Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months</li> <li>Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months</li> <li>Dietary supplement with ω 3 or ω 6 according to investigator's judgement</li> <li>Having undergone any form of ablation therapy for AF</li> <li>Patient trea</li></ol> |
|---|---|
| | <ul> <li>Other criteria:</li> <li>20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion</li> <li>21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection</li> <li>22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints</li> <li>23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator</li> <li>24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship</li> <li>25. Breastfeeding female patient</li> </ul> |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV) ECV will be performed in patients without dyskalemia If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280 Soft Capsules Arm with 1g of F273280 |
| Dose: Mode of Administration: | Arm with 1g of F373280 Oral, one capsule each evening with dinner. |
| | [ Oral one cancille each evening with dinner |

Final version 492/1185

| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
|---|---|
| Reference Therapy | Placebo soft capsules |
| Mode of Administration: | Placebo will be administered in the same conditions as the tested product. Oral, one capsule each evening with dinner |
| | , , |
| Evaluation Criteria: | Efficacy evaluation variables: Primary evaluation variable: Time to first Atrial Fibrillation recurrence defined by the first episode of AF lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit). Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24. For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5). Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM. All ECG traces will be evaluated by a Central Reading Laboratory. Secondary evaluation variables: During the 7-day continuous ECG monitoring, Numbers of AF episodes Duration of AF episodes Uning the whole study: Number of recurrence of symptomatic AF episodes EHRA score Hospitalization for cardiovascular events Hospitalization for thromboembolic stroke All causes of hospitalization Cardioversion: Assessment of spontaneous cardioversion Assessment of spontaneous cardioversion Assessment of patients needing an other cardioversion after the initial ECV Other: Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial |
| | <ul> <li>diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA(mL/m²), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))</li> <li>Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).</li> </ul> |
| | <ul> <li>Safety criteria: <ul> <li>Adverse events (observed and / or spontaneously reported)</li> <li>Vital signs (Blood pressure (supine and standing), heart rate</li> <li>Physical examination (body weight)</li> <li>Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized)</li> <li>Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets</li> <li>Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)</li> </ul> </li> </ul> |

Final version 493/1185

| | - <b>Coagulation parameters:</b> Activated partial thromboplastin time (aPTT), thrombin cle time (TCT), INR <i>(local laboratory)</i> , Prothrombine Time <i>(PT)</i> |
|---|---|
| Statistical Methods: | Sample Size: Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. Primary Efficacy Analysis The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model. Secondary Analyses All secondary efficacy criteria will be described and compared using appropriate tests on the FAS. Safety Analyses Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment). |

Final version 494/1185

## STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | X | Х | Х | Х | Х | Х | Х | Х |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | X | X | X | | Х | Х | Х | Х | Х |
| Echocardiography | X | X | | X | | х | | | Х |
| Eligibility criteria check | X | X | | | | | | | |
| Blood pressure, heart rate | X | X | X | X | Х | Х | X | X | X |
| 12-Lead ECG Recording | X | X | X | | x | x | X | X | X |
| INR | <b>\</b> | | (2) | | Х | Х | Х | Х | X |
| aPTT, TCT | Х | X | X | | Х | Х | Х | Х | X |
| Biochemistry | Х | | | | | | | | X |
| Hematology | Х | | X | | | Х | | | X |
| Urinary pregnancy test | | X | | | | | | | X |
| Red Blood Cell concentrations of DHA | | X | X | | | x | | | X |
| Treatment allocation | | X | | | | X | | | |
| IVRS/IWRS | Х | X | | | | Х | | | |
| ECV (3) | | | X | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | x | Х | x | Х | Х | Х | Х | Х |
| Holter ECG | <b>←</b> (4) | | <b>←</b> | (5) | | | | | |
| TTEM (6) | | | | + | | | | | <b>—</b> |

Final version 495/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of AVK introduction: INR 2 to 3 times a week, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) TTEM: everyday from week 6 to week 8;. then every 2 days from week 9 to week 24; at any time in case of AF symptoms. In case of AF recurrence for at least 10 minutes and if the patient does not stop the study treatment, then TTEM once a week

## LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK : Anti-vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

Final version 496/1185

HDL : High density lipoprotein

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 497/1185

## 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

Final version 498/1185

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of

Final version 499/1185

functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

## 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

Final version 500/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

## 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

## 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

Final version 501/1185

#### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus 637  $\pm$  196 sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and 79  $\pm$  51 sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of

Final version 502/1185

DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases

plasma level of DHA, it could be estimated that the compound may exert a similar protective

effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 503/1185

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

Final version 504/1185
## Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 505/1185

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic heart failure.

#### 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common (>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000), not known (cannot be estimated from the available data).

Final version 506/1185

- The reported adverse events are:

• Infection and infestations:

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

• Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Final version 507/1185

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

Final version 508/1185

## 2. STUDY OBJECTIVES

## 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

#### 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the

Final version 509/1185

included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (anti-vitamin K), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with anti-vitamin K (AVK) for at least 3 weeks before ECV
- ECV in patients with stabilized INR (i.e. values between 2 and 3;sp to ) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV). Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Final version 510/1185

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1 g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit
- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

Final version 511/1185

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Persistent AF history (less than three years) with a duration of the current episode from 7 days to 6 months.
- a moderately abnormal systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- a Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

Final version 512/1185

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmic class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before ECV. According to guidelines for the management of AF [6], AVK should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Final version 513/1185

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

## 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/mL and 60 to 90 mg/mL, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports an once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

# 5.1. INCLUSION CRITERIA

# Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whomelectrical cardioversion is warranted

Final version 514/1185

- 3. History of first documented persistent AF less than 3 years
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

# • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- documented as surgically sterilized

## • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

## Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

## 5.2. NON INCLUSION CRITERIA

# Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 3 years,
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),

Final version 515/1185

- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Oral amiodarone:
  - 13a Previous treatment with oral amiodarone within 4 months prior to inclusion
  - 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion
- 14. Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection.
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship.
- 25. Breastfeeding female patient.

#### 5.3. NUMBER OF PATIENTS

76 x 2 patients (taking into account 15 % of non evaluable patients).

Final version 516/1185

#### 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
- have the patient's decision written on the consent form
- obtain the reason(s) for withdrawal and report it/them in the case report form
- evaluate the patient's clinical condition
- if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event
  occurs and is considered by the Investigator liable to threaten the health of the patient. The
  monitor will be informed by phone or fax and a letter or report explaining the withdrawal
  will be forwarded to the monitor as soon as possible.

Final version 517/1185

- Erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion/non inclusion criteria will immediately be withdrawn and an appropriate treatment will be given by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with AVK for at least 3 weeks before ECV.
- Patients who will not have a stabilized INR between 2 and 3 on at least 3 consecutive weekly tests.
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 weeks for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early relapse within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence that would require, at the investigator's judgement, a
  cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or
  uncomfortable clinical symptoms for instance.

## 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

# 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the

Final version 518/1185

Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.

- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

• F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

Final version 519/1185

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number, and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date

Final version 520/1185

- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

#### 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

Final version 521/1185

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once patient's eligibility is confirmed at selection visit (V1):

- The Investigator:
  - Contacts the IVRS/IWRS
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment according to the same process as described above.

Final version 522/1185

#### 6.5. DRUG ADMINISTRATION

## **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

Final version 523/1185

## 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

Final version 524/1185

## 7.1. ANTI-VITAMIN K TREATMENT

AVK should be given for at least 3 weeks before ECV and continued for the whole study duration. The AVK used will be left to the decision of the each Investigator according to his/her local practice.

## 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
- Class IA: Disopyramide, Procainamide, Quinidine
- Class IB: Lidocaine, Mexiletine
- Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any anticoagulant treatment other than AVK: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

Final version 525/1185

# 8. EVALUATION CRITERIA

## 8.1. PRIMARY EFFICACY CRITERION

## **8.1.1.** Time to the first Atrial Fibrillation Recurrence

# 8.1.1.1. Definition

Time to first AF recurrence is defined by the first episode of AF (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from visit 4 (week 5) to visit 5 (week 8). Then every two days from visit 5 (week 8) to visit 9 (week 24 – End of study).

Moreover, if patient experiences AF symptoms during this TTEM period, it should be documented using the TTEM.

Final version 526/1185

In case of AF recurrence and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

## 8.1.2. Secondary Efficacy Criteria

## 8.1.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

# 8.1.2.1.1. *Definition*

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

# 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

#### 8.1.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

Final version 527/1185

# 8.1.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

## 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episode.

## 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

## 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

# 8.1.2.3. Clinical parameters evaluation

#### 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

Final version 528/1185

## 8.1.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

#### 8.1.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during all the study period.

# 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

# 8.1.2.3.3. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

## 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)
  - Number of patients needing another cardioversion after initial ECV

# 8.1.2.5. Evolution of echocardiographic parameters

# 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), LVEF (%), Left ventricular end diastolic volume/BSA (mL/m<sup>2</sup>), Left ventricular end systolic volume/BSA (mL/m<sup>2</sup>), Left

Final version 529/1185

ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL).

#### 8.1.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.2.2. Blood samples

# 8.2.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

Final version 530/1185

# 8.2.2.2. Technical handling

Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

## **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as µg/g for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

## 8.3. SAFETY ASSESSMENT

#### 8.3.1. Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the

Final version 531/1185

Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

# 8.3.2. Laboratory Investigations

#### 8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 mL.

## 8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: hematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and absolute), reticulocytes, platelets.

Chemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L]

in women:

Final version 532/1185

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

#### 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

Final version 533/1185

# 8.3.5. Electrocardiogram (ECG)

## 8.3.5.1. *Schedule*

An ECG will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

#### 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

• 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

## **8.3.6.** Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV
- INR every 4 weeks after ECV

Final version 534/1185

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by AVK should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial, can be found in section 7.

## 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit, the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

## 9. STUDY PROCEDURES

## Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history

Final version 535/1185

- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory. The Central Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

Final version 536/1185

The patient will receive from the investigational centre the study card to be kept for the duration

of the study.

**Visit 2 - Inclusion Visit (Day 1)** 

If the patient's behaviour during the selection period and/or the result of complementary

examinations particularly the confirmation of the presence of persistent AF by the Central

Reading Laboratory during this period, the INR and laboratory tests, are compatible with the

inclusion criteria, the patient will be assessed for the following:

Adverse events

• Concomitant treatments (authorised, disallowed)

• Laboratory examination: red blood cell concentrations of DHA and coagulation

parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time

(aPTT), Thrombin Clotting Time (TCT)

Global Physical examination/bodyweight

Vital signs

• Echocardiography using a two-dimensional echocardiography

• 12-lead ECG

• Urine pregnancy test for women of child bearing potential

If the results of the above assessments are compatible with the inclusion criteria, the patient will

be included and allocated a treatment number using the IVRS/IWRS.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to

paragraph 8.3.6) in order to ensure that the INR is stable (between 2 to 3 before electrical

cardioversion).

At the end of the visit, the Investigator will organise the appointment for the next visit and will

give the treatment for the next 4-week period.

Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Final version 537/1185

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE performed in the same day (and before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

Final version 538/1185

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

## Visit 4 (Week 5: D35 -2/+7 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Body weight (body weight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms, additional transmissions may be performed.

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) – Visit 7 (Week 16: D112  $\pm$  7 days) – Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of

Final version 539/1185

discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT

should be stopped.

• Global Physical examination/bodyweight

Vital signs

• 12-lead ECG

The cardiac monitoring will be continued using a TTEM device. The device will be given

to the patient who will be requested to perform daily transmission from week 6 to week 8,

then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms, additional

transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused

capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give

the treatment to be taken during the next 4-week treatment period.

In addition:

- at visit 6:

• the investigator will contact the IVRS/IWRS to obtain the treatment unit number to

be dispensed at visit 6 for the last 12-week period.

• an echocardiography will be performed, an haematology examination will be done

and the RBC concentration of DHA will be measured.

End-of-Study Visit - Visit 9 (Week 24: D168  $\pm$  7 days)

Patient will be assessed for the following:

Adverse events

• Concomitant treatments (authorised, disallowed)

Final version 540/1185
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused soft capsules.

# 10. ADVERSE EVENTS: DEFINITION AND REPORTING

#### 10.1. ADVERSE EVENTS

#### **10.1.1.** Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

Final version 541/1185

# **10.1.2.** Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

# **10.1.3.** Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

# 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

Final version 542/1185

\* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:

- planned (as per protocol) medical/surgical procedure
- preparation for routine health assessment/procedure (e.g. routine colonoscopy)
- planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
- administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

# 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

## HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

#### 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

Final version 543/1185

# **10.2.4. SAE Occurring After the Study**

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

## 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

#### 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Final version 544/1185

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

Final version 545/1185

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

#### 11.2. STUDY MONITORING

# 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

Final version 546/1185

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
- has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

#### 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

Final version 547/1185

# 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

# 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

Final version 548/1185

#### 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

Final version 549/1185

The Sponsor Clinical Development Physician will validate the coding.

#### 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

#### 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

Final version 550/1185

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

# 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

• The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.

Final version 551/1185

- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

## **13.5.1.** Dropouts

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

# 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

#### 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- <u>Quantitative parameters</u> will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Final version 552/1185

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

# 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

# 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

# 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

Final version 553/1185

# 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

# 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

## 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

Final version 554/1185

# 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs
- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

Final version 555/1185

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (for all patients).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

#### 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration

Final version 556/1185

assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)

Final version 557/1185

- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

Final version 558/1185

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

## 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

#### 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by the rapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

### 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated \_actual \_consumption}{Theoretical \_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Final version 559/1185

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

#### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

## 14. GENERAL ETHICAL CONSIDERATIONS

#### 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

# 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

Final version 560/1185

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi

Final version 561/1185

Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

# 15. ADMINISTRATIVE PROCEDURES

#### 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

# 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

Final version 562/1185

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not.
- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

# 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

# 15.3.2. Early Study Termination

#### 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety

Final version 563/1185

• Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

Final version 564/1185

#### 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

# 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

Final version 565/1185

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 566/1185

#### 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 567/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

# [14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 568/1185

# [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

#### [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

# [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

## [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

#### [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 569/1185

# 17. APPENDICES

Final version 570/1185

#### 17.1. DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 571/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 572/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 573/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 574/1185

# 17.2. SAE REPORT FORM

Final version 575/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE CORPORATE VIGILANCES DIVISION |
|---|
| TO BE TRANSMITTED TO THE CORPORATE VIGILANCES DIVISION BY E-MAIL WITHIN 24H TO HQ.pharmacovigilance@pierre-fabre.com OR BY FAX WITHIN 24H – Fax N°: 33 (0) 1.49.10.80.90 |
| Transmission date (ddmmyyyy) Country: |
| SAE N° |
| > SUBJECT CHARACTERISTICS |
| Birth date |
| Gender1=M, 2=F Height cm Weight ·kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: |
| ■ Pregnancy exposure Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE arget data |
| AE onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| • Date of first study treatment administration |
| • Date of last study treatment administration before the occurence of SAE |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 576/1185
| SAE N° | | | FIRST NOTIFICA | FOL | LOW-UP | N° |
|---|---|---|---|---|---|---|
| > CONCOMITANT MEDICATION SINCE TRIAL INITIATION and UP UNTIL THE OCCURRENCE OF THE SAE (EXCEPT THE TREATMENTS GIVEN FOR THE SAE) | | | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAK | EN FOLLOWIN | NG THE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage modification, specify: Modification Date:// | | | | | | |
| ☐ Temporarily | ☐ Temporarily discontinued Readministration date :// | | | | | |
| ☐ Withdrawn | | End date :/ | | | | |
| ☐ Not applical | ble | | | | | |

Transmission date

Final version 577/1185

| • The event led to: | | | | | | |
|---|---|---|---|---|---|---|
| ☐ Prescription | of corrective or sy | mptomatic treatments | : | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Discontinuat | ion of concomitan | t treatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, speci | fy: | | | | | |
| > OUTCOME | | | | | | |
| ☐ Not recovered/l | Not resolved | ☐ Recovering/R | esolving $\square$ | Recovered/Resolved | | |
| ☐ Recovered/Reso | olved with sequela | e 🖵 Fatal | □ U | nknown | | |
| In case of dea | ath, has an autopsy | been conducted? | □ Yes □ No | | | |
| > INVESTIGATOR ( | CAUSALITY AS | SESSMENT (investi | gator's assessment | to be done as soon as | possible) | |
| Study drug: | | Relate | ed to study protocol: | | | |
| □ Not Suspected □ Suspected □ Not Suspected □ Suspected | | | | | | |
| Comments: | | | | | | |

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

Final version 578/1185

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|---|---|---|---|---|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| TO THE TOTAL | Protein | g/1 | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | рН | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/1 | | N x (30/95) |

N = upper limit of normal range

Final version 579/1185

<sup>(

)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

# **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | Decrease of at least 2g/dl and value < 10 g/dl whatever the baseline value If missing baseline : value <10g/dl |
| NEUTRO | PHILS | $\bullet$ < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline:</li> <li>TB &gt; 1.5 N</li> <li>If abnormal baseline:</li> <li>TB &gt; 2 N</li> </ul> |

## N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 580/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg}$ and increase $\ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \leq 50$ mmHg and decrease $\geq 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| , G , | | , | ge from Baseline | to the | |
|---|---|---|---|---|---|
| Post-baseline Va | alue | | Minimum Post-b | paseline Value | |
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| ≥ 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | - | Classes for the Minimum Post-baseline Value for each parameter | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤50 | ≤90 | ≤ 50 | ≤50 |
| [120;140] | [80;90[ | <i>[50 ;75]</i> | [90 ;120] | [50;80[ | [50;75] |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | SBP < 90 or DBP < 50 |
| or DBP [90;100[ and SBP < 160 | 3B1 ≥ 90 01 DB1 ≥ 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

Table 5: Definition of orthostatic hypotension

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq$ 20 mmHg or DBP Decrease $\geq$ 10 mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 581/1185

16.1.1.6. Protocol and appendices (version 06: 02 December 2013)

Final version 582/1185

F 373280 CA 2 01

Final version 583/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

# CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE - Centre de

R&D Pierre Fabre - BP 13562 3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 69 69

E-mail:gaelle.alcaraz@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

**Associate Professor of Cardiology** 

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>; nodari@med.unibs.it

### Version 6-02DEC2013

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 584/1185

# **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

# **Clinical Study Manager (Monitor)**

Gaëlle ALCARAZ

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien

31035 TOULOUSE Cedex 1, FRANCE

Phone: +33 5 34 50 62 16 Fax: +33 5 34 50 69 69

E-mail: gaelle.alcaraz@pierre-

fabre.com

# **Medical Director**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 69 69

E-mail: richard.roche@pierre-

fabre.com

Final version 585/1185

## CONTRACT RESEARCH ORGANISATIONS

# For Feasibility, Monitoring and Regulatory issues:

# Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

# For Feasibility, Monitoring and Regulatory issues (in Spain):

# Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

## For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6, Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

# For Centralised Reading of Holder ECG and TTEM and equipment supply:

# **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

### For intra erythrocyte DHA dosage:

# Agrocampus Ouest

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER – FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 586/1185

# For refund of patients expenses linked to the study (in France):

**CLINACT** 

6-10 rue TROYON 92310 SEVRES – FRANCE

Phone: +33 1 46 90 27 27 - Fax: +33 1 46 23 01 56

Email: sebastien.beaumont@clinact.com

Final version 587/1185

# Protocol F 373280 CA 2 01

### APPROVAL FORM

Protocol Version 6-02 DEC 2013

Sponsor's Representative:

Medical Director: Richard ROCHE, MD Date: 02/12/2013 Signature:

Study Coordinating Investigator: Savina NODARI, MD

Date:

Signature:

# Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

# **Protocol Version 6 – 02 DEC 2013**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 589/1185

### Protocol F 373280 CA 2 01

### INVESTIGATOR SIGNATURE FORM

Protocol Version 6 – 02 DEC 2013

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 02 December 2013 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * To be adapted |
|-----------------|
|-----------------|

| Date: Si | ignature |
|----------|----------|
|----------|----------|

Final version 590/1185

# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|-------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 24 |
| 1.2.1. | Chemical and pharmaceutical characteristics. | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1.2 | 7 | |
| 1.2.2. | | |
| 1.2.2. | $\mathcal{C}$ | |
| 1.2.2.3 | | |
| 1.2.2.4 | C, 1 | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 33 |
| 2.1. | PRIMARY OBJECTIVE | 33 |
| 2.2. | SECONDARY OBJECTIVES | |
| <b>3.</b> 1 | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 35 |
| 4.1. | OVERALL DESCRIPTION | 35 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | 38 |
| 5.2. | NON INCLUSION CRITERIA | 39 |
| 5.3. | NUMBER OF PATIENTS | 40 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 41 |
| 5.6. | WITHDRAWAL CRITERIA | 41 |
| 5.7. | REPLACEMENT OF PATIENTS | 42 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 42 |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | 42 |

| 6. | STUDY TREATMENT | 43 |
|---|---|---|
| 6.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL | 42 |
| 6.2. | PRODUCTPACKAGING AND LABELLING | |
| 6.2.1.<br>6.2.2. | PackagingLabelling | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | |
| 6.5. | DRUG ADMINISTRATION | |
| 6.5.1. | Duration of Treatment | |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration | |
| 6.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 47 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| 7. ( | CONCOMITANT TREATMENTS | 48 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | |
| 7.3. | AUTHORISED TREATMENTS | |
| <b>8.</b> ] | EVALUATION CRITERIA | |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence | 50 |
| 8.1.1. | 1. Definition | 50 |
| 8.1.1.2 | | |
| 8.1.1.í<br>8.1.2. | | |
| 8.1.2.<br>8.1.2. | Secondary Efficacy Criteria | |
| 8.1.2. | | |
| 8.1.2. | 1 | |
| 8.1.2.4 | | |
| 8.1.2.: | | 53 |
| 8.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA | 5.1 |
| 8.2.1. | Definition | |
| 8.2.1.<br>8.2.2. | Blood samples | |
| 8.2.2. | | |
| 8.2.2.2 | 2. Technical handling | 55 |
| 8.2.3. | DHA concentration measurement | |
| 8.3. | SAFETY ASSESSMENT | |
| 8.3.1. | Adverse Events | |
| 8.3.2. | Laboratory Investigations | 56 |

| 8.3.2.1. Schedule | 56 |
|----------------------------------------------------------------|----------|
| 8.3.2.2. Technical Procedures and Parameters | 56 |
| 8.3.3. Global Physical Examination | 57 |
| 8.3.4. Vital Signs | 57 |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.3.7. Concomitant Treatments | |
| 8.4. COMPLIANCE | 59 |
| 9. STUDY PROCEDURES | 59 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 65 |
| 10.1. ADVERSE EVENTS | 65 |
| 10.1.1. Definition of Adverse Events | 65 |
| 10.1.2. Grading of Adverse Events | 66 |
| 10.1.3. Reporting of Adverse Events | 66 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 66 |
| 10.2.1. Definition | 66 |
| 10.2.2. Reporting of SAE | |
| 10.2.3. Follow-up of SAE | 67 |
| 10.2.4. SAE Occurring After the Study | 68 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 68 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 68 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | |
| 11. DATA COLLECTION AND STUDY MONITORING | 69 |
| 11.1. DATA COLLECTION | 69 |
| 11.1.1 Casa Panort Form | 60 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | |
| 11.2.1. Monitoring visits | |
| 11.2.1.1 Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | |
| 12. DATA MANAGEMENT | 73 |
| 12.1. DATA ENTRY | |
| 12.2 DATA CLEANING | 73<br>73 |

| 12.3. DATA CODING | 73 |
|---|---|
| 12.4. DATA STORAGE | 74 |
| 12.5. DATABASE LOCK | 74 |
| 13. STATISTICAL ANALYSIS | 74 |
| 13.1. GENERAL CONSIDERATIONS | 74 |
| 13.2. SAMPLE SIZE | 75 |
| 13.4. DATA SETS ANALYSED | 75 |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | 76 |
| 13.5.1. Dropouts | 76 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 13.7. EFFICACY ANALYSIS | 77 |
| 13.7.1. Primary Criterion | |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2.1 Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 84 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 84 |
| 14.1. ETHICAL CONDITIONS | 84 |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 84 |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 85 |
| 14.4. PERSONAL DATA PROTECTION | 85 |

| 14.5. INSURANCE POLICY | 86 |
|---|---|
| 15. ADMINISTRATIVE PROCEDURES | 86 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 86 |
| 15.3. END OF THE STUDY | 87 |
| 15.3.1. Definition of the End of Study | 87 |
| 15.3.2. Early Study Termination | |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | 88 |
| 15.4. AUDIT | 88 |
| 15.5. INSPECTION | 88 |
| 15.6. CONFIDENTIALITY | 88 |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 89 |
| 15.9. STUDY RESULTS PUBLICATION | 89 |
| 16. REFERENCES | 91 |
| 17. APPENDICES | 94 |
| 17.1. DECLARATION OF HELSINKI | 95 |
| 17.2. SAE REPORT FORM | 99 |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | |

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | International, multicentric, randomised, double-blind, placebo controlled study Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing.[1] Moreover, the effectiveness of PolyUnsaturated Fatty Acid (PUFA) has been proven in the following conditions: - prevention of AF recurrence in patients with persistent AF, in co-administration with amiodarone (add on therapy) [2] - Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – January 2015 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>Safety and tolerability of F373280</li> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> </ul> |
| Study Schedule | <ul> <li>Treatment duration: 24 weeks</li> <li>9 visits will be scheduled:</li> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to</li> </ul> |

Final version 596/1185

| | clinical practice of the centre) (installation of the Holter device) - V4/ W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM) |
|---|---|
| | <ul> <li>V5/ W8 (D56± 7 days): follow-up visit</li> <li>V6/ W12 (D84 ± 7 days): follow-up visit</li> <li>V7/ W16 (D112 ± 7 days): follow-up visit</li> <li>V8/ W20 (D140 ± 7 days): follow-up visit</li> <li>V9/ W24 (D168 ± 7 days): final study visit</li> </ul> |
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | <ol> <li>Inclusion Criteria:</li> <li>Demographic Characteristics and Other Baseline Characteristics:</li> <li>Men or women aged more than 18 years (inclusive)</li> <li>Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted</li> <li>History of first documented persistent AF less than 3 years.</li> <li>History of ischemic or non ischemic heart failure</li> <li>NYHA class I or II chronic heart failure at selection and at inclusion</li> <li>Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion</li> <li>On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers</li> <li>Left atrial area ≤ 40 cm² at selection and at inclusion</li> <li>Patients treated or having to be treated by anti-vitamin K</li> </ol> |
| | <ul> <li>For female patient of child-bearing potential: <ul> <li>in all the countries except Italy: <ul> <li>use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment</li></ul></li></ul></li></ul> |

- the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

## Non-Inclusion Criteria:

Criteria related to pathologies:

- History of first documented episode of persistent AF more than 3 years
- More than two successful cardioversions (electrical or pharmacological) in the last 6

Final version 597/1185

| | <ul> <li>months</li> <li>Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)</li> <li>NYHA class III or IV heart failure at selection or at inclusion</li> <li>Thyroid disease uncontrolled by treatment: TSH ± T4L ± T3L to be checked in case of treatment for thyroid disease</li> <li>Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection</li> <li>Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate &lt; 30 mL/min) at selection</li> <li>Bradycardia (HR ≤ 50 bpm)</li> <li>Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection</li> <li>Cardiac surgery within 3 months before selection or planned during the study duration</li> <li>Criteria related to treatments:</li> <li>Previously ineffective pharmacological or electrical cardioversion</li> <li>Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers</li> <li>Oral amiodarone:</li> </ul> |
|---|---|
| | <ul> <li>13a Previous treatment with oral amiodarone within 4 months prior to inclusion 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion</li> <li>14. Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion</li> <li>15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months</li> <li>16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months</li> <li>17. Dietary supplement with ω 3 or ω 6 according to investigator's judgement</li> <li>18. Having undergone any form of ablation therapy for AF</li> <li>19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel</li> </ul> |
| | <ul> <li>Other criteria:</li> <li>20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion</li> <li>21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection</li> <li>22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints</li> <li>23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator</li> <li>24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship</li> <li>25. Breastfeeding female patient</li> </ul> |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV) ECV will be performed in patients without dyskalemia If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280<br>Soft Capsules<br>Arm with 1g of F373280 |
| Dose: Mode of Administration: | Oral, one capsule each evening with dinner. |

Final version 598/1185

| Duration of Treatment: | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
|---|---|
| Reference Therapy | Placebo soft capsules Placebo will be administrated in the same conditions as the tested product. |
| Mode of Administration: | Placebo will be administered in the same conditions as the tested product. Oral, one capsule each evening with dinner |
| | · · · · · · |
| Evaluation Criteria: | Efficacy evaluation variables: Primary evaluation variables: - Time to first Atrial Fibrillation recurrence defined by the first episode of AF lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit). Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24. For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5). Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM. All ECG traces will be evaluated by a Central Reading Laboratory. Secondary evaluation variables: During the 7-day continuous ECG monitoring, Numbers of AF episodes During the whole study: Number of AF episodes Clinical parameters: During the whole study: Number of recurrence of symptomatic AF episodes EHRA score Hospitalization for cardiovascular events Hospitalization for thromboembolic stroke All causes of hospitalization Cardioversion: Assessment of spontaneous cardioversion Assessment of successful cardioversion Number of patients needing an other cardioversion after the initial ECV Other: Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial |
| | <ul> <li>diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA(mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))</li> <li>Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).</li> </ul> |
| | <ul> <li>Safety criteria:</li> <li>Adverse events (observed and / or spontaneously reported)</li> <li>Vital signs (Blood pressure (supine and standing), heart rate</li> <li>Physical examination (body weight)</li> <li>Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized)</li> <li>Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets</li> <li>Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)</li> </ul> |

Final version 599/1185

| | - <b>Coagulation parameters:</b> Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR <i>(local laboratory)</i> , Prothrombine Time <i>(PT)</i> |
|---|---|
| Statistical Methods: | Sample Size: Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. Primary Efficacy Analysis The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model. Secondary Analyses All secondary efficacy criteria will be described and compared using appropriate tests on the FAS. Safety Analyses Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment). |

Final version 600/1185

# STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | х | X | х | | X | X | X | Х | X |
| Echocardiography | Х | Х | | Х | | Х | | | Х |
| Eligibility criteria check | Х | X | | | | | | | |
| Blood pressure, heart rate | X | X | Х | X | X | Х | X | x | X |
| 12-Lead ECG Recording | Х | X | Х | | Х | Х | Х | Х | Х |
| INR | ← | | (2) | | Х | Х | Х | Х | X |
| aPTT, TCT | Х | Х | Х | | Х | Х | Х | Х | Х |
| Biochemistry | Х | | | | | | | | X |
| Hematology | Х | | Х | | | Х | | | Х |
| Urinary pregnancy test | | Х | | | | | | | X |
| Red Blood Cell concentrations of DHA | | Х | Х | | | X | | | X |
| Treatment allocation | | X | | | | Х | | | |
| IVRS/IWRS | Х | Х | | | | X | | | |
| ECV (3) | | | x | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | х | Х | X | Х | Х | Х | Х | Х |
| Holter ECG | <b>←</b> (4) | | <b>+</b> | (5) | | | | | |
| TTEM (6) | | | | <b>—</b> | <b>—</b> | | | | <del></del> |

Final version 601/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of AVK introduction: INR 2 to 3 times a week, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) TTEM: everyday from week 6 to week 8;. then every 2 days from week 9 to week 24; at any time in case of AF symptoms. In case of AF recurrence for at least 10 minutes and if the patient does not stop the study treatment, then TTEM once a week

# LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK : Anti-vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

Final version 602/1185

HDL : High density lipoprotein

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 603/1185

# 1. INTRODUCTION AND STUDY RATIONALE

### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

Final version 604/1185

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of

Final version 605/1185

functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p < 0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

# 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

Final version 606/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

# 1.2.1. Chemical and pharmaceutical characteristics

# 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

# 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

Final version 607/1185

### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

# 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an  $IC_{50}$  value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus 637  $\pm$  196 sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and 79  $\pm$  51 sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of

Final version 608/1185

DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases

plasma level of DHA, it could be estimated that the compound may exert a similar protective

effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 609/1185

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

Final version 610/1185

## Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 611/1185

### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic heart failure.

### 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common (>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000), not known (cannot be estimated from the available data).

Final version 612/1185
- The reported adverse events are:

• Infection and infestations:

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

• Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Final version 613/1185

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

Final version 614/1185

## 2. STUDY OBJECTIVES

## 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

#### 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the

Final version 615/1185

included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (anti-vitamin K), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with anti-vitamin K (AVK) for at least 3 weeks before ECV
- ECV in patients with stabilized INR (i.e. values between 2 and 3;sp to ) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV). Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Final version 616/1185

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1 g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit
- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

Final version 617/1185

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Persistent AF history (less than three years) with a duration of the current episode from 7 days to 6 months.
- a moderately abnormal systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- a Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

# 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

Final version 618/1185

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmic class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before ECV. According to guidelines for the management of AF [6], AVK should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Final version 619/1185

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

## 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/mL and 60 to 90 mg/mL, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports an once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

## 5.1. INCLUSION CRITERIA

## Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whomelectrical cardioversion is warranted

Final version 620/1185

- 3. History of first documented persistent AF less than 3 years
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

# • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- documented as surgically sterilized

## • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

## Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

## 5.2. NON INCLUSION CRITERIA

# Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 3 years,
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),

Final version 621/1185

- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Oral amiodarone:
  - 13a Previous treatment with oral amiodarone within 4 months prior to inclusion
  - 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion
- 14. Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection.
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship.
- 25. Breastfeeding female patient.

#### 5.3. NUMBER OF PATIENTS

76 x 2 patients (taking into account 15 % of non evaluable patients).

Final version 622/1185

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
- have the patient's decision written on the consent form
- obtain the reason(s) for withdrawal and report it/them in the case report form
- evaluate the patient's clinical condition
- if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.

Final version 623/1185

- Erroneous inclusion according to the study protocol. Any inclusion not respecting inclusion/non inclusion criteria will immediately be withdrawn and an appropriate treatment will be given by the investigator under his/her responsibility. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with AVK for at least 3 weeks before ECV.
- Patients who will not have a stabilized INR between 2 and 3 on at least 3 consecutive weekly tests.
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 weeks for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early relapse within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence that would require, at the investigator's judgement, a
  cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or
  uncomfortable clinical symptoms for instance.

## 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

# 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the

Final version 624/1185

Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.

- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

• F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

Final version 625/1185

# 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number, and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date

Final version 626/1185

- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

#### 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

Final version 627/1185

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once patient's eligibility is confirmed at selection visit (V1):

- The Investigator:
  - Contacts the IVRS/IWRS
- Answers the questions relating to the patient
- In return, the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment according to the same process as described above.

Final version 628/1185

## 6.5. DRUG ADMINISTRATION

## **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

Final version 629/1185

## 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

Final version 630/1185

## 7.1. ANTI-VITAMIN K TREATMENT

AVK should be given for at least 3 weeks before ECV and continued for the whole study duration. The AVK used will be left to the decision of the each Investigator according to his/her local practice.

## 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
- Class IA: Disopyramide, Procainamide, Quinidine
- Class IB: Lidocaine, Mexiletine
- Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any anticoagulant treatment other than AVK: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

Final version 631/1185

# 8. EVALUATION CRITERIA

## 8.1. PRIMARY EFFICACY CRITERION

## **8.1.1.** Time to the first Atrial Fibrillation Recurrence

# 8.1.1.1. Definition

Time to first AF recurrence is defined by the first episode of AF (symptomatic or not) lasting for at least 10 minutes.

### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from visit 4 (week 5) to visit 5 (week 8). Then every two days from visit 5 (week 8) to visit 9 (week 24 – End of study).

Moreover, if patient experiences AF symptoms during this TTEM period, it should be documented using the TTEM.

Final version 632/1185

In case of AF recurrence and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be faxed to the site. The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

## 8.1.2. Secondary Efficacy Criteria

## 8.1.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

# 8.1.2.1.1. *Definition*

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

# 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

### 8.1.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

Final version 633/1185

# 8.1.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

# 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episode.

## 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

## 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

# 8.1.2.3. Clinical parameters evaluation

#### 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

Final version 634/1185

## 8.1.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

#### 8.1.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during all the study period.

# 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

# 8.1.2.3.3. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

## 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shock distribution (1, 2 or 3 shocks)
  - Number of patients needing another cardioversion after initial ECV

# 8.1.2.5. Evolution of echocardiographic parameters

# 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), LVEF (%), Left ventricular end diastolic volume/BSA (mL/m<sup>2</sup>), Left ventricular end systolic volume/BSA (mL/m<sup>2</sup>), Left

Final version 635/1185

ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL).

#### 8.1.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

## 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.2.2. Blood samples

# 8.2.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

Final version 636/1185

# 8.2.2.2. Technical handling

Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored at +4°C (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

## **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as µg/g for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

## 8.3. SAFETY ASSESSMENT

#### 8.3.1. Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the

Final version 637/1185

Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

## **8.3.2.** Laboratory Investigations

### 8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 mL.

## 8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: hematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and absolute), reticulocytes, platelets.

Chemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L]

in women:

Final version 638/1185

GFR (mL/min) = [(140-age)] x weight / 7.2 x serum creatinine in mg/L] x 0.85

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

#### 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

Final version 639/1185

# 8.3.5. Electrocardiogram (ECG)

## *8.3.5.1. Schedule*

An ECG will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

#### 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

## **8.3.6.** Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV
- INR every 4 weeks after ECV

Final version 640/1185

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by AVK should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### **8.3.7.** Concomitant Treatments

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial, can be found in section 7.

## 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit, the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

## 9. STUDY PROCEDURES

## Visit 1 - Selection Visit (Week -4 to Week -1)

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history

Final version 641/1185

- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

- A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory. The Central Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.
- The patient will enter the selection period in which anticoagulant (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

Final version 642/1185

The patient will receive from the investigational centre the study card to be kept for the duration

of the study.

Visit 2 - Inclusion Visit (Day 1)

If the patient's behaviour during the selection period and/or the result of complementary

examinations particularly the confirmation of the presence of persistent AF by the Central

Reading Laboratory during this period, the INR and laboratory tests, are compatible with the

inclusion criteria, the patient will be assessed for the following:

Adverse events

• Concomitant treatments (authorised, disallowed)

Laboratory examination: red blood cell concentrations of DHA and coagulation

parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time

(aPTT), Thrombin Clotting Time (TCT)

Global Physical examination/bodyweight

Vital signs

Echocardiography using a two-dimensional echocardiography

12-lead ECG

Urine pregnancy test for women of child bearing potential

If the results of the above assessments are compatible with the inclusion criteria, the patient will

be included and allocated a treatment number using the IVRS/IWRS.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to

paragraph 8.3.6) in order to ensure that the INR is stable (between 2 to 3 before electrical

cardioversion).

At the end of the visit, the Investigator will organise the appointment for the next visit and will

give the treatment for the next 4-week period.

Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Final version 643/1185 Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE performed in the same day (and before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

Final version 644/1185

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

## Visit 4 (Week 5: D35 -2/+7 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Body weight (body weight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms, additional transmissions may be performed.

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) – Visit 7 (Week 16: D112  $\pm$  7 days) – Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of

Final version 645/1185

discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT

should be stopped.

Global Physical examination/bodyweight

Vital signs

• 12-lead ECG

• The cardiac monitoring will be continued using a TTEM device. The device will be given

to the patient who will be requested to perform daily transmission from week 6 to week 8,

then every 2 days from week 9 to week 24. Moreover, in case of AF symptoms, additional

transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused

capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give

the treatment to be taken during the next 4-week treatment period.

In addition:

- at visit 6:

• the investigator will contact the IVRS/IWRS to obtain the treatment unit number to

be dispensed at visit 6 for the last 12-week period.

• an echocardiography will be performed, an haematology examination will be done

and the RBC concentration of DHA will be measured.

End-of-Study Visit - Visit 9 (Week 24: D168  $\pm$  7 days)

Patient will be assessed for the following:

Adverse events

• Concomitant treatments (authorised, disallowed)

Final version 646/1185

- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused soft capsules.

## 10. ADVERSE EVENTS: DEFINITION AND REPORTING

#### 10.1. ADVERSE EVENTS

#### **10.1.1.** Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

Final version 647/1185

## **10.1.2.** Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

## **10.1.3.** Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

# 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

Final version 648/1185
\* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:

- planned (as per protocol) medical/surgical procedure
- preparation for routine health assessment/procedure (e.g. routine colonoscopy)
- planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
- administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

## 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

## HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

#### 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

Final version 649/1185

## **10.2.4. SAE Occurring After the Study**

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

## 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Final version 650/1185

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

## 11. DATA COLLECTION AND STUDY MONITORING

## 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

Final version 651/1185

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

## 11.2. STUDY MONITORING

## 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

Final version 652/1185

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
  - has received the technical protocol, administrative and financial agreement signed by all parties
  - has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed curriculum vitae of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

Final version 653/1185

## 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

## 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

#### 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

Final version 654/1185

## 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

Final version 655/1185

The Sponsor Clinical Development Physician will validate the coding.

## 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

## 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

## 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

Final version 656/1185

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

## 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

• The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.

Final version 657/1185

- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

## 13.5. HANDLING OF DROPOUTS AND MISSING DATA

## **13.5.1.** Dropouts

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

## 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

## 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- Quantitative parameters will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Final version 658/1185

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

## 13.7. EFFICACY ANALYSIS

## 13.7.1. Primary Criterion

## 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

## 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

## 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

## 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

Final version 659/1185

# 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

# 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

## 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

## 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

Final version 660/1185

## 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs
- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

Final version 661/1185

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (for all patients).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

## 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration

Final version 662/1185

assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)

Final version 663/1185

- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

## 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

## 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

## 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

Final version 664/1185

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

## 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

## 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by the rapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

## 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Final version 665/1185

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

#### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

## 14. GENERAL ETHICAL CONSIDERATIONS

#### 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

# 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

Final version 666/1185

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi

Final version 667/1185

Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

## 15. ADMINISTRATIVE PROCEDURES

#### 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

## 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

Final version 668/1185

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not.
- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

## 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

## 15.3.2. Early Study Termination

## 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety

Final version 669/1185

• Stopping of the development ...

## 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

## 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

Final version 670/1185

## 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

## 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

Final version 671/1185

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 672/1185

## 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 673/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

[14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 674/1185

# [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

## [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

## [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

## [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

## [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 675/1185

# 17. APPENDICES

Final version 676/1185

#### 17.1. DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 677/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 678/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 679/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 680/1185

# 17.2. SAE REPORT FORM

Final version 681/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE CORPORATE VIGILANCES DIVISION |
|---|
| TO BE TRANSMITTED TO THE CORPORATE VIGILANCES DIVISION BY E-MAIL WITHIN 24H TO HQ.pharmacovigilance@pierre-fabre.com OR BY FAX WITHIN 24H – Fax N°: 33 (0) 1.49.10.80.90 |
| Transmission date (ddmmyyyy) Country: |
| SAE N° |
| > SUBJECT CHARACTERISTICS |
| Birth date |
| Gender1=M, 2=F Height cm Weight ·kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Congenital abnormality or abnormal pregnancy outcome ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: |
| ■ Pregnancy exposure Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE arget data |
| AE onset date |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| • Date of first study treatment administration |
| • Date of last study treatment administration before the occurence of SAE |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 682/1185

| Transmission date | | | (ddmmyyyy) | Country: | | |
|---|---|---|---|---|---|---|
| SAE N° | FIRST NOTIFICATION G FOLLOW-UP N° | | | | | |
| > CONCOMITANT MEDICATION SINCE TRIAL INITIATION and UP UNTIL THE OCCURRENCE OF THE SAE (EXCEPT THE TREATMENTS GIVEN FOR THE SAE) | | | | | | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAKEN FOLLOWING THE SAE | | | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | | |
| ☐ Dosage modification, specify: | | | Modi | fication Date : | / | |
| ☐ Temporarily discontinued | | | Readministration date: | | / | _/ |
| ☐ Withdrawn | | | | End date : | / | / |
| ☐ Not applica | ble | | | | | |

Final version 683/1185

| • The event led to: | | | | | | |
|---|---|---|---|---|---|---|
| ☐ Prescription of corrective or symptomatic treatments: | | | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Discontinuation of concomitant treatments: | | | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, specify: | | | | | | |
| > OUTCOME | | | | | | |
| □ Not recovered/Not resolved □ Recovering/Resolving □ Recovered/Resolved | | | | | | |
| ☐ Recovered/Resolved with sequelae ☐ Fatal ☐ Unknown | | | | | | |
| In case of death, has an autopsy been conducted? Yes No | | | | | | |
| > INVESTIGATOR CAUSALITY ASSESSMENT (investigator's assessment to be done as soon as possible) | | | | | | |
| Study drug: Related to study protocol: | | | | | | |
| ☐ Not Suspected | ☐ Suspected | d □ Not Suspected □ Suspected | | | | |
| Comments: | | | | | | |

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

Final version 684/1185
# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|---|---|---|---|---|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| 1,0111111111111111111111111111111111111 | Protein | g/l | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pН | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/1 | - | N x (23/36) |
| | ALAT (SGPT) | U/1 | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 685/1185

<sup>(

)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

#### **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | Decrease of at least 2g/dl and value < 10 g/dl whatever the baseline value If missing baseline : value <10g/dl |
| NEUTRO | PHILS | $\bullet$ < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline:</li> <li>TB &gt; 1.5 N</li> <li>If abnormal baseline:</li> <li>TB &gt; 2 N</li> </ul> |

#### N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 686/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90$ mmHg and decrease $\ge 20$ mmHg |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \leq 50$ mmHg and decrease $\geq 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>paseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the Minimum Post-baseline Value for each parameter | | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤50 | ≤90 | ≤50 | ≤50 |
| [120;140] | [80;90[ | <i>[50;75]</i> | [90 ;120] | [50;80] | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3B1 ≥ 90 01 DB1 ≥ 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

Table 5: Definition of orthostatic hypotension

| Orthostatic Hypotension * |
|---|
| SBP Decrease ≥ 20 mmHg or DBP Decrease ≥ 10 mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 687/1185

16.1.1.7. Protocol amendment n° PA04
General and non-substantial dated on 03 June
2014 linked to Protocol and appendices
(version 7: 03 June 2014)

Final version 688/1185

CLINICAL STUDY PROTOCOL AMENDMENT n° PA04 Version 1 (General – Non Substantial)

Final version 689/1185

Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne, France

#### CLINICAL STUDY PROTOCOL AMENDMENT n° PA04 Version 1

(General – Non Substantial)

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Pierre Fabre Study Code: F373280 CA 2 01

**EudraCT Number or equivalent:** 2012-003487-48

Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE

Sponsor's Representative: Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien 31035 TOULOUSE Cedex 1

Pr Savina NODARI

Department of Clinical and Surgical Specialities, Radiological Science and

Public Health

Section of Cardiovascular Diseases

Study Coordinating Investigator: University Medical School and Spedali Civili Hospital of Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

**Date of amendment PA04:** 03 Jun 2014

Final version 690/1185



Study code: F373280 CA 2 01


#### APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

### Clinical Study Protocol Amendment no PA04 Version 1

(General – Non Substantial)
Dated: 03JUN2014

| Sponsor's representative(s) | | | |
|---|---|---|---|
| · Medical Director | Dr Richard ROCHE | Date: 06/06/20 | Signature: |
| · Clinical Study Manager: | Gaëlle ALCARAZ | Date: OF JUN 814 | Signature: Reason |
| Study Coordinating Investigator | : | Date: | Signature: |
| | Pr Savina NODARI | | |

Clinical study protocol amendment no PA04 Version 1 (General – Non Substantial)

Date: 03JUN2014




Study code: F373280 CA 2 01


#### APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

### Clinical Study Protocol Amendment n° PA04 Version 1

(General – Non Substantial)

Dated: 03JUN2014

| Sponsor's representative(s) | | | |
|---|---|---|---|
| · Medical Director | | Date: | Signature: |
| | Dr Richard ROCHE | E | |
| · Clinical Study Manager : | | Date: | Signature: |
| | Gaëlle ALCARAZ | | |
| Study Coordinating Investigator | ; | Date: | Signature: |
| | Pr Savina NODAR | 11/06/2014 | Sonae Moder |

Clinical study protocol amendment n° PA04 Version 1 (General – Non Substantial)

Date: 03JUN2014


#### COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

## Clinical Study Protocol Amendment n° PA04 Version 1

(General – Non Substantial)
Dated: 03JUN2014

| <b>Country Coordinating Investigator:</b> | Date: | Signature: |
|-------------------------------------------|-------|------------|

Final version 693/1185

#### **INVESTIGATOR SIGNATURE FORM**

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

## Clinical Study Protocol Amendment nº PA04 Version 1

 $(General-Non\ Substantial)$ 

Dated: 03JUN2014

| By my signature below, I, Dr | , hereby confirm that I have read, taker |
|---|---|
| note of (and will apply) the modifications brou- | ight by the protocol amendment n° PA04 and I will |
| conduct the trial according to these new modalities | es. |
| Date: | Signature: |

Final version 694/1185

### HISTORY OF AMENDMENTS

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| NA | NA | General | NA | Following French CA request (ANSM) and leading to protocol version 2: - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 |
| PA01 | Substantial | Local (Italy) | 01MAR2013 | Corresponding to Protocol Version 3: - Integration of the modification included in the protocol version 2 - Harmonisation of the protocol and the Informed Consent Form: * adjustment of the selection criteria n°10 related to the contraception method * addition of a letter that is given by the patient to his/her general practitioner (GP) * precision that the sponsor can not collect a copy of the Informed Consent Form * precision that the patient card is in Italian language only (without any English mention) |
| PA02 | Non<br>Substantial | General | 28MAR2013 | Corresponding to Protocol Version 4: - change of Sponsor's Representative (Clinical Study Manager), - modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed, - precision on the function and address of the International Study Coordinator Pr Nodari, - add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study), - adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage", - precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee), - correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized) addition of the changes included in the local italian substantial protocol amendment (i.e: contraception method, letter to General Practionner, patient card in Italian and no collection of the consent form by the sponsor in Italy). |

Final version 695/1185

| PA03 | Substantial | General | 23OCT2013 | Corresponding to Protocol Version 5: |
|---|---|---|---|---|
| | | | | - Fax modification of the sponsor's representatives |
| | | | | <ul> <li>Planned end of study postponed to January 2015.</li> <li>The authorized history of the first documented persistent atrial fibrillation is less than 3 years.</li> <li>At selection a hyperkalemia or a hypokalemia is better defined by the standards of the local laboratories.</li> <li>Regarding previous treatments by amiodarone the non inclusion criteria of the protocol are adapted as follow: <ul> <li>Previous treatment with oral amiodarone within 4 months prior to inclusion</li> <li>Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion</li> <li>Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion.</li> <li>For male with a child-bearing potential partner (in Italy only): taking into account the duration of spermatogenesis the absolute abstention from sexual intercourse or the use of double barrier contraception method are extended to 3 months after the end of the study.</li> <li>Ranolazine is an antiarrhythmic treatment added to the prohibited treatments.</li> <li>Update of Serious Adverse Events (SAEs) form: Main change is the SAE sending: SAEs have to be reported to the Corporate Vigilance Department, and not anymore to the clinical study manager. Also SAEs can be sent by email and by fax.</li> <li>Addition of Alpha Bioresearch as CRO involved for Feasibility, Monitoring and Regulatory issues in Spain.</li> <li>Correction of some minor typographic errors</li> </ul> </li> </ul> |

#### 1. AMENDMENT RATIONALE

The purpose of this non-substantial amendment is to clarify or specify some points of the protocol. Theses changes do not affect the balance of the risk and benefits in the study nor change the specific aims or design of the study.

Final version 696/1185

### 2. CHANGES DESCRIPTION

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| SYNOPSIS | SYNOPSIS |
| Study Schedule: [] - V2/ D1: Inclusion visit (start of treatment) | Study Schedule: [] - V2/ D1: Inclusion visit (start of study treatment) |
| Evaluation Criteria: | Evaluation Criteria: |
| Efficacy evaluation variables: [] Cardioversion: | Efficacy evaluation variables: [] Cardioversion: |
| Other: • Evolution of echocardiographic parameters (from V4 to V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA(mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL) | Other: Evolution of echocardiographic parameters (at V4, V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA(mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL)) [] |
| Safety criteria: - Adverse events (observed and / or spontaneously reported) - Vital signs (Blood pressure (supine and standing), heart rate) - Physical examination (body weight) - Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns (ECG not centralized) | Safety criteria: - Adverse events (observed and / or spontaneously reported) - Vital signs (Blood pressure (supine and standing), heart rate) - Physical examination (body weight, body surface area) - Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns (ECG not centralized) Concomitant treatments |
| | Compliance |

Final version 697/1185

#### 4. STUDY DESIGN

#### 4.1 OVERALL DESCRIPTION

[...]

After a 1 to 4-week of run-in period without treatment, patients will be randomised into one of the following treatment groups: F373280 1 g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of treatment)

# 4. STUDY DESIGN OVERALL DESCRIPTION

[...]

After a 1 to 4-week of run-in period without **study** treatment, patients will be randomised into one of the following treatment groups: F373280 1 g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of **study** treatment)

# 8. EVALUATION CRITERIA PRIMARY EFFICACY CRITERION

# Time to the first Atrial Fibrillation Recurrence

#### 8.1.1.3. Evaluation Methods

[...]

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from visit 4 (week 5) to visit 5 (week 8). Then every two days from visit 5 (week 8) to visit 9 (week 24 – End of study).

[...]

The cardiologist interpretation will be faxed to the site.

#### 8. EVALUATION CRITERIA

#### 8.1 PRIMARY EFFICACY CRITERION

# 8.1.1 Time to the first Atrial Fibrillation Recurrence

#### 8.1.1.3 Evaluation Methods

[...]

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from **the day after visit 4 (week 6)** to visit 5 (week 8). Then every two days from **the day after visit 5** (week 9) to visit 9 (week 24 – End of study).

[...]

The cardiologist interpretation will be emailed to the site (or per fax on request of the site).

#### 8.1.2.4. Cardioversion assessment

[...]

Shock distribution (1, 2 or 3 shocks)

#### 8.1.2.4. Cardioversion assessment

[...]

• Shocks distribution (1, 2 or 3 shocks)

Final version 698/1185

## 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.2 Blood samples

#### 8.2.2.2. Technical handling

Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored at +4°C (<u>no freezing will be allowed</u>) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### 8.3. SAFETY ASSESSMENT

#### 8.3.3 Global physical examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

#### 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An ECG will be recorded at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

#### 8.3.5.2. Technical Procedure and Parameters

Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), repolarisation patterns will be reported in the e-CRF.

## 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.2 Blood samples

#### 8.2.2.2 Technical handling

Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored **between +2°C/+8°C** in a **fridge** (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### 8.3. SAFETY ASSESSMENT

#### 8.3.3 Global physical examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The Body surface area (BSA) will be calculated at the same visits using Mostellers' formula:

BSA =  $[(Weight x Height)/3600]^{1/2}$ (Weight in kg, height in cm)

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

#### 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An ECG will be recorded **after at least 10 minutes of rest** at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

#### 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns will be reported in the e-CRF.

Final version 699/1185

#### 8.3.7. Concomitant Treatments

#### 8.4. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit, the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

#### 8.4. CONCOMITANT TREATMENTS

#### 8.5. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit (except at visit 4), the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

#### 9. STUDY PROCEDURES

Visit 4 (Week 5: D35 -2/+7 days)

[...]

The patient will be requested to performed daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24.

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

[...]

The cardiac monitoring will be continued using a TTEM device. The device will be given to the patient who will be requested to perform daily transmission from week 6 to week 8, then every 2 days from week 9 to week 24.

#### 9. STUDY PROCEDURES

Visit 4 (Week 5: D35 -2/+7 days)

[...]

The patient will be requested to **perform** daily transmission from **the day after visit 4 (week 6) to visit 5 (week 8),** then every two days from **the day after visit 5 (week 9) to visit 9 (week 24 – End of study)**.

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

[...]

The cardiac monitoring will be continued using a TTEM device. The device will be given to the patient who will be requested to perform daily transmission from the day after visit 4 (week 6) to visit 5 (week 8), then every two days from the day after visit 5 (week 9) to visit 9 (week 24 – End of study).

Final version 700/1185

# 13. STATISTICAL ANALYSIS 13.11. INTERIM ANALYSIS AND DATA MONITORING

No interim analysis is planned.

# 13. STATISTICAL ANALYSIS 13.11. INTERIM ANALYSIS AND DATA MONITORING

No analyses of efficacy data are planned for IDMC that ensures that the overall probability of type I error is controlled. No Type I error and sample size adjustments are necessary. Any recommendations of the IDMC to alter study conduct will be based on safety, so IDMC monitoring of the study will not affect the statistical operating characteristics of the final analysis. The IDMC will review, three times during the study period (after the first 30 subjects will have been randomized, when the first 80 subjects will have terminated their study participation and when 130 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable.

Final version 701/1185

F 373280 CA 2 01

Final version 702/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

#### CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 69 69

E-mail:gaelle.alcaraz@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

Associate Professor of Cardiology

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: <a href="mailto:savinanodari@gmail.com">savinanodari@gmail.com</a>; nodari@med.unibs.it

#### **Version 7 – 03JUN2014**

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 703/1185

#### **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

### **Clinical Study Manager (Monitor)**

Gaëlle ALCARAZ

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 62 16 Fax: +33 5 34 50 69 69

E-mail: gaelle.alcaraz@pierre-

fabre.com

#### **Medical Director**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 69 69

E-mail: richard.roche@pierre-

fabre.com

Final version 704/1185

#### CONTRACT RESEARCH ORGANISATIONS

#### For Feasibility, Monitoring and Regulatory issues:

#### Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: www.psnglobal.org

#### For Feasibility, Monitoring and Regulatory issues (in Spain):

#### Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

#### For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6, Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

#### For Centralised Reading of Holder ECG and TTEM and equipment supply:

#### **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage:

#### Agrocampus Ouest

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

#### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER – FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 705/1185

## For refund of patients expenses linked to the study (in France):

**CLINACT** 

6-10 rue TROYON 92310 SEVRES – FRANCE

Phone: +33 1 46 90 27 27 - Fax: +33 1 46 23 01 56

Email: sebastien.beaumont@clinact.com

Final version 706/1185

# Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 7 – 03 JUN2014

| Sponsor's Representative: Medical Director: Richard ROCHE, MD | Date: <b>06</b> / 6 | 9611 014 Signature: |
|---|---|---|
| Study Coordinating Investigator:<br>Savina NODARI, MD | Date: | Signature: |

# Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 7 - 03 JUN2014

| Sponsor's Representative: | | | |
|----------------------------------------|---|------------|------------|
| Medical Director:<br>Richard ROCHE, MD | | Date: | Signature: |
| Savina NODARI, MD | | Date: | Signature: |
| | ¥ | 11/06/2014 | Some noder |

#### Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

### **Protocol Version 7 – 03 JUN 2014**

| Country: | | |
|--------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator</b> : | | |
| "Name" | Date: | Signature: |

Final version 709/1185

#### Protocol F 373280 CA 2 01

#### **INVESTIGATOR SIGNATURE FORM**

Protocol Version 7 – 03 JUN 2014

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 03 June 2014 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * To be adapted | |
|-----------------|---|
| | T |

| Date: Si | ignature |
|----------|----------|
|----------|----------|

Final version 710/1185

## TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|-------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | 24 |
| 1.2.1. | Chemical and pharmaceutical characteristics. | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1.2 | 7 | |
| 1.2.2. | | |
| 1.2.2. | $\mathcal{C}$ | |
| 1.2.2.3 | | |
| 1.2.2.4 | C, 1 | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 33 |
| 2.1. | PRIMARY OBJECTIVE | 33 |
| 2.2. | SECONDARY OBJECTIVES | |
| <b>3.</b> 1 | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 35 |
| 4.1. | OVERALL DESCRIPTION | 35 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | 38 |
| 5.2. | NON INCLUSION CRITERIA | 39 |
| 5.3. | NUMBER OF PATIENTS | 40 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 41 |
| 5.6. | WITHDRAWAL CRITERIA | 41 |
| 5.7. | REPLACEMENT OF PATIENTS | 42 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | 42 |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | 42 |

| 6. | STUDY TREATMENT | 43 |
|---|---|---|
| 6.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 43 |
| 6.2. | PACKAGING AND LABELLING | |
| 6.2.1. | | |
| 6.2.2. | | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 6.5. | DRUG ADMINISTRATION | 47 |
| 6.5.1. | Duration of Treatment | 47 |
| 6.5.2. | | |
| 6.5.3. | | 47 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | 48 |
| 7. | CONCOMITANT TREATMENTS | 48 |
| 7.1. | ANTI-VITAMIN K TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | |
| 7.3. | AUTHORISED TREATMENTS | |
| 8. | EVALUATION CRITERIA | |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence. | 50 |
| 8.1.1. | | |
| 8.1.1. | | |
| 8.1.1. | | |
| 8.1.2. | j j | |
| 8.1.2.<br>8.1.2. | $\mathcal{E}$ | |
| 8.1.2.<br>8.1.2. | | |
| 8.1.2. | 1 | |
| 8.1.2. | | |
| 8.2. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF | |
| | DHA | 54 |
| 8.2.1. | Definition | 54 |
| 8.2.2. | Blood samples | 54 |
| 8.2.2. | 1. Collection schedule | 54 |
| 8.2.2. | $\boldsymbol{c}$ | |
| 8.2.3. | DHA concentration measurement | 55 |
| 8.3. | SAFETY ASSESSMENT | 55 |
| 8.3.1. | | |
| 8.3.2. | Laboratory Investigations | 56 |

| 8.3.2.1. Schedule | 56 |
|----------------------------------------------------------------|----|
| 8.3.2.2. Technical Procedures and Parameters | 56 |
| 8.3.3. Global Physical Examination | 57 |
| 8.3.4. Vital Signs | 57 |
| 8.3.4.1. Schedule | |
| 8.3.4.2. Technical Procedure and Parameters | |
| 8.3.5. Electrocardiogram (ECG) | |
| 8.3.5.1. Schedule | |
| 8.3.5.2. Technical Procedure and Parameters | |
| 8.3.6. Coagulation parameters | |
| 8.4. CONCOMITANT TREATMENTS | |
| 8.5. COMPLIANCE | 59 |
| 9. STUDY PROCEDURES | 59 |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 65 |
| 10.1. ADVERSE EVENTS | 65 |
| 10.1.1. Definition of Adverse Events | 65 |
| 10.1.2. Grading of Adverse Events | 66 |
| 10.1.3. Reporting of Adverse Events | 66 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 66 |
| 10.2.1. Definition | 66 |
| 10.2.2. Reporting of SAE | 67 |
| 10.2.3. Follow-up of SAE | 68 |
| 10.2.4. SAE Occurring After the Study | 68 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 68 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 68 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | 69 |
| 11. DATA COLLECTION AND STUDY MONITORING | 69 |
| 11.1. DATA COLLECTION | 69 |
| 11.1.1. Case Report Form | 69 |
| 11.1.2. Source Documents | |
| 11.2. STUDY MONITORING | 71 |
| 11.2.1. Monitoring visits | |
| 11.2.1.1 Site Preselection Visit | |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | 73 |
| 12. DATA MANAGEMENT | 73 |
| 12.1. DATA ENTRY | 73 |
| 12.2 DATA CI FANING | 73 |

| 12.3. DATA CODING | 74 |
|---|---|
| 12.4. DATA STORAGE | 74 |
| 12.5. DATABASE LOCK | 74 |
| 13. STATISTICAL ANALYSIS | 74 |
| 13.1. GENERAL CONSIDERATIONS | 75 |
| 13.2. SAMPLE SIZE | 75 |
| 13.4. DATA SETS ANALYSED | 76 |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | 76 |
| 13.5.1. Dropouts | 76 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 13.7. EFFICACY ANALYSIS | |
| 13.7.1. Primary Criterion | |
| 13.7.1.1. Primary Analysis | |
| 13.7.2. Secondary Criteria | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| 13.8.4.1. Vital Sign Measurements Over Time | |
| 13.8.4.2. Body weight | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | |
| 14. GENERAL ETHICAL CONSIDERATIONS | 84 |
| 14.1. ETHICAL CONDITIONS | 84 |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | |
| 14.4. PERSONAL DATA PROTECTION | 86 |

| 14.5. INSURANCE POLICY | 86 |
|---|---|
| 15. ADMINISTRATIVE PROCEDURES | 87 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 87 |
| 15.3. END OF THE STUDY | 88 |
| 15.3.1. Definition of the End of Study | 88 |
| 15.3.2. Early Study Termination | 88 |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | 88 |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | 88 |
| 15.4. AUDIT | 88 |
| 15.5. INSPECTION | 89 |
| 15.6. CONFIDENTIALITY | 89 |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 89 |
| 15.9. STUDY RESULTS PUBLICATION | 90 |
| 16. REFERENCES | 91 |
| 17. APPENDICES | 94 |
| 17.1. DECLARATION OF HELSINKI | 95 |
| 17.2. SAE REPORT FORM | 99 |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTI CLINICALLY SIGNIFICANT CHANGES AND VALUES | |

## **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|
| Name of Finished Product: | Not applicable |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. |
| Abbreviated Title: | International, multicentric, randomised, double-blind, placebo controlled study Not applicable |
| Study Coordinating Investigator: | Pr Savina NODARI |
| Study Centres: | International, multicentric |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing.[1] Moreover, the effectiveness of PolyUnsaturated Fatty Acid (PUFA) has been proven in the following conditions: — prevention of AF recurrence in patients with persistent AF, in co-administration with amiodarone (add on therapy) [2] — Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. |
| Planned Study Period: | January 2013 – January 2015 Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>INR 2-3 anti-vitamin K should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> <li>Cardiac monitoring: <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms</li> </ul> </li> <li>Treatment duration: 24 weeks</li> </ul> |
| Study Schedule: | <ul> <li>9 visits will be scheduled:</li> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of study treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to</li> </ul> |

Final version 716/1185

| | <ul> <li>clinical practice of the centre) (installation of the Holter device)</li> <li>V4/ W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V5/ W8 (D56± 7 days): follow-up visit</li> <li>V6/ W12 (D84 ± 7 days): follow-up visit</li> <li>V7/ W16 (D112 ± 7 days): follow-up visit</li> </ul> |
|---|---|
| | - V8/ W20 (D140 ± 7 days): follow-up visit<br>- V9/ W24 (D168 ± 7 days): final study visit |
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | <ol> <li>Inclusion Criteria:</li> <li>Demographic Characteristics and Other Baseline Characteristics:</li> <li>Men or women aged more than 18 years (inclusive)</li> <li>Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted</li> <li>History of first documented persistent AF less than 3 years.</li> <li>History of ischemic or non ischemic heart failure</li> <li>NYHA class I or II chronic heart failure at selection and at inclusion</li> <li>Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion</li> <li>On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers</li> <li>Left atrial area ≤ 40 cm² at selection and at inclusion</li> <li>Patients treated or having to be treated by anti-vitamin K</li> </ol> |
| | <ul> <li>For female patient of child-bearing potential: <ul> <li>in all the countries except Italy: <ul> <li>use of an effective method of contraception (hormonal contraception or intrauterine device) assessed by the investigator, for at least 2 months before the selection in the study, and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment</li></ul></li></ul></li></ul> |

- the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

- History of first documented episode of persistent AF more than 3 years
- More than two successful cardioversions (electrical or pharmacological) in the last 6

Final version 717/1185

| Mode of Administration; | , |
|---|---|
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| Dose: | Soft Capsules Arm with 1g of F373280 |
| Test Product: | F373280 |
| Exclusion criteria before V3: | Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV) ECV will be performed in patients without dyskalemia If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days. |
| Exclusion criteria before V3. | selection 10. Cardiac surgery within 3 months before selection or planned during the study duration Criteria related to treatments: 11. Previously ineffective pharmacological or electrical cardioversion 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calcium-blockers 13. Oral amiodarone: 13a Previous treatment with oral amiodarone within 4 months prior to inclusion 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion 14. Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months 17. Dietary supplement with ω 3 or ω 6 according to investigator's judgement 18. Having undergone any form of ablation therapy for AF 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel Other criteria: 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion 21. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints 23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship 25. Breastfeeding female patient |
| | rate < 30 mL/min) at selection 8. Bradycardia (HR ≤ 50 bpm) 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at |
| | <ul> <li>coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection</li> <li>7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration</li> </ul> |
| | treatment for thyroid disease 6. Myocardial infarction or unstable angina or presence of unstable ischemic |
| | <ul> <li>IV)</li> <li>NYHA class III or IV heart failure at selection or at inclusion</li> <li>Thyroid disease uncontrolled by treatment: TSH ± T4L ± T3L to be checked in case of</li> </ul> |
| | months 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to |

Final version 718/1185

| Duration of Treatment: | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
|---|---|
| Reference Therapy | Placebo soft capsules |
| Mode of Administration: | Placebo will be administered in the same conditions as the tested product. Oral, one capsule each evening with dinner |
| | Efficacy evaluation variables: |
| Evaluation Criteria: | Primary evaluation variable: Time to first Atrial Fibrillation recurrence defined by the first episode of AF lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 (ECV visit). Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24. For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5). Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM. All ECG traces will be evaluated by a Central Reading Laboratory. Secondary evaluation variables: During the 7-day continuous ECG monitoring, Numbers of AF episodes Duration of AF episodes |
| | Clinical parameters: During the whole study: Number of recurrence of symptomatic AF episodes EHRA score Hospitalization for cardiovascular events Hospitalization for thromboembolic stroke All causes of hospitalization Cardioversion: Assessment of spontaneous cardioversion Assessment of successful cardioversion Shocks distribution (1, 2 or 3 shocks) Number of patients needing an other cardioversion after the initial ECV |
| | <ul> <li>Other:</li> <li>Evolution of echocardiographic parameters (at V4, V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (mL), Left atrial volume/BSA (mL/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (mL/m²), Left ventricular end systolic volume/BSA(mL/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (mL))</li> <li>Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).</li> </ul> |
| | <ul> <li>Safety criteria:</li> <li>Adverse events (observed and / or spontaneously reported)</li> <li>Vital signs (Blood pressure (supine and standing), heart rate)</li> <li>Physical examination (body weight, body surface area)</li> <li>Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), QTcB. (ms), QTcF. (ms), repolarisation patterns (ECG not centralized)</li> <li>Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets</li> <li>Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol</li> </ul> |

Final version 719/1185

| | <ul> <li>(HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)</li> <li>Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR (local laboratory), Prothrombine Time (PT)</li> <li>Concomitant treatments</li> <li>Compliance</li> </ul> |
|---|---|
| Statistical Methods: | Sample Size: Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. Primary Efficacy Analysis The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model. Secondary Analyses All secondary efficacy criteria will be described and compared using appropriate tests on the FAS. Safety Analyses Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment). |

Final version 720/1185
## STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | X | Х | Х | Х | Х | Х | Х | Х |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | X | X | X | | Х | Х | Х | Х | Х |
| Echocardiography | X | X | | X | | х | | | X |
| Eligibility criteria check | X | X | | | | | | | |
| Blood pressure, heart rate | X | X | X | X | Х | Х | Х | X | X |
| 12-Lead ECG Recording | X | X | X | | x | x | X | X | X |
| INR | <b>\</b> | | (2) | | Х | Х | Х | Х | X |
| aPTT, TCT | Х | X | X | | Х | Х | Х | Х | X |
| Biochemistry | Х | | | | | | | | Х |
| Hematology | Х | | X | | | Х | | | X |
| Urinary pregnancy test | | X | | | | | | | Х |
| Red Blood Cell concentrations of DHA | | X | X | | | x | | | X |
| Treatment allocation | | X | | | | х | | | |
| IVRS/IWRS | Х | X | | | | Х | | | |
| ECV (3) | | | X | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | x | Х | x | Х | Х | Х | Х | Х |
| Holter ECG | <b>←</b> (4) | | <b>←</b> | (5) | | | | | |
| TTEM (6) | | | | + | | | | | <b>—</b> |

Final version

721/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of AVK introduction: INR 2 to 3 times a week, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) TTEM: everyday from week 6 to week 8;. then every 2 days from week 9 to week 24; at any time in case of AF symptoms. In case of AF recurrence for at least 10 minutes and if the patient does not stop the study treatment, then TTEM once a week

## LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

AVK : Anti-vitamin K

βHCG : beta human chorionic gonadotrophinBLQ : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Trans-esophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

Final version 722/1185

HDL : High density lipoprotein

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set

QTcB QT interval using Bazett's correction formula QTcF QT interval using Fridericia's correction formula

RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

T0 : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 723/1185

## 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

Final version 724/1185

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of

Final version 725/1185

functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61 +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

## 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

Final version 726/1185

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 Investigator's Brochure. [1]

#### 1.2.1. Chemical and pharmaceutical characteristics

#### 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

#### 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

## Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

Final version 727/1185

#### 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus 637  $\pm$  196 sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and 79  $\pm$  51 sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of

Final version 728/1185

DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases

plasma level of DHA, it could be estimated that the compound may exert a similar protective

effect [1].

1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the

central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively

detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were

performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low

circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and

in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat

toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on

changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical

pharmacokinetic profile of F373280 is not associated with particular alerts concerning the

proposed clinical phase IIa study.

1.2.3. Clinical data

Part A: single dose

Final version 729/1185

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

Final version 730/1185

#### Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

Final version 731/1185

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic heart failure.

#### 1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common (>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000), not known (cannot be estimated from the available data).

Final version 732/1185

- The reported adverse events are:

• Infection and infestations:

Uncommon: gastroenteritis

• Immune system disorders:

Uncommon: hypersensitivity

• Metabolism and nutrition disorders:

Rare: hyperglycaemia

• Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

• Vascular disorders:

Very rare: hypotension

• Respiratory thoracic and mediastinal disorders:

Very rare: nasal dryness

• Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

• Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Final version 733/1185

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene® (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

Final version 734/1185

## 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

#### 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form.

A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the

Final version 735/1185

included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (anti-vitamin K), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with anti-vitamin K (AVK) for at least 3 weeks before ECV
- ECV in patients with stabilized INR (i.e. values between 2 and 3;sp to ) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE (trans-esophageal echocardiograph) performed in the same day (before ECV). Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Final version 736/1185

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without study treatment, patients will be randomised into one of the following treatment groups: F373280 1 g or placebo for 24 weeks.

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit
- Visit 9 (V9): W24 (D168  $\pm$  7D): final study visit

### 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

Final version 737/1185

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Persistent AF history (less than three years) with a duration of the current episode from 7 days to 6 months.
- a moderately abnormal systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.
- a Left Atrial Area (LAA) not severely abnormal (less than 40 cm² as defined in the report from the American Society of Echocardiography's Guideline). According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personnal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

Final version 738/1185

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmic class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Eligible participants will enter a selection phase in which anticoagulant treatment (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before ECV. According to guidelines for the management of AF [6], AVK should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Final version 739/1185

Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

#### 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/mL and 60 to 90 mg/mL, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough fluctuation (baseline corrected) was around 0.3. This value supports an once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

## Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whomelectrical cardioversion is warranted

Final version 740/1185

- 3. History of first documented persistent AF less than 3 years
- 4. History of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion
- 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers
- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by anti-vitamin K
- 10. For female patient of child-bearing potential:

## • in all the countries except Italy:

- use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- documented as surgically sterilized

#### • in Italy only:

- absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical /legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. History of first documented episode of persistent AF more than 3 years,
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),

Final version 741/1185

- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 mL/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Oral amiodarone:
  - 13a Previous treatment with oral amiodarone within 4 months prior to inclusion
  - 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion
- 14. Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatted Acid within the last 3 months Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection.
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship.
- 25. Breastfeeding female patient.

#### 5.3. NUMBER OF PATIENTS

76 x 2 patients (taking into account 15 % of non evaluable patients).

Final version 742/1185

#### 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

#### 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

#### 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
- have the patient's decision written on the consent form
- obtain the reason(s) for withdrawal and report it/them in the case report form
- evaluate the patient's clinical condition
- if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.

Final version 743/1185

- Erroneous inclusion according to the study protocol. Any inclusion not respecting
  inclusion/non inclusion criteria will immediately be withdrawn and an appropriate
  treatment will be given by the investigator under his/her responsibility. Erroneous
  inclusions will not be paid to the investigator.
- Patients who could not be treated with AVK for at least 3 weeks before ECV.
- Patients who will not have a stabilized INR between 2 and 3 on at least 3 consecutive weekly tests.
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 weeks for whom a trans-oesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early relapse within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence that would require, at the investigator's judgement, a
  cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or
  uncomfortable clinical symptoms for instance.

#### 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

#### 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate to another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the

Final version 744/1185

Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.

- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

### 6. STUDY TREATMENT

The Clinical Pharmacy Department of the *Institut de Recherche Pierre Fabre (IRPF)* will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

• F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the *IRPF* according to European Directive and local requirements.

Final version 745/1185

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number, and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date

Final version 746/1185

- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

#### 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the *IRPF* will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection.

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

Final version 747/1185

#### 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

Practically, once patient's eligibility is confirmed at selection visit (V1):

- The Investigator:
  - Contacts the IVRS/IWRS
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment according to the same process as described above.

Final version 748/1185

#### 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

#### 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

#### 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

Final version 749/1185

#### 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

### 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

Final version 750/1185

#### 7.1. ANTI-VITAMIN K TREATMENT

AVK should be given for at least 3 weeks before ECV and continued for the whole study duration. The AVK used will be left to the decision of the each Investigator according to his/her local practice.

#### 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I
- Class IA: Disopyramide, Procainamide, Quinidine
- Class IB: Lidocaine, Mexiletine
- Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any anticoagulant treatment other than AVK: thrombin inhibitor such as Dabigatran or antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel
- Dietary supplement with Omega 3 or Omega 6

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

#### 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

Final version 751/1185

## 8. EVALUATION CRITERIA

#### 8.1. PRIMARY EFFICACY CRITERION

### **8.1.1.** Time to the first Atrial Fibrillation Recurrence

## 8.1.1.1. Definition

Time to first AF recurrence is defined by the first episode of AF (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. *Schedule*

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

#### 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from the day after visit 4 (week 6) to visit 5 (week 8). Then every two days from the day after visit 5 (week 9) to visit 9 (week 24 – End of study).

Moreover, if patient experiences AF symptoms during this TTEM period, it should be documented using the TTEM.

Final version 752/1185

In case of AF recurrence and provided that the patient does not required a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

## 8.1.2. Secondary Efficacy Criteria

## 8.1.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

## 8.1.2.1.1. *Definition*

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

## 8.1.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

#### 8.1.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

Final version 753/1185

## 8.1.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

## 8.1.2.2.1. *Definition*

Duration of AF episodes will consist in the sum of duration of each AF episode.

#### 8.1.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

### 8.1.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

## 8.1.2.3. Clinical parameters evaluation

#### 8.1.2.3.1. EHRA score assessment

#### 8.1.2.3.1.1. Definition

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

Final version 754/1185

#### 8.1.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

#### 8.1.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during all the study period.

## 8.1.2.3.2. Number of recurrence of symptomatic AF

It consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

## 8.1.2.3.3. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
  - Hospitalization for AF treatment
  - Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

#### 8.1.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

## 8.1.2.5. Evolution of echocardiographic parameters

## 8.1.2.5.1. *Definition*

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm<sup>2</sup>), Left atrial volume (mL), Left atrial volume/BSA (mL/m<sup>2</sup>), LVEF (%), Left ventricular end diastolic volume/BSA (mL/m<sup>2</sup>), Left ventricular end systolic volume/BSA (mL/m<sup>2</sup>), Left

Final version 755/1185

ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (mL), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (mL).

#### 8.1.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.1.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.2.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.2.2. Blood samples

## 8.2.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

Final version 756/1185
# 8.2.2.2. Technical handling

Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored between +2°C/+8°C in a fridge (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between +2°C and +8°C). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### **8.2.3.** DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent) and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as µg/g for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

#### 8.3. SAFETY ASSESSMENT

#### 8.3.1. Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the

Final version 757/1185

Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

# 8.3.2. Laboratory Investigations

#### 8.3.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kaliemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 mL.

#### 8.3.2.2. Technical Procedures and Parameters

The following tests will be performed:

Haematology: hematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and absolute), reticulocytes, platelets.

Chemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinin, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (mL/min) = [(140-age) x weight / (7.2 x serum creatinine in mg/L)]

in women:

Final version 758/1185

GFR (mL/min) =  $[(140\text{-age}) \times \text{weight} / (7.2 \times \text{serum creatinine in mg/L})] \times 0.85$ 

- with serum creatinine expressed as µmol/l:

GFR (mL/min) =  $[(140\text{-age}) \text{ x weight / serum creatinine in } \mu\text{mol/l}] \text{ x k,where } k = 1.23 \text{ for men, } 1.04 \text{ for women.}$ 

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

# 8.3.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

The Body surface area (BSA) will be calculated at the same visits using Mostellers' formula:

 $BSA = [(Weight x Height)/3600]^{1/2}$ 

(Weight in kg, height in cm)

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

# 8.3.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

# 8.3.4.1. Schedule

Vital signs will be measured at each visit.

#### 8.3.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

Final version 759/1185

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

# 8.3.5. Electrocardiogram (ECG)

# 8.3.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

#### 8.3.5.2. Technical Procedure and Parameters

• Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns will be reported in the e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

• 24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

# 8.3.6. Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

Final version 760/1185

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

- INR 2-3 times a week for the first week of treatment
- INR weekly up to ECV
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by AVK should be given at least 3 weeks before ECV and continued for the whole study duration.

The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

#### 8.4. CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial, can be found in section 7.

# 8.5. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit (except at visit 4), the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

#### 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week -4 to Week -1)

Final version 761/1185

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate

If the results of the above assessments are compatible with the selection criteria

A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed
on the patient to monitor the patient heart rhythm. The patient will be requested to bring
back the device after the termination of 24 hours recording. The recording will be
transmitted from the Investigational site to the Central Reading Laboratory. The Central

Final version 762/1185

Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.

• The patient will enter the selection period in which anticoagulant (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

# **Visit 2 - Inclusion Visit (Day 1)**

If the patient's behaviour during the selection period and/or the result of complementary examinations particularly the confirmation of the presence of persistent AF by the Central Reading Laboratory during this period, the INR and laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Urine pregnancy test for women of child bearing potential

Final version 763/1185

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and allocated a treatment number using the IVRS/IWRS.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.3.6) in order to ensure that the INR is stable (between 2 to 3 before electrical cardioversion).

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period.

#### Visit 3 (Week 4: D28 -2/+7 days) cardioversion

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target international normalized ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE performed in the same day (and before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of

Final version 764/1185

sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge. Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

# Visit 4 (Week 5: D35 -2/+7 days)

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Body weight (body weight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to perform daily transmission from the day after visit 4 (week 6) to visit 5 (week 8), then every two days from the day after visit 5 (week 9) to visit 9 (week 24 – End of study). Moreover, in case of AF symptoms, additional transmissions may be performed.

Final version 765/1185

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial
  Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of
  discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT
  should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- The cardiac monitoring will be continued using a TTEM device. The device will be given to the patient who will be requested to perform daily transmission from the day after visit 4 (week 6) to visit 5 (week 8), then every two days from the day after visit 5 (week 9) to visit 9 (week 24 End of study). Moreover, in case of AF symptoms, additional transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week treatment period.

In addition:

- at visit 6:

• the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.

Final version 766/1185

• an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

# End-of-Study Visit - Visit 9 (Week 24: D168 ± 7 days)

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.
- Urine pregnancy test for women of childbearing potential
- Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused soft capsules.

# 10. ADVERSE EVENTS: DEFINITION AND REPORTING

#### 10.1. ADVERSE EVENTS

# 10.1.1. Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, *i.e.* any subjective signs and symptoms or change in a concomitant disease present at the Selection Visit considered or not related to the treatment.

Final version 767/1185

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should be repeated until the values return to normal or to a stable status. Abnormal results are defined as those falling out of the laboratory normal ranges and that are clinically significant. The frequency of such checks should be defined by the Investigator according to the degree of abnormality.

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

# **10.1.2.** Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

# **10.1.3.** Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

#### 10.2. SERIOUS ADVERSE EVENTS (SAE)

# 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*

Final version 768/1185

• Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

- \* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:
  - planned (as per protocol) medical/surgical procedure
  - preparation for routine health assessment/procedure (e.g. routine colonoscopy)
  - planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
  - administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

#### 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

# HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

Final version 769/1185

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

# 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

The serious adverse events must be followed up until resolution or stabilisation.

# 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

#### 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

Final version 770/1185

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

# 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Final version 771/1185

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF.

Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation.

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

Final version 772/1185

# 11.2. STUDY MONITORING

# 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
- has received the technical protocol, administrative and financial agreement signed by all parties
- has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

Final version 773/1185

The CRA has also to provide training on the study protocol requirements and study specific procedures.

# 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

# 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

Final version 774/1185

# 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

# 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

Final version 775/1185

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate the coding.

#### 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

# 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

Final version 776/1185

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

Final version 777/1185

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

#### 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3.
   This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

# **13.5.1. Dropouts**

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

#### 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

#### 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

Final version 778/1185

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- Quantitative parameters will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

# 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

Final version 779/1185

# 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

# 13.7.2.1. Numbers of Atrial Fibrillation Episodes

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

# 13.7.2.2. Duration of Atrial Fibrillation Episodes

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

# 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

#### 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

Final version 780/1185

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

#### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs

Final version 781/1185

- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (<u>for all patients</u>).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study

Final version 782/1185

treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

# 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

Final version 783/1185

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

Final version 784/1185

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

#### 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

#### 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by the rapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

Final version 785/1185

#### 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

#### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No analyses of efficacy data are planned for IDMC that ensures that the overall probability of type I error is controlled. No Type I error and sample size adjustments are necessary. Any recommendations of the IDMC to alter study conduct will be based on safety, so IDMC monitoring of the study will not affect the statistical operating characteristics of the final analysis. The IDMC will review, three times during the study period (after the first 30 subjects will have been randomized, when the first 80 subjects will have terminated their study participation and when 130 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable.

# 14. GENERAL ETHICAL CONSIDERATIONS

#### 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

Final version 786/1185

# 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

Final version 787/1185

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor *Pierre Fabre Médicament*, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

Final version 788/1185

# 15. ADMINISTRATIVE PROCEDURES

#### 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

# 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all patients included in the trial or not.
- Retains a list of the patient's names, addresses (and/or number of medical file), code
   numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

Final version 789/1185

#### 15.3. END OF THE STUDY

# 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

# 15.3.2. Early Study Termination

# 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at *Pierre Fabre Médicament* and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

Final version 790/1185

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

#### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

#### 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

#### 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

Final version 791/1185

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 792/1185
#### 16. REFERENCES

- [1] F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2] NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L.

  Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy

  J. Am. Coll. Cardiol. 2011;57;870-879
- [4] MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study

  \*American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5
- [5] GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6] CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct; 31(19):2369-429
- [7] KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 793/1185

[8] BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9] OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10] BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11] TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12] LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13] METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr* (2007); 85 : 1225.

[14] ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83 : 1469-1473S.

[15] TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16] SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6): 652-9.

Final version 794/1185

## [17] LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human *Lipids*, 2010, 45, 11-19.

#### [18] HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

#### [19] ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion *World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain* 

[20] KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G. Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association. *Europace* 2007, 9, 1006-1023

#### [21] EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter. *EMA/CHMA/EWP/213056/2010* 

#### [22] OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955-961

[23] ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

Final version 795/1185

### 17. APPENDICES

Final version 796/1185

#### 17.1. DECLARATION OF HELSINKI

#### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

Final version 797/1185

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

- 11. It is the duty of physicians who participate in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research.
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.

Final version 798/1185

- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.

Final version 799/1185

- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

## C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 800/1185

### 17.2. SAE REPORT FORM

Final version 801/1185

| | RSE EVENT (SAE) OR PREGNANCY<br>RATE VIGILANCES DIVISION |
|---|---|
| TO BE TRANSMITTED TO THE CORPORATE V<br>HQ.pharmacovigilance@pierre-fabre.com OR BY FAX WITHIN | VIGILANCES DIVISION BY E-MAIL WITHIN 24H TO<br>I 24H – Fax N°: 33 (0) 1.49.10.80.90 |
| Transmission date | (ddmmyyyy) Country: |
| SAE N° | IRST NOTIFICATION ☐ FOLLOW-UP ☐ N° |
| > SUBJECT CHARACTERISTICS | |
| | Birth date |
| Gender 1=M, 2=F Height | cm Weight kg |
| > DESCRIPTION OF THE EVENT | <del></del> |
| | ☐ Congenital abnormality or abnormal pregnancy outcome |
| The serious adverse event resulted in: Death (whatever may be the cause) | ☐ Cancer |
| Hospitalisation (*) or extension thereof | ☐ Other (any other serious clinical or laboratory event |
| Life threatening | according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) |
| DI CE CECE | Other fact to be notified: |
| | ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the m | |
| AE onset date _ (ddmmyyyy) | |
| Seriousness onset date (ddmmyyyy) | |
| Summary description (if clinical cause, significant history, progressi | on of event available laboratory results etc. ): |
| wasting description (in chinear cause, significant motory, progress) | on or event, available modulatory results, etc). |
| (*) Except hospitalisations with durations and goals planned in the pro | tocol |
| > THE SAE IN RELATION TO THE TRIAL | |
| TREATMENT NUMBER | |
| • Time of occurrence of SAE | |
| ☐ <b>During</b> the selection or run-in period | |
| ☐ <b>During</b> the administration phase of the study treatment | |
| ☐ After the administration phase of the study treatment | |
| Date of first study treatment administration | _ |
| Date of last study treatment administration | |
| before the occurence of SAE | |
| • Was the blind broken? | cable |
| Conditions of administration (cycles(s), daily dose(s), route(s) of | of administration_etc_): |
| Conditions of administration (cycles(s), daily dose(s), foute(s) | ,, william structure, ctc |

Final version 802/1185

| Transmission date | (ddmmyyyy) Country: | | | | | |
|---|---|---|---|---|---|---|
| SAE N° | SAE N° | | | | | |
| > CONCOMITANT M<br>(EXCEPT THE TRE | IEDICATION SING<br>ATMENTS GIVEN | CE TRIAL INITIATION <i>FOR THE SAE)</i> | ON and UP UNTIL TH | E OCCURRENCE O | F THE SAE | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAKE | N FOLLOWING T | HE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | , , | |
| □ Dosage modi | fication, specify : | | Modification D | ate: | //_ | |
| ☐ Temporarily | discontinued | | Readministration date | e: | //_ | |
| ☐ Withdrawn | | | End date | : | // | |
| ☐ Not applicabl | le | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription o | of corrective or symp | otomatic treatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| \ / | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Discontinuati | on of concomitant tr | reatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | / | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, specif | fy: | | | | • | |
| > OUTCOME | | | | | | |
| ☐ Not recovered/No. ☐ Recovered/Resol | lved with sequelae | ☐ Recovering/Resolvi ☐ Fatal | ing □ Recovered □ Unknown | d/Resolved | | |
| In case of deat | h, has an autopsy be | en conducted? | es 🗆 No | | | |
| > INVESTIGATOR C | AUSALITY ASSES | SSMENT (investigator | 's assessment to be don | e as soon as possible) | | |
| Study drug: | | | | | | |
| □ Not Suspected □ Suspected □ Not Suspected □ Suspected | | | | | | |

Final version 803/1185

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

## 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values (xxx)

| PARAMETERS | | UNIT | | PSC |
|---|---|---|---|---|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | - | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| 1,61141101,112 | Protein | g/1 | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pН | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 804/1185

<sup>(¤)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

#### **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | <ul> <li>Decrease of at least 2g/dl and value &lt; 10 g/dl whatever the baseline value</li> <li>If missing baseline: value &lt;10g/dl</li> </ul> |
| NEUTRO | PHILS | $\bullet$ < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC<br>(if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline: <ul> <li>TB &gt; 1.5 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>TB &gt; 2 N</li> </ul> </li> </ul> |

#### N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 805/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | HR ≥ 110 bpm and increase ≥ 10 bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>paseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| ≥ 0 | ≥ 0 | > 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the Minimum Post-baseline Value for each parameter | | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤50 | ≤90 | ≤50 | ≤50 |
| [120;140] | [80;90[ | <i>[50;75]</i> | [90 ;120] | [50;80] | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3BI 2 90 01 DBI 2 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

Table 5: Definition of orthostatic hypotension

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq$ 20 mmHg or DBP Decrease $\geq$ 10 mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 806/1185

16.1.1.8. Protocol amendment n° PA05 - General and substantial dated on 22 October 2014 linked to Protocol and appendices (version 8: 22 October 2014)

Final version 807/1185

## CLINICAL STUDY PROTOCOL AMENDMENT n° PA05 (General – Substantial)

Final version 808/1185

Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne, France

#### CLINICAL STUDY PROTOCOL AMENDMENT n° PA05

(General – Substantial)

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Pierre Fabre Study Code: F373280 CA 2 01

**EudraCT Number or equivalent:** 2012-003487-48

Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE

Sponsor's Representative: Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien 31035 TOULOUSE Cedex 1

**Pr Savina NODARI** 

Department of Clinical and Surgical Specialities, Radiological Science

and Public Health

Section of Cardiovascular Diseases

Study Coordinating Investigator: University Medical School and Spedali Civili Hospital of Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

**Date of amendment PA05:** 22OCT2014

Final version 809/1185



Study code: F373280 CA 2 01

#### APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Clinical Study Protocol Amendment nº PA05

(General – Substantial) Dated: 22OCT2014

| Sponsor's representative(s) | |
|---|---|
| Medical Director Dr Richard ROCH | Date: Signature: |
| Clinical Study Manager: Gaëlle ALCARAZ | Date; Signature: |
| Study Coordinating Investigator: Pr Savina NODAR | Date: Signature: Sorre On U |

Clinical study protocol amendment no PA05 (General - Substantial)

Date: 220CT2014


#### COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

### Clinical Study Protocol Amendment no PA05

(General – Substantial)
Dated: 22OCT2014

| <b>Country Coordinating Investigator</b> : | Date: | Signature: |
|--------------------------------------------|-------|------------|

Final version 811/1185

#### **INVESTIGATOR SIGNATURE FORM**

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

#### Clinical Study Protocol Amendment no PA05

(General – Substantial) Dated: 22OCT2014

| By my signature below, I, Dr | , hereby confirm that I have read |
|---|---|
| taken note of (and will apply) the modifications | brought by the protocol amendment n° PA05 and |
| will conduct the trial according to these new mod | dalities. |
| _ | |
| Date: | Signature: |

Final version 812/1185

#### HISTORY OF AMENDMENTS

| N° | ТҮРЕ | APPLICATION | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | AREA | | |
| NA | NΑ | General | NA | Corresponding to Protocol Version 2: Following French CA request (ANSM) and leading to protocol version 2: - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 |
| PA01 | Substantial | Local (Italy) | 01MAR2013 | Corresponding to Protocol Version 3: - Integration of the modification included in the protocol version 2 - Harmonisation of the protocol and the Informed Consent Form: • adjustment of the selection criteria n°10 related to the contraception method • addition of a letter that is given by the patient to his/her general practitioner (GP) • precision that the sponsor can not collect a copy of the Informed Consent Form • precision that the patient card is in Italian language only (without any English mention) |
| PA02 | Non<br>Substantial | General | 28MAR2013 | Corresponding to Protocol Version 4: - change of Sponsor's Representative (Clinical Study Manager), - modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed, - precision on the function and address of the International Study Coordinator Pr Nodari, - add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study), - adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage", - precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee), - correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized). - addition of the changes included in the local italian substantial protocol amendment (i.e: contraception method, letter to General Practionner, patient card |

Final version 813/1185

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | | | in Italian and no collection of the consent form by the sponsor in Italy). |
| PA03 | Substantial | General | 23OCT2013 | Corresponding to Protocol Version 5: - Fax modification of the sponsor's representatives |
| | | | | - Planned end of study postponed to January 2015. |
| | | | | - The authorized history of the first documented persistent atrial fibrillation is less than 3 years. |
| | | | | - At selection a hyperkalemia or a hypokalemia is better defined by the standards of the local laboratories. |
| | | | | - Regarding previous treatments by amiodarone the non inclusion criteria of the protocol are adapted as follow: |
| | | | | Previous treatment with oral amiodarone within 4 months prior to inclusion |
| | | | | <ul> <li>Intake of oral amiodarone for more than 1<br/>month within 4 to 12 months before<br/>inclusion</li> </ul> |
| | | | | <ul> <li>Previous treatment with intravenous<br/>amiodarone within 4 weeks prior to<br/>inclusion.</li> </ul> |
| | | | | - For male with a child-bearing potential partner (in Italy only): taking into account the duration of spermatogenesis the absolute abstention from sexual intercourse or the use of double barrier contraception method are extended to 3 months after the end of the study. |
| | | | | - Ranolazine is an antiarrhythmic treatment added to the prohibited treatments. |
| | | | | - Update of Serious Adverse Events (SAEs) form: Main change is the SAE sending: SAEs have to be reported to the Corporate Vigilance Department, and not anymore to the clinical study manager. Also SAEs can be sent by e-mail and by fax. |
| | | | | - Addition of Alpha Bioresearch as CRO involved for Feasibility, Monitoring and Regulatory issues in Spain. |
| | | | | - Correction of some minor typographic errors |
| PA04 | Non | General | 03JUN2014 | Corresponding to protocol V7: |
| | Substantial | | | <ul> <li>Precision on the temperature storage of DHA samples</li> <li>Precision on the BSA formula</li> <li>Addition of QTcB and QTcF</li> <li>Precision on TTEM recording timelines</li> <li>Clarification of the section Interim analysis and data monitoring (13.11)</li> <li>Clarifications and specifications on some</li> </ul> |
| | | | | minor points |

Final version 814/1185

#### 1. AMENDMENT RATIONALE

The purpose of this amendment is mainly to clarify some points of the protocol regarding the management of vitamin K antagonist (VKA) treatment and to decrease constraints of the study for patients.

This amendment relates also to a precision regarding the primary efficacy criterion, to an adjustment of some selection criteria in order to improve the feasibility of the study and relates to minor changes as typographical errors or style.

The clinical study protocol is updated with the following changes:

- Due to a recruitment rate lower than expected the planned end of study is postponed to April 2016.
- In order to have a better harmonization between the centres in the management of treatment with VKA some clarifications are incorporated in Chapter 8.4.6 Coagulation parameters.
- Atrial fibrillation and Atrial flutter are not the same rhythm disorder, but they are very similar and both are the expression of abnormal electrical impulses starting in the atria. So regarding the definition of the primary criterion, the atrial flutter emergence should be considered as having the same meaning as a recurrence in persistent AF. This primary criterion will be more precisely defined by the time to the first Atrial Fibrillation recurrence or Atrial Flutter emergence.
- To reduce constraints of patients follow-up, the number of scheduled visits passes from 9 to 7 and the TTEM will be weekly transmitted from week 6 to the end of the study instead of to be transmitted daily from week 6 to week 8 and then every two days from week 9 to week 24. These changes do not affect the overall risk of the study. The frequency of visits remains what is usually done in daily practice. A weekly TTEM has no impact on patient safety because on one hand patients are treated with an anticoagulant throughout the study and on the other hand a TTEM can be performed at any time in case of AF or atrial flutter symptoms.
- Patients must have a previous history of a first documented persistent Atrial Fibrillation without limitation in time instead of no longer than 3 years. This modification will expand the target population without changing the characteristics of the selected patients by enabling the management of patients who could experience a long period without AF relapse nor atrial flutter emergence.
- Patients must have a systolic heart failure defined by a reduced ventricular ejection fraction and or defined also through other echocardiographic parameters mentioned in the ESC guidelines for the diagnosis and treatment of acute and chronic heart failure (2012).
- Regarding previous prohibited treatments by amiodarone or droderanone, the non inclusion criteria of the protocol are adapted as follow:
  - Concomitant treatment with oral amiodarone or dronedarone from selection
  - Concomitant treatment with intravenous amiodarone from selection

Final version 815/1185

Despite the long half life of amiodarone, these time limits relating to its non-use before inclusion should not interfere in a major way with the assessment of the product 6 months after inclusion.

Final version 816/1185

#### 2. CHANGES DESCRIPTION

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| CLINICAL RESEARCH ORGANISATIONS | CLINICAL RESEARCH ORGANISATIONS |
| For Feasibility, Monitoring and Regulatory issues: Pharmaceutical Service Network (PSN) Rufino Gonzalez 28 037 Madrid - SPAIN Phone: +34 91 375 6930 - Fax: +34 91 375 6931 E-mail: www.psnglobal.org | For Feasibility, Monitoring and Regulatory issues (in Hungary, Czech Republic and Italy): Pharmaceutical Service Network (PSN) Rufino Gonzalez 28 037 Madrid - SPAIN Phone: +34 91 375 6930 - Fax: +34 91 375 6931 E-mail: rzurita@psnglobal.org |
| For refund of patients expenses linked to the study (in France): CLINACT 6-10 rue TROYON 92310 SEVRES – FRANCE Phone: +33 1 46 90 27 27 - Fax: +33 1 46 23 01 56 Email: sebastien.beaumont@clinact.com | For refund of patients expenses linked to the study (in France): CLINACT 6-10 rue TROYON 92310 SEVRES — FRANCE Phone: +33 1 46 90 27 27 — Fax: +33 1 46 23 01 56 Email: sebastien.beaumont@clinact.com |
| SYNOPSIS | SYNOPSIS |

Planned Study Period: January 2013 – January 2015

#### Methodology:

- Start of treatment 4 weeks before ECV
  - Condition to ECV:
  - INR 2-3 (anti-vitamin K should be given at least 3 weeks before ECV)
  - No spontaneous cardioversion before ECV
- Cardiac monitoring:
  - TTEM: daily transmission from week 6 to week 8; then every two days from week 9 to week 24, and in case of AF symptoms.

#### **Study Schedule:**

9 visits will be scheduled:

- V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)
- V2/D1: Inclusion visit (start of study treatment)
- V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to clinical

Planned Study Period: January 2013 – April 2016

#### Methodology:

- Start of treatment 4 weeks before ECV
  - Condition to ECV:
  - Ideally INR 2-3 (vitamin K antagonist should be given at least 3 weeks before ECV)
  - No spontaneous cardioversion before ECV
- Cardiac monitoring:
- TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms.

#### **Study Schedule:**

7 visits will be scheduled:

- V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)
- V2/D1: Inclusion visit (start of study treatment)
- V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to clinical practice of the

Final version 817/1185

#### PREVIOUS VERSION

practice of the centre) (installation of the Holter device)

- V4/W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)
- V5/W8 (D56± 7 days): follow-up visit
- V6/W12 (D84  $\pm$  7 days): follow-up visit
- V7/W16 (D112  $\pm$  7 days): follow-up visit
- V8/W20 (D140  $\pm$  7 days): follow-up visit
- V9/W24 (D168  $\pm$  7 days): final study visit

#### **Diagnosis and Criteria for Inclusion:**

#### **Inclusion Criteria:**

Demographic Characteristics and Other Baseline Characteristics:

[...]

- 3. History of first documented persistent AF less than 3 years.
- 4. History of ischemic or non ischemic heart failure

[...]

6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion

[...]

#### **MODIFIED VERSION**

centre) (installation of the Holter device)

- V4/W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)
- V5/W8 (D56± 7 days): follow up visit
- V6/W12 (D84  $\pm$  7 days): follow-up visit
- V7/W16 (D112  $\pm$  7 days): follow-up visit
- $\frac{V8}{W20}$  (D140 ± 7 days): follow up visit
- V9/W24 (D168  $\pm$  7 days): final study visit

#### **Diagnosis and Criteria for Inclusion:**

#### **Inclusion Criteria:**

Demographic Characteristics and Other Baseline Characteristics:

[...]

- Previous history of first documented episode of persistent AF
- 4. **Previous** history of ischemic or non ischemic heart failure

[...]

- 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF)  $\geq$  30% and  $\leq$  45% or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size  $(diameter \geq 60~mm~and/or > 32~mm/m^2~and/or~volume > 97~ml/m^2)$
  - and/or an increased left ventricular endsystolic size

(diameter > 45 mm and/or > 25 mm/m $^2$  and/or volume > 43 ml/m $^2$ )

• and/or a reduced left ventricular outflow tract velocity time integral < 15 cm

[...]

Final version 818/1185

#### PREVIOUS VERSION MODIFIED VERSION Non-Inclusion Criteria: Non-Inclusion Criteria: Criteria related to pathologies: Criteria related to pathologies: 1. History of first documented episode of persistent AF 1. No previous history of first documented episode of more than 3 years persistent AF [...] [...] Criteria related to treatments: Criteria related to treatments: 12. Concomitant treatment with ranolazine or any 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calciumexcept amiodarone, dronedarone and stable dose of blockers digoxin, betablockers, calcium-blockers 13. Oral amiodarone: 13. Concomitant treatment with oral amiodarone or 13a Previous treatment with oral amiodarone within dronedarone from selection 4 months prior to inclusion 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion 14. Previous treatment with intravenous amiodarone 14. Concomitant treatment within 4 weeks prior to inclusion

[...]

19. Patient treated with other anticoagulant treatment than antivitamin K: thrombin inhibitor such as Dabigatran or treated with antiaggregant P2Y12 inhibitors such as Clopidogrel or Prasugrel

#### **Exclusion criteria before V3:**

Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO -TE (trans-esophageal echocardiograph) performed in the same day (before ECV)

ECV will be performed in patients without dyskalemia

with intravenous

[...]

19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel

#### **Exclusion criteria before V3:**

amiodarone from selection

Patients without dyskalemia who will not have INR values  $\geq 2$  on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study.

However, if only 2 INR values are  $\geq$  2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal echocardiography) performed on the

Final version 819/1185

#### PREVIOUS VERSION

If necessary for obtaining stabilized INR between 2 and 3, the ECV (and following visits) could be postponed by 7 days.

[...]

#### **Evaluation Criteria:**

#### **Efficacy evaluation variables:**

Primary evaluation variable:

 Time to first Atrial Fibrillation recurrence defined by the first episode of AF lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 – ECV visit).

Handling of AF recurrences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: daily transmission from week 6 to week 8. Then, every two days from week 9 to week 24.

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

Moreover, during this TTEM period, if patient experiences any AF symptoms, it should be recorded and documented using the TTEM.

All ECG traces will be evaluated by a Central Reading Laboratory.

[...]

#### **Statistical Methods:**

#### **Sample Size:**

Assuming an AF recurrence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per

#### **MODIFIED VERSION**

same day (before ECV) and the patient can continue the study.

If necessary, **for meeting these INR conditions**, the ECV (and following visits) could be postponed by 7 days.

[...]

#### **Evaluation Criteria:**

#### **Efficacy evaluation variables:**

Primary evaluation variable:

- Time to first Atrial Fibrillation recurrence **or atrial flutter emergence** defined by the **time to** first episode of AF **or atrial flutter** lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 – ECV visit).

Handling of AF recurrences or atrial flutter emergences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5).

Moreover, during this TTEM period, if patient experiences any AF **or atrial flutter** symptoms, it should be recorded and documented using the TTEM.

All ECG (Holter and TTEM) will be evaluated by a Central Reading Laboratory.

[...]

#### **Statistical Methods:**

#### **Sample Size:**

Assuming an AF recurrence or atrial flutter emergence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76

Final version 820/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. | randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%. |
| STUDY FLOW CHART | STUDY FLOW CHART |

#### STUDY FLOW CHART

Please see flow-chart of previous version in appendix 1

#### 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

[...]

During the study, in case of AF recurrence that would require cardioversion or the introduction of an antiarrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped.

[...]

- ECV in patients with stabilized INR (i.e. values between 2 and 3;sp to ) on at least 3 consecutive weekly tests performed. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests performed before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO -TE (trans-esophageal echocardiograph) performed in the same day (before ECV). Patients who do not revert to sinus rhythm or present an early relapse within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be scheduled at least every month. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored between visits using daily, then every 2 days Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

[...]

## Please see flow-chart of modified version in appendix 2

ETHICAL CONSIDERATIONS RELATING

[...]

TO THE STUDY

During the study, in case of AF recurrence or atrial flutter emergence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped.

[...]

- ECV will be performed in patients with AF and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values  $\geq 2$  on the 3 last tests performed before ECV are required. However, if only 2 INR values are  $\geq$  2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Patients who do not revert to sinus rhythm or present an early AF relapse or an early atrial flutter emergence within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be performed throughout the study period. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored once a week between visits using Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading

Final version 821/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|------------------|------------------|
| | Laboratory. |
| | [] |

#### 4. STUDY DESIGN

#### 4.1 OVERALL DESCRIPTION

[...]

Nine visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow-up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140  $\pm$  7D): follow-up visit
- Visit 9 (V9): W24 (D168 ± 7D): final study visit
   [...]

#### 4.2. DISCUSSION OF THE STUDY DESIGN

#### 4.2.1. Choice of the Study Population

[...]

The study aim is to investigate the product effect in patients with:

- Persistent AF history (less than three years) with a duration of the current episode from 7 days to 6 months.
- a moderately abnormal systolic heart failure (Left Ventricular Ejection Fraction (LVEF) between 30 to 45% as defined in the report from the American Society of Echocardiography's Guideline).

#### 4. STUDY DESIGN

#### 4.1 OVERALL DESCRIPTION

[...]

**Seven** visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28 -2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)
- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 5 (V5): W8 (D56  $\pm$  7D): follow up visit
- Visit 6 (V6): W12 (D84  $\pm$  7D): follow-up visit
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 8 (V8): W20 (D140 ± 7D): follow up visit
- Visit 9 (V9): W24 (D168 ± 7D): final study visit
   [...]

#### 4.2. DISCUSSION OF THE STUDY DESIGN

#### 4.2.1. Choice of the Study Population

[...]

The study aim is to investigate the product effect in patients with:

- **Previous history of persistent AF** with duration of the current episode from 7 days to 6 months.
- A systolic heart failure defined by a reduced left ventricular ejection fraction (≥ 30% and ≤ 45%) or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size
     (diameter ≥ 60 mm and/or > 32 mm/m² and/or

Final version 822/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| [] - a Left Atrial Area (LAA) not severely abnormal (less than 40 cm2 as defined in the report from the American Society of Echocardiography's Guideline). | <ul> <li>volume &gt; 97 ml/m²),</li> <li>and/or an increased left ventricular end-systolic size (diameter &gt; 45 mm and/or &gt; 25 mm/m² and/or volume &gt; 43 ml/m²),</li> <li>and/or a reduced left ventricular outflow tract velocity time integral &lt; 15 cm [23, 24].</li> <li>[]</li> <li>A Left Atrial Area (LAA) not severely abnormal (no greater than 40 cm2 as defined in the report from the American Society of Echocardiography's Guideline) [23].</li> </ul> |
| 4.2.2. Choice of the Study Design | 4.2.2. Choice of the Study Design |
| [] According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF since cardioversion. To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit. Eligible participants will enter a selection phase in which anticoagulant treatment (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2.0 to 3.0 before ECV. According to guidelines for the management of AF [6], AVK should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion. [] | According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF (or emergence of atrial flutter) since cardioversion. To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit. Eligible participants will enter a selection phase in which anticoagulant treatment (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) of 2 to 3 before ECV. According to guidelines for the management of AF [6], VKA should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion. [] |
| Finally, during the study, patients will be scheduled for a clinical visit every month (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters. | Finally, during the study, patients will be scheduled for a clinical visit every <b>4 weeks or 8 weeks</b> (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety |

Final version 823/1185

[...]

parameters.

[...]

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 5. STUDY POPULATION 5.1 INCLUSION CRITERIA | 5. STUDY POPULATION 5.1 INCLUSION CRITERIA |
| Demographic Characteristics and Other Baseline Characteristics: | Demographic Characteristics and Other Baseline Characteristics: |
| <ul> <li>[]</li> <li>3. History of first documented persistent AF less than 3 years</li> <li>4. History of ischemic or non ischemic heart failure</li> <li>[]</li> </ul> | <ul> <li>[]</li> <li>3. Previous history of first documented episode of persistent AF</li> <li>4. Previous history of ischemic or non ischemic heart failure</li> </ul> |
| 6. Reduced left ventricular ejection fraction between 30% and 45% inclusive (using the two-dimensional echocardiography biplane Simpson's rule) at selection and at inclusion [] | <ul> <li>[]</li> <li>6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF) ≥ 30% and ≤ 45% or for patients with a LVEF &gt; 45%:</li> <li>• an increased left ventricular end-diastolic size (diameter ≥ 60 mm and/or &gt; 32 mm/m² and/or volume &gt; 97 ml/m²)</li> <li>• and/or an increased left ventricular end-systolic size (diameter &gt; 45 mm and/or &gt; 25 mm/m² and/or volume &gt; 43 ml/m²)</li> </ul> |
| | and/or a reduced left ventricular outflow tract velocity<br>time integral < 15 cm [] |

Final version 824/1185

#### PREVIOUS VERSION MODIFIED VERSION 5.2 NON INCLUSION CRITERIA 5.2 NON INCLUSION CRITERIA Criteria related to pathologies: Criteria related to pathologies: 1. History of first documented episode of persistent AF 1. No previous history of first documented episode more than 3 years, of persistent Atrial Fibrillation [...] [...] Criteria related to treatments: Criteria related to treatments: [...] [...] 12. Concomitant treatment with ranolazine or any 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), antiarrhythmic drug (within 7 days prior to selection), except stable dose of digoxin, betablockers, calciumexcept amiodarone, dronedarone and stable dose of blockers digoxin, betablockers, calcium-blockers 13. Oral amiodarone: 13. Concomitant treatment with oral amiodarone or 13a Previous treatment with oral amiodarone within dronedarone from selection 4 months prior to inclusion 13b Intake of oral amiodarone for more than 1 month within 4 to 12 months before inclusion 14. Previous treatment with intravenous amiodarone 14. Concomitant treatment with intravenous within 4 weeks prior to inclusion amiodarone from selection [...] [...] 19. Patient treated with oral anticoagulant treatment other 19. Patient treated with other anticoagulant treatment than than vitamin K antagonist: new oral anticoagulants antivitamin K: thrombin inhibitor such as Dabigatran (dabigatran, rivaroxaban, apixaban), or treated with or treated with antiaggregant P2Y12 inhibitors such as irreversible antiplatelet agents P2Y12 inhibitors such as Clopidogrel or Prasugrel ticlopidine, clopidogrel or prasugrel 5.6 WITHDRAWAL CRITERIA 5.6 WITHDRAWAL CRITERIA [...] [...] • Erroneous inclusion according to the study protocol. Erroneous inclusion according to the study protocol.

Final version 825/1185

Any inclusion not respecting inclusion/non inclusion

criteria will immediately be withdrawn and an

appropriate treatment will be given by the investigator

The decision to maintain or not the patient in the

study will be taken jointly by the investigator and the

sponsor. Erroneous inclusions will not be paid to the

#### PREVIOUS VERSION

under his/her responsibility. Erroneous inclusions will not be paid to the investigator.

- Patients who could not be treated with AVK for at least 3 weeks before ECV.
- Patients who will not have a stabilized INR between 2 and 3 on at least 3 consecutive weekly tests.
- Patients with only 2 consecutives INR tests between 2 and 3 in the last 3 weeks for whom a transoesophagoal echocardiography can not be performed before ECV or for whom a trans-oesophagoal echocardiography shows a thrombus in the atria.
- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early relapse within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance.

[...]

#### **MODIFIED VERSION**

investigator.

- Patients who could not be treated with VKA for at least
   3 weeks before ECV or who will experience a VKA intolerance during the study.
- Patients without dyskalemia who will not have INR values ≥ 2 on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study. However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study.
- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early AF relapse or early atrial flutter emergence within the observation period after ECV will be considered to have finished follow-up.
- Occurrence of AF recurrence or atrial flutter emergence that would require, at the investigator's judgement, a cardioversion or an introduction of an antiarrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance.

[...]

#### 6. STUDY TREATMENT

#### 6.2. PACKAGING AND LABELLING

#### 6.2.1. Packaging

[...]

The Investigator will provide the patient with the treatment according to the following schedule:

At Inclusion Visit (V2): a 12-week treatment unit will contain 3 cases, each case containing:

- 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

At Visit 6 (V6): a 12-week treatment unit will contain 3 cases, each case containing:

#### 6. STUDY TREATMENT

#### 6.2. PACKAGING AND LABELLING

#### 6.2.1. Packaging

[...]

**Two** 12-week treatment units will contain 3 cases, each case of **4-week treatment** containing: 10 blister packs of four 1 g F373280 soft capsules or **1 g** placebo soft capsules each.

[...]

Final version 826/1185

# PREVIOUS VERSION - 10 blister packs of four 1 g F373280 soft capsules or placebo soft capsules each.

#### **MODIFIED VERSION**

[...]

## 6.4 ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

[...]

Practically, once patient's eligibility is confirmed at selection visit (V1):

- The Investigator:
  - Contacts the IVRS/IWRS
  - Answers the questions relating to the patient
  - In return, the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

[...]

The Investigator will dispense to the patient the case which label indicates the treatment number and the administration period.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment according to the same process as described above.

## 6.4 ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

[...]

At selection visit (V1), practically, once patient's eligibility is confirmed:

- The Investigator:
  - Contacts the IVRS/IWRS
  - Answers the questions related to the patient

[...]

At inclusion visit (V2), the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment according to the same process as described above.

The Investigator will dispense to the patient the 4-week treatment cases (one or two according to the visit) which label indicates the treatment number and the administration period.

#### 7. CONCOMITANT TREATMENTS

#### 7.1. ANTI-VITAMIN K TREATMENT

AVK should be given for at least 3 weeks before ECV and continued for the whole study duration. The AVK used will be left to the decision of the each Investigator according to his/her local practice.

#### 7. CONCOMITANT TREATMENTS

#### 7.1. <u>VITAMIN K ANTAGONIST</u> TREATMENT

VKA should be given for at least 3 weeks before ECV and continued for the whole study duration. However, VKA should be stopped in case of occurrence of VKA intolerance during the study and the patient should be withdrawn from the study. The VKA used will be left to the decision of each Investigator according to his/her local practice.

Final version 827/1185

#### PREVIOUS VERSION MODIFIED VERSION 7.2. PROHIBITED TREATMENTS 7.2. PROHIBITED TREATMENTS Any anticoagulant treatment other than AVK: thrombin Any oral anticoagulant treatment other than VKA: new inhibitor such as Dabigatran or antiaggregant P2Y12 anticoagulants oral (dabigatran, rivaroxaban. inhibitors such as Clopidogrel or Prasugrel apixaban), or irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel [...] [...]

#### 8. EVALUATION CRITERIA

#### 8.1 PRIMARY EFFICACY CRITERIA

## 8.1.1. Time to the first Atrial Fibrillation Recurrence 8.1.1.1. Definition

Time to first AF recurrence is defined by the first episode of AF (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. Schedule

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF will be assessed after visit 3 (week 5).

#### 8.1.1.3. Evaluation Methods

[...]

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: daily transmission from the day after visit 4 (week 6) to visit 5 (week 8). Then every two days from the day after visit 5 (week 9) to visit 9 (week 24 – End of study).

Moreover, if patient experiences AF symptoms during this TTEM period, it should be documented using the TTEM. In case of AF recurrence and provided that the patient does not require a cardioversion or an introduction of an anti-

#### 8. EVALUATION CRITERIA

#### 8.1 PRIMARY EFFICACY CRITERIA

8.1.1. Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence

#### **8.1.1.1. Definition**

Time to first AF recurrence **or atrial flutter emergence** is defined by the **time to** first episode of AF **or atrial flutter** (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. Schedule

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5).

#### 8.1.1.3. Evaluation Methods

[...]

• Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM.

Moreover, if patient experiences AF **or atrial flutter** symptoms during this TTEM period, it should be documented using the TTEM.

Final version 828/1185
arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

The TTEM will be centralized by the Central Reading Laboratory. The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM. The TTEM will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign this document.

The TTEM process will be fully described in a separate document.

#### **MODIFIED VERSION**

In case of AF recurrence **or atrial flutter emergence** and provided that the patient does not require a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

• Process of centralisation of ECG (Holter and TTEM)

**ECG** (Holter and TTEM) will be centralized by the Central Reading Laboratory. The **ECG** will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign these documents.

The **Holter and** TTEM process will be fully described in separate documents.

Final version 829/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| 8.1.2 Secondary Efficacy Criteria | 8. 2 SECONDARY EFFICACY CRITERIA |
| 8.1.2.3. Clinical parameters evaluation | 8.2.3. Clinical parameters evaluation |
| 8.1.2.3.1. EHRA score assessment | 8.2.3.1. EHRA score assessment |
| 8.1.2.3.1.3. Evaluation Methods | 8.2.3.1.3. Evaluation Methods |
| EHRA evaluation will be collected by Central Reading | EHRA evaluation will be collected by Central Reading |
| Laboratory during all the study period. | Laboratory during TTEM period. |
| | 8.2.3.2. Time to first AF recurrence less than 10 minutes Time to first AF recurrence less than 10 minutes will be assessed during TTEM period. |
| 8.1.2.3.2. Number of recurrence of symptomatic AF | 8.2.3.3 Recurrence of symptomatic AF |
| It consists of the number of AF recurrences associated with | Recurrence of symptomatic AF will be assessed during |
| a symptom (palpitation, fatigue, dizziness, dyspnea, chest | TTEM period. |
| pain and anxiety) and confirmed by an ECG. | The number of recurrences of symptomatic AF consists |
| pain and annety) and committee by an 200. | of the number of AF recurrences associated with a |
| | symptom (palpitation, fatigue, dizziness, dyspnea, chest |
| | pain and anxiety) and confirmed by an ECG. |
| | The time to first symptomatic AF recurrence is defined |
| | by the time to first episode of symptomatic AF. |
| 8.2. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA 8.2.2 Blood samples | 8.3. BIOMARKER ASSESSMENT: RED BLOOD<br>CELL CONCENTRATIONS OF DHA<br>8.3.2 Blood samples |
| 8.2.2.2. Technical handling | 8.3.2.2. Technical handling |
| Two blood samples (4 ml) will be collected in EDTA tubes. They will be gently shaken, stored between +2°C/+8°C in a fridge (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions | Two blood samples (2 x 4 ml) will be collected in EDTA tubes. They will be homogenized slowly by inverting the tube without shaking, stored between +2°C/+8°C in a fridge (no freezing will be allowed) and sent to Analytical |
| (between +2°C and +8°C). | Centre in refrigerated conditions (between +2°C and +8°C). |
| [] | [] |

Final version 830/1185

[...]

#### PREVIOUS VERSION MODIFIED VERSION 8.3 SAFETY ASSESSMENT **8.4 SAFETY ASSESSMENT 8.3.2** Laboratory Investigations 8.4.2 Laboratory Investigations 8.3.2.2 Technical Procedures and Parameters 8.4.2.2 Technical Procedures and Parameters [...] Haematology: hematocrit, haemoglobin, RBC count, Haematology: haematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC white blood cells (WBC) count, WBC differential counts (% and absolute), differential counts (% and/or absolute), reticulocytes, platelets. reticulocytes, platelets. Chemistry: [...] **Biochemistry** [...] Additional tests may be done at the Investigator's Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal discretion, in the patient's interest. In case of any abnormal or clinically significant results, the Investigator will order and/or clinically significant results, the Investigator should laboratory control tests. order laboratory control tests. 8.3.3. Global Physical Examination 8.4.3. Global Physical Examination A global physical examination including the measurement A global physical examination including the measurement of body weight will be carried out on each body system at of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 1, visit 2, visit 3, visit 4, visit 5, visit 6, visit 7, visit 8 visit 9. and visit 9 [...] [...].

# 8.3.5. Electrocardiogram (ECG)

#### 8.3.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

[...]

#### 8.3.6 Coagulation parameters

[...]

During the pre-cardioversion period, if the anticoagulation by AVK should be initiated, then the INR monitoring will be as follow:

INR 2-3 times a week for the first week of treatment

Electrocardiogram (ECG)

### 8.4.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9 using an usual standardised 12-lead cardiograph.

[...]

8.4.5.

#### 8.4.6 Coagulation parameters

[...]

The recommendations for the controls of INR are the following [25, 26]:

1) During the pre-cardioversion period, if the anticoagulation by VKA has to be initiated, the treatment must be initiated at least 3 weeks prior to

Final version 831/1185

- INR weekly up to ECV
- INR every 4 weeks after ECV

For patients already treated with AVK, INR monitoring will be as follow:

- INR weekly up to ECV
- INR every 4 weeks after ECV

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9.

Anti-coagulation by AVK should be given at least 3 weeks before ECV and continued for the whole study duration. The quantity of blood samples collected at each time for coagulation parameters will be 2 mL.

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal or clinically significant results, the Investigator will order laboratory control tests.

[...]

#### MODIFIED VERSION

cardioversion then the INR will be monitored as follow:

- The adjustment of the dosage of VKA should be performed stepwise by controlling INR 2 to 3 times a week until stabilization within the target range (2 - 3) on 2 successive tests.
- When the INR is within the target range (2 3) on 2 successive tests, the dose of VKA should be maintained. Then the controls of INR will be progressively spaced within a few weeks.
- When INR is stabilized, at least one test should be performed each week.
- In all cases, an INR control must be performed within 24 h before ECV.
- 2) During the pre-cardioversion period, if the anticoagulation by VKA was already initiated, the INR will be monitored as follow:
  - One INR per week up to ECV
  - An INR control must be performed within 24 h before ECV
- 3) After cardioversion : one INR each month
- 4) Throughout the duration of the study if INR > 3 the advocated actions are:
- No transesophageal echocardiography before cardioversion
- For asymptomatic patients:
  - 3 < INR < 4: no omission of VKA (dose adjustment if required), no vitamin K
  - $4 \le INR < 6$ : omit one dose of VKA, no vitamin K
  - 6 ≤ INR < 10: interrupt VKA, vitamin K 2 mg orally
  - INR  $\geq$  10: interrupt VKA, vitamin K 5 mg orally

For INR  $\geq$  6, an adverse event has to be reported (asymptomatic overdose).

Anti-coagulation by **VKA** should be given at least 3 weeks before ECV and continued for the whole study duration.

Final version 832/1185

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| | aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 5, visit 6, visit 7, visit 8 and visit 9. The quantity of blood samples collected at each time for coagulation parameters will be 2 ml. |
| | Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests. [] |
| 9.4 CONCOMITANT TOEATMENTS | 9.5. CONCOMITANT THE ATMENTS |

#### 8.4 CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements relating to patient's concomitant treatments started before screening visit and continued throughout the trial, or started during the trial, can be found in section 7.

#### 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week - 4 to Week -1):

[...]

• The patient will enter the selection period in which anticoagulant (AVK) will be adjusted to achieve an International Normalized Ratio (INR) of 2 to 3 before ECV.

[...]

The patient will receive from the investigational centre the study card to be kept for the duration of the study.

#### Visit 2 - Inclusion Visit (Day 1)

If the patient's behaviour during the selection period and/or the result of complementary examinations, particularly the confirmation of the presence of persistent AF by the

#### 8.5 CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements related to patient's concomitant treatments started before **selection** visit and continued throughout the trial, or started during the trial, can be found in section 7.

#### 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week - 4 to Week -1):

[...]

• The patient will enter the selection **and precardioversion** periods in which anticoagulant **(VKA)** will be adjusted to achieve **ideally** an International Normalized Ratio (INR) **in the range** of 2 to 3 before ECV.

[...]

The patient will receive from the investigational centre the **participant** card to be kept for **all** the duration of the study.

#### Visit 2 - Inclusion Visit (Day 1):

If the patient's behaviour during the selection period and/or the result of complementary examinations, particularly the confirmation of the presence of persistent AF by the Central

Final version 833/1185

Central Reading Laboratory during this period, the INR and laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

[...]

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and allocated a treatment number using the IVRS/IWRS.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.3.6) in order to ensure that the INR is stable (between 2 to 3 before electrical cardioversion).

[...]

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period.

#### Vist 3 (Week 4: D28 -2/+7 days) cardioversion

[...]

Electrocardioversion (ECV): ECV has to be scheduled 4 weeks after randomization and after target International Normalized Ratio levels will be stabilized (between 2 and 3) on at least 3 consecutive weekly tests in patients with AF. Patients not stabilized for INR (i.e. values not between 2 and 3) on at least 3 consecutive weekly tests before ECV will be excluded from the study, unless the presence of atrial thrombosis may be excluded with ECHO –TE performed in the same day (and before ECV). ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia.

[...]

Patients who will not revert to sinus rhythm or with early relapse within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

[...]

#### **MODIFIED VERSION**

Reading Laboratory during this period, the INR and the laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

[...]

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 2 for the first 12-week period.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.4.6) in order to fulfil the ECV conditions (refer to paragraph 3).

[...]

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period (one case of treatment).

#### Vist 3 (Week 4: D28 -2/+7 days) cardioversion

[...]

Electrocardioversion (ECV): ECV has to be performed 4 weeks after randomization in patients with AF. ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values  $\geq 2$  on the 3 last tests performed before ECV are required. However, if only 2 INR values are  $\geq 2$  among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study.

[...]

Patients who will not revert to sinus rhythm or with early AF relapse or early atrial flutter emergence within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-

Final version 834/1185

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week period.

[...]

#### Visit 4 (Week 5: D35 -2/+7 days)

[...]

The patient will be requested to perform daily transmission from the day after visit 4 (week 6) to visit 5 (week 8), then every two days from the day after visit 5 (week 9) to visit 9 (week 24 – End of study). Moreover, in case of AF symptoms, additional transmissions may be performed.

[...]

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days)

[...]

Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV, the monitoring of INR, aPTT and TCT should be stopped.

[...]

• The cardiac monitoring will be continued using a TTEM device. The device will be given to the patient who will be requested to perform daily transmission from the day after visit 4 (week 6) to visit 5 (week 8), then every two days from the day after visit 5 (week

#### **MODIFIED VERSION**

up.

[...]

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 8-week period (two cases of treatment).

[...]

Visit 4 (Week 5: D35 -2/+7 days)

[...]

The patient will be requested to perform one transmission per week from this visit (initial call to perform with the patient) to the visit 9 (week 24 – end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

[...]

Visit 5 (Week 8: D56  $\pm$  7 days) – Visit 6 (Week 12: D84  $\pm$  7 days) - Visit 7 (Week 16: D112  $\pm$  7 days) - Visit 8 (Week 20: D140  $\pm$  7 days):

[...]

Laboratory examination: Prothrombin Time/INR
 (PT/INR), Activated Partial Thromboplastin Time
 (aPTT), Thrombin Clotting Time (TCT). However, in
 case of discontinuation of anticoagulation after ECV
 due to occurrence of VKA intolerance, the
 monitoring of INR, aPTT and TCT should be stopped.

[...]

The cardiac monitoring will be continued using the TTEM device through one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may

Final version 835/1185

9) to visit 9 (week 24 – End of study). Moreover, in case of AF symptoms, additional transmissions may be performed.

[...]

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 4-week treatment period.

In addition,:

- at visit 6:
- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

[...]

End-of-Study Visit - Visit 9 (Week 24: D168  $\pm$  7 days):

[...]

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused soft capsules

[...]

#### **MODIFIED VERSION**

be performed.

[...]

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

In addition, at visit 6:

- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

At the end of each visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next treatment period: one case at visit 6 and two cases at visit 7.

[...]

Visit 9 - End-of-Study Visit (Week 24: D168  $\pm$  7 days):

[...

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused soft capsules.

The total volume of blood collected should be about 90 mL for the study duration (30 mL for the total volume of haematology and biochemistry, 2 mL for each blood samples for coagulations parameters and 4 mL for each blood samples of DHA).

[...]

Final version 836/1185

#### PREVIOUS VERSION MODIFIED VERSION 13. STATISTICAL ANALYSIS 13. STATISTICAL ANALYSIS 13.2. SAMPLE SIZE 13.2. SAMPLE SIZE Assuming an AF recurrence or flutter emergence rate of Assuming an AF recurrence or atrial flutter emergence 85% under placebo and 65% under active group, i.e. a rate of 85% under placebo and 65% under active group, i.e. clinically relevant difference $\Delta$ of 20%, a sample size of 64 a clinically relevant difference $\Delta$ of 20%, a sample size of assessable patients per group is required, using a log-rank 64 assessable patients per group is required, using a logtest of survival curves with a 80 % power and a 5 % tworank test of survival curves with a 80 % power and a 5 % sided significance level. two-sided significance level. 13.7. EFFICACY ANALYSIS 13.7. EFFICACY ANALYSIS 13.7.1. Primary Criterion 13.7.1. Primary Criterion 13.7.1.1. Primary Analysis 13.7.1.1. Primary Analysis The primary criteria, time to first recurrence, will be The primary criteria, time to first recurrence of AF or analysed using the Kaplan Meier method and compared atrial flutter emergence, will be analysed using the with the Log rank test. Hazard ratios and 95% confidence Kaplan Meier method and compared with the Log rank test. intervals will be estimated with the Cox regression model. Hazard ratios and 95% confidence intervals will be [...] estimated with the Cox regression model. [...] 13.7.2. Secondary Criteria 13.7.2. Secondary Criteria 13.7.2.1. Numbers of Atrial Fibrillation Episodes 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the [...] first week following V3 [...] 13.7.2.2. Duration of Atrial Fibrillation Episodes [...] 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3 [...] 16. REFERENCES 3 added references: [24]. **JOHN** J.V. MCMURRAY, **STAMATIS** ADAMOPOULOS, STEFAN D. ANKER, ANGELO AURICCHIO, MICHAEL BÖHM, KENNETH DICKSTEIN, VOLKMAR FALK, GERASIMOS FILIPPATOS, CÂNDIDA FONSECA, MIGUEL ANGEL GOMEZ-SANCHEZ, TINY JAARSMA. LARS KØBER, GREGORY Y.H. LIP, ALDO **PIETRO** MAGGIONI. ALEXANDER BURKERT M. PARKHOMENKO, PIESKE.

Final version 837/1185

BOGDAN A. POPESCU, PER K. RØNNEVIK, FRANS H. RUTTEN, JUERG SCHWITTER, PETAR SEFEROVIC, JANINA STEPINSKA, PEDRO T.

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| | TRINDADE, ADRIAAN A. VOORS, FAIEZ<br>ZANNAD, ANDREAS ZEIHER |
| | ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012 European Heart Journal (2012) 33, 1787–1847 |
| | [25]. AGENCE NATIONALE DE SECURITE DU MEDICAMENT ET DES PRODUITS DE SANTE (ANSM). |
| | Bon usage des médicaments antivitamine K (AVK) Actualisation – Juillet 2012 |
| | [26]. GILLES PERNOD, ANNE GODIER, CLAIRE<br>GOZALO, BENJAMIN TREMEY, PIERRE SIE |
| | French clinical practice guidelines on the management of patients on vitamin K antagonists in at-risk situations (overdose, risk of bleeding, and active bleeding) Thrombosis Research 126 (2010) e167–e174 |

Final version 838/1185

# ANNEXE 1 STUDY FLOW-CHART FROM PROTOCOL VERSION 7

Final version 839/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W8<br>(56+/-7D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W20<br>(140+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | X | X | x | Х | X | Х | Х | X | Х |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | X | X | Х | | Х | х | x | X | Х |
| Echocardiography | Х | X | | Х | | Х | | | Х |
| Eligibility criteria check | Х | X | | | | | | | |
| Blood pressure, heart rate | Х | X | Х | Х | Х | Х | Х | Х | Х |
| 12-Lead ECG Recording | Х | X | Х | | X | Х | Х | Х | Х |
| INR | | | (2) | | Х | Х | Х | Х | Х |
| aPTT, TCT | х | X | х | | Х | х | х | x | Х |
| Biochemistry | X | | | | | | | | X |
| Hematology | Х | | х | | | Х | | | Х |
| Urinary pregnancy test | | X | | | | | | | Х |
| Red Blood Cell concentrations of DHA | | X | Х | | | х | | | X |
| Treatment allocation | | X | | | | Х | | | |
| IVRS/IWRS | Х | X | | | | Х | | | |
| ECV (3) | | | x | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | x | x | x | Х | Х | Х | Х | Х |
| Holter ECG | <b>←</b> → <sup>(4)</sup> | | <b>←</b> | (5) | | | | | |
| TTEM (6) | | | | + | | | | | |

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of AVK introduction: INR 2 to 3 times a week, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(6) 24-</sup>hour Holter ECG
(6) 7-day Holter ECG
(6) TTEM: everyday from week 6 to week 8; then every 2 days from week 9 to week 24; at any time in case of AF symptoms. In case of AF recurrence for at least 10 minutes and if the patient does not stop the study treatment, then TTEM once a week

# ANNEXE 2 STUDY FLOW-CHART FROM PROTOCOL VERSION 8

Final version 841/1185

| F373280 CA 201 | V1 | V2 | V3 | V4 | V6 | V7 | V9 |
|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | W12<br>(84+/-7D) | W16<br>(112+/-7D) | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | |
| Informed consent | Х | | | | | | |
| Demographic characteristics | х | | | | | | |
| Medico-surgical history | х | | | | | | |
| Concomitant disease | х | | | | | | |
| Concomitant treatment | х | Х | Х | Х | Х | Х | Х |
| Habits | х | | | | | | |
| Global physical examination (body weight) | х | Х | Х | | Х | Х | Х |
| Echocardiography | х | Х | | х | Х | | Х |
| Eligibility criteria check | х | х | | | | | |
| Blood pressure, heart rate | х | Х | Х | х | Х | х | Х |
| 12-Lead ECG Recording | x | X | X | | Х | x | X |
| INR | <b>←</b> | | | | | | (2) |
| aPTT, TCT | х | х | х | | Х | Х | Х |
| Biochemistry | х | | | | | | Х |
| Haematology | х | | х | | Х | | Х |
| Urinary pregnancy test | | х | | | | | Х |
| Red Blood Cell concentrations of DHA | | х | х | | Х | | Х |
| Treatment number allocation | | Х | | | Х | | |
| IVRS/IWRS | х | х | | | Х | | |
| ECV (3) | | | Х | | | | |
| Drug administration | | <b>←</b> | | | | | |
| Adverse events recording | | x | Х | х | Х | Х | X |
| Holter ECG | <b>←</b> → <sup>(4)</sup> | | <b>←</b> | (5) | | | |
| TTEM (6) | | | | <b>←</b> | | | <b>→</b> |

Final version

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of VKA introduction: INR 2 to 3 times a week until stabilization, then weekly until the ECV, then every 4 weeks after ECV
(3) In patients with AF
(4) 24-hour Holter ECG
(5) 7-day Holter ECG
(6) T-Tay Holter ECG
(6) TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms.
TTEM once a week even in case of AF recurrence or atrial flutter emergence for at least 10 minutes.

Final version 843/1185

F 373280 CA 2 01

Final version 844/1185



Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

# CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Gaëlle ALCARAZ

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 62 16 Fax:+33 5 34 50 69 69

E-mail:gaelle.alcaraz@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

Associate Professor of Cardiology

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: savinanodari@gmail.com; nodari@med.unibs.it

#### **Version 8 – 22OCT2014**

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 845/1185

# **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

# **Clinical Study Manager (Monitor)**

Gaëlle ALCARAZ

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 62 16 Fax: +33 5 34 50 69 69

E-mail: gaelle.alcaraz@pierre-

fabre.com

# **Medical Director**

Richard ROCHE, MD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 61 94 Fax: +33 5 34 50 69 69

E-mail: richard.roche@pierre-

fabre.com

Final version 846/1185

#### CONTRACT RESEARCH ORGANISATIONS

# For Feasibility, Monitoring and Regulatory issues (in Hungary, Czech Republic and Italy):

#### Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: rzurita@psnglobal.org

# For Feasibility, Monitoring and Regulatory issues (in Spain):

# Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

#### For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6. Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

# For Centralised Reading of Holder ECG and TTEM and equipment supply:

#### **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage:

#### **Agrocampus Ouest**

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

#### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER - FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 847/1185

# Protocol F 373280 CA 2 01

#### APPROVAL FORM

Protocol Version 8 - 22OCT2014

Sponsor's Representative:

Medical Director: Richard ROCHE, MD Date: 12/10/2014

Signature:

Study Coordinating Investigator:

Savina NODARI, MD

Date:

Signature:

# Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR

# **SIGNATURE FORM**

# **Protocol Version 8 – 22OCT2014**

| Country: | | |
|-------------------------------------------|-------|------------|
| <b>Country Coordinating Investigator:</b> | | |
| "Name" | Date: | Signature: |

Final version 849/1185

#### Protocol F 373280 CA 2 01

#### INVESTIGATOR SIGNATURE FORM

#### Protocol Version 8 – 22OCT2014

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 22OCT2014 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

# Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * ' | То | be | ad | lap | ted |
|-----|----|----|----|-----|-----|

| Date: | Signature: |
|-------|------------|
| | 2-6 |

Final version 850/1185

# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|------------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | |
| 1.2.1. | Chemical and pharmaceutical characteristics | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1. | $\mathcal{L}$ | |
| 1.2.2. | | |
| 1.2.2.<br>1.2.2. | $\mathcal{E}$ 1 | |
| 1.2.2. | | |
| 1.2.2. | | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | 29 |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 32 |
| 2.1. | PRIMARY OBJECTIVE | 32 |
| 2.2. | SECONDARY OBJECTIVES | 32 |
| 3. | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 34 |
| 4.1. | OVERALL DESCRIPTION | 34 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 40 |
| 5.3. | NUMBER OF PATIENTS | 41 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 42 |
| 5.6. | WITHDRAWAL CRITERIA | 42 |
| 5.7. | REPLACEMENT OF PATIENTS | 43 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | |
| 6. | STUDY TREATMENT | 44 |

| 6.1. | SOURCE, PRESENTATION AND COMPOSITION OF INVESTIGATIONAL PRODUCT | 44 |
|---|---|---|
| 6.2. | PACKAGING AND LABELLING | 44 |
| 6.2.1. | Packaging | |
| 6.2.2. | Labelling | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 6.5. | DRUG ADMINISTRATION | 47 |
| 6.5.1. | Duration of Treatment | 47 |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration | 47 |
| 6.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF INVESTIGATIONAL PRODUCT | 48 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| | CONCOMITANT TREATMENTS | |
| 7.1. | VITAMIN K ANTAGONIST TREATMENT | |
| 7.2. | PROHIBITED TREATMENTS | |
| 7.3. | AUTHORISED TREATMENTS | 50 |
| 8. I | EVALUATION CRITERIA | 50 |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence | 50 |
| 8.1.1.1 | | |
| 8.1.1.2 | | |
| 8.1.1.3 | | |
| 8.2. | SECONDARY EFFICACY CRITERIA | 51 |
| 8.2.1. | F | |
| 8.2.1.1 | | |
| 8.2.1.2 | | |
| 8.2.1.3 | | |
| 8.2.2. | Duration of AF episodes in the first week following visit 3 (ECV visit) | |
| 8.2.2.1<br>8.2.2.2 | | |
| 8.2.2.3 | | |
| 8.2.3. | Clinical parameters evaluation | |
| 8.2.3.1 | <u>.</u> | |
| 8.2.3.2 | | |
| 8.2.3.3 | | |
| 8.2.3.4 | , 1 | |
| 8.2.4. | Cardioversion assessment | 54 |
| 8.2.5. | Evolution of echocardiographic parameters | 54 |
| 8.2.5.1 | Definition | 54 |

Final version 852/1185

| 3.2.5.2. Schedule | 54 |
|----------------------------------------------------------------|----|
| 3.2.5.3. Evaluation method | 54 |
| BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA | 55 |
| 3.3.1. Definition | |
| 8.3.2. Blood samples | |
| 3.3.2.2. Technical handling | |
| 3.3.3. DHA concentration measurement | |
| 3.4. SAFETY ASSESSMENT | |
| 8.4.1. Adverse Events | 56 |
| 3.4.2. Laboratory Investigations | |
| 8.4.2.1. Schedule | |
| 3.4.2.2. Technical Procedures and Parameters | 56 |
| 3.4.3. Global Physical Examination | 57 |
| 8.4.4. Vital Signs | |
| 3.4.4.1. Schedule | |
| 3.4.4.2. Technical Procedure and Parameters | |
| 8.4.5. Electrocardiogram (ECG) | |
| 8.4.5.1. Schedule | |
| 3.4.6. Coagulation parameters | |
| 3.5. CONCOMITANT TREATMENTS | |
| 8.6. COMPLIANCE | |
| O. STUDY PROCEDURES | |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | |
| 10.1. ADVERSE EVENTS | |
| 10.1.1. Definition of Adverse Events | 66 |
| 10.1.2. Grading of Adverse Events | |
| 10.1.3. Reporting of Adverse Events | |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 67 |
| 10.2.1. Definition | 67 |
| 10.2.2. Reporting of SAE | 68 |
| 10.2.3. Follow-up of SAE | |
| 10.2.4. SAE Occurring After the Study | 69 |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 69 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 69 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | 70 |
| 11. DATA COLLECTION AND STUDY MONITORING | 70 |
| 11.1. DATA COLLECTION | 70 |
| 11.1.1 Case Report Form | 70 |

| 11.1.2. Source Documents | 71 |
|---|---|
| 11.2. STUDY MONITORING | 71 |
| 11.2.1. Monitoring visits | 71 |
| 11.2.1.1. Site Preselection Visit | 72 |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | |
| 12. DATA MANAGEMENT | 74 |
| 12.1. DATA ENTRY | 74 |
| 12.2. DATA CLEANING | 74 |
| 12.3. DATA CODING | 74 |
| 12.4. DATA STORAGE | 75 |
| 12.5. DATABASE LOCK | 75 |
| 13. STATISTICAL ANALYSIS | |
| 13.1. GENERAL CONSIDERATIONS | |
| 13.2. SAMPLE SIZE | |
| 13.3. PROTOCOL DEVIATIONS | |
| 13.4. DATA SETS ANALYSED | |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 77 |
| 13.7. EFFICACY ANALYSIS | |
| 13.7.1. Primary Criterion | 78 |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2. Secondary Criteria | 78 |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | 79 |
| 13.8. SAFETY ANALYSIS | 79 |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | |
| 13.8.3. Global Physical Examination | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | 83 |

| 13.8.4.1. Vital Sign Measurements Over Time | 83 |
|---|---|
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | 84 |
| 13.10. COMPLIANCE | 84 |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 84 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 85 |
| 14.1. ETHICAL CONDITIONS | 85 |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 85 |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 86 |
| 14.4. PERSONAL DATA PROTECTION | 86 |
| 14.5. INSURANCE POLICY | 87 |
| 15. ADMINISTRATIVE PROCEDURES | 87 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 87 |
| 15.3. END OF THE STUDY | |
| 15.3.1. Definition of the End of Study | 88 |
| 15.3.2. Early Study Termination | 88 |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | |
| 15.4. AUDIT | 89 |
| 15.5. INSPECTION | 89 |
| 15.6. CONFIDENTIALITY | 89 |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 90 |
| 15.9. STUDY RESULTS PUBLICATION | 90 |
| 16. REFERENCES | 92 |
| 17. APPENDICES | 96 |
| 17.1. DECLARATION OF HELSINKI | 97 |
| 17.2. SAE REPORT FORM | 101 |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 104 |

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented by the Institut de Recherche Pierre Fabre (IRPF) | |
|---|---|---|
| Name of Finished Product: | Not applicable | |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) | |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. International, multicentric, randomised, double-blind, placebo controlled study | |
| Abbreviated Title: | Not applicable | |
| Study Coordinating Investigator: | Pr Savina NODARI | |
| <b>Study Centres:</b> | International, multicentric | |
| Publication / Rationale: | of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study pduration of AF induced by burst pacing. Moreover, the effectiveness of PolyUns following conditions: - prevention of AF recurrence with amiodarone (add on them - Improvement of ventricular final hospitalisation in patients with Taking into account these studies, it see treatment of patients with both persisten This phase IIa study is designed to ass | in patients with persistent AF, in co-administration apy) [2] unctional parameters, morbi-mortality and duration of a heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the t atrial fibrillation and chronic heart failure. less the efficacy and the safety of the investigational sinus rhythm after electrical cardioversion (ECV) in |
| Planned Study Period: | January 2013 – April 2016 | Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 | |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>Ideally INR 2-3 (vitamin K antagonist should be given at least 3 weeks before ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit) <ul> <li>Condition: successful ECV or spontaneous CV</li> </ul> </li> </ul> | |
| | - Cardiac monitoring: | |

Final version 856/1185

| | <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: one transmission per week from the day of visit 4 (end of week 5) to (week 24) and at any time in case of AF or atrial flutter symptoms.</li> </ul> |
|---|---|
| | - Treatment duration: 24 weeks |
| Study Schedule: | <ul> <li>7 visits will be scheduled:</li> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of study treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter device)</li> <li>V4/W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V6/W12* (D84 ± 7 days): follow-up visit</li> <li>*see amendment PA05 dated 22OCT2014</li> <li>V7/W16 (D112 ± 7 days): final study visit</li> <li>V9/W24* (D168 ± 7 days): final study visit</li> <li>*see amendment PA05 dated 22OCT2014</li> </ul> |
| Number of Patients: | 76 x 2 patients |
| Diagnosis and Criteria for Inclusion: | Inclusion Criteria: |
| | Demographic Characteristics and Other Baseline Characteristics: |
| | 1. Men or women aged more than 18 years (inclusive) |
| | 2. Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted |
| | 3. Previous history of first documented episode of persistent AF. |
| | 4. Previous history of ischemic or non ischemic heart failure |
| | 5. NYHA class I or II chronic heart failure at selection and at inclusion |
| | 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF) ≥ 30% and ≤ 45% or for patients with a LVEF > 45%: |
| | an increased left ventricular end-diastolic size |
| | (diameter $\geq 60 \text{ mm}$ and/or $> 32 \text{ mm/m}^2$ and/or volume $> 97 \text{ ml/m}^2$ ) |
| | <ul> <li>and/or an increased left ventricular end-systolic size</li> </ul> |
| | (diameter $> 45$ mm and/or $> 25$ mm/m <sup>2</sup> and/or volume $> 43$ ml/m <sup>2</sup> ) |
| | • and/or a reduced left ventricular outflow tract velocity time integral < 15 cm |
| | 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers |
| | 8. Left atrial area ≤ 40 cm² at selection and at inclusion |
| | 9. Patients treated or having to be treated by vitamin K antagonist |
| | 10. For female patient of child-bearing potential: |
| | In all the countries except Italy: |
| | <ul> <li>Use of an effective method of contraception (hormonal contraception or intra-<br/>uterine device) assessed by the investigator, for at least 2 months before the<br/>selection in the study, and agreement to go on using it during the whole duration of<br/>the study and up to 1 month after the last dose of the study treatment</li> </ul> |
| | - Documented as surgically sterilized |
| | • In Italy only: |
| | <ul> <li>Absolute abstention from sexual intercourse during the whole duration of the study<br/>and for a month after the end of the study or</li> </ul> |
| | - Use of double barrier contraception method (use of effective medical contraception |

Final version 857/1185

- method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical / legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent AF
- More than two successful cardioversions (electrical or pharmacological) in the last 6 months
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine  $\geq$  25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- 8. Bradycardia (HR ≤ 50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, betablockers, calcium-blockers
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months
- 17. Dietary supplement with  $\omega$  3 or  $\omega$  6 according to investigator's judgement
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible

Final version 858/1185

| | antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel |
|---|---|
| | Other criteria: |
| | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion |
| | 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection |
| | 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints |
| | 23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator |
| | 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship |
| | 25. Breastfeeding female patient |
| Exclusion criteria before V3: | Patients without dyskalemia who will not have INR values $\geq 2$ on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study. |
| | However, if only 2 INR values are $\geq$ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. |
| | If necessary, for meeting these INR conditions, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280<br>Soft Capsules |
| Dose: | Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules Placebo will be administered in the same conditions as the tested product. |
| Mode of Administration: | Oral, one capsule each evening with dinner |
| Evaluation Criteria: | Efficacy evaluation variables: |
| | Primary evaluation variable: |
| | - Time to first Atrial Fibrillation recurrence or atrial flutter emergence defined by the time to first episode of AF or atrial flutter lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 – ECV visit). |
| | Handling of AF recurrences or atrial flutter emergences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24). |
| | For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5). Moreover, during this TTEM period, if patient experiences any AF or atrial flutter symptoms, it should be recorded and documented using the TTEM. |
| | All ECG (Holter and TTEM) will be evaluated by a Central Reading Laboratory. |
| | Secondary evaluation variables: |
| | During the 7-day continuous ECG monitoring, |

Final version 859/1185

- Numbers of AF episodes
- Duration of AF episodes

#### Clinical parameters:

During the whole study:

- Number of recurrence of symptomatic AF episodes
- EHRA score
- Hospitalization for cardiovascular events
- Hospitalization for thromboembolic stroke
- All causes of hospitalization

#### Cardioversion:

- Assessment of spontaneous cardioversion
- Assessment of successful cardioversion
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing an other cardioversion after the initial ECV

#### Other:

- Evolution of echocardiographic parameters (at V4, V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA(ml/m²), Left ventricular end diastolic volume (ml) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (ml))
- Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).

#### Safety criteria:

- Adverse events (observed and / or spontaneously reported)
- Vital signs (Blood pressure (supine and standing), heart rate)
- Physical examination (body weight, body surface area)
- Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns (ECG not centralized)
- Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets
- Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)
- Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR *(local laboratory)*, Prothrombine Time *(PT)*.

#### **Concomitant treatments**

#### Compliance

#### Statistical Methods:

#### Sample Size:

Assuming an AF recurrence or atrial flutter emergence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%.

### **Primary Efficacy Analysis**

Final version 860/1185

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### **Secondary Analyses**

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

#### Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment).

Final version 861/1185

# STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | | V6 | <b>V</b> 7 | | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | | W12<br>(84+/-7D) | W16<br>(112+/-7D) | | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | Х | Х | X | X | Х | Х | X | Х |
| Habits | X | | | | | | | | |
| Global physical examination (body weight) | Х | х | Х | | X | Х | Х | X | Х |
| Echocardiography | х | х | | X | | Х | | | Х |
| Eligibility criteria check | X | X | | | | | | | |
| Blood pressure, heart rate | X | X | Х | X | X | Х | х | X | X |
| 12-Lead ECG Recording | Х | Х | Х | | X | Х | Х | X | X |
| INR | <b>+</b> | | | | X | | | X | (2) |
| aPTT, TCT | х | х | Х | | X | Х | х | X | Х |
| Biochemistry | X | | | | | | | | X |
| Haematology | Х | | Х | | | Х | | | Х |
| Urinary pregnancy test | | Х | | | | | | | X |
| Red Blood Cell concentrations of DHA | | Х | Х | | | Х | | | Х |
| Treatment number allocation | | X | | | | Х | | | |
| IVRS/IWRS | X | X | | | | Х | | | |
| ECV (3) | | | Х | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | х | Х | X | X | Х | Х | X | X |
| Holter ECG | <b>←</b> → <sup>(4)</sup> | | <b>+</b> | (5) | | | | | |
| TTEM (6) | | | | <b>←</b> | | | | | <b></b> |

Final version 862/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of VKA introduction: INR 2 to 3 times a week until stabilization, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) T-EM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms. TTEM once a week even in case of AF recurrence or atrial flutter emergence for at least 10 minutes.

# LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

βHCG : beta human chorionic gonadotrophinBLO : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

C<sub>max</sub> : Maximum concentration C<sub>min</sub> : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC : "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Transesophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL : High density lipoprotein

Final version 863/1185

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH : International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
 IRPF : Institut de Recherche Pierre Fabre
 IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC : "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set

QTcB : QT interval using Bazett's correction formula QTcF : QT interval using Fridericia's correction formula

RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

To : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

VKA : Vitamin K Antagonist WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 864/1185
## 1. INTRODUCTION AND STUDY RATIONALE

## 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced

Final version 865/1185

canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95%] confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage

Final version 866/1185

of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61
   +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p < 0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

## 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

Final version 867/1185

# 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

# 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

## 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

Final version 868/1185

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus 637  $\pm$  196 sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and 79  $\pm$  51 sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the compound may exert a similar protective effect [1].

Final version 869/1185

# 1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

## 1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

#### 1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical pharmacokinetic profile of F373280 is not associated with particular alerts concerning the proposed clinical phase IIa study.

#### 1.2.3. Clinical data

## Part A: Single dose

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of

Final version 870/1185

an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

## Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Final version 871/1185

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Final version 872/1185

Taking into account these studies, it seems that DHA might be of therapeutic interest in the

treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product

(F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic

heart failure.

1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular

diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor

contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for

hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial

infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common

(>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000),

not known (cannot be estimated from the available data).

- The reported adverse events are:

Infection and infestations:

Uncommon: gastroenteritis

Immune system disorders:

Uncommon: hypersensitivity

Metabolism and nutrition disorders:

Rare: hyperglycaemia

Uncommon: dizziness, dysgeusia

Rare: headache

Nervous system disorders:

Vascular disorders:

Very rare: hypotension

Respiratory thoracic and mediastinal disorders:

Final version 873/1185 Very rare: nasal dryness

• Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

• Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene<sup>®</sup> (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after

Final version 874/1185

administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

## 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

Final version 875/1185

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form. A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (vitamin K antagonist, VKA), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence or atrial flutter emergence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with vitamin K antagonist (VKA) for at least 3 weeks before ECV
- ECV will be performed in patients with AF and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values  $\geq 2$  on the 3 last

Final version 876/1185

tests performed before ECV are required. However, if only 2 INR values are  $\geq 2$  among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Patients who do not revert to sinus rhythm or present an early AF relapse or an early atrial flutter emergence within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be performed throughout the study period. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored once a week between visits using Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without study treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Seven visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28-2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)

Final version 877/1185

- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 6\* (V6): W12 (D84 ± 7D): follow-up visit
   \*see amendment PA05 dated 22OCT2014
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 9\* (V9): W24 (D168 ± 7D): final study visit
   \*see amendment PA05 dated 22OCT2014

# 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Previous history of persistent AF with duration of the current episode from 7 days to 6 months.
- A systolic heart failure defined by a reduced left ventricular ejection fraction (≥ 30% and ≤ 45%) or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size (diameter ≥ 60 mm and/or > 32 mm/m² and/or volume > 97 ml/m²),
  - and/or an increased left ventricular end-systolic size (diameter > 45 mm and/or > 25 mm/m² and/or volume > 43 ml/m²),
  - and/or a reduced left ventricular outflow tract velocity time integral < 15 cm [23, 24].</li>

Final version 878/1185

According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.

- A Left Atrial Area (LAA) not severely abnormal (no greater than 40 cm<sup>2</sup> as defined in the report from the American Society of Echocardiography's Guideline) [23]. According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF (or emergence of atrial flutter) since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Final version 879/1185

Eligible participants will enter a selection phase in which anticoagulant treatment (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) of 2 to 3 before ECV. According to guidelines for the management of AF [6], VKA should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every 4 weeks or 8 weeks (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

## 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/ml and 60 to 90 mg/ml, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough

Final version 880/1185

fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

## 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted
- 3. Previous history of first documented episode of persistent AF
- 4. Previous history of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF)  $\geq$  30% and  $\leq$  45% or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size

 $(diameter \ge 60 \text{ mm and/or} > 32 \text{ mm/m}^2 \text{ and/or volume} > 97 \text{ ml/m}^2)$ 

• and/or an increased left ventricular end-systolic size

(diameter  $> 45 \text{ mm and/or} > 25 \text{ mm/m}^2 \text{ and/or volume} > 43 \text{ ml/m}^2$ )

- and/or a reduced left ventricular outflow tract velocity time integral < 15 cm
- On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers

Final version 881/1185

- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by vitamin K antagonist
- 10. For female patient of child-bearing potential:

## • In all the countries except Italy:

- Use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- Documented as surgically sterilized

## • In Italy only:

- Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- Use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

## Ethical /legal considerations:

13. Having signed his/her written informed consent,

Final version 882/1185

14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent Atrial Fibrillation
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment: TSH  $\pm$  T4L  $\pm$  T3L to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months

Final version 883/1185

- 16. Treatment with any Polyunsaturated Fatty Acid within the last 3 months
- 17. Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship,
- 25. Breastfeeding female patient.

#### **5.3. NUMBER OF PATIENTS**

76 x 2 patients (taking into account 15 % of non evaluable patients).

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

Final version 884/1185

## 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form
  - obtain the reason(s) for withdrawal and report it/them in the case report form
  - evaluate the patient's clinical condition
  - if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.
- Erroneous inclusion according to the study protocol. The decision to maintain or not the patient in the study will be taken jointly by the investigator and the sponsor. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with VKA for at least 3 weeks before ECV or who will
  experience a VKA intolerance during the study.
- Patients without dyskalemia who will not have INR values ≥ 2 on the 3 last tests
  performed before ECV should not have an ECV and will be excluded from the study.
  However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed
  if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal

Final version 885/1185

echocardiography) performed on the same day (before ECV) and the patient can continue the study.

- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early AF
  relapse or early atrial flutter emergence within the observation period after ECV will be
  considered to have finished follow-up.
- Occurrence of AF recurrence or atrial flutter emergence that would require, at the investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance.

## 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate in another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.
- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

Final version 886/1185

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the Institut de Recherche Pierre Fabre (IRPF) will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the IRPF according to European Directive and local requirements.

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

Two 12-week treatment units will contain 3 cases, each case of 4-week treatment containing: 10 blister packs of four 1 g F373280 soft capsules or 1 g placebo soft capsules each.

# 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

Final version 887/1185

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

## 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the IRPF will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection

Final version 888/1185

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

## 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

At selection visit (V1), practically, once patient's eligibility is confirmed:

- The Investigator:
- Contacts the IVRS/IWRS

Final version 889/1185

- Answers the questions related to the patient
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

At inclusion visit (V2), the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment.

The Investigator will dispense to the patient the 4-week treatment cases (one or two according to the visit) which label indicates the treatment number and the administration period.

## 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

## 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

Final version 890/1185


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

#### 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

Final version 891/1185

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

#### 7.1. VITAMIN K ANTAGONIST TREATMENT

VKA should be given for at least 3 weeks before ECV and continued for the whole study duration. However, VKA should be stopped in case of occurrence of VKA intolerance during the study and the patient should be withdrawn from the study. The VKA used will be left to the decision of each Investigator according to his/her local practice.

#### 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I:
    - o Class IA: Disopyramide, Procainamide, Quinidine
    - o Class IB: Lidocaine, Mexiletine
    - o Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any oral anticoagulant treatment other than VKA: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel
- Dietary supplement with Omega 3 or Omega 6

Final version 892/1185

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

## 8. EVALUATION CRITERIA

## 8.1. PRIMARY EFFICACY CRITERION

## 8.1.1. Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence

# 8.1.1.1. Definition

Time to first AF recurrence or atrial flutter emergence is defined by the time to first episode of AF or atrial flutter (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. Schedule

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

Final version 893/1185

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

## • Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM.

Moreover, if patient experiences AF or atrial flutter symptoms during this TTEM period, it should be documented using the TTEM.

In case of AF recurrence or atrial flutter emergence and provided that the patient does not require a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

## • Process of centralisation of ECG (Holter and TTEM)

ECG (Holter and TTEM) will be centralized by the Central Reading Laboratory. The ECG will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign these documents.

The Holter and TTEM process will be fully described in separate documents.

## 8.2. SECONDARY EFFICACY CRITERIA

## 8.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.1.1. *Definition*

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

Final version 894/1185

### 8.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

#### 8.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

## 8.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.2.1. Definition

Duration of AF episodes will consist in the sum of duration of each AF episode.

## 8.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

## 8.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

## 8.2.3. Clinical parameters evaluation

#### 8.2.3.1. EHRA score assessment

# 8.2.3.1.1. *Definition*

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

Final version 895/1185

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

#### 8.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

## 8.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during TTEM period.

## 8.2.3.2. Time to first AF recurrence less than 10 minutes

Time to first AF recurrence less than 10 minutes will be assessed during TTEM period.

## 8.2.3.3. Recurrence of symptomatic AF

Recurrence of symptomatic AF will be assessed during TTEM period.

The number of recurrences of symptomatic AF consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

The time to first symptomatic AF recurrence is defined by the time to first episode of symptomatic AF.

## 8.2.3.4. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
- Hospitalization for AF treatment

Final version 896/1185

- Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

#### **8.2.4.** Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

# 8.2.5. Evolution of echocardiographic parameters

# 8.2.5.1. Definition

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), LVEF (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA (ml/m²), Left ventricular end diastolic volume (ml), Left ventricular end systolic volume (ml), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (ml).

## 8.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European

Final version 897/1185

Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

# 8.3. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.3.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.3.2. Blood samples

#### 8.3.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

## 8.3.2.2. Technical handling

Two blood samples (2 x 4 ml) will be collected in EDTA tubes. They will be homogenized slowly by inverting the tube without shaking, stored between  $+2^{\circ}\text{C}/+8^{\circ}\text{C}$  in a fridge (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between  $+2^{\circ}\text{C}$  and  $+8^{\circ}\text{C}$ ). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### 8.3.3. DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent)

Final version 898/1185

and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

## **8.4. SAFETY ASSESSMENT**

#### **8.4.1.** Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

## 8.4.2. Laboratory Investigations

#### 8.4.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kalemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 ml.

#### 8.4.2.2. Technical Procedures and Parameters

The following tests will be performed:

Final version 899/1185

<u>Haematology</u>: haematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and/or absolute), reticulocytes, platelets.

<u>Biochemistry</u>: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (ml/min) =  $[(140\text{-age}) \times \text{weight} / (7.2 \times \text{serum creatinine in mg/L})]$ 

in women:

GFR (ml/min) =  $[(140\text{-age}) \times \text{weight} / (7.2 \times \text{serum creatinine in mg/L})] \times 0.85$ 

- with serum creatinine expressed as µmol/l:

GFR (ml/min) = [(140-age) x weight / serum creatinine in  $\mu$ mol/l] x k,where k = 1.23 for men, 1.04 for women.

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

## 8.4.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

Final version 900/1185
The Body surface area (BSA) will be calculated at the same visits using Mostellers' formula:

 $BSA = [(Weight x Height)/3600]^{1/2}$ 

(Weight in kg, height in cm)

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

# 8.4.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

#### 8.4.4.1. Schedule

Vital signs will be measured at each visit.

## 8.4.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

# 8.4.5. Electrocardiogram (ECG)

## 8.4.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9 using a usual standardised 12-lead cardiograph.

# 8.4.5.2. Technical Procedure and Parameters

## • Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns will be reported in the

Final version 901/1185

e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

# **8.4.6.** Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

The recommendations for the controls of INR are the following [25, 26]:

- 1) During the pre-cardioversion period, if the anticoagulation by VKA has to be initiated, the treatment must be initiated at least 3 weeks prior to cardioversion then the INR will be monitored as follow:
  - The adjustment of the dosage of VKA should be performed stepwise by controlling INR 2
     to 3 times a week until stabilization within the target range (2 3) on 2 successive tests.
  - When the INR is within the target range (2 3) on 2 successive tests, the dose of VKA should be maintained. Then the controls of INR will be progressively spaced within a few weeks.
  - When INR is stabilized, at least one test should be performed each week.
  - In all cases, an INR control must be performed within 24 h before ECV.
- 2) During the pre-cardioversion period, if the anticoagulation by VKA was already initiated, the INR will be monitored as follow:
  - One INR per week up to ECV
  - An INR control must be performed within 24 h before ECV
- 3) After cardioversion : one INR every 4 weeks
- 4) Throughout the duration of the study if INR > 3 the advocated actions are:

Final version 902/1185

- No transesophageal echocardiography before cardioversion
- For asymptomatic patients:
  - 3 < INR < 4: no omission of VKA (dose adjustment if required), no vitamin K
  - $4 \le INR < 6$ : omit one dose of VKA, no vitamin K
  - $6 \le INR < 10$ : interrupt VKA, vitamin K 2 mg orally
  - INR ≥ 10: interrupt VKA, vitamin K 5 mg orally
     For INR ≥ 6, an adverse event has to be reported (asymptomatic overdose).

Anti-coagulation by VKA should be given at least 3 weeks before ECV and continued for the whole study duration.

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

The quantity of blood samples collected at each time for coagulation parameters will be 2 ml. Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

#### 8.5. CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements related to patient's concomitant treatments started before selection visit and continued throughout the trial, or started during the trial, can be found in section 7.

#### 8.6. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit (except at visit 4), the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

## 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week - 4 to Week -1):

Final version 903/1185

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate If the results of the above assessments are compatible with the selection criteria:
  - A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory. The Central Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.

Final version 904/1185

• The patient will enter the selection and pre-cardioversion periods in which anticoagulant (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) in the range of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

The patient will receive from the investigational centre the participant card to be kept for all the duration of the study.

# Visit 2 - Inclusion Visit (Day 1):

If the patient's behaviour during the selection period and/or the result of complementary examinations, particularly the confirmation of the presence of persistent AF by the Central Reading Laboratory during this period and the laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Urine pregnancy test for women of child bearing potential

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 2 for the first 12-week period.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.4.6) in order to fulfil the ECV conditions (refer to paragraph 3).

Final version 905/1185

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period (one case of treatment).

# Visit 3 (Week 4: D28 -2/+7 days) cardioversion:

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be performed 4 weeks after randomization in patients with AF. ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values ≥ 2 on the 3 last tests performed before ECV are required. However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge.

Final version 906/1185

Patients who will not revert to sinus rhythm or with early AF relapse or early atrial flutter emergence within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 8-week period (two cases of treatment).

## Visit 4 (Week 5: D35 -2/+7 days):

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Bodyweight (bodyweight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to perform one transmission per week from this visit (initial call to perform with the patient) to the visit 9 (week 24 – end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

## Visit 6\* (Week 12: D84 $\pm$ 7 days) - Visit 7 (Week 16: D112 $\pm$ 7 days) :

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following criteria:

Adverse events

Final version 907/1185

- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV due to occurrence of VKA intolerance, the monitoring of INR, aPTT and TCT should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- The cardiac monitoring will be continued using the TTEM device through one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

In addition, at visit 6:

- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

At the end of each visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next treatment period: one case at visit 6 and two cases at visit 7.

# Visit 9\* - End-of-Study Visit (Week 24: D168 $\pm$ 7 days):

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight

Final version 908/1185

Vital signs

• 12-lead ECG

 Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time

(aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.

• Urine pregnancy test for women of childbearing potential

Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused

soft capsules.

The total volume of blood collected should be about 90 ml for the study duration (30 ml for the

total volume of haematology and biochemistry, 2 ml for each blood samples for coagulations

parameters and 4 ml for each blood samples of DHA).

10. ADVERSE EVENTS: DEFINITION AND REPORTING

10.1. ADVERSE EVENTS

**10.1.1.** Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, i.e. any subjective signs and

symptoms or change in a concomitant disease present at the Selection Visit considered or not

related to the treatment.

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for

vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should

be repeated until the values return to normal or to a stable status. Abnormal results are defined as

those falling out of the laboratory normal ranges and that are clinically significant. The frequency

of such checks should be defined by the Investigator according to the degree of abnormality.

Final version 909/1185

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

## 10.1.2. Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

# 10.1.3. Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

# 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Final version 910/1185

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

- \* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:
  - planned (as per protocol) medical/surgical procedure
  - preparation for routine health assessment/procedure (e.g. routine colonoscopy)
  - planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
  - administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

# 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

## HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

# 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

Final version 911/1185

The serious adverse events must be followed up until resolution or stabilisation.

# 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Final version 912/1185

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

# 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF. Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

Final version 913/1185

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

#### 11.2. STUDY MONITORING

## 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

Final version 914/1185

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
- has received the technical protocol, administrative and financial agreement signed by all parties
- has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

Final version 915/1185

## 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

## 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

Final version 916/1185

## 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

## 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate the coding.

Final version 917/1185

#### 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

# 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence or atrial flutter emergence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients

Final version 918/1185

per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4). A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the

Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

#### 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol

Final version 919/1185

deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

# **13.5.1. Dropouts**

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

# 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

# 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- <u>Quantitative parameters</u> will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

Final version 920/1185

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

# 13.7.1. Primary Criterion

# 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence of AF or atrial flutter emergence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

# 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

## 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

## 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

# 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

Final version 921/1185

# 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

# 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

# 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

#### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

## 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

Final version 922/1185

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event.
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs
- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Final version 923/1185

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (reported in 1% patients in any group) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (for all patients).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

# 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Final version 924/1185

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

# 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

Final version 925/1185

# 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

# 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

# 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

Final version 926/1185

# 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

## 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

#### 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

#### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No analyses of efficacy data are planned for IDMC that ensures that the overall probability of type I error is controlled. No Type I error and sample size adjustments are necessary. Any recommendations of the IDMC to alter study conduct will be based on safety, so IDMC monitoring of the study will not affect the statistical operating characteristics of the final analysis.

Final version 927/1185

The IDMC will review, three times during the study period (after the first 30 subjects will have been randomized, when the first 80 subjects will have terminated their study participation and when 130 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable.

# 14. GENERAL ETHICAL CONSIDERATIONS

#### 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

# 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

Final version 928/1185

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

## 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

Final version 929/1185

## 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor Pierre Fabre Médicament, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

## 15. ADMINISTRATIVE PROCEDURES

# 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities.

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

## 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all
  patients included in the trial or not.

Final version 930/1185

- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

# 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

# 15.3.2. Early Study Termination

# 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

# 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

Final version 931/1185

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at Pierre Fabre Médicament and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

#### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

## 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

#### 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

Final version 932/1185

## 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

## 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

Final version 933/1185

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 934/1185

## 16. REFERENCES

- [1]. F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2]. NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- [3]. NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L. Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy *J. Am. Coll. Cardiol.* 2011;57;870-879
- [4]. MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study *American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5*
- [5]. GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6]. CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct;31(19):2369-429
- [7]. KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 935/1185

[8]. BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9]. OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10]. BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11]. TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12]. LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13]. METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr (2007); 85 : 1225.* 

[14]. ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15]. TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16]. SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6):652-9.

[17]. LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

Final version 936/1185
The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human. *Lipids*, 2010, 45, 11-19.

[18]. HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

[19]. ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion

World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain

[20]. KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G.

Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association.

Europace 2007, 9, 1006-1023

#### [21]. EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter.

EMA/CHMA/EWP/213056/2010

#### [22]. OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955–961

[23]. ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

[24]. JOHN J.V. McMURRAY, STAMATIS ADAMOPOULOS, STEFAN D. ANKER, ANGELO AURICCHIO, MICHAEL BÖHM, KENNETH DICKSTEIN, VOLKMAR FALK, GERASIMOS FILIPPATOS, CÂNDIDA FONSECA, MIGUEL ANGEL GOMEZ-SANCHEZ, TINY JAARSMA, LARS KØBER, GREGORY Y.H. LIP, ALDO PIETRO MAGGIONI, ALEXANDER PARKHOMENKO, BURKERT

Final version 937/1185

# M. PIESKE, BOGDAN A. POPESCU, PER K. RØNNEVIK, FRANS H. RUTTEN, JUERG SCHWITTER, PETAR SEFEROVIC, JANINA STEPINSKA, PEDRO T. TRINDADE, ADRIAAN A. VOORS, FAIEZ ZANNAD, ANDREAS ZEIHER

ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012 European Heart Journal (2012) 33, 1787–1847

[25]. AGENCE NATIONALE DE SECURITE DU MEDICAMENT ET DES PRODUITS DE SANTE (ANSM).

Bon usage des médicaments antivitamine K (AVK) Actualisation – Juillet 2012

[26]. GILLES PERNOD, ANNE GODIER, CLAIRE GOZALO, BENJAMIN TREMEY, PIERRE SIE

French clinical practice guidelines on the management of patients on vitamin K antagonists in at-risk situations (overdose, risk of bleeding, and active bleeding) *Thrombosis Research 126 (2010) e167–e174* 

Final version 938/1185

# 17. APPENDICES

Final version 939/1185

#### 17.1. DECLARATION OF HELSINKI

### WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

11. It is the duty of physicians who participate in medical research to protect the life, health, dignity,

Final version 940/1185

- integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.
- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be

Final version 941/1185

- enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

Final version 942/1185

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 943/1185

# 17.2. SAE REPORT FORM

Final version 944/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE CORPORATE VIGILANCES DIVISION |
|---|
| TO BE TRANSMITTED TO THE CORPORATE VIGILANCES DIVISION BY E-MAIL WITHIN 24H TO HQ.pharmacovigilance@pierre-fabre.com OR BY FAX WITHIN 24H – Fax N°: 33 (0) 1.49.10.80.90 |
| Transmission date (ddmmyyyy) Country: |
| SAE N° |
| > SUBJECT CHARACTERISTICS |
| Birth date |
| Gender1=M, 2=F Height cm Weight · kg |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: □ Death (whatever may be the cause) □ Hospitalisation (*) or extension thereof □ Life threatening □ Invalidity or disability □ Congenital abnormality or abnormal pregnancy outcome □ Cancer □ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) Other fact to be notified: □ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date (ddmmyyyy) |
| Seriousness onset date |
| <b>Summary description</b> (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER |
| • Time of occurrence of SAE |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| Date of first study treatment administration (ddmmyyyy) |
| Date of last study treatment administration before the occurrence of SAE |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |
| $\mathbf{i}$ |

Final version 945/1185

| Transmission date | n date (ddmmyyyy) Country: | | | | | |
|---|---|---|---|---|---|---|
| SAE N° | SAE N° FIRST NOTIFICATION ☐ FOLLOW-UP ☐ N° | | | | | |
| > CONCOMITANT MI<br>(EXCEPT THE TREA | EDICATION SING<br>ATMENTS GIVEN | CE TRIAL INITIATION FOR THE SAE) | ON and UP UNTIL TH | E OCCURRENCE O | F THE SAE | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAKEN | FOLLOWING T | HE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | / / | |
| □ Dosage modified | ication, specify : | | Modification D | ate: | //_ | |
| ☐ Temporarily d | iscontinued | | Readministration date | e: | //_ | |
| ☐ Withdrawn | | | End date | : | // | |
| ☐ Not applicable | | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription of | f corrective or symp | tomatic treatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| , | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Discontinuation | on of concomitant tr | eatments: | <u>.</u> | | | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, specify | y: | | | | | |
| > OUTCOME | | | | | | |
| □ Not recovered/Not resolved □ Recovering/Resolving □ Recovered/Resolved □ Recovered/Resolved □ Unknown In case of death, has an autopsy been conducted ? □ Yes □ No | | | | | | |
| > INVESTIGATOR CAUSALITY ASSESSMENT (investigator's assessment to be done as soon as possible) | | | | | | |
| Study drug: | | | study protocol: | P | | |
| □ Not Suspected □ Suspected □ Suspected □ Suspected □ Suspected | | | | | | |

Final version 946/1185

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values<sup>(\mathridge{m})</sup>

| PARAMETERS | | UNIT | PSC | |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | _ | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| TO THE TOTAL | Protein | g/l | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pH | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 947/1185

<sup>(¤)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

### **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| НАЕМО | GLOBIN | Decrease of at least 2g/dl and value < 10 g/dl whatever the baseline value If missing baseline : value <10g/dl |
| NEUTRO | NEUTROPHILS • < 1 500/mm <sup>3</sup> whatever the baseline value | |
| WBC (if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline: <ul> <li>TB &gt; 1.5 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>TB &gt; 2 N</li> </ul> </li> </ul> |

### N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 948/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg}$ and increase $\ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110 \text{ bpm}$ and increase $\ge 10 \text{ bpm}$ |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>paseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | > 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | | Classes for the for each parame | Minimum Post-bo<br>ter | aseline Value |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤ <i>50</i> | ≤90 | ≤50 | ≤50 |
| [120;140] | [80;90[ | <i>[50 ;75]</i> | [90 ;120] | [50;80] | <i>[50 ;75]</i> |
| [140;160[ | [90;100[ | [75;100[ | [120;140[ | [80;90[ | [75;100[ |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3BI 2 90 01 DBI 2 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq 20$ mmHg or DBP Decrease $\geq 10$ mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 949/1185

16.1.1.9. Protocol amendment n° PA06 General and non-substantial dated on 06 June 2016)

Final version 950/1185

# CLINICAL STUDY PROTOCOL AMENDMENT n° PA06 (GENERAL – Non Substantial)

Final version 951/1185

Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne, France

#### CLINICAL STUDY PROTOCOL AMENDMENT n° PA06

(GENERAL – Non-Substantial)

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Pierre Fabre Study Code: F373280 CA 2 01

**EudraCT Number or equivalent:** 2012-003487-48

Karim KEDDAD

INSTITUT DE RECHERCHE PIERRE FABRE

**Sponsor's Representative:** Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien

31035 TOULOUSE Cedex 1, FRANCE

**Pr Savina NODARI** 

Department of Clinical and Surgical Specialities, Radiological Science

and Public Health

Section of Cardiovascular Diseases

Study Coordinating Investigator: University Medical School and Spedali Civili Hospital of Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

**Date of amendment PA06:** 06JUN2016

The information contained in this document is confidential and is the property of the sponsor Pierre Fabre Médicament. This information is given for the needs of the trial and must not be disclosed without prior written consent of the sponsor Pierre Fabre Médicament. Persons to whom this information is given for the needs of the trial must be informed that it is confidential and must be disclosed.

Final version 952/1185



Study code: F373280 CA 2 01

#### APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

#### Clinical Study Protocol Amendment no PA06

(GENERAL - Non-Substantial)

Dated: 06JUN2016

| Sponsor's | renresen | tative(s) |
|-----------|-------------|-----------|
| SDOMEOU 9 | I CDI CSCII | tative(5) |

Head of Medical Unit

Date:

Signature:

Dr Karim KEDDAD

**Study Coordinating Investigator:** 

Date: 20/06/2016 Signature:

Pr Savina NODARI



Study code: F373280 CA 2 01

#### COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

#### Clinical Study Protocol Amendment no PA06

(GENERAL - Non-Substantial)

Dated: 06JUN2016

**Country Coordinating Investigator:** 

Date: 20/06/20(6 Signature:

Version 1

#### **INVESTIGATOR SIGNATURE FORM**

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

### Clinical Study Protocol Amendment no PA06

(GENERAL – Non-Substantial)

Dated: 06JUN2016

| By my signature below, I, Dr | , hereby confirm that I have read, |
|---|---|
| taken note of (and will apply) the modifications b | brought by the protocol amendment n° PA06 and I |
| will conduct the trial according to these new mod | alities. |
| D | 0. |
| Date: | Signature: |

Final version 955/1185

# HISTORY OF AMENDMENTS

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| NA | NA | General | NA | Corresponding to Protocol Version 2: Following French CA request (ANSM) and leading to protocol version 2: - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 |
| PA01 | Substantial | Local (Italy) | 01MAR2013 | Corresponding to Protocol Version 3: Integration of the modification included in the protocol version 2 Harmonisation of the protocol and the Informed Consent Form: adjustment of the selection criteria n°10 related to the contraception method addition of a letter that is given by the patient to his/her GENERAL practitioner (GP) precision that the sponsor can not collect a copy of the Informed Consent Form precision that the patient card is in Italian language only (without any English mention) |
| PA02 | Non<br>Substantial | General | 28MAR2013 | Corresponding to Protocol Version 4: - change of Sponsor's Representative (Clinical Study Manager), - modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed, - precision on the function and address of the International Study Coordinator Pr Nodari, - add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study), - adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage", - precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee), - correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized). - addition of the changes included in the local italian |

Final version 956/1185

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | | | substantial protocol amendment (i.e: contraception method, letter to GENERAL Practionner, patient card in Italian and no collection of the consent form by the sponsor in Italy). |
| PA03 | Substantial | General | 23OCT2013 | Corresponding to Protocol Version 5: Fax modification of the sponsor's representatives Planned end of study postponed to January 2015. The authorized history of the first documented persistent atrial fibrillation is less than 3 years. At selection a hyperkalemia or a hypokalemia is better defined by the standards of the local laboratories. Regarding previous treatments by amiodarone the non inclusion criteria of the protocol are adapted as follow: Previous treatment with oral amiodarone within 4 months prior to inclusion Previous treatment with intravenous amiodarone within 4 to 12 months before inclusion Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion. For male with a child-bearing potential partner (in Italy only): taking into account the duration of spermatogenesis the absolute abstention from sexual intercourse or the use of double barrier contraception method are extended to 3 months after the end of the study. Ranolazine is an antiarrhythmic treatment added to the prohibited treatments. Update of Serious Adverse Events (SAEs) form: Main change is the SAE sending: SAEs have to be reported to the Corporate Vigilance Department, and not anymore to the clinical study manager. Also SAEs can be sent by e-mail and by fax. Addition of Alpha Bioresearch as CRO involved for Feasibility, Monitoring and Regulatory issues in Spain. Correction of some minor typographic errors |
| PA04 | Non<br>Substantial | General | 03JUN2014 | Corresponding to protocol V7: - Precision on the temperature storage of DHA samples - Precision on the BSA formula - Addition of QTcB and QTcF - Precision on TTEM recording timelines - Clarification of the section Interim analysis and data monitoring (13.11) - Clarifications and specifications on some |

Final version 957/1185

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | | | minor points |
| PA05 | Substantial | General | 22OCT2014 | Corresponding to protocol V8: - Planned end of study postponed to April 2016 - Clarifications regarding the management of VKA treatment - Precision regarding the primary efficacy criterion (the time to the first Atrial Fibrillation recurrence or Atrial Flutter emergence) - Deletion of Visit 5 and Visit 8 - Previous history of a first documented persistent Atrial Fibrillation without limitation in time instead of no longer than 3 years - Patients must have a systolic heart failure defined by a reduced ventricular ejection fraction and or defined also through other echocardiographic parameters mentioned in the ESC guidelines for the diagnosis and treatment of acute and chronic heart failure (2012) - Regarding previous prohibited treatments by amiodarone or droderanone, the non inclusion criteria of the protocol are adapted as follow: • Concomitant treatment with oral amiodarone or dronedarone from selection • Concomitant treatment with intravenous amiodarone from selection |

Final version 958/1185

#### 1. AMENDMENT RATIONALE

This amendment is written to update the Sponsor Personnel list following changes in the Clinical team and to extend the planned end date of the study:

- The previous Clinical Study Manager left the team: Gaëlle Alcaraz, and one new Clinical Study Manager has joined the team: Marine Fagard
- Dr Richard Roche (Medical Director) is replaced by Dr Karim Keddad (Head of medical Unit)
- Due to a recruitment rate lower than expected the planned end of study is postponed to September 2017.

#### 2. CHANGES DESCRIPTION

31035 TOULOUSE Cedex 1, France

Phone: +33 5 34 50 61 94

Fax: +33 5 34 50 69 69

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| Sponsor Personnel, page 2 & page 3 | |
| Clinical Study Manager (Monitor) | Clinical Study Manager (Monitor) |
| Gaëlle ALCARAZ | Marine FAGARD |
| Institut de Recherche Pierre Fabre | Institut de Recherche Pierre Fabre |
| Centre de R&D Pierre Fabre | Centre de R&D Pierre Fabre |
| BP 13 562 | BP 13 562 |
| 3, Avenue Hubert Curien | 3, Avenue Hubert Curien |
| 31035 TOULOUSE Cedex 1, France | 31035 TOULOUSE Cedex 1, France |
| Phone: +33 5 34 50 62 16 | Phone: +33 (0)5 34 50 63 54 |
| Fax: + 33 5 34 50 69 69 | Fax: +33 (0)5 34 50 65 92 |
| E-mail: gaelle.alcaraz@pierre-fabre.com | E-mail: marine.fagard@pierre-fabre.com |
| Sponsor Personnel, page 2, page 3 & page 5 | |
| <b>Medical Director</b> | <b>Head of Medical Unit</b> |
| Richard ROCHE, MD | Karim KEDDAD, MD, PhD |
| Institut de Recherche Pierre Fabre | Institut de Recherche Pierre Fabre |
| Centre de R&D Pierre Fabre | Centre de R&D Pierre Fabre |
| BP 13 562 | BP 13 562 |
| 3, Avenue Hubert Curien | 3, Avenue Hubert Curien |

Final version 959/1185

31035 TOULOUSE Cedex 1, France

Phone: +33 5 34 50 61 69

Fax: +33 (0)5 34 50 65 92

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| E-mail: richard.roche@pierre-fabre.com | E-mail: karim.keddad@pierre-fabre.com |
| SYNOPSIS, page 13 Planned Study Period: January 2013 – April 2016 | Planned Study Period: January 2013 – September 2017 |

Final version 960/1185

16.1.1.10. Protocol amendment n° PA07
General and substantial dated on 28 September 2016
linked to Protocol and appendices
(version 9: 28 September 2016)

Final version 961/1185

# CLINICAL STUDY PROTOCOL AMENDMENT n° PA07 (GENERAL –SUBSTANTIAL)

Final version 962/1185

Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne, France

#### CLINICAL STUDY PROTOCOL AMENDMENT n° PA07

(GENERAL – SUBSTANTIAL)

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Pierre Fabre Study Code: F373280 CA 2 01

**EudraCT Number or equivalent:** 2012-003487-48

Karim KEDDAD

INSTITUT DE RECHERCHE PIERRE FABRE

Centre de R&D Pierre Fabre - BP 13562

**Sponsor's Representative:** 3 avenue Hubert Curien

31035 TOULOUSE Cedex 1, FRANCE

Pr Savina NODARI

Department of Clinical and Surgical Specialities, Radiological Science

and Public Health

Section of Cardiovascular Diseases

Study Coordinating Investigator: University Medical School and Spedali Civili Hospital of Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

**Date of amendment PA07:** 28SEP16

The information contained in this document is confidential and is the property of the sponsor Pierre Fabre Médicament. This information is given for the needs of the trial and must not be disclosed without prior written consent of the sponsor Pierre Fabre Médicament. Persons to whom this information is given for the needs of the trial must be informed that it is confidential and must be disclosed.

Final version 963/1185



Study code: F373280 CA 2 01

#### APPROVAL FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Clinical Study Protocol Amendment nº PA07

(GENERAL - SUBSTANTIAL)

Dated: 28SEP16

| Sponsor | s represen | tative(s) |
|---------|------------|-----------|

· Head of Medical Unit

Date

Signature

Dr Karim KEDDAD

**Study Coordinating Investigator:** 

Date:

Signature:

Pr Savina NODARI

ld 10/2016




Study code: F373280 CA 2 01

#### COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

Clinical Study Protocol Amendment no PA07

(GENERAL – SUBSTANTIAL)

Dated: 28SEP16

**Country Coordinating Investigator:** 

Date:

10/2016

Signature:

#### **INVESTIGATOR SIGNATURE FORM**

STUDY: Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

# Clinical Study Protocol Amendment n° PA07 (GENERAL –SUBSTANTIAL)

Dated: 28SEP16

| By my signature below, I, Dr | , hereby confirm that I have read |
|---|---|
| taken note of (and will apply) the modifications | brought by the protocol amendment n° PA07 and l |
| will conduct the trial according to these new modalities. | |
| _ | |
| Date: | Signature: |

Final version 966/1185

# HISTORY OF AMENDMENTS

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| NA | NA | General | NA | Corresponding to Protocol Version 2: Following French CA request (ANSM) and leading to protocol version 2: - Add of a non inclusion criteria: "Breast-feeding female patient" - Add of haematology examination at visit 3 and 6 |
| PA01 | Substantial | Local (Italy) | 01MAR2013 | Corresponding to Protocol Version 3: Integration of the modification included in the protocol version 2 Harmonisation of the protocol and the Informed Consent Form: adjustment of the selection criteria n°10 related to the contraception method addition of a letter that is given by the patient to his/her GENERAL practitioner (GP) precision that the sponsor can not collect a copy of the Informed Consent Form precision that the patient card is in Italian language only (without any English mention) |
| PA02 | Non<br>Substantial | General | 28MAR2013 | Corresponding to Protocol Version 4: - change of Sponsor's Representative (Clinical Study Manager), - modification of the technical handling of the blood samples for determination of red blood cells concentration of DHA: the centrifugation is no more needed, - precision on the function and address of the International Study Coordinator Pr Nodari, - add of address and contacts details of two CRO newly involved in the study: Theradis (in charge of transportation of blood samples to the Analytical centre and material supply) and "Clinact" (in charge of refund of patients expenses linked to the study), - adjustment of the wording, in agreement with the commitment to the French Ethics Committee. In the paragraphe 8.3.2.1, the wording "hematology examination" is replaced by "standard hematologic dosage", - precision of the full title in the study synopsis (in agreement with the commitment to the Spanish Ethics Committee), - correction of a mistake in section 8.1.1.3 (related to TTEM transmission) and sections 3, 9 and study synopsis (related to the definition of INR not stabilized). - addition of the changes included in the local italian |

Final version 967/1185

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | | | substantial protocol amendment (i.e: contraception method, letter to GENERAL Practionner, patient card in Italian and no collection of the consent form by the sponsor in Italy). |
| PA03 | Substantial | General | 23OCT2013 | Corresponding to Protocol Version 5: Fax modification of the sponsor's representatives Planned end of study postponed to January 2015. The authorized history of the first documented persistent atrial fibrillation is less than 3 years. At selection a hyperkalemia or a hypokalemia is better defined by the standards of the local laboratories. Regarding previous treatments by amiodarone the non inclusion criteria of the protocol are adapted as follow: Previous treatment with oral amiodarone within 4 months prior to inclusion Previous treatment with intravenous amiodarone within 4 to 12 months before inclusion Previous treatment with intravenous amiodarone within 4 weeks prior to inclusion. For male with a child-bearing potential partner (in ltaly only): taking into account the duration of spermatogenesis the absolute abstention from sexual intercourse or the use of double barrier contraception method are extended to 3 months after the end of the study. Ranolazine is an antiarrhythmic treatment added to the prohibited treatments. Update of Serious Adverse Events (SAEs) form: Main change is the SAE sending: SAEs have to be reported to the Corporate Vigilance Department, and not anymore to the clinical study manager. Also SAEs can be sent by e-mail and by fax. Addition of Alpha Bioresearch as CRO involved for Feasibility, Monitoring and Regulatory issues in Spain. Correction of some minor typographic errors |
| PA04 | Non<br>Substantial | General | 03JUN2014 | Corresponding to protocol V7: - Precision on the temperature storage of DHA samples - Precision on the BSA formula - Addition of QTcB and QTcF - Precision on TTEM recording timelines - Clarification of the section Interim analysis and data monitoring (13.11) - Clarifications and specifications on some |

Final version 968/1185

| N° | ТҮРЕ | APPLICATION<br>AREA | DATE | MODIFICATIONS |
|---|---|---|---|---|
| | | | | minor points |
| PA05 | Substantial | General | 22OCT2014 | - Planned end of study postponed to April 2016 - Clarifications regarding the management of VKA treatment - Precision regarding the primary efficacy criterion (the time to the first Atrial Fibrillation recurrence or Atrial Flutter emergence) - Deletion of Visit 5 and Visit 8 - Previous history of a first documented persistent Atrial Fibrillation without limitation in time instead of no longer than 3 years - Patients must have a systolic heart failure defined by a reduced ventricular ejection fraction and or defined also through other echocardiographic parameters mentioned in the ESC guidelines for the diagnosis and treatment of acute and chronic heart failure (2012) - Regarding previous prohibited treatments by amiodarone or droderanone, the non inclusion criteria of the protocol are adapted as follow: • Concomitant treatment with oral amiodarone or dronedarone from selection • Concomitant treatment with intravenous amiodarone from selection |
| PA06 | Non<br>substantial | General | 06JUN2016 | Corresponding to protocol V8 Change of sponsor Clinical Study Manager and Clinical Development Physician Planned end of study postponed to September 2017 |

Final version 969/1185

#### 1. AMENDMENT RATIONALE

The F373280 CA 201 planned initially to recruit 152 patients over 6 months across 50 sites in Europe.

Since May 2013, only 134 patients have been randomised and 1 patient is currently enrolled. Due to very slow recruitment over more than 3 years, and, in the absence of any possibility to plan a reliable date for completion of recruitment, the Sponsor has decided to stop the recruitment of patients as of September 23, 2016. This population of maximum 135 randomised patients will be taken into account for efficacy and safety analyses. Despite the loss of power, statistical analyses planned in the protocol are maintained.

There is no unexpected safety signal on the current population, therefore, enrolled patients may continue receiving treatment and participate in the study, as planned by the protocol.

In this context, the purpose of this amendment is limited to the change of the number of patients, the number of IDMC meetings and the planned study period.

This change does apply to all relevant sections of the protocol. Furthermore, all enrolled patients will be informed of this change of recruited patient number.

Final version 970/1185

# 2. CHANGES DESCRIPTION

| PREVIOUS VERSION | MODIFIED VERSION |
|---|---|
| Synopsis Planned Study Period: January 2013 – September 2017 (according to amendment PA06) Number of Patients: 76 x 2 patients | Synopsis Planned Study Period: January 2013 – April 2017 Number of Patients: maximum 135 patients |
| 13.11 INTERIM ANALYSIS AND DATA MONITORING The IDMC will review, three times during the study period (after the first 30 subjects will have been randomized, when the first 80 subjects will have terminated their study participation and when 130 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable. | 13.11 INTERIM ANALYSIS AND DATA MONITORING The IDMC will review, two times during the study period (after the first 30 subjects will have been randomized and when the first 80 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable. |

Final version 971/1185

F 373280 CA 2 01

Final version 972/1185


Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

## CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

Sponsor's Representative: Marine FAGARD

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 63 54 Fax:+33 5 34 50 65 92

E-mail:marine.fagard@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

Associate Professor of Cardiology

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: savinanodari@gmail.com; nodari@med.unibs.it

#### **Version 9 – 28SEP2016**

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 973/1185

## **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

## **Clinical Study Manager (Monitor)**

## Marine FAGARD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 63 54 Fax: +33 5 34 50 65 92

E-mail: marine.fagard@pierre-

fabre.com

## **Head of Medical Unit**

## Karim KEDDAD, MD, PhD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE

Phone: +33 5 34 50 61 69 Fax: +33 5 34 50 65 29

E-mail: karim.keddad@pierre-

fabre.com

Final version 974/1185

#### CONTRACT RESEARCH ORGANISATIONS

## For Feasibility, Monitoring and Regulatory issues (in Hungary, Czech Republic and Italy):

## Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: rzurita@psnglobal.org

## For Feasibility, Monitoring and Regulatory issues (in Spain):

## Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

## For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6. Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

## For Centralised Reading of Holder ECG and TTEM and equipment supply:

## **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

## For intra erythrocyte DHA dosage:

## **Agrocampus Ouest**

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

## For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

#### Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER - FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 975/1185

## Protocol F 373280 CA 2 01 APPROVAL FORM

Protocol Version 9 – 28SEP2016

| Sponsor's Representative | e: |
|--------------------------|----|
|--------------------------|----|

<u>Head of Medical Unit:</u> Karim KEDDAD, MD, PhD Date: 29/00/50

Signature:

Study Coordinating Investigator:

Savina NODARI, MD

Date:

Signature:

20/10/2016

## Protocol F 373280 CA 2 01

## COUNTRY COORDINATING INVESTIGATOR SIGNATURE FORM

**Protocol Version 9 – 28SEP2016** 

| Country | | | | | | | | | | I | - | | 1 | 7 | 4 | 1 | - | L | _( | 4 | / | , | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Country: | • | • | • | • | • | • | • | • | • | • | • | • | | • | • | • | • | • | ٠ | / | • | • | • | • | • | • |

**Country Coordinating Investigator:** 

SAVINA NODARI

"Name"

Data:

Signature:

#### Protocol F 373280 CA 2 01

## INVESTIGATOR SIGNATURE FORM

Protocol Version 9 – 28SEP2016

By my signature below, I, Dr / Pr "

", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 28SEP2016 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

## Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

| * | | Γο | he | ad | lan | ted |
|---|---|----|----|----|-----|-----|
| | _ | | - | uv | ιαρ | icu |

| Date: | Signature: |
|-------|--------------|
| Dute. | Digitatai C. |

Final version 978/1185

## TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|------------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | |
| 1.2.1. | Chemical and pharmaceutical characteristics | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1. | $\mathcal{L}$ | |
| 1.2.2. | | |
| 1.2.2.<br>1.2.2. | $\mathcal{E}$ 1 | |
| 1.2.2. | | |
| 1.2.2. | | |
| 1.2.3. | | |
| 1.3. | STUDY RATIONALE | 29 |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 32 |
| 2.1. | PRIMARY OBJECTIVE | 32 |
| 2.2. | SECONDARY OBJECTIVES | 32 |
| 3. | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 34 |
| 4.1. | OVERALL DESCRIPTION | 34 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 40 |
| 5.3. | NUMBER OF PATIENTS | 41 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 42 |
| 5.6. | WITHDRAWAL CRITERIA | 42 |
| 5.7. | REPLACEMENT OF PATIENTS | 43 |
| 5.8. | POST-STUDY EXCLUSION PERIOD | |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | |
| 6. | STUDY TREATMENT | 44 |

|---|---|---|
| 6.2. | PACKAGING AND LABELLING | 44 |
| 6.2.1. | Packaging | |
| 6.2.2. | Labelling | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 6.5. | DRUG ADMINISTRATION | 47 |
| 6.5.1. | Duration of Treatment | 47 |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration. | 47 |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| 7. ( | CONCOMITANT TREATMENTS | |
| 7.1. | VITAMIN K ANTAGONIST TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | |
| 7.3. | AUTHORISED TREATMENTS | |
| 8. I | EVALUATION CRITERIA | |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence | 50 |
| 8.1.1.1 | • | |
| 8.1.1.2 | | |
| 8.1.1.3 | B. Evaluation Methods | 50 |
| 8.2. | SECONDARY EFFICACY CRITERIA | 51 |
| 8.2.1. | F | |
| 8.2.1.1 | | |
| 8.2.1.2 | | |
| 8.2.1.3 | | |
| 8.2.2. | Duration of AF episodes in the first week following visit 3 (ECV visit) | |
| 8.2.2.1<br>8.2.2.2 | | |
| 8.2.2.3 | | |
| 8.2.3. | Clinical parameters evaluation | |
| 8.2.3.1 | • | |
| 8.2.3.2 | | |
| 8.2.3.3 | | |
| 8.2.3.4 | , <u>,</u> | |
| 8.2.4. | Cardioversion assessment. | |
| 8.2.5. | Evolution of echocardiographic parameters | |
| 8.2.5.1 | | |

Final version 980/1185

| 8.2.5.2. Schedule | 54 |
|---------------------------------------------------------------|---------|
| 8.2.5.3. Evaluation method | 54 |
| 8.3. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONAL DHA | |
| 8.3.1. Definition | |
| 8.3.2. Blood samples | |
| 8.3.2.1. Collection schedule | |
| 8.3.2.2. Technical handling | 55 |
| 8.3.3. DHA concentration measurement | 55 |
| 8.4. SAFETY ASSESSMENT | 56 |
| 8.4.1. Adverse Events | 56 |
| 8.4.2. Laboratory Investigations | 56 |
| 8.4.2.1. Schedule | |
| 8.4.2.2. Technical Procedures and Parameters | |
| 8.4.3. Global Physical Examination | |
| 8.4.4. Vital Signs | |
| 8.4.4.1. Schedule | |
| 8.4.4.2. Technical Procedure and Parameters | |
| 8.4.5. Electrocardiogram (ECG) | |
| 8.4.5.2. Technical Procedure and Parameters | |
| 8.4.6. Coagulation parameters | |
| 8.5. CONCOMITANT TREATMENTS | |
| 8.6. COMPLIANCE | |
| 9. STUDY PROCEDURES | |
| 10. ADVERSE EVENTS: DEFINITION AND REPORTING | 66 |
| 10.1. ADVERSE EVENTS | 66 |
| 10.1.1. Definition of Adverse Events | 66 |
| 10.1.2. Grading of Adverse Events | 67 |
| 10.1.3. Reporting of Adverse Events | 67 |
| 10.2. SERIOUS ADVERSE EVENTS (SAE) | 67 |
| 10.2.1. Definition. | 67 |
| 10.2.2. Reporting of SAE | 68 |
| 10.2.3. Follow-up of SAE | |
| 10.2.4. SAE Occurring After the Study | |
| 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR | 69 |
| 10.4. REPORTING OF PREGNANCY TO THE SPONSOR | 69 |
| 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURI | POSES70 |
| 11. DATA COLLECTION AND STUDY MONITORING | 70 |
| 11.1. DATA COLLECTION | 70 |
| 11.1.1 Case Report Form | 70 |

| 11.1.2. Source Documents | 71 |
|---|---|
| 11.2. STUDY MONITORING | 71 |
| 11.2.1. Monitoring visits | 71 |
| 11.2.1.1. Site Preselection Visit | 72 |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE 12. DATA MANAGEMENT | |
| 12.1. DATA ENTRY | |
| 12.2. DATA CLEANING | |
| 12.3. DATA CODING | |
| 12.4. DATA STORAGE | |
| 12.5. DATABASE LOCK | 75 |
| 13. STATISTICAL ANALYSIS | 75 |
| 13.1. GENERAL CONSIDERATIONS | 75 |
| 13.2. SAMPLE SIZE | 75 |
| 13.4. DATA SETS ANALYSED | 76 |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | 77 |
| 13.5.1. Dropouts | 77 |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 13.7. EFFICACY ANALYSIS | 78 |
| 13.7.1. Primary Criterion | |
| 13.7.1.1. Primary Analysis | 78 |
| 13.7.1.2. Supportive Analysis | |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | 79 |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | |
| 13.8.1. Adverse Events | |
| <ul><li>13.8.2. Clinical Laboratory Evaluation</li><li>13.8.3. Global Physical Examination</li></ul> | |
| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | |
| | _ |

| 13.8.4.1. Vital Sign Measurements Over Time | 83 |
|---|---|
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | 84 |
| 13.10. COMPLIANCE | 84 |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 84 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 85 |
| 14.1. ETHICAL CONDITIONS | 85 |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 85 |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 86 |
| 14.4. PERSONAL DATA PROTECTION | 86 |
| 14.5. INSURANCE POLICY | 87 |
| 15. ADMINISTRATIVE PROCEDURES | 87 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 87 |
| 15.3. END OF THE STUDY | 88 |
| 15.3.1. Definition of the End of Study | 88 |
| 15.3.2. Early Study Termination | |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | |
| 15.4. AUDIT | |
| 15.5. INSPECTION | 89 |
| 15.6. CONFIDENTIALITY | 89 |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 90 |
| 15.9. STUDY RESULTS PUBLICATION | 90 |
| 16. REFERENCES | 92 |
| 17. APPENDICES | 96 |
| 17.1. DECLARATION OF HELSINKI | 97 |
| 17.2. SAE REPORT FORM | 101 |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES | 104 |

## **SYNOPSIS**

| cardioversion in patients with persistent International, multicentric, randomised, Not applicable Pr Savina NODARI International, multicentric F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study puration of AF induced by burst pacing. Moreover, the effectiveness of PolyUn following conditions: — prevention of AF recurrence with amiodarone (add on them— improvement of ventricular following into account these studies, it see | IA delivery (pro-drug) developed for the maintenance ersion in persistent atrial fibrillation (AF) patients with performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the in patients with persistent AF, in co-administration apy) [2] functional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
|---|---|
| Efficacy and safety study of F373280 cardioversion in patients with persistent International, multicentric, randomised, Not applicable Pr Savina NODARI International, multicentric F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study puration of AF induced by burst pacing. Moreover, the effectiveness of PolyUm following conditions: — prevention of AF recurrence with amiodarone (add on them— Improvement of ventricular failures) in patients with Taking into account these studies, it see | Atrial Fibrillation and Chronic Heart Failure. Adouble-blind, placebo controlled study IA delivery (pro-drug) developed for the maintenance ersion in persistent atrial fibrillation (AF) patients with performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the erin patients with persistent AF, in co-administration appy) [2] functional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| cardioversion in patients with persistent International, multicentric, randomised, Not applicable Pr Savina NODARI International, multicentric F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study puration of AF induced by burst pacing. Moreover, the effectiveness of PolyUn following conditions: — prevention of AF recurrence with amiodarone (add on them— improvement of ventricular following into account these studies, it see | Atrial Fibrillation and Chronic Heart Failure. Adouble-blind, placebo controlled study IA delivery (pro-drug) developed for the maintenance ersion in persistent atrial fibrillation (AF) patients with performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the erin patients with persistent AF, in co-administration appy) [2] functional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| Pr Savina NODARI International, multicentric F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study puration of AF induced by burst pacing. Moreover, the effectiveness of PolyUnfollowing conditions: — prevention of AF recurrence with amiodarone (add on there with a miodarone). — Improvement of ventricular for hospitalisation in patients with Taking into account these studies, it see | performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the in patients with persistent AF, in co-administration apy) [2] unctional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| International, multicentric F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study place duration of AF induced by burst pacing. Moreover, the effectiveness of PolyUnfollowing conditions: - prevention of AF recurrence with amiodarone (add on there hospitalisation in patients witl Taking into account these studies, it see | person in persistent atrial fibrillation (AF) patients with performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the in patients with persistent AF, in co-administration apy) [2] functional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| F373280 is a new therapy based on DH of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study place duration of AF induced by burst pacing. Moreover, the effectiveness of PolyUnfollowing conditions: - prevention of AF recurrence with amiodarone (add on there hospitalisation in patients witl Taking into account these studies, it see | performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the in patients with persistent AF, in co-administration apy) [2] unctional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| of sinus rhythm after electrical cardiove chronic heart failure. The results of a pharmacological study pluration of AF induced by burst pacing. Moreover, the effectiveness of PolyUnfollowing conditions: - prevention of AF recurrence with amiodarone (add on them.) - Improvement of ventricular following into account these studies, it see | performed in animals evidenced that DHA reduces the [1] saturated Fatty Acid (PUFA) has been proven in the in patients with persistent AF, in co-administration apy) [2] unctional parameters, morbi-mortality and duration of h heart failure [3, 4, 5] ems that DHA might be of therapeutic interest in the |
| of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing.[1] Moreover, the effectiveness of PolyUnsaturated Fatty Acid (PUFA) has been proven in the | |
| January 2013 – April 2017 | Clinical Phase: IIa |
| <ul> <li>International, multicentre, randomised</li> <li>Selection period</li> <li>Start of treatment 4 weeks before EC</li> <li>Condition to ECV:</li> <li>Ideally INR 2-3 (vitamin K ECV)</li> <li>No spontaneous cardioversion</li> </ul> | V antagonist should be given at least 3 weeks before n before ECV V visit) |
| | <ul> <li>Efficacy of F373280 on the efficience</li> <li>Effect of F373280 on echocardiograph</li> <li>Safety and tolerability of F373280</li> <li>International, multicentre, randomise</li> <li>Selection period</li> <li>Start of treatment 4 weeks before EC</li> <li>Condition to ECV:</li> <li>Ideally INR 2-3 (vitamin K ECV)</li> </ul> |

Final version 984/1185

| | <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms.</li> </ul> |
|---|---|
| | - Treatment duration: 24 weeks |
| Study Schedule: | <ul> <li>7 visits will be scheduled: <ul> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of study treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter device)</li> <li>V4/W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V6/W12* (D84 ± 7 days): follow-up visit <ul> <li>*see amendment PA05 dated 22OCT2014</li> <li>V7/W16 (D112 ± 7 days): follow-up visit</li> <li>V9/W24* (D168 ± 7 days): final study visit</li> <li>*see amendment PA05 dated 22OCT2014</li> </ul> </li> </ul></li></ul> |
| Number of Patients: | Maximum 135 patients |
| Diagnosis and Criteria for Inclusion: | Inclusion Criteria: |
| | Demographic Characteristics and Other Baseline Characteristics: |
| | 1. Men or women aged more than 18 years (inclusive) |
| | 2. Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted |
| | 3. Previous history of first documented episode of persistent AF. |
| | 4. Previous history of ischemic or non ischemic heart failure |
| | 5. NYHA class I or II chronic heart failure at selection and at inclusion |
| | 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF) ≥ 30% and ≤ 45% or for patients with a LVEF > 45%: |
| | an increased left ventricular end-diastolic size |
| | (diameter $\geq 60 \text{ mm and/or} > 32 \text{ mm/m}^2 \text{ and/or volume} > 97 \text{ ml/m}^2$ ) |
| | <ul> <li>and/or an increased left ventricular end-systolic size</li> </ul> |
| | (diameter > 45 mm and/or > 25 mm/m <sup>2</sup> and/or volume > 43 ml/m <sup>2</sup> ) |
| | • and/or a reduced left ventricular outflow tract velocity time integral < 15 cm |
| | 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers |
| | 8. Left atrial area ≤ 40 cm² at selection and at inclusion |
| | 9. Patients treated or having to be treated by vitamin K antagonist |
| | 10. For female patient of child-bearing potential: |
| | In all the countries except Italy: |
| | - Use of an effective method of contraception (hormonal contraception or intra-<br>uterine device) assessed by the investigator, for at least 2 months before the<br>selection in the study, and agreement to go on using it during the whole duration of<br>the study and up to 1 month after the last dose of the study treatment |
| | - Documented as surgically sterilized |
| | • In Italy only: |
| | <ul> <li>Absolute abstention from sexual intercourse during the whole duration of the study<br/>and for a month after the end of the study or</li> </ul> |
| | - Use of double barrier contraception method (use of effective medical contraception |

Final version 985/1185

- method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical / legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### Non-Inclusion Criteria:

Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent AF
- More than two successful cardioversions (electrical or pharmacological) in the last 6 months
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine  $\geq$  25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- 8. Bradycardia (HR ≤ 50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, betablockers, calcium-blockers
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months
- 17. Dietary supplement with  $\omega$  3 or  $\omega$  6 according to investigator's judgement
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible

Final version 986/1185

| | antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel |
|---|---|
| | Other criteria: |
| | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion |
| | 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection |
| | 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints |
| | 23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator |
| | 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship |
| | 25. Breastfeeding female patient |
| Exclusion criteria before V3: | Patients without dyskalemia who will not have INR values $\geq 2$ on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study. |
| | However, if only 2 INR values are $\geq$ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. |
| | If necessary, for meeting these INR conditions, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280<br>Soft Capsules |
| Dose: | Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules Placebo will be administered in the same conditions as the tested product. |
| Mode of Administration: | Oral, one capsule each evening with dinner |
| Evaluation Criteria: | Efficacy evaluation variables: |
| | Primary evaluation variable: |
| | - Time to first Atrial Fibrillation recurrence or atrial flutter emergence defined by the time to first episode of AF or atrial flutter lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 – ECV visit). |
| | Handling of AF recurrences or atrial flutter emergences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24). |
| | For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5). Moreover, during this TTEM period, if patient experiences any AF or atrial flutter symptoms, it should be recorded and documented using the TTEM. |
| | All ECG (Holter and TTEM) will be evaluated by a Central Reading Laboratory. |
| | Secondary evaluation variables: |
| | During the 7-day continuous ECG monitoring, |

Final version 987/1185

- Numbers of AF episodes
- Duration of AF episodes

#### Clinical parameters:

During the whole study:

- Number of recurrence of symptomatic AF episodes
- EHRA score
- Hospitalization for cardiovascular events
- Hospitalization for thromboembolic stroke
- All causes of hospitalization

#### Cardioversion:

- Assessment of spontaneous cardioversion
- Assessment of successful cardioversion
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing an other cardioversion after the initial ECV

#### Other:

- Evolution of echocardiographic parameters (at V4, V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA(ml/m²), Left ventricular end diastolic volume (ml) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (ml))
- Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).

#### Safety criteria:

- Adverse events (observed and / or spontaneously reported)
- Vital signs (Blood pressure (supine and standing), heart rate)
- Physical examination (body weight, body surface area)
- Standard 12-lead ECG: heart rate (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns (ECG not centralized)
- Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets
- Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)
- Coagulation parameters: Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR *(local laboratory)*, Prothrombine Time *(PT)*.

#### **Concomitant treatments**

#### Compliance

#### Statistical Methods:

#### Sample Size:

Assuming an AF recurrence or atrial flutter emergence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%.

## **Primary Efficacy Analysis**

Final version 988/1185

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

#### **Secondary Analyses**

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

#### Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment).

Final version 989/1185

## STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | | V6 | <b>V</b> 7 | | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | | W12<br>(84+/-7D) | W16<br>(112+/-7D) | | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | Х | Х | х | X | Х | Х | X | Х |
| Habits | X | | | | | | | | |
| Global physical examination (body weight) | Х | Х | Х | | X | Х | Х | X | Х |
| Echocardiography | х | Х | | х | | Х | | | Х |
| Eligibility criteria check | Х | Х | | | | | | | |
| Blood pressure, heart rate | X | Х | X | X | X | Х | х | X | Х |
| 12-Lead ECG Recording | Х | Х | X | | X | Х | Х | X | Х |
| INR | <b>+</b> | | | | X | | | X | (2) |
| aPTT, TCT | х | х | х | | X | Х | х | X | Х |
| Biochemistry | Х | | | | | | | | Х |
| Haematology | Х | | х | | | Х | | | Х |
| Urinary pregnancy test | | Х | | | | | | | Х |
| Red Blood Cell concentrations of DHA | | Х | х | | | Х | | | Х |
| Treatment number allocation | | Х | | | | Х | | | |
| IVRS/IWRS | Х | Х | | | | Х | | | |
| ECV (3) | | | Х | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b>—</b> |
| Adverse events recording | | х | x | х | X | Х | Х | X | Х |
| Holter ECG | <b>←</b> → <sup>(4)</sup> | | <b>←</b> | (5) | | | | | |
| TTEM (6) | | | | <b>-</b> | | | | | <b>—</b> |

Final version

990/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of VKA introduction: INR 2 to 3 times a week until stabilization, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) T-EM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms. TTEM once a week even in case of AF recurrence or atrial flutter emergence for at least 10 minutes.

## LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

βHCG : beta human chorionic gonadotrophinBLO : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

 $C_{max}$  : Maximum concentration  $C_{min}$  : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC : "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Transesophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL : High density lipoprotein

Final version 991/1185

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH : International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
IRPF : Institut de Recherche Pierre Fabre
IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC : "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set

QTcB : QT interval using Bazett's correction formula QTcF : QT interval using Fridericia's correction formula

RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

To : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

VKA : Vitamin K Antagonist WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 992/1185

## 1. INTRODUCTION AND STUDY RATIONALE

## 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced

Final version 993/1185

canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95%] confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage

Final version 994/1185

of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61
   +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p <0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

## 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

Final version 995/1185

## 1.2.1. Chemical and pharmaceutical characteristics

## 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

## 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

## 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

Final version 996/1185

## 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an  $IC_{50}$  value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus  $637 \pm 196$  sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and  $79 \pm 51$  sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the compound may exert a similar protective effect [1].

Final version 997/1185

## 1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

## 1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

#### 1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical pharmacokinetic profile of F373280 is not associated with particular alerts concerning the proposed clinical phase IIa study.

#### 1.2.3. Clinical data

## Part A: Single dose

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of

Final version 998/1185

an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

## Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Final version 999/1185

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Final version 1000/1185

Taking into account these studies, it seems that DHA might be of therapeutic interest in the

treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product

(F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic

heart failure.

1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular

diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor

contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for

hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial

infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common

(>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000),

not known (cannot be estimated from the available data).

- The reported adverse events are:

Infection and infestations:

Uncommon: gastroenteritis

Immune system disorders:

Uncommon: hypersensitivity

Metabolism and nutrition disorders:

Rare: hyperglycaemia

Uncommon: dizziness, dysgeusia

Rare: headache

Nervous system disorders:

Vascular disorders:

Very rare: hypotension

Respiratory thoracic and mediastinal disorders:

Final version 1001/1185 Very rare: nasal dryness

Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

• Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene<sup>®</sup> (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after

Final version 1002/1185

administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

## 2. STUDY OBJECTIVES

## 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

Final version 1003/1185

## 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form. A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (vitamin K antagonist, VKA), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence or atrial flutter emergence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with vitamin K antagonist (VKA) for at least 3 weeks before ECV
- ECV will be performed in patients with AF and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values  $\geq 2$  on the 3 last

Final version 1004/1185

tests performed before ECV are required. However, if only 2 INR values are  $\geq 2$  among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Patients who do not revert to sinus rhythm or present an early AF relapse or an early atrial flutter emergence within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be performed throughout the study period. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored once a week between visits using Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

## 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 152 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without study treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Seven visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28-2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)

Final version 1005/1185

- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 6\* (V6): W12 (D84 ± 7D): follow-up visit
   \*see amendment PA05 dated 22OCT2014
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 9\* (V9): W24 (D168 ± 7D): final study visit
   \*see amendment PA05 dated 22OCT2014

## 4.2. DISCUSSION OF THE STUDY DESIGN

## 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Previous history of persistent AF with duration of the current episode from 7 days to 6 months.
- A systolic heart failure defined by a reduced left ventricular ejection fraction (≥ 30% and ≤ 45%) or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size (diameter ≥ 60 mm and/or > 32 mm/m² and/or volume > 97 ml/m²),
  - and/or an increased left ventricular end-systolic size (diameter > 45 mm and/or > 25 mm/m² and/or volume > 43 ml/m²),
  - and/or a reduced left ventricular outflow tract velocity time integral < 15 cm [23, 24].</li>

Final version 1006/1185

According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.

- A Left Atrial Area (LAA) not severely abnormal (no greater than 40 cm<sup>2</sup> as defined in the report from the American Society of Echocardiography's Guideline) [23]. According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

## 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF (or emergence of atrial flutter) since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Final version 1007/1185

Eligible participants will enter a selection phase in which anticoagulant treatment (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) of 2 to 3 before ECV. According to guidelines for the management of AF [6], VKA should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every 4 weeks or 8 weeks (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

## 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/ml and 60 to 90 mg/ml, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough

Final version 1008/1185
fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

## 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted
- 3. Previous history of first documented episode of persistent AF
- 4. Previous history of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF)  $\geq$  30% and  $\leq$  45% or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size

 $(diameter \ge 60 \text{ mm and/or} > 32 \text{ mm/m}^2 \text{ and/or volume} > 97 \text{ ml/m}^2)$ 

• and/or an increased left ventricular end-systolic size

(diameter  $> 45 \text{ mm and/or} > 25 \text{ mm/m}^2 \text{ and/or volume} > 43 \text{ ml/m}^2$ )

- and/or a reduced left ventricular outflow tract velocity time integral < 15 cm
- On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers

Final version 1009/1185

- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by vitamin K antagonist
- 10. For female patient of child-bearing potential:

## • In all the countries except Italy:

- Use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- Documented as surgically sterilized

## • In Italy only:

- Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- Use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

## Ethical /legal considerations:

13. Having signed his/her written informed consent,

Final version 1010/1185

14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent Atrial Fibrillation
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment: TSH  $\pm$  T4L  $\pm$  T3L to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months

Final version 1011/1185

- 16. Treatment with any Polyunsaturated Fatty Acid within the last 3 months
- 17. Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship,
- 25. Breastfeeding female patient.

#### **5.3. NUMBER OF PATIENTS**

76 x 2 patients (taking into account 15 % of non evaluable patients).

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

Final version 1012/1185

## 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form
  - obtain the reason(s) for withdrawal and report it/them in the case report form
  - evaluate the patient's clinical condition
  - if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.
- Erroneous inclusion according to the study protocol. The decision to maintain or not the patient in the study will be taken jointly by the investigator and the sponsor. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with VKA for at least 3 weeks before ECV or who will
  experience a VKA intolerance during the study.
- Patients without dyskalemia who will not have INR values ≥ 2 on the 3 last tests
  performed before ECV should not have an ECV and will be excluded from the study.
  However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed
  if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal

Final version 1013/1185

echocardiography) performed on the same day (before ECV) and the patient can continue the study.

- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early AF
  relapse or early atrial flutter emergence within the observation period after ECV will be
  considered to have finished follow-up.
- Occurrence of AF recurrence or atrial flutter emergence that would require, at the
  investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because
  of intolerable and/or uncomfortable clinical symptoms for instance.

## 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate in another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.
- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

Final version 1014/1185

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the Institut de Recherche Pierre Fabre (IRPF) will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the IRPF according to European Directive and local requirements.

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

Two 12-week treatment units will contain 3 cases, each case of 4-week treatment containing: 10 blister packs of four 1 g F373280 soft capsules or 1 g placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

Final version 1015/1185

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

## 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the IRPF will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection

Final version 1016/1185

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

## 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

At selection visit (V1), practically, once patient's eligibility is confirmed:

- The Investigator:
- Contacts the IVRS/IWRS

Final version 1017/1185

- Answers the questions related to the patient
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

At inclusion visit (V2), the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment.

The Investigator will dispense to the patient the 4-week treatment cases (one or two according to the visit) which label indicates the treatment number and the administration period.

## 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

## 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

Final version 1018/1185


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

#### 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

Final version 1019/1185

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

#### 7.1. VITAMIN K ANTAGONIST TREATMENT

VKA should be given for at least 3 weeks before ECV and continued for the whole study duration. However, VKA should be stopped in case of occurrence of VKA intolerance during the study and the patient should be withdrawn from the study. The VKA used will be left to the decision of each Investigator according to his/her local practice.

#### 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I:
    - o Class IA: Disopyramide, Procainamide, Quinidine
    - o Class IB: Lidocaine, Mexiletine
    - o Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any oral anticoagulant treatment other than VKA: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel
- Dietary supplement with Omega 3 or Omega 6

Final version 1020/1185

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

## 8. EVALUATION CRITERIA

## 8.1. PRIMARY EFFICACY CRITERION

## 8.1.1. Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence

## 8.1.1.1. Definition

Time to first AF recurrence or atrial flutter emergence is defined by the time to first episode of AF or atrial flutter (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. Schedule

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

Final version 1021/1185

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

## • Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM.

Moreover, if patient experiences AF or atrial flutter symptoms during this TTEM period, it should be documented using the TTEM.

In case of AF recurrence or atrial flutter emergence and provided that the patient does not require a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

## • Process of centralisation of ECG (Holter and TTEM)

ECG (Holter and TTEM) will be centralized by the Central Reading Laboratory. The ECG will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign these documents.

The Holter and TTEM process will be fully described in separate documents.

## 8.2. SECONDARY EFFICACY CRITERIA

## 8.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.1.1. *Definition*

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

Final version 1022/1185

#### 8.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

#### 8.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

## 8.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.2.1. Definition

Duration of AF episodes will consist in the sum of duration of each AF episode.

## 8.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

## 8.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

## 8.2.3. Clinical parameters evaluation

#### 8.2.3.1. EHRA score assessment

## 8.2.3.1.1. *Definition*

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

Final version 1023/1185

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

#### 8.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

## 8.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during TTEM period.

## 8.2.3.2. Time to first AF recurrence less than 10 minutes

Time to first AF recurrence less than 10 minutes will be assessed during TTEM period.

## 8.2.3.3. Recurrence of symptomatic AF

Recurrence of symptomatic AF will be assessed during TTEM period.

The number of recurrences of symptomatic AF consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

The time to first symptomatic AF recurrence is defined by the time to first episode of symptomatic AF.

## 8.2.3.4. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
- Hospitalization for AF treatment

Final version 1024/1185

- Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

## 8.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

## 8.2.5. Evolution of echocardiographic parameters

## 8.2.5.1. **Definition**

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), LVEF (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA (ml/m²), Left ventricular end diastolic volume (ml), Left ventricular end systolic volume (ml), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (ml).

## 8.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European

Final version 1025/1185

Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

## 8.3. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.3.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.3.2. Blood samples

#### 8.3.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

## 8.3.2.2. Technical handling

Two blood samples (2 x 4 ml) will be collected in EDTA tubes. They will be homogenized slowly by inverting the tube without shaking, stored between  $+2^{\circ}\text{C}/+8^{\circ}\text{C}$  in a fridge (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between  $+2^{\circ}\text{C}$  and  $+8^{\circ}\text{C}$ ). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### 8.3.3. DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent)

Final version 1026/1185

and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

## **8.4. SAFETY ASSESSMENT**

#### **8.4.1.** Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

## **8.4.2.** Laboratory Investigations

#### 8.4.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kalemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 ml.

#### 8.4.2.2. Technical Procedures and Parameters

The following tests will be performed:

Final version 1027/1185

<u>Haematology</u>: haematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and/or absolute), reticulocytes, platelets.

Biochemistry: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft- Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (ml/min) = [(140-age) x weight / (7.2 x serum creatinine in mg/L)]

in women:

GFR (ml/min) =  $[(140\text{-age}) \times \text{weight} / (7.2 \times \text{serum creatinine in mg/L})] \times 0.85$ 

- with serum creatinine expressed as µmol/l:

GFR (ml/min) = [(140-age) x weight / serum creatinine in  $\mu$ mol/l] x k,where k = 1.23 for men, 1.04 for women.

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

## 8.4.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

Final version 1028/1185

The Body surface area (BSA) will be calculated at the same visits using Mostellers' formula:

 $BSA = [(Weight x Height)/3600]^{1/2}$ 

(Weight in kg, height in cm)

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.4.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

#### 8.4.4.1. Schedule

Vital signs will be measured at each visit.

## 8.4.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

## 8.4.5. Electrocardiogram (ECG)

#### 8.4.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9 using a usual standardised 12-lead cardiograph.

## 8.4.5.2. Technical Procedure and Parameters

## • Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns will be reported in the

Final version 1029/1185

e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

## **8.4.6.** Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

The recommendations for the controls of INR are the following [25, 26]:

- 1) During the pre-cardioversion period, if the anticoagulation by VKA has to be initiated, the treatment must be initiated at least 3 weeks prior to cardioversion then the INR will be monitored as follow:
  - The adjustment of the dosage of VKA should be performed stepwise by controlling INR 2
     to 3 times a week until stabilization within the target range (2 3) on 2 successive tests.
  - When the INR is within the target range (2 3) on 2 successive tests, the dose of VKA should be maintained. Then the controls of INR will be progressively spaced within a few weeks.
  - When INR is stabilized, at least one test should be performed each week.
  - In all cases, an INR control must be performed within 24 h before ECV.
- 2) During the pre-cardioversion period, if the anticoagulation by VKA was already initiated, the INR will be monitored as follow:
  - One INR per week up to ECV
  - An INR control must be performed within 24 h before ECV
- 3) After cardioversion : one INR every 4 weeks
- 4) Throughout the duration of the study if INR > 3 the advocated actions are:

Final version 1030/1185

- No transesophageal echocardiography before cardioversion
- For asymptomatic patients:
  - 3 < INR < 4: no omission of VKA (dose adjustment if required), no vitamin K
  - $4 \le INR < 6$ : omit one dose of VKA, no vitamin K
  - $6 \le INR < 10$ : interrupt VKA, vitamin K 2 mg orally
  - INR ≥ 10: interrupt VKA, vitamin K 5 mg orally
     For INR ≥ 6, an adverse event has to be reported (asymptomatic overdose).

Anti-coagulation by VKA should be given at least 3 weeks before ECV and continued for the whole study duration.

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

The quantity of blood samples collected at each time for coagulation parameters will be 2 ml. Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

#### 8.5. CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements related to patient's concomitant treatments started before selection visit and continued throughout the trial, or started during the trial, can be found in section 7.

#### 8.6. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit (except at visit 4), the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

## 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week - 4 to Week -1):

Final version 1031/1185

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate If the results of the above assessments are compatible with the selection criteria:
  - A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory. The Central Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.

Final version 1032/1185

• The patient will enter the selection and pre-cardioversion periods in which anticoagulant (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) in the range of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

The patient will receive from the investigational centre the participant card to be kept for all the duration of the study.

## Visit 2 - Inclusion Visit (Day 1):

If the patient's behaviour during the selection period and/or the result of complementary examinations, particularly the confirmation of the presence of persistent AF by the Central Reading Laboratory during this period and the laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Urine pregnancy test for women of child bearing potential

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 2 for the first 12-week period.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.4.6) in order to fulfil the ECV conditions (refer to paragraph 3).

Final version 1033/1185

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period (one case of treatment).

## Visit 3 (Week 4: D28 -2/+7 days) cardioversion:

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be performed 4 weeks after randomization in patients with AF. ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values ≥ 2 on the 3 last tests performed before ECV are required. However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge.

Final version 1034/1185

Patients who will not revert to sinus rhythm or with early AF relapse or early atrial flutter emergence within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 8-week period (two cases of treatment).

## Visit 4 (Week 5: D35 -2/+7 days):

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Bodyweight (bodyweight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to perform one transmission per week from this visit (initial call to perform with the patient) to the visit 9 (week 24 – end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

## Visit 6\* (Week 12: D84 $\pm$ 7 days) - Visit 7 (Week 16: D112 $\pm$ 7 days) :

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following criteria:

Adverse events

Final version 1035/1185

- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV due to occurrence of VKA intolerance, the monitoring of INR, aPTT and TCT should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- The cardiac monitoring will be continued using the TTEM device through one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

In addition, at visit 6:

- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

At the end of each visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next treatment period: one case at visit 6 and two cases at visit 7.

## Visit 9\* - End-of-Study Visit (Week 24: D168 $\pm$ 7 days):

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight

Final version 1036/1185

Vital signs

• 12-lead ECG

• Laboratory examination: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time

(aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.

• Urine pregnancy test for women of childbearing potential

• Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused

soft capsules.

The total volume of blood collected should be about 90 ml for the study duration (30 ml for the

total volume of haematology and biochemistry, 2 ml for each blood samples for coagulations

parameters and 4 ml for each blood samples of DHA).

10. ADVERSE EVENTS: DEFINITION AND REPORTING

10.1. ADVERSE EVENTS

10.1.1. Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, i.e. any subjective signs and

symptoms or change in a concomitant disease present at the Selection Visit considered or not

related to the treatment.

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for

vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should

be repeated until the values return to normal or to a stable status. Abnormal results are defined as

those falling out of the laboratory normal ranges and that are clinically significant. The frequency

of such checks should be defined by the Investigator according to the degree of abnormality.

Final version 1037/1185

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

## 10.1.2. Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

## 10.1.3. Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

## 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Final version 1038/1185

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

- \* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:
  - planned (as per protocol) medical/surgical procedure
  - preparation for routine health assessment/procedure (e.g. routine colonoscopy)
  - planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
  - administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

## 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

## HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

## 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

Final version 1039/1185

The serious adverse events must be followed up until resolution or stabilisation.

## 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Final version 1040/1185

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

## 11. DATA COLLECTION AND STUDY MONITORING

## 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF. Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

Final version 1041/1185

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

#### 11.2. STUDY MONITORING

## 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

Final version 1042/1185

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
- has received the technical protocol, administrative and financial agreement signed by all parties
- has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

Final version 1043/1185

## 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

## 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

Final version 1044/1185
#### 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

#### 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

#### 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

#### 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate the coding.

Final version 1045/1185

#### 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

#### 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

#### 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

#### 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

#### 13.2. SAMPLE SIZE

Assuming an AF recurrence or atrial flutter emergence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients

Final version 1046/1185

per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

#### 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4). A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the

Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

#### 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol

Final version 1047/1185

deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

#### 13.5. HANDLING OF DROPOUTS AND MISSING DATA

#### **13.5.1. Dropouts**

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

#### 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

#### 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

#### 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- <u>Quantitative parameters</u> will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- <u>Qualitative parameters</u> will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

Final version 1048/1185

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

#### 13.7. EFFICACY ANALYSIS

#### 13.7.1. Primary Criterion

#### 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence of AF or atrial flutter emergence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

#### 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

#### 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

#### 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

#### 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

Final version 1049/1185

#### 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

#### 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

#### 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

#### 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

Final version 1050/1185

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event.
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs
- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity
- And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Final version 1051/1185

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (reported in 1% patients in any group) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (for all patients).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

#### 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Final version 1052/1185

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

#### 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

Final version 1053/1185

#### 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

#### 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

#### 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

#### 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

#### 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

Final version 1054/1185

#### 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

#### 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

#### 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

### 13.11. INTERIM ANALYSIS AND DATA MONITORING

No analyses of efficacy data are planned for IDMC that ensures that the overall probability of type I error is controlled. No Type I error and sample size adjustments are necessary. Any recommendations of the IDMC to alter study conduct will be based on safety, so IDMC monitoring of the study will not affect the statistical operating characteristics of the final analysis.

Final version 1055/1185

The IDMC will review, two times during the study period (after the first 30 subjects will have been randomized and when the first 80 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable.

#### 14. GENERAL ETHICAL CONSIDERATIONS

#### 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

#### 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

Final version 1056/1185

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

#### 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

Final version 1057/1185

#### 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor Pierre Fabre Médicament, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

#### 15. ADMINISTRATIVE PROCEDURES

#### 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities.

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

#### 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all
  patients included in the trial or not.

Final version 1058/1185

- Retains a list of the patient's names, addresses (and/or number of medical file), code numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

#### 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

## 15.3.2. Early Study Termination

#### 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

### 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

Final version 1059/1185

#### **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at Pierre Fabre Médicament and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

#### 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

#### 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

#### 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

Final version 1060/1185

#### 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

#### 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

Final version 1061/1185

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 1062/1185

#### 16. REFERENCES

- [1]. F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2]. NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- [3]. NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L. Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy *J. Am. Coll. Cardiol.* 2011;57;870-879
- [4]. MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study *American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5*
- [5]. GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6]. CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct;31(19):2369-429
- [7]. KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 1063/1185

[8]. BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9]. OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10]. BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11]. TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12]. LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13]. METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr (2007); 85 : 1225.* 

[14]. ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15]. TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? *J. Am. Coll. Cardiol.* 1998;31;167-173

[16]. SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6):652-9.

[17]. LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

Final version 1064/1185

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human. *Lipids*, 2010, 45, 11-19.

[18]. HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

[19]. ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion

World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain

[20]. KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G.

Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association.

Europace 2007, 9, 1006-1023

#### [21]. EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter.

EMA/CHMA/EWP/213056/2010

#### [22]. OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955–961

[23]. ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

[24]. JOHN J.V. McMURRAY, STAMATIS ADAMOPOULOS, STEFAN D. ANKER, ANGELO AURICCHIO, MICHAEL BÖHM, KENNETH DICKSTEIN, VOLKMAR FALK, GERASIMOS FILIPPATOS, CÂNDIDA FONSECA, MIGUEL ANGEL GOMEZ-SANCHEZ, TINY JAARSMA, LARS KØBER, GREGORY Y.H. LIP, ALDO PIETRO MAGGIONI, ALEXANDER PARKHOMENKO, BURKERT

Final version 1065/1185

# M. PIESKE, BOGDAN A. POPESCU, PER K. RØNNEVIK, FRANS H. RUTTEN, JUERG SCHWITTER, PETAR SEFEROVIC, JANINA STEPINSKA, PEDRO T. TRINDADE, ADRIAAN A. VOORS, FAIEZ ZANNAD, ANDREAS ZEIHER

ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012 European Heart Journal (2012) 33, 1787–1847

[25]. AGENCE NATIONALE DE SECURITE DU MEDICAMENT ET DES PRODUITS DE SANTE (ANSM).

Bon usage des médicaments antivitamine K (AVK) Actualisation – Juillet 2012

[26]. GILLES PERNOD, ANNE GODIER, CLAIRE GOZALO, BENJAMIN TREMEY, PIERRE SIE

French clinical practice guidelines on the management of patients on vitamin K antagonists in at-risk situations (overdose, risk of bleeding, and active bleeding) *Thrombosis Research 126 (2010) e167–e174* 

Final version 1066/1185

# 17. APPENDICES

Final version 1067/1185

#### 17.1. DECLARATION OF HELSINKI

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

#### B. PRINCIPLES FOR ALL MEDICAL RESEARCH

11. It is the duty of physicians who participate in medical research to protect the life, health, dignity,

Final version 1068/1185

- integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.
- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be

Final version 1069/1185

- enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

Final version 1070/1185

# C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 1071/1185

# 17.2. SAE REPORT FORM

Final version 1072/1185

| NOTIFICATION OF SERIOUS ADVERSE EVENT (SAE) OR PREGNANCY TO PIERRE FABRE CORPORATE VIGILANCES DIVISION |
|---|
| TO BE TRANSMITTED TO THE CORPORATE VIGILANCES DIVISION BY E-MAIL WITHIN 24H TO HQ.pharmacovigilance@pierre-fabre.com OR BY FAX WITHIN 24H – Fax N°: 33 (0) 1.49.10.80.90 |
| Transmission date (ddmmyyyy) Country: |
| SAE N° FIRST NOTIFICATION FOLLOW-UP N° |
| > SUBJECT CHARACTERISTICS |
| Birth date |
| Gender |
| > DESCRIPTION OF THE EVENT |
| The serious adverse event resulted in: ☐ Death (whatever may be the cause) ☐ Hospitalisation (*) or extension thereof ☐ Life threatening ☐ Invalidity or disability ☐ Cancer ☐ Other (any other serious clinical or laboratory event according to the investigator or the protocol, overdosage meeting seriousness criteria, suicide attempts) ☐ Other fact to be notified: ☐ Pregnancy exposure |
| Nature of the event (if clinical nature, indicate the diagnosis or the major symptom): |
| AE onset date (ddmmyyyy) |
| <b>Seriousness onset date</b> _ _ _ _ (ddmmyyyy) |
| Summary description (if clinical cause, significant history, progression of event, available laboratory results, etc): |
| (*) Except hospitalisations with durations and goals planned in the protocol |
| > THE SAE IN RELATION TO THE TRIAL |
| TREATMENT NUMBER • Time of occurrence of SAE |
| _ |
| ☐ During the selection or run-in period ☐ During the administration phase of the study treatment ☐ After the administration phase of the study treatment |
| • Date of first study treatment administration |
| • Date of last study treatment administration before the occurence of SAE |
| Was the blind broken? □ Yes □ No □ Not applicable If yes, or if this is an open study, drug(s) administered: |
| Conditions of administration (cycles(s), daily dose(s), route(s) of administration, etc): |

Final version 1073/1185

| Transmission date | (ddmmyyyy) Country: | | | | | |
|---|---|---|---|---|---|---|
| SAE N° | FIRST NOTIFICATION G FOLLOW-UP N° | | | | | |
| > CONCOMITANT MI<br>(EXCEPT THE TREA | EDICATION SING<br>TIMENTS GIVEN | CE TRIAL INITIATION FOR THE SAE) | ON and UP UNTIL TH | E OCCURRENCE O | F THE SAE | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| > MEASURES TAKEN | FOLLOWING T | HE SAE | | | | |
| • Study treatment | | | | | | |
| ☐ No change | | | | | 1 1 | |
| ☐ Dosage modifi | ication, specify : | | Modification D | ate: | //_ | |
| □ Temporarily d | iscontinued | | Readministration date | e : | //_ | |
| ■ Withdrawn | | | End date | : | // | |
| ☐ Not applicable | ; | | | | | |
| • The event led to: | | | | | | |
| ☐ Prescription of | f corrective or symp | otomatic treatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| (Of Invity) | | / / | | / / | | |
| | | / / | | / / | | |
| | | / / | | / / | | |
| ☐ Discontinuation | on of concomitant tr | reatments: | | | | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, specify | y : | | | | | |
| > OUTCOME | | | | | | |
| □ Not recovered/No □ Recovered/Resolv | ved with sequelae | □ Recovering/Resolvi □ Fatal | ☐ Unknown | d/Resolved | | |
| | , has an autopsy be | | | | | |
| > INVESTIGATOR CA | AUSALITY ASSES | | | e as soon as possible) | | |
| Study drug: ☐ Not Suspected | Related to study protocol: Suspected Suspected Suspected | | | | | |

Final version 1074/1185

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values<sup>(\mathridge{m})</sup>

| PARAMETERS | | UNIT | PSC | |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | _ | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| TO THE TOTAL | Protein | g/l | 11 | 10 |
| | Cholesterol | mmol/l | - | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | pH | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/l | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 1075/1185

<sup>(¤)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

# **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| PARAMETERS | | CNALV |
|---|---|---|
| | | <ul> <li>Decrease of at least 2g/dl and value &lt; 10 g/dl whatever the baseline value</li> <li>If missing baseline: value &lt;10g/dl</li> </ul> |
| NEUTRO | PHILS | • < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing | g value for neutrophils) | • < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> <li>if baseline value &gt; 2.5 N:</li> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline: <ul> <li>AP &gt; 1.25 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>AP &gt; 2 N</li> </ul> </li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline: <ul> <li>TB &gt; 1.5 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>TB &gt; 2 N</li> </ul> </li> </ul> |

## N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 1076/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \le 50$ mmHg and decrease $\ge 10$ mmHg |
| HR | Increase ≥ 10 bpm | HR ≥ 110 bpm and increase ≥ 10 bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>paseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| > 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | Talue Classes for the Minimum Post-baseline Value for each parameter | | | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤ <i>50</i> | ≤90 | ≤ 50 | ≤50 |
| [120;140] | [80;90[ | <i>[50;75]</i> | [90 ;120] | [50;80[ | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3BI 2 90 01 DBI 2 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq$ 20 mmHg or DBP Decrease $\geq$ 10 mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 1077/1185

#### **Title of the study**:

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

An international, multicentric, randomised, double-blind, placebo controlled study.

Dear patient,

You are currently or you have been taking part of the above-named research study evaluating the effect of F373280 on the maintenance of normal cardiac rhythm after direct electrical cardioversion in patients with persistent Atrial Fibrillation and cardiac failure.

The purpose of this letter it is to provide you with new information about the study.

In fact, as it was explained to you at the beginning of your participation in the trial, it was planned to involve in the study 152 male or female patients suffering from persistent Atrial Fibrillation, aged more than 18 years, in several countries.

However, since May 2013, only 88% of needed patients have been involved in the study. Therefore, due to very slow recruitment over more than 3 years, the Sponsor, Pierre Fabre Médicament, has decided to stop prematurely the recruitment of patients. There will be a maximum of 135 patients involved in this trial.

This decision is not related to any new safety information linked to the product. Ongoing patients may therefore, continue being involved in the study, receiving treatment; and, analyses of all collected data are maintained.

All the other information that were given to you previously remain unchanged

#### **CONTACT FOR FURTHER INFORMATION**

If you feel that you would need more information or should there be anything that is not clear, don't hesitate to ask your investigator (doctor in charge of the study):

| Dr | Telephone number : |
|----|--------------------|

We thank you for your participation in this study.

Final version 1078/1185

16.1.1.11. Protocol amendment n° PA07 Local (Italy) and substantial dated on 06 December 2016 linked to Protocol and appendices (version 9: 06 December 2016)

Final version 1079/1185

F 373280 CA 2 01

Final version 1080/1185


Pierre Fabre Médicament Represented by: Institut de Recherche Pierre Fabre 45, Place Abel Gance F-92100 Boulogne

# CLINICAL STUDY PROTOCOL

Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure.

International, multicentric, randomised, double-blind, placebo controlled study

F373280 / Soft Capsules / 1g

Pierre Fabre Study Code: F 373280 CA 2 01 EudraCT Number: 2012 – 003487 - 48

**Sponsor's Representative:** Marine FAGARD

INSTITUT DE RECHERCHE PIERRE FABRE -

Centre de R&D Pierre Fabre - BP 13562

3 avenue Hubert Curien

31035 TOULOUSE Cédex 1, FRANCE

Phone: +33 5 34 50 63 54 Fax:+33 5 34 50 65 92

E-mail:marine.fagard@pierre-fabre.com

Study Coordinating Investigator Pr Savina NODARI

Associate Professor of Cardiology

Department of Clinical and Surgical Specialities,

Radiological Science and Public Health Section of Cardiovascular Diseases

University Medical School and Spedali Civili Hospital of

Brescia

c/o Spedali Civili di Brescia Piazzale Spedali Civili, 1 25123 - BRESCIA, ITALY

Phone: +39 030 3996 587 - +39 030 393849

Fax: +39 030 3700 359

E-mail: savinanodari@gmail.com; nodari@med.unibs.it

#### **Version 9 – 06DEC2016**

The information contained in this document is confidential and is the property of the Sponsor, Pierre Fabre Medicament. This information is given for the needs of the study and must not be disclosed without prior written consent of the Sponsor Pierre Fabre Medicament. Persons to whom this information is given for the needs of the study must be informed that it is confidential and must not be disclosed.

Final version 1081/1185

# **SPONSOR PERSONNEL**

# PIERRE FABRE MEDICAMENT represented by Institut de Recherche Pierre Fabre

# **Clinical Study Manager (Monitor)**

#### Marine FAGARD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE Phone: +33 5 34 50 63 54 Fax: +33 5 34 50 65 92

E-mail: marine.fagard@pierre-

fabre.com

# **Head of Medical Unit**

# Karim KEDDAD, MD, PhD

Institut de Recherche Pierre Fabre Centre de R&D Pierre Fabre BP 13 562 3, Avenue Hubert Curien 31035 TOULOUSE Cedex 1, FRANCE

Phone: +33 5 34 50 61 69 Fax: +33 5 34 50 65 29

E-mail: karim.keddad@pierre-

fabre.com

Final version 1082/1185

#### CONTRACT RESEARCH ORGANISATIONS

# For Feasibility, Monitoring and Regulatory issues (in Hungary, Czech Republic and Italy):

#### Pharmaceutical Service Network (PSN)

Rufino Gonzalez

28 037 Madrid - SPAIN

Phone: +34 91 375 6930 - Fax: +34 91 375 6931

E-mail: rzurita@psnglobal.org

# For Feasibility, Monitoring and Regulatory issues (in Spain):

# Alpha Bioresearch

Paseo de la Castellana, 163 - 2º Izquierda

28 046 Madrid - SPAIN

Phone: +34 91 745 2520 - Fax: +34 91 745 0653 E-mail: teresa.bricio@alphabioresearch.com

#### For Centralised Randomisation and Electronic Case Report Form

#### S-Clinica

6, Chaussée de Boondael

B-1050 Brussels - BELGIUM

Phone: +32 2 645 0567 - Fax: +32 2 645 0569

E-mail: irena.seredina@s-clinica.com

# For Centralised Reading of Holter ECG and TTEM and equipment supply:

# **Biomedical System**

1945 Chaussée de Wavre

B-1160 Brussels - BELGIUM

Phone: +32 2 661 20 70 - Fax: +32 2 661 20 71

E-mail: sjacobs@biomedsys.com

#### For intra erythrocyte DHA dosage:

#### **Agrocampus Ouest**

Laboratoire de Biochimie

65 rue de Saint Brieuc – CS 84215

35042 RENNES Cedex - FRANCE

Phone: +33 2 23 48 55 49 - Fax: +33 2 23 48 55 50 E-mail: daniel.catheline@agrocampus-ouest.fr

# For transportation of blood sample to the Analytical centre (Agrocampus) and material supply:

# Theradis Pharma

41, chemin des Presses

06800 CAGNES-SUR-MER - FRANCE

Phone: +33 (0)4 97 02 07 07 - Fax: +33 (0)4 97 10 08 78

E-mail: chantal.raffy@theradis.pharma.com

Final version 1083/1185

# Protocol F 373280 CA 2 01

#### APPROVAL FORM

Protocol Version 9 - 06DEC2016

| S | ponsor <sup>,</sup> | S | Re | presenta | tive: |
|---|---------------------|---|----|----------|-------|

Head of Medical Unit:

Karim KEDDAD, MD, PhD

Date:

Signature:

Study Coordinating Investigator:

Savina NODARI, MD

Date:

13/Dec/2016 Sorrie

Signature:

# Protocol F 373280 CA 2 01

# COUNTRY COORDINATING INVESTIGATOR

### **SIGNATURE FORM**

Protocol Version 9 – 06DEC2016

| | TTALY | 0 |
|----------|-------|---|
| Country: | | |

**Country Coordinating Investigator:** 

"Name"

Date:

Signature:

SAJINA NODARI

13/Dec/2016

# Protocol F 373280 CA 2 01

# INVESTIGATOR SIGNATURE FORM

Protocol Version 9 – 06DEC2016

By my signature below, I, Dr / Pr " SAVINA WODEN", hereby confirm that I agree:

- to conduct the trial described in the protocol F 373280 CA 2 01, dated 06DEC2016 in compliance with GCP, with applicable regulatory requirements and with the protocol agreed upon by the Sponsor Pierre Fabre Médicament and given approval / favourable\* opinion by the Ethics Committee;
- to document the delegation of significant study-related tasks and to notify the Sponsor of changes in site personnel involved in the study;
- · to comply with the procedure for data recording and reporting;
- to allow monitoring, auditing and inspection;
- to retain the trial-related essential documents until the Sponsor informs that these documents are no longer needed.

Furthermore, I hereby confirm that I will have and will use the available adequate resources, personnel and facilities for conduct this trial.

I have been informed that certain regulatory authorities require the Sponsor Pierre Fabre Médicament to obtain and supply details about the investigator's ownership interest in the Sponsor or the study drug, and more generally about his/her financial relationships with the Sponsor. The Sponsor will use and disclose the information solely for the purpose of complying with regulatory requirements.

#### Hence I agree:

- to supply the Sponsor with any information regarding ownership interest and financial relationships with the Sponsor (including those of my spouse and dependent children);
- to promptly update this information if any relevant changes occur during the course of the study and for 1 year following completion of the study;
- that the Sponsor may disclose this information about such ownership interests and financial relationships to regulatory authorities.

\* To be adapted

13/Dec/2016

Signature:

# TABLE OF CONTENTS OF CLINICAL STUDY PROTOCOL

| 1. | INTRODUCTION AND STUDY RATIONALE | 22 |
|------------------|---------------------------------------------------|----|
| 1.1. | TARGET PATHOLOGY AND THERAPY | 22 |
| 1.2. | INFORMATION ON THE TEST PRODUCT | |
| 1.2.1. | Chemical and pharmaceutical characteristics | 25 |
| 1.2.1. | 1. Nomenclature and structure | 25 |
| 1.2.1. | $\mathcal{L}$ | |
| 1.2.2. | | |
| 1.2.2.<br>1.2.2. | $\mathcal{E}$ 1 | |
| 1.2.2. | J F | |
| 1.2.2. | 6, 1 | |
| 1.2.3. | Clinical data | 27 |
| 1.3. | STUDY RATIONALE | 29 |
| 1.4. | OVERALL RISK AND BENEFIT ASSESSMENT | 30 |
| 2. | STUDY OBJECTIVES | 32 |
| 2.1. | PRIMARY OBJECTIVE | 32 |
| 2.2. | SECONDARY OBJECTIVES | 32 |
| 3. | ETHICAL CONSIDERATIONS RELATING TO THE STUDY | 33 |
| 4. | STUDY DESIGN | 34 |
| 4.1. | OVERALL DESCRIPTION | 34 |
| 4.2. | DISCUSSION OF THE STUDY DESIGN | 35 |
| 4.2.1. | Choice of the Study Population | 35 |
| 4.2.2. | | |
| 4.2.3. | | |
| 4.2.4. | Choice of the Sample Size | 38 |
| 5. | STUDY POPULATION | 38 |
| 5.1. | INCLUSION CRITERIA | |
| 5.2. | NON INCLUSION CRITERIA | 40 |
| 5.3. | NUMBER OF PATIENTS | 41 |
| 5.4. | RECRUITMENT MODALITIES | 41 |
| 5.5. | PATIENT IDENTIFICATION | 42 |
| 5.6. | WITHDRAWAL CRITERIA | 42 |
| 5.7. | REPLACEMENT OF PATIENTS | |
| 5.8. | POST-STUDY EXCLUSION PERIOD | |
| 5.9. | STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S) | |
| 6. | STUDY TREATMENT | 44 |

|---|---|---|
| 6.2. | PACKAGING AND LABELLING | 44 |
| 6.2.1. | Packaging | 44 |
| 6.2.2. | Labelling | |
| 6.3. | DISTRIBUTION TO CENTRE AND STORAGE | 45 |
| 6.4. | ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT | 46 |
| 6.5. | DRUG ADMINISTRATION | 47 |
| 6.5.1. | Duration of Treatment | 47 |
| 6.5.2. | Dose Schedule | |
| 6.5.3. | Route and Conditions of Administration. | 47 |
| 6.6. | ACCOUNTABILITY ON SITE AND RETURN/DESTRUCTION OF | 40 |
| - <b>-</b> | INVESTIGATIONAL PRODUCT | |
| 6.7. | RECALL OF INVESTIGATIONAL PRODUCTS | |
| 7. | CONCOMITANT TREATMENTS | 48 |
| 7.1. | VITAMIN K ANTAGONIST TREATMENT | 49 |
| 7.2. | PROHIBITED TREATMENTS | 49 |
| 7.3. | AUTHORISED TREATMENTS | 50 |
| 8. 1 | EVALUATION CRITERIA | 50 |
| 8.1. | PRIMARY EFFICACY CRITERION | 50 |
| 8.1.1. | Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence | 50 |
| 8.1.1.1 | | |
| 8.1.1.2 | | |
| 8.1.1.3 | | |
| 8.2. | SECONDARY EFFICACY CRITERIA | 51 |
| 8.2.1. | F | |
| 8.2.1.1 | | |
| 8.2.1.2 | | |
| 8.2.1.3 | | |
| 8.2.2.<br>8.2.2.1 | Duration of AF episodes in the first week following visit 3 (ECV visit) Definition | |
| 8.2.2.2 | | |
| 8.2.2.3 | | |
| 8.2.3. | Clinical parameters evaluation | |
| 8.2.3.1 | <u>.</u> | |
| 8.2.3.2 | 2. Time to first AF recurrence less than 10 minutes | 53 |
| 8.2.3.3 | J = 1 | |
| 8.2.3.4 | 1 | |
| 8.2.4. | Cardioversion assessment | |
| 8.2.5. | Evolution of echocardiographic parameters | |
| 8.2.5.1 | Definition | 54 |

Final version 1088/1185

| 8.2.5.2 | 2. Schedule | 54 |
|---|---|---|
| 8.2.5.3 | B. Evaluation method | 54 |
| 8.3. | BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA | 55 |
| 021 | Definition | |
| 8.3.1.<br>8.3.2. | Blood samples | |
| 8.3.2.1 | 1 | |
| 8.3.2.2 | | |
| 8.3.3. | DHA concentration measurement | |
| 8.4. | SAFETY ASSESSMENT | 56 |
| 8.4.1. | Adverse Events | 56 |
| 8.4.2. | Laboratory Investigations | |
| 8.4.2.1 | | |
| 8.4.2.2 | | |
| 8.4.3. | Global Physical Examination | |
| 8.4.4.<br>8.4.4.1 | Vital Signs | |
| 8.4.4.2 | | |
| 8.4.5. | Electrocardiogram (ECG) | |
| 8.4.5.1 | | |
| 8.4.5.2 | 2. Technical Procedure and Parameters | 58 |
| 8.4.6. | Coagulation parameters | 59 |
| 8.5. | CONCOMITANT TREATMENTS | |
| 8.6. | COMPLIANCE | 60 |
| 9. 8 | STUDY PROCEDURES | 60 |
| <b>10.</b> A | ADVERSE EVENTS: DEFINITION AND REPORTING | 66 |
| 10.1. | ADVERSE EVENTS | 66 |
| 10.1.1 | . Definition of Adverse Events | 66 |
| 10.1.2 | | |
| 10.1.3 | | |
| 10.2. | SERIOUS ADVERSE EVENTS (SAE) | |
| 10.2.1 | | |
| 10.2.2 | | |
| 10.2.3 | 1 | |
| | SAE Occurring After the Study | |
| 10.3. | REPORTING OF OVERDOSAGE TO THE SPONSOR | |
| 10.4.<br>10.5. | SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES | |
| | DATA COLLECTION AND STUDY MONITORING | |
| 11.1. | DATA COLLECTION | |
| 11.1.1. | . Case Report Form | 70 |

| 11.1.2. Source Documents | 71 |
|---|---|
| 11.2. STUDY MONITORING | 71 |
| 11.2.1. Monitoring visits | 71 |
| 11.2.1.1. Site Preselection Visit | 72 |
| 11.2.1.2. Initiation Visit | |
| 11.2.1.3. Follow-up Visits | |
| 11.2.1.4. Closing Visit | |
| 11.2.2. Direct Access to Source Documents | |
| 11.3. INDEPENDENT DATA MONITORING COMMITTEE | |
| 12. DATA MANAGEMENT | 74 |
| 12.1. DATA ENTRY | 74 |
| 12.2. DATA CLEANING | 74 |
| 12.3. DATA CODING | 74 |
| 12.4. DATA STORAGE | 75 |
| 12.5. DATABASE LOCK | 75 |
| 13. STATISTICAL ANALYSIS | |
| 13.1. GENERAL CONSIDERATIONS | |
| 13.2. SAMPLE SIZE | |
| 13.3. PROTOCOL DEVIATIONS | |
| 13.4. DATA SETS ANALYSED | |
| 13.5. HANDLING OF DROPOUTS AND MISSING DATA | |
| 13.5.1. Dropouts | |
| 13.5.2. Repositioning of Visits | |
| 13.5.3. Missing Data | |
| 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 77 |
| 13.7. EFFICACY ANALYSIS | |
| 13.7.1. Primary Criterion | 78 |
| 13.7.1.1. Primary Analysis | |
| 13.7.1.2. Supportive Analysis | |
| 13.7.1.3. Additional Analysis | 78 |
| 13.7.2. Secondary Criteria | 78 |
| 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3 | |
| 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic | |
| 13.7.2.4. Clinical parameters evaluation | |
| 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA | |
| 13.8. SAFETY ANALYSIS | 79 |
| 13.8.1. Adverse Events | |
| 13.8.2. Clinical Laboratory Evaluation | 81 |
| 13.8.3. Global Physical Examination | 82 |

| 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety | 83 |
|---|---|
| 13.8.4.1. Vital Sign Measurements Over Time | 83 |
| 13.8.4.2. Body weight | |
| 13.8.4.3. Individual Patient Changes | |
| 13.8.5. ECG | |
| 13.8.6. Coagulation parameters | |
| 13.9. CONCOMITANT TREATMENTS | |
| 13.10. COMPLIANCE | |
| 13.11. INTERIM ANALYSIS AND DATA MONITORING | 84 |
| 14. GENERAL ETHICAL CONSIDERATIONS | 85 |
| 14.1. ETHICAL CONDITIONS | |
| 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS | 85 |
| 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM | 86 |
| 14.4. PERSONAL DATA PROTECTION | 86 |
| 14.5. INSURANCE POLICY | 87 |
| 15. ADMINISTRATIVE PROCEDURES | 87 |
| 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE | 87 |
| 15.3. END OF THE STUDY | |
| 15.3.1. Definition of the End of Study | 88 |
| 15.3.2. Early Study Termination | 88 |
| 15.3.2.1. Early Study Termination Decided by the Sponsor | |
| 15.3.2.2. Early Study Termination Decided by the Competent Authorities | 88 |
| 15.4. AUDIT | 89 |
| 15.5. INSPECTION | 89 |
| 15.6. CONFIDENTIALITY | 89 |
| 15.7. CLINICAL STUDY REPORT | 89 |
| 15.8. STUDY RESULTS COMMUNICATION | 90 |
| 15.9. STUDY RESULTS PUBLICATION | 90 |
| 16. REFERENCES | 92 |
| 17. APPENDICES | |
| 17.1. DECLARATION OF HELSINKI | 97 |
| 17.2. SAE REPORT FORM | |
| 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY | |
| CLINICALLY SIGNIFICANT CHANGES AND VALUES | 104 |

Final version 1091/1185

# **SYNOPSIS**

| Name of Sponsor: | Pierre Fabre Médicament represented | by the Institut de Recherche Pierre Fabre (IRPF) |
|---|---|---|
| Name of Finished Product: | Not applicable | |
| Name of Active Substance: | F373280 (Panthenyl-Ester of DHA) | |
| Title of the Study: | Efficacy and safety study of F373280 for maintenance of sinus rhythm after electrical cardioversion in patients with persistent Atrial Fibrillation and Chronic Heart Failure. International, multicentric, randomised, double-blind, placebo controlled study | |
| Abbreviated Title: | Not applicable | |
| Study Coordinating Investigator: | Pr Savina NODARI | |
| <b>Study Centres:</b> | International, multicentric | |
| Publication / Rationale: | F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after electrical cardioversion in persistent atrial fibrillation (AF) patients with chronic heart failure. The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing.[1] Moreover, the effectiveness of PolyUnsaturated Fatty Acid (PUFA) has been proven in the following conditions: — prevention of AF recurrence in patients with persistent AF, in co-administration with amiodarone (add on therapy) [2] — Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5] Taking into account these studies, it seems that DHA might be of therapeutic interest in the treatment of patients with both persistent atrial fibrillation and chronic heart failure. This phase IIa study is designed to assess the efficacy and the safety of the investigational product (F373280) for maintenance of sinus rhythm after electrical cardioversion (ECV) in patients with persistent atrial fibrillation and chronic heart failure. | |
| Planned Study Period: | January 2013 – April 2017 | Clinical Phase: IIa |
| Objectives: | Primary: - Efficacy of F373280 on the maintenance of sinus rhythm after direct electrical cardioversion in patients with persistent atrial fibrillation and chronic heart failure Secondary: - Efficacy of F373280 on the efficiency of direct electrical cardioversion - Effect of F373280 on echocardiographic parameters - Safety and tolerability of F373280 | |
| Methodology: | <ul> <li>International, multicentre, randomised, double-blind, placebo-controlled</li> <li>Selection period</li> <li>Start of treatment 4 weeks before ECV</li> <li>Condition to ECV: <ul> <li>Ideally INR 2-3 (vitamin K antagonist should be given at least 3 weeks bet ECV)</li> <li>No spontaneous cardioversion before ECV</li> </ul> </li> <li>Follow-up 20 weeks after visit 3 (ECV visit)</li> <li>Condition: successful ECV or spontaneous CV</li> </ul> | |
| | - Cardiac monitoring: | |

Final version 1092/1185

| | <ul> <li>7-days continuous ECG ambulatory recording (Holter ECG) between visit 3 (ECV visit) and visit 4 (week 5) in patients with sinusal rhythm</li> <li>TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms.</li> </ul> |
|---|---|
| | - Treatment duration: 24 weeks |
| Study Schedule: | <ul> <li>7 visits will be scheduled:</li> <li>V1/W-4 to W-1: selection visit (7 to 28 days before the inclusion visit)</li> <li>V2/D1: Inclusion visit (start of study treatment)</li> <li>V3/W4 (D28 -2/+7 days): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter device)</li> <li>V4/W5 (D35 -2/+7 days): follow-up visit (removing of the Holter device and installation of the TTEM)</li> <li>V6/W12* (D84 ± 7 days): follow-up visit</li> <li>*see amendment PA05 dated 22OCT2014</li> <li>V7/W16 (D112 ± 7 days): follow-up visit</li> <li>V9/W24* (D168 ± 7 days): final study visit</li> <li>*see amendment PA05 dated 22OCT2014</li> </ul> |
| Number of Patients: | Maximum 135 patients |
| Diagnosis and Criteria for Inclusion: | Inclusion Criteria: |
| | Demographic Characteristics and Other Baseline Characteristics: |
| | 1. Men or women aged more than 18 years (inclusive) |
| | 2. Patients with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted |
| | 3. Previous history of first documented episode of persistent AF. |
| | 4. Previous history of ischemic or non ischemic heart failure |
| | 5. NYHA class I or II chronic heart failure at selection and at inclusion |
| | 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF) ≥ 30% and ≤ 45% or for patients with a LVEF > 45%: |
| | an increased left ventricular end-diastolic size |
| | (diameter $\geq 60 \text{ mm}$ and/or $> 32 \text{ mm/m}^2$ and/or volume $> 97 \text{ ml/m}^2$ ) |
| | <ul> <li>and/or an increased left ventricular end-systolic size</li> </ul> |
| | (diameter $> 45$ mm and/or $> 25$ mm/m <sup>2</sup> and/or volume $> 43$ ml/m <sup>2</sup> ) |
| | <ul> <li>and/or a reduced left ventricular outflow tract velocity time integral &lt; 15 cm</li> </ul> |
| | 7. On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers |
| | 8. Left atrial area ≤ 40 cm² at selection and at inclusion |
| | 9. Patients treated or having to be treated by vitamin K antagonist |
| | 10. For female patient of child-bearing potential: |
| | • In all the countries except Italy: |
| | <ul> <li>Use of an effective method of contraception (hormonal contraception or intra-<br/>uterine device) assessed by the investigator, for at least 2 months before the<br/>selection in the study, and agreement to go on using it during the whole duration of<br/>the study and up to 1 month after the last dose of the study treatment</li> </ul> |
| | - Documented as surgically sterilized |
| | • In Italy only: |
| | <ul> <li>Absolute abstention from sexual intercourse during the whole duration of the study<br/>and for a month after the end of the study or</li> </ul> |
| | - Use of double barrier contraception method (use of effective medical contraception |

Final version 1093/1185

- method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

#### Ethical / legal considerations:

- 13. Having signed his/her written informed consent,
- 14. Affiliated to a social security system, or is beneficiary (if applicable in the national regulation)

#### **Non-Inclusion Criteria**:

Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent AF
- More than two successful cardioversions (electrical or pharmacological) in the last 6 months
- Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV)
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment:  $TSH \pm T4L \pm T3L$  to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine  $\geq$  25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- Bradycardia (HR ≤ 50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any antiarrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, betablockers, calcium-blockers
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months
- 16. Treatment with any Polyunsaturated Fatty Acid (PUFA) within the last 3 months
- 17. Dietary supplement with  $\omega$  3 or  $\omega$  6 according to investigator's judgement
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible

Final version 1094/1185

| | antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel |
|---|---|
| | Other criteria: |
| | 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion |
| | 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection |
| | 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself/herself to its constraints |
| | 23. Patient family member or work associate (secretary, nurse, technician,) of the Investigator |
| | 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship |
| | 25. Breastfeeding female patient |
| Exclusion criteria before V3: | Patients without dyskalemia who will not have INR values $\geq 2$ on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study. |
| | However, if only 2 INR values are $\geq$ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. |
| | If necessary, for meeting these INR conditions, the ECV (and following visits) could be postponed by 7 days. |
| Test Product: | F373280<br>Soft Capsules |
| Dose: | Arm with 1g of F373280 |
| Mode of Administration: | Oral, one capsule each evening with dinner. |
| <b>Duration of Treatment:</b> | 24 weeks of treatment exposure with F373280 (25 weeks if ECV postponed by 1 week) |
| Reference Therapy | Placebo soft capsules Placebo will be administered in the same conditions as the tested product. |
| Mode of Administration: | Oral, one capsule each evening with dinner |
| Evaluation Criteria: | Efficacy evaluation variables: |
| | Primary evaluation variable: |
| | - Time to first Atrial Fibrillation recurrence or atrial flutter emergence defined by the time to first episode of AF or atrial flutter lasting for at least 10 minutes (Follow up of 20 weeks after visit 3 – ECV visit). |
| | Handling of AF recurrences or atrial flutter emergences: 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) between visit 3 (ECV visit) and visit 4 (week 5). Then, the follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24). |
| | For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5). Moreover, during this TTEM period, if patient experiences any AF or atrial flutter symptoms, it should be recorded and documented using the TTEM. |
| | All ECG (Holter and TTEM) will be evaluated by a Central Reading Laboratory. |
| | Secondary evaluation variables: |
| | During the 7-day continuous ECG monitoring, |

Final version 1095/1185

- Numbers of AF episodes
- Duration of AF episodes

#### Clinical parameters:

During the whole study:

- Number of recurrence of symptomatic AF episodes
- EHRA score
- Hospitalization for cardiovascular events
- Hospitalization for thromboembolic stroke
- All causes of hospitalization

#### Cardioversion:

- Assessment of spontaneous cardioversion
- Assessment of successful cardioversion
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing an other cardioversion after the initial ECV

#### Other:

- Evolution of echocardiographic parameters (at V4, V6 and V9) (Left atrial diameter (mm), Left atrial area (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), Left ventricular ejection fraction (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA(ml/m²), Left ventricular end diastolic diameter (mm), Left ventricular end diastolic volume (ml) Left ventricular end systolic diameter (mm), Left ventricular end systolic volume (ml))
- Evolution of omega 3 index and intra erythrocyte DHA (For this assessment samples will be centralized).

#### Safety criteria:

- Adverse events (observed and / or spontaneously reported)
- Vital signs (Blood pressure (supine and standing), heart rate)
- Physical examination (body weight, body surface area)
- **Standard 12-lead ECG**: heart rate (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns (ECG not centralized)
- Haematology: haematocrit, haemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, WBC differential count, reticulocytes, platelets
- **Biochemistry:** sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT, albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose, total cholesterol, cholesterol (HDL, LDL), triglycerides, creatin phosphokinase (CPK) fibrinogen (local laboratory)
- **Coagulation parameters:** Activated partial thromboplastin time (aPTT), thrombin clotting time (TCT), INR *(local laboratory)*, Prothrombine Time *(PT)*.

#### **Concomitant treatments**

#### Compliance

#### Statistical Methods:

#### Sample Size:

Assuming an AF recurrence or atrial flutter emergence rate under placebo of 85%, a power of 80%, an alpha risk of 5% and a rate of not assessable patients of 15%, 76 randomised patients per group will be necessary, using a log-rank test of survival curves, a difference between groups of 20%.

# **Primary Efficacy Analysis**

Final version 1096/1185

The primary analysis, performed on the Full Analysis Set (FAS: all randomised patients with at least one dose of treatment and with a successful cardioversion observed at visit 3), will be a survival analysis using the Kaplan Meier method and Cox regression model.

# **Secondary Analyses**

All secondary efficacy criteria will be described and compared using appropriate tests on the FAS.

#### Safety Analyses

Descriptive statistics will be performed on the Safety Set (all randomised patients with at least one dose of treatment).

Final version 1097/1185

# STUDY FLOW-CHART

| F373280 CA 201 | V1 | V2 | V3 | V4 | | V6 | <b>V</b> 7 | | V9 |
|---|---|---|---|---|---|---|---|---|---|
| Weeks | W-4 to W-1 | D1 | W4<br>(28 -2D/+7 D) | W5<br>(35 -2D/+7 D) | | W12<br>(84+/-7D) | W16<br>(112+/-7D) | | W24<br>(168+/-7D) |
| Outpatient or Hospitalization (1) | | | Х | | | | | | |
| Informed consent | Х | | | | | | | | |
| Demographic characteristics | Х | | | | | | | | |
| Medico-surgical history | Х | | | | | | | | |
| Concomitant disease | Х | | | | | | | | |
| Concomitant treatment | Х | Х | Х | Х | X | Х | Х | X | Х |
| Habits | Х | | | | | | | | |
| Global physical examination (body weight) | X | X | X | | X | Х | х | X | X |
| Echocardiography | Х | Х | | Х | | Х | | | Х |
| Eligibility criteria check | X | X | | | | | | | |
| Blood pressure, heart rate | X | X | X | X | X | X | x | X | X |
| 12-Lead ECG Recording | X | X | X | | X | X | X | X | Х |
| INR | ◆ | | | | X | | | X | (2) |
| aPTT, TCT | Х | Х | Х | | X | Х | Х | X | Х |
| Biochemistry | Х | | | | | | | | Х |
| Haematology | Х | | X | | | Х | | | X |
| Urinary pregnancy test | | X | | | | | | | Х |
| Red Blood Cell concentrations of DHA | | X | X | | | X | | | X |
| Treatment number allocation | | X | | | | X | | | |
| IVRS/IWRS | Х | X | | | | X | | | |
| ECV (3) | | | X | | | | | | |
| Drug administration | | <b>←</b> | | | | | | | <b></b> |
| Adverse events recording | | x | x | х | X | Х | Х | X | Х |
| Holter ECG | <b>←</b> → <sup>(4)</sup> | | <b>←</b> | (5) | | | | | |
| TTEM (6) | | | | <b>—</b> | | | | | <b>—</b> |

Final version 1098/1185

<sup>(1)</sup> Outpatient or hospitalization according to clinical practice of the centre (less or more than 24 hours)
(2) In case of VKA introduction: INR 2 to 3 times a week until stabilization, then weekly until the ECV, then every 4 weeks after ECV

<sup>(3)</sup> In patients with AF

<sup>(4) 24-</sup>hour Holter ECG

<sup>(6) 7-</sup>day Holter ECG
(6) T-EM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24) and at any time in case of AF or atrial flutter symptoms. TTEM once a week even in case of AF recurrence or atrial flutter emergence for at least 10 minutes.

# LIST OF ABBREVIATIONS

aPTT : Activated partial thromboplastin time

AE : Adverse event
AF : Atrial fibrillation
ALA : Alpha-linoleic acid
ALT : Alanine aminotransferase
AST : Aspartate aminotransferase

AUC : Area under the plasma concentration versus time curve AUC<sub>inf</sub> : Total area under the curve extrapolated to infinity

βHCG : beta human chorionic gonadotrophinBLO : Below the limit of quantification

BMI : Body mass index
BP : Blood pressure
BSA : Body Surface Area

CEP : Protocol evaluation committee

CHMP : Committee for medicinal products for human use

 $C_{max}$  : Maximum concentration  $C_{min}$  : Minimum concentration

CNALV : Clinically noteworthy abnormal laboratory value

CPK : Creatin phosphokinase

CPP : Comité de protection des personnes

CRA : Clinical research associate

CRT : Cardiac resynchronization therapy

CSC : "Clinically Significant Change", i.e., Predefined potentially clinically significant

change leading to a potentially clinically significant value (vital signs)

CV : Coefficient of variation
DBP : Diastolic blood pressure
DHA : Docosahexaenoic acid
EC : Ethics committee
ECG : Electrocardiogram

ECHO – TE : Transesophageal echocardiograph

ECV : Electrical cardioversion

EHRA : European heart rhythm association

EPA : Eicosapentaenoic acid e-CRF : Electronic case report form

FAS : Full analysis set

Fe : Fraction of the administered drug excreted in urine

GCP : Good clinical practice GFR : Glomerular Filtration Rate

HBs : Hepatitis B antigen HCV : Hepatitis C virus

HDL : High density lipoprotein

Final version 1099/1185

HF : Heart failure

HIV : Human immunodeficiency virus

HR : Heart rate

ICH : International conference on harmonisation of technical requirements for

registration of pharmaceuticals for human use

IDMC : Independent data monitoring committee

INR : International normalized ratio
 IRPF : Institut de Recherche Pierre Fabre
 IVRS : Interactive voice response system

LAA : Left atrial area

LC/MS-MS : Liquid chromatography with tandem mass spectrometry

LDL : Low density lipoprotein LOQ : Limit of quantification

LVEF : Left ventricular ejection fraction

MedDRA : Medical dictionary for regulatory activities

MR : Mineralocorticoid receptor
MR perfusion : Magnetic Resonance perfusion
MTD : Maximum tolerated dose

N : Number of determinations or replicates

NOAEL : No observed adverse effect level NYHA : New York heart association

od : Once a day

PC : "Predefined Change", i.e., Predefined potentially clinically significant change (lab

or vital signs)

PCA : PC leading to an out-of-range value (lab values)

PFB : Pierre Fabre Biométrie

PSC : Potentially Clinically Significant Change PSCV : Potentially Clinically Significant Value

PUFA : PolyUnsaturated fatty acid

p.o. : Per os

PP : Per protocol data set

QTcB : QT interval using Bazett's correction formula QTcF : QT interval using Fridericia's correction formula

RBC : Red blood cells

SAE : Serious adverse event
SBP : Systolic blood pressure
SD : Standard deviation
T<sub>1/2</sub> : Terminal half-life

To : Time of drug administration

 $T_{max}$ : Time to reach the maximal concentration

TCT : Thrombin clotting time

TEAEs : Treatment emergent adverse events
TTEM : TransTelephonic ECG monitoring

VKA : Vitamin K Antagonist WBC : White blood cells

WHO-DRUG: World health organization drug reference list

Final version 1100/1185

#### 1. INTRODUCTION AND STUDY RATIONALE

#### 1.1. TARGET PATHOLOGY AND THERAPY

Atrial Fibrillation (AF) is a supraventricular arrhythmia characterized by uncoordinated atrial electric activity with consequent deterioration of atrial mechanical function. It is the most common sustained cardiac rhythm disorder, increasing in prevalence with age. Haemodynamic impairment and thromboembolic events related to AF result in significant morbidity and mortality [7].

In 2009, Decision Resources estimated that there were 7.8 million diagnosed prevalent cases of AF in US, Europe and Japan. This age-related pathology should increase to 9.4 million cases in 2019.

Except for the conventional class I and class III anti-arrhythmic agents, the Polyunsaturated Fatty Acids (PUFAs) constitute one emerging antiarrhythmic therapy. These compounds potently address the AF substrate by directly targeting both the electrical and the structural remodelling of the deficient atria. The n-3 PUFAs, essential for human, are alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). First, PUFAs specifically modulate ionic channels by fastening their inactivating mode which renders these compounds selective for pathological situations (such as AF) without any major effect in normal conditions. PUFAs are "open K<sub>v1.5</sub> channel blockers" leading to a lengthening of atrial action potential duration and are "persistent Na<sub>v1.5</sub> channel blockers" leading to hyperpolarization of diastolic resting potential. Second, PUFAs influence structural remodelling through their anti-inflammatory effects as they directly compete with arachidonic acid in the production of inflammatory eicosanoids. In summary, PUFAs share unique, well-tolerated antiarrhythmic potential by interacting with the electrical and structural remodelling during sustained AF. In animal studies, it was recently demonstrated that DHA is particularly effective in pathologic conditions such as ischemia and/or AF.

The potential anti-arrythmic effects of a PUFA were previously developed in AF: nicotinyl ester of DHA (pro-drug based on DHA delivery) was assessed in a two-week ventricular tachypaced

Final version 1101/1185

canine model. Dogs were subjected to 4 weeks of medication prior to undergoing an electrophysiology study, and received either placebo or nicotinyl ester of DHA. Dogs were tachypaced at 240 beats per min for the final two weeks of the treatment plan. The results showed that the tested PUFA reduced the duration of AF induced by burst pacing, and the incidence of sustained AF, compared to dogs treated with the placebo [1].

In clinical practice, Nodari and coll [2] assessed n-3 PUFAs in the prevention of AF recurrences after electrical cardioversion (ECV). All included patients were treated with amiodarone and a renin-angiotensin-aldosterone system inhibitor. The 199 patients were assigned either to placebo or n-3 PUFAs 2 g/d and then underwent direct ECV 4 weeks later. The primary end point was the maintenance of sinus rhythm at 1 year after cardioversion. At the 1-year follow up, the maintenance of sinus rhythm was significantly higher in the n-3 PUFAs treated patients compared with the placebo group (hazard ratio, 0.62 [95% confidence interval, 0.52 to 0.72] and 0.36 [95% confidence interval, 0.26 to 0.46], respectively; p = 0.0001). The study concludes that in patients with persistent AF on amiodarone and a renin-angiotensin-aldosterone system inhibitor, the addition of n-3 PUFAs 2 g/d improves the probability of the maintenance of sinus rhythm after direct current cardioversion. Previously, during the World Congress of Cardiology in 2006, an abstract reported the effectiveness of PUFAs on top of traditional treatment (amiodarone, beta blockers, renin-angiotensin-aldosterone system inhibitor) in the prevention of AF relapses in patients having undergone ECV. In the PUFA group, AF relapses were significantly lower than in the placebo group at 1 month (3.3% vs 10%; p = 0.043), at 3 months (10% vs 25%; p = 0.004) and at 6 months (13.3% vs 40%; p < 0.0001) [19].

In contrast, in the general AF population (paroxystic atrial fibrillation and persistent atrial fibrillation), PUFAs failed to prove their efficacy [7] because of the absence of cardiac remodelling or because of a short pre-treatment duration before ECV (1 week) [8]. The effects of PUFAs were only observed in patients with persistent AF on add on therapy and after a sufficient pre-treatment before ECV. Persistent AF is commonly associated to heart failure. Previous studies performed in heart failure population demonstrated the benefit of PUFAs on the improvement of functional ventricular parameters and morbi-mortality, and on the reduction of hospitalisation [3, 4, 5].

Nodari and coll [3] performed a trial in patients with chronic heart failure (NYHA I to III and LVEF< 45%). After a treatment of 133 patients with PUFAs (n=67) or placebo (n=66) at a dosage

Final version 1102/1185

of 5 g/day for 1 month, then 2 g/day for 11 months, the n-3 PUFAs group and the placebo group differed significantly (p <0.001) in regard to:

- LVEF (increased by 10.4% and decreased by 5.0%, respectively)
- peak VO<sub>2</sub> (increased by 6.2% and decreased by 4.5%, respectively)
- exercise duration (increased by 7.5% and decreased by 4.8%, respectively)
- mean New York Heart Association functional class (decreased from 1.88+/- 0.33 to 1.61
   +/- 0.49 and increased from 1.83+/- 0.38 to 2.14 +/- 0.65, respectively).

The hospitalization rates for patients with HF were 6% in the n-3 PUFAs and 30% in the placebo group (p < 0.0002).

Moertl and coll [4] performed a dose-ranging study in patients with a more severe chronic heart failure (NYHA III and IV and LVEF < 35%). It was a double-blind, randomised, controlled pilot trial in 43 patients treated with PUFAs or placebo for 3 months (1 g/d n3-PUFA (n = 14), 4 g/d n3-PUFA (n = 13), or placebo (n = 16)). After treatment, left ventricular ejection fraction increased in a dose-dependent manner (p = 0.01 for linear trend) in the 4 g/d (baseline vs 3 months [mean  $\pm$  SD]: 24%  $\pm$  7% vs 29%  $\pm$  8%, p = 0.005) and 1 g/d treatment groups (24%  $\pm$  8% vs 27%  $\pm$  8%, p = 0.02).

No changes in any investigated parameters were noted with placebo.

Taking into account these studies performed with PUFAs, it seems that the best target for DHA is persistent AF in patients with heart failure. The aim of this proof of concept study is to assess in stand alone therapy (without association of other anti-arrhythmic treatments), the effect of F373280 in patients with persistent AF and heart failure in the maintenance of sinus rhythm after ECV.

#### 1.2. INFORMATION ON THE TEST PRODUCT

F373280 or panthenyl ester of DHA is the mono-ester of panthotenic alcohol and DHA, selected to be developed for the management of AF.

F373280 is a prodrug of DHA.

A brief summary of F373280 known characteristics is presented in this section. For further details, please refer to the F373280 *Investigator's Brochure*. [1]

Final version 1103/1185

# 1.2.1. Chemical and pharmaceutical characteristics

### 1.2.1.1. Nomenclature and structure

Chemical name (IUPAC):

(4Z,7Z,10Z,13Z,16Z,19Z)-3-((R)-2,4-dihydroxy-3,3-diméthylbutanamido) propyl docosa-4,7,10,13,16,19-hexaenoate

Structural formula:

Laboratory code: F373280

Molecular formula: C<sub>31</sub>H<sub>49</sub>NO<sub>5</sub>

Molecular mass: 515.7

# 1.2.1.2. Physical and chemical general properties

Appearance: Clear oily viscous liquid

Solubilities:

Water: Practically insoluble

Alcohol: Very soluble

- Trimethylpentane: Slightly soluble

# 1.2.2. Non-clinical Data

Non-clinical data are exhaustively detailed in the Investigator's brochure [1]. A brief summary is provided below.

Final version 1104/1185

# 1.2.2.1. Pharmacological profile

F373280 (mono-ester of panthotenic alcohol and DHA) is a novel pro-drug of DHA which exerts antiarrhythmic properties by interacting with the electrical and structural remodelling of the atria.

Experimental investigations were conducted in HEK293 cell line transfected with human Kv1.5 channel using the whole cell patch clamp technique to evaluate whether F373280 could block the sustained component of  $I_{Kv1.5}$ . F373280 concentration-dependently reduced Kv1.5 channel activity with an IC<sub>50</sub> value of 13.7  $\mu$ M.

The effects of F373280 on atrial effective refractory period were investigated in anesthetized pig using a conventional pacing protocol through epicardial electrodes placed on the left atrium. F373280 administered as a bolus and an infusion (10 mg/kg) significantly increased atrial effective refractory period (23.8  $\pm$  2.2 ms versus -7.3  $\pm$  11.5 ms in the presence of vehicle, p < 0.05). In addition, F373280 was devoid of significant effect on the hemodynamic and the electrocardiogram (ECG) intervals.

Proof of the pharmacological concept was performed with a different DHA derivative named: Nicotinyl ester of DHA (pro-drug based on DHA delivery). Ventricular tachypacing-induced congestive heart failure provides a clinically-relevant animal model of AF associated with structural remodelling, as is often seen clinically. It has been shown that sustained oral PUFA administration suppresses congestive heart failure-induced AF-promotion and fibrosis in the ventricular tachypacing canine model. Nicotinyl ester of DHA was tested in this model, at 1 g/day and 5 g/day, during 4 weeks, to prevent congestive heart failure-related atrial structural remodelling and AF promotion in dogs. Nicotinyl ester of DHA dose dependently reduced heart failure-induced increases in AF duration (989  $\pm$  111 sec, n=5 in the presence of placebo versus 637  $\pm$  196 sec, n=5 in the presence of 1 g/kg/d Nicotinyl ester of DHA and 79  $\pm$  51 sec, n=5, in the presence of 5 g/kg/d Nicotinyl ester of DHA). The protective effect of Nicotinyl ester of DHA was associated with a marked increase of plasma level of DHA and important incorporation of DHA in the left atrial tissue. Because F373280 similarly to Nicotinyl ester of DHA increases plasma level of DHA, it could be estimated that the compound may exert a similar protective effect [1].

Final version 1105/1185

# 1.2.2.2. Safety pharmacology

A battery of safety pharmacology studies was performed to evaluate the effects of F373280 on the central nervous, cardiovascular and respiratory systems. Data of these studies are exhaustively detailed in the Investigator's brochure [1].

No particular alerts were evidenced with F373280.

# 1.2.2.3. Toxicology profile

Concerning the toxicological data, 4-week and 26-week repeat-dose studies in rat and dog were performed. Compared to the high administered doses of F373280 (500 to 2000 mg/kg/day), low circulating concentrations of F373280 were measured.

During these toxicity studies, no toxicity was observed in rat after 4 and 26 weeks of dosing and in dog after 4 weeks of dosing. A NOAEL of 2000 mg/kg/day was established in these repeat toxicity studies.

During the 26-week toxicity study in dogs, the NOAEL was set at 1000 mg/kg/day based on changes observed on red blood cell parameters.

Based on toxicological profiles, F373280 is considered to support the proposed clinical trial.

#### 1.2.2.4. Pharmacokinetic data

According to animal studies described in the Investigator's brochure [1], the non-clinical pharmacokinetic profile of F373280 is not associated with particular alerts concerning the proposed clinical phase IIa study.

#### 1.2.3. Clinical data

#### Part A: Single dose

Six consecutive single ascending doses were tested (0.5 g, 1 g, 2 g, 4 g, 8 g and 16 g) on 6 independent cohorts of 8 subjects (6 verum + 2 placebo). 49 subjects were treated and 48 completed the study.

No Serious Adverse Events (SAE) occurred in the course of the study.

Regarding the reported Treatment Emergent Adverse Events (TEAEs) that were judged by the Investigator as having a causal relationship with the study drug administration in the absence of

Final version 1106/1185

an alternative explanation, 3 TEAEs were observed in the placebo group (palpitation, dizziness in standing position, symptomatic orthostatic hypotension without loss of consciousness) and 4 in the group of F373280 at the dosage of 16 g (meteorism, liquid stool, symptomatic orthostatic hypotension and dizziness in standing position). None of these adverse events (AE) were reported in the groups of F373280 at the dosages of 0.5 g, 1 g, 2 g, 4 g and 8 g.

After a single administration of the different tested doses no difference between the tested product and placebo has been reported, regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters (related to coagulation: platelets and fibrinogen) and coagulation parameters (bleeding time, prothrombin time/INR, activated partial thromboplastin time, thrombin clotting time). Variations of these parameters were within the physiological ranges.

After single oral administration of F373280 from 0.5 g to 16 g in 36 young healthy male subjects (6 per dose level), the following was observed:

- **F373280**: Whatever the tested dose there is no circulating F373280 in plasma: only few, sparse and non consecutive samples with quantifiable level of F373280 close to LOQ were observed. This confirms that F373280 is a prodrug.
- **Panthenol**: Cmax and AUC increased with the administered dose between 0.5 and 16 g. Panthenol concentrations were rapidly cleared from plasma with a mean terminal half-life around 2 hours.
- **DHA:** after 0.5 and 1 g, low increased in DHA plasma concentrations compared to the baseline levels led to a high inter-individual variability of the corresponding Pharmacokinetics parameters. Plasma exposure in DHA increased with the administered dose between 2 and 16 g with no departure from proportionality (baseline corrected parameters).

#### Part B: Multiple doses

Three consecutive repeated ascending doses (1, 2 and 4 g) were tested on 3 independent cohorts of 12 subjects (9 verum + 3 placebo, double blind). 36 subjects completed the study. Each treatment was administered over a period of 28 days. Pharmacokinetic parameters were assessed over a period of 14 days.

Final version 1107/1185

Among the TEAE judged by the investigator as suspected to F373280, 5/9 TEAEs were classified according the System Organ Class in vascular system disorder with orthostatic hypotension (2 in the 1 g group, 1 in the 2 g group and 2 in the 4 g group) and 4/9 were classified in nervous system disorder with 3 dizziness (2 in the 2 g group and 1 in the 4 g group) and 1 migraine (in the 1 g group). These TEAEs have already been reported with PUFAs and are commonly observed in phase I studies.

After a repeated administration of the different tested doses, no difference between the tested products and placebo was reported regarding vital signs (heart rate, systolic blood pressure and diastolic blood pressure), biological parameters. The assessment of coagulation parameters and platelet function after administration of repeated dose of F373280 did not report any bleeding issue. The reported changes in coagulation parameters and platelet function were within physiological ranges.

After a 14-day repeated oral administration of F373280 from 1 g to 4 g, the following was observed:

- ✓ **Panthenol**: Cmax and AUC increased with the administered dose between 1 and 4 g. No accumulation of panthenol in plasma was observed.
- ✓ **DHA**: Plasma exposure increased with dose. A 2-fold accumulation in total plasma exposure of DHA was observed after 14 days of administration, whatever the administered dose.

#### 1.3. STUDY RATIONALE

F373280 is a new therapy based on DHA delivery (pro-drug) developed for the maintenance of sinus rhythm after ECV in persistent AF patients with chronic heart failure.

The results of a pharmacological study performed in animals evidenced that DHA reduces the duration of AF induced by burst pacing [1].

Moreover, the effectiveness of PUFAs has been proven in the following conditions:

- Prevention of AF recurrence in patients with persistent AF in co-administration with amiodarone (add on therapy) [2],
- Improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

Final version 1108/1185

Taking into account these studies, it seems that DHA might be of therapeutic interest in the

treatment of patients with both persistent AF and chronic heart failure.

This phase IIa study is designed to assess the efficacy and the safety of the investigational product

(F373280) for maintenance of sinus rhythm after ECV in patients with persistent AF and chronic

heart failure.

1.4. OVERALL RISK AND BENEFIT ASSESSMENT

F373280 is a new pro-drug of DHA.

DHA is a well-known long chain PUFAs with a long-term clinical experience in cardiovascular

diseases. DHA is contained in several medicinal products such as Omacor®, (1 g of Omacor

contains about 320 mg of DHA acid) marketed by Laboratoires Pierre Fabre for

hypertriglyceridemia and as an adjuvant treatment for secondary prevention after myocardial

infarction. According to the summary product characteristics of Omacor® [9]:

- The frequencies of adverse reactions are ranked according to the following: common

(>1/100, <1/10); uncommon (>1/1000, <1/100); rare (>1/10000, <1/1000); very rare (<1/10000),

not known (cannot be estimated from the available data).

- The reported adverse events are:

Infection and infestations:

Uncommon: gastroenteritis

Immune system disorders:

Uncommon: hypersensitivity

Metabolism and nutrition disorders:

Rare: hyperglycaemia

Nervous system disorders:

Uncommon: dizziness, dysgeusia

Rare: headache

Vascular disorders:

Very rare: hypotension

Respiratory thoracic and mediastinal disorders:

Final version 1109/1185 Very rare: nasal dryness

• Gastrointestinal disorders:

Common: dyspepsia, nausea

Uncommon: abdominal pain, gastrointestinal disorders, gastritis, abdominal pain upper

Rare: gastrointestinal pain

Very rare: lower gastrointestinal haemorrhage

• Hepatobiliary disorders:

Rare: hepatic disorders

• Skin and subcutaneous tissue disorders:

Rare: acne, rash pruritic

Very rare: urticaria

• General disorders and administration site conditions:

Rare: malaise sensation

• Investigations:

Very rare: white blood count increased, blood lactate dehydrogenase increased

Moderate elevation of transaminases has been reported in patients with hypertriglyceridaemia.

Panthenol is a well-known substance with a long-term experience in medical, nutraceutic and cosmetic uses. According to the summary product characteristics of a product such as Bépanthene<sup>®</sup> (tablet indicated in alopecia) which contains panthenol (100 mg), adverse event observed are rare cases of urticaria and erythema [10]. Panthenol is metabolised in panthotenic acid, i.e. B5 vitamin.

Concerning toxicological studies performed results can support the administration of F373280 in the proposed clinical phase II study without particular alert [1].

Any safety warning was reported during a phase I study performed with F373280 administered to 84 healthy volunteers in single dose in a range between 500 mg and 16 g or in repeated dose during 28 days in a range between 1 g and 4 g. Adverse events reported and related to study treatment were minor to moderate. The adverse events were palpitations, orthostatic hypotension, dizziness, meteorism and liquid stool. Most were reported in both groups (placebo and F373280) without a dose relationship. The assessment of coagulation parameters and platelet function after

Final version 1110/1185

administration of repeated dose of F373280 did not report any bleeding concern: the reported changes in coagulation parameters and platelet function were within physiological ranges.

Moreover, DHA has been associated with anticoagulant products in AF studies [2, 8]. The range of PUFAs doses tested was between 2 g to 3 g (640 mg to 960 mg of DHA) and the range of study durations between 6 to 12 months. This association did not report a significant side effect of bleeding.

DHA has already been used in HF patients in several studies without safety concern [3, 4, 5]. The range of PUFAs doses tested was between 1 g to 5 g (1 g of the tested PUFAs contains about 320 mg of DHA acid) and the range of study durations was between 3 months to 3.9 years.

Thus, inclusion of patients with no specific antiarrhythmic treatment is acceptable. They will receive an anticoagulant treatment to prevent the thrombo-embolic complications of AF (particularly stroke) and the adequate treatments to control the heart rate and heart failure.

In conclusion, the overall available data allow in safe conditions the treatment of patients with persistent AF and chronic heart failure with F373280 in safe conditions.

# 2. STUDY OBJECTIVES

# 2.1. PRIMARY OBJECTIVE

The primary objective of the study is to assess the efficacy of F373280 on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

# 2.2. SECONDARY OBJECTIVES

The secondary objectives of the study are to assess:

- the efficacy of F373280 on the efficiency of direct ECV
- the effect of F373280 on echocardiographic parameters
- the safety and tolerability of F373280

Final version 1111/1185

# 3. ETHICAL CONSIDERATIONS RELATING TO THE STUDY

The trial is conducted according to Good Clinical Practices (CPMP/ICH/135/95), the National regulations and the Declaration of Helsinki and its subsequent amendments (see Appendix 17.1). This protocol and the informed consent form will be submitted for approval to independent local or national Institutional Review Boards/Ethics Committees before the study set up, according to national regulation.

All the protocol amendments or critical events liable to increase the risks incurred by the patients or to compromise the validity of the study or patients' rights will be submitted to the coordinator and to the Ethics Committees.

After being informed orally and in writing of all potential risks and constraints of the trial, as well as their freedom to withdraw their participation at any time, patients will then sign a consent form. A time of reflection will be given to the patients, before giving a written consent and starting the study procedures.

The use of a placebo is in accordance with EMA Addendum to the guideline on antiarrhythmics on AF and atrial flutter (EMA/CHMP/EWP/213056/2010) [21] and is acceptable because the included patients will remain under the standard treatment of AF and chronic heart failure. Except antiarrythmics, they will receive anticoagulant (vitamin K antagonist, VKA), rate control treatment, chronic heart failure treatment. During the study, in case of AF recurrence or atrial flutter emergence that would require cardioversion or the introduction of an anti-arrhythmic because of intolerable and/or uncomfortable clinical symptoms for instance, patients will be withdrawn and the tested product stopped. These patients will be considered as treatment failure.

In this study, patients will be carefully screened, particularly for their cardiac condition, with ECG, 24-hour holter monitor and echocardiographic data, and their biologic and coagulation condition.

The study will be addressed only to patients requiring an ECV due to their persistent AF, in the following conditions:

- ECV in patients not presenting a contra-indication
- Anticoagulation with vitamin K antagonist (VKA) for at least 3 weeks before ECV
- ECV will be performed in patients with AF and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values  $\geq 2$  on the 3 last

Final version 1112/1185

tests performed before ECV are required. However, if only 2 INR values are  $\geq 2$  among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Patients who do not revert to sinus rhythm or present an early AF relapse or an early atrial flutter emergence within the observation period after ECV will be withdrawn and the tested product stopped.

During the whole study, patients will remain under medical control: visits in cardiology units will be performed throughout the study period. This follow up will include clinical signs, ECG, biological and coagulation parameters. Moreover, patient's cardiac rhythm will be monitored once a week between visits using Trans Telephonic ECG Monitoring (TTEM) reviewed by a Central Reading Laboratory.

Patients may withdraw from the study at any time without having to give a reason and can expect to receive regular conventional therapy.

#### 4. STUDY DESIGN

#### 4.1. OVERALL DESCRIPTION

This phase IIa trial will be conducted as an international, multicentric, 24 weeks, double-blind, placebo-controlled, randomised, parallel group design, trial in 135 patients suffering from persistent AF and chronic heart failure.

After a 1 to 4-week of run-in period without study treatment, patients will be randomised into one of the following treatment groups: F373280 1g or placebo for 24 weeks.

Seven visits are planned for the study:

- Visit 1 (V1): W-4 to W-1: Selection visit (7 to 28 days before the Inclusion Visit)
- Visit 2 (V2): D1: Inclusion visit (start of study treatment)
- Visit 3 (V3): W4 (D28-2/+7D): cardioversion visit (outpatient or hospitalization according to clinical practice of the centre) (installation of the Holter ECG device)

Final version 1113/1185

- Visit 4 (V4): W5 (D35 -2/+7D): follow-up visit (removing of Holter ECG device and installation of the TTEM)
- Visit 6\* (V6): W12 (D84 ± 7D): follow-up visit
   \*see amendment PA05 dated 22OCT2014
- Visit 7 (V7): W16 (D112  $\pm$  7D) : follow-up visit
- Visit 9\* (V9): W24 (D168 ± 7D): final study visit
   \*see amendment PA05 dated 22OCT2014

# 4.2. DISCUSSION OF THE STUDY DESIGN

# 4.2.1. Choice of the Study Population

The target indication of F373280 will be the maintenance of sinus rhythm after cardioversion of patients with persistent AF and chronic heart failure. In the present proof of concept study, the evaluation will focus on patients within this indication. This target population is justified by:

- The proved efficacy of PUFAs in patients with persistent AF with or without heart failure in co-administration with amiodarone (add on therapy) [2]
- The proved efficacy of PUFAs on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5]

The study aim is to investigate the product effect in patients with:

- Previous history of persistent AF with duration of the current episode from 7 days to 6 months.
- A systolic heart failure defined by a reduced left ventricular ejection fraction (≥ 30% and ≤ 45%) or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size (diameter ≥ 60 mm and/or > 32 mm/m² and/or volume > 97 ml/m²),
  - and/or an increased left ventricular end-systolic size (diameter > 45 mm and/or > 25 mm/m² and/or volume > 43 ml/m²),
  - and/or a reduced left ventricular outflow tract velocity time integral < 15 cm [23, 24].</li>

Final version 1114/1185

According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would be effective to prevent recurrence of AF after cardioversion in patients with moderately abnormal LVEF.

- A Left Atrial Area (LAA) not severely abnormal (no greater than 40 cm<sup>2</sup> as defined in the report from the American Society of Echocardiography's Guideline) [23]. According to a sub-group analysis performed in patients with persistent AF associated to heart failure (Nodari S. personal data), PUFAs would not be effective to prevent recurrence of AF after cardioversion of patients with severely abnormal LAA.

For the successful rate of ECV, patients should have a stable medical treatment of heart failure and should not have any myocardial infarction or unstable angina or unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection.

# 4.2.2. Choice of the Study Design

As the target indication would be the prevention of AF recurrence after ECV, the study design meets the requirements of EMA guideline on antiarrhythmics in AF (EMA/CHMP/EWP/213056/2010) [21].

As F373280 aims to be a safe treatment for the prevention of AF recurrence, it will not be tested as an add-on therapy during the study. To avoid any interaction with the tested product, antiarrhythmics class I and III will be forbidden during the study.

The study design is defined in order to avoid methodological bias. A double blind study is appropriate to assess the efficacy and safety of the use of F373280 to prevent recurrence of AF episodes. Moreover, this study design is similar to the design of almost all trials that have assessed intervention for rhythm control [2, 8, 11, 12].

According to the target indication, only patients with persistent AF and requiring an ECV will be included in order to assess the time to first documented recurrence of AF (or emergence of atrial flutter) since cardioversion.

To confirm the persistent nature of AF, a 24-hour holter monitoring will be performed during the selection visit.

Final version 1115/1185

Eligible participants will enter a selection phase in which anticoagulant treatment (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) of 2 to 3 before ECV. According to guidelines for the management of AF [6], VKA should be given at least 3 weeks before cardioversion because of risk of thrombo-embolism due to post-cardioversion.

Experimental data suggest that the maximal incorporation of n-3 PUFAs in the myocardial cell membrane takes up to 28 days to occur [22]. In addition, as shown in Nodari's study [2], the duration of pre-treatment with PUFAs before cardioversion appears to be a contributing factor in success. Therefore, before starting follow up for the assessment of AF recurrence, treatment with F373280 should be started 28 days before ECV.

Detection of AF recurrence will be performed using systematic (scheduled) ECG recording, thus allowing detection of asymptomatic (about 50% of episodes) as well as symptomatic AF episodes. According to previous studies, most of AF recurrences occurred during the first days after cardioversion [11, 15]. So that, the heart rhythm will be closely monitored during the first week after successful cardioversion using an ambulatory continuous 7-day holter ECG recording in order to increase sensibility to detect asymptomatic AF episodes. Thereafter, to improve patient compliance, this follow up will be continued using an easier device to carry and to use, i.e. a TTEM.

Finally, during the study, patients will be scheduled for a clinical visit every 4 weeks or 8 weeks (with an additional visit 7 days after visit 3 (ECV visit)) in order to ensure a close medical monitoring and to assess efficacy and safety parameters.

# 4.2.3. Choice of the Dose

According to a previous study in patients with AF [2], the tested PUFA product (Omacor®) at the dose of 2 g (i.e. 640 mg of DHA acid) was effective in the prevention of AF after cardioversion. Moreover, PUFAs at dosage of 1 g and 2 g were also effective on the improvement of ventricular functional parameters, morbi-mortality and duration of hospitalisation in patients with heart failure [3, 4, 5].

From the F373280 phase I study, after a 14-day repeated administration of F373280 (1 g/day), observed plasma concentrations of DHA measured before treatment (Cmin) were similar to that of an effective dose of Omacor® at 2 g/day (60 to 95 mg/ml and 60 to 90 mg/ml, respectively) (phase I study of F373280 and [16]). With regard to the rhythm of administration, mean peak/trough

Final version 1116/1185
fluctuation (baseline corrected) was around 0.3. This value supports a once-daily administration allowing a 24-hour plasma exposure in DHA. Therefore, a 1 g daily dose of F373280 is considered to be appropriate for this proof of concept study.

## 4.2.4. Choice of the Sample Size

See chapter 13.

## 5. STUDY POPULATION

Each patient fulfilling all the inclusion criteria and none of the non inclusion criteria will be eligible.

#### 5.1. INCLUSION CRITERIA

#### Demographic Characteristics and Other Baseline Characteristics:

- 1. Men or women aged more than 18 years (inclusive)
- 2. Patient with current episode of persistent AF between 7 days and 6 months duration for whom electrical cardioversion is warranted
- 3. Previous history of first documented episode of persistent AF
- 4. Previous history of ischemic or non ischemic heart failure
- 5. NYHA class I or II chronic heart failure at selection and at inclusion
- 6. Left ventricular systolic dysfunction defined at selection and at inclusion by a reduced left ventricular ejection fraction (LVEF)  $\geq$  30% and  $\leq$  45% or for patients with a LVEF > 45%:
  - an increased left ventricular end-diastolic size

 $(diameter \ge 60 \text{ mm and/or} > 32 \text{ mm/m}^2 \text{ and/or volume} > 97 \text{ ml/m}^2)$ 

• and/or an increased left ventricular end-systolic size

(diameter  $> 45 \text{ mm and/or} > 25 \text{ mm/m}^2 \text{ and/or volume} > 43 \text{ ml/m}^2$ )

- and/or a reduced left ventricular outflow tract velocity time integral < 15 cm
- On appropriate, stable medical treatments for heart failure, including a diuretic and/or angiotensin-converting enzyme, and/or angiotensin-receptor blocker and/or mineralocorticoid receptor (MR) antagonists, and/or betablockers

Final version 1117/1185

- 8. Left atrial area  $\leq 40 \text{ cm}^2$  at selection and at inclusion
- 9. Patient treated or having to be treated by vitamin K antagonist
- 10. For female patient of child-bearing potential:

## • In all the countries except Italy:

- Use of an effective method of contraception (hormonal contraception or intra-uterine device) assessed by the investigator for at least 2 months before the selection in the study and agreement to go on using it during the whole duration of the study and up to 1 month after the last dose of the study treatment or
- Documented as surgically sterilized

## • In Italy only:

- Absolute abstention from sexual intercourse during the whole duration of the study and for a month after the end of the study or
- Use of double barrier contraception method (use of effective medical contraception method) from at least 2 months before the start of the study to the entire duration of the study and for a month after the end of the study or
- Documented as surgically sterilized
- 11. For female patient of child-bearing potential: negative urine pregnancy test at inclusion
- 12. For male with a child-bearing potential partner (In Italy only):
  - Absolute abstention from sexual intercourse during the whole duration of the study and for 3 months after the end of the study or
  - Use of double barrier contraception method (use of condom for male and effective contraception method for the partner) from the entire duration of the study to 3 months after the end of the study.

## Ethical /legal considerations:

13. Having signed his/her written informed consent,

Final version 1118/1185

14. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

#### 5.2. NON INCLUSION CRITERIA

## Criteria related to pathologies:

- 1. No previous history of first documented episode of persistent Atrial Fibrillation
- 2. More than two successful cardioversions (electrical or pharmacological) in the last 6 months,
- 3. Secondary Atrial Fibrillation due to alcohol or severe valvular heart disease (grade III to IV),
- 4. NYHA class III or IV heart failure at selection or at inclusion
- 5. Thyroid disease uncontrolled by treatment: TSH  $\pm$  T4L  $\pm$  T3L to be checked in case of treatment for thyroid disease
- 6. Myocardial infarction or unstable angina or presence of unstable ischemic coronaropathy assessed by coronarography or cardiac stress test (Echo stress, exercise stress test, nuclear or MR perfusion evaluation methods) within 6 months before selection
- 7. Severe chronic kidney disease (creatinine ≥ 25 mg/L or estimated glomerular filtration rate < 30 ml/min) at selection
- 8. Bradycardia (HR  $\leq$  50 bpm)
- 9. Hyperkalemia or hypokalemia (according to the standards of local laboratories) at selection
- 10. Cardiac surgery within 3 months before selection or planned during the study duration

#### Criteria related to treatments:

- 11. Previously ineffective pharmacological or electrical cardioversion
- 12. Concomitant treatment with ranolazine or any anti-arrhythmic drug (within 7 days prior to selection), except amiodarone, dronedarone and stable dose of digoxin, beta-blockers, calcium-blockers.
- 13. Concomitant treatment with oral amiodarone or dronedarone from selection
- 14. Concomitant treatment with intravenous amiodarone from selection
- 15. Patient requiring a cardiac resynchronization therapy (CRT) or having undergone CRT implantation within the last 6 months

Final version 1119/1185

- 16. Treatment with any Polyunsaturated Fatty Acid within the last 3 months
- 17. Dietary supplement with  $\omega 3$  or  $\omega 6$  according to investigator's judgment
- 18. Having undergone any form of ablation therapy for AF
- 19. Patient treated with oral anticoagulant treatment other than vitamin K antagonist: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or treated with irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel

#### Others criteria:

- 20. Patient liable not to comply with protocol instructions and/or with treatment, in the investigator's opinion,
- 21. Patient having taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of selection,
- 22. Patient linguistically or mentally unable to understand the nature, objectives and possible consequences of the trial, or refusing to patient himself / herself to its constraints,
- 23. Patient family member or work associate (secretary, nurse, technician...) of the Investigator,
- 24. Patient having forfeited his / her freedom by administrative or legal award or being under guardianship,
- 25. Breastfeeding female patient.

#### **5.3. NUMBER OF PATIENTS**

Maximum 135 patients (taking into account 15% of non-evaluable patients).

## 5.4. RECRUITMENT MODALITIES

Patients will be recruited within the medical consultation of each centre involved in the study. If necessary and when authorized by local and national regulation, some specific supports or tools will be used to improve the recruitment (announcement, mailing to general practitioners, leaflet, website including ClinicalTrials.gov, CRO...).

Before implementation, the documents will be submitted to and approved by the Ethics Committee.

Final version 1120/1185

## 5.5. PATIENT IDENTIFICATION

Patient's code will contain 7 digits: the 2 first digits corresponding to the country number, the following 2 digits corresponding to the centre number and the last 3 digits corresponding to the patient's chronological order once having signed the written informed consent.

## 5.6. WITHDRAWAL CRITERIA

Reasons for a patient's premature withdrawal from the study may be the following:

- Patient's decision. A patient who wishes to withdraw from the study for any reason may
  do so at any time but must inform the investigator. In all cases, the Investigator should
  attempt to contact the patient as soon as possible for a final assessment in order to:
  - have the patient's decision written on the consent form
  - obtain the reason(s) for withdrawal and report it/them in the case report form
  - evaluate the patient's clinical condition
  - if necessary, take appropriate therapeutic measures: management of an adverse effect or concomitant disease, prescription of another treatment.
- Investigator's decision in the patient's interest, particularly if a serious adverse event occurs and is considered by the Investigator liable to threaten the health of the patient. The monitor will be informed by phone or fax and a letter or report explaining the withdrawal will be forwarded to the monitor as soon as possible.
- Erroneous inclusion according to the study protocol. The decision to maintain or not the patient in the study will be taken jointly by the investigator and the sponsor. Erroneous inclusions will not be paid to the investigator.
- Patients who could not be treated with VKA for at least 3 weeks before ECV or who will
  experience a VKA intolerance during the study.
- Patients without dyskalemia who will not have INR values ≥ 2 on the 3 last tests performed before ECV should not have an ECV and will be excluded from the study. However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO-TE (transesophageal

Final version 1121/1185

echocardiography) performed on the same day (before ECV) and the patient can continue the study.

- Patients who will not revert to sinus rhythm (i.e. unsuccessful ECV) or with early AF
  relapse or early atrial flutter emergence within the observation period after ECV will be
  considered to have finished follow-up.
- Occurrence of AF recurrence or atrial flutter emergence that would require, at the
  investigator's judgement, a cardioversion or an introduction of an anti-arrhythmic because
  of intolerable and/or uncomfortable clinical symptoms for instance.

## 5.7. REPLACEMENT OF PATIENTS

Withdrawn patients will not be replaced.

## 5.8. POST-STUDY EXCLUSION PERIOD

Patients will not be allowed to participate in another clinical trial during 3 months following the study termination.

## 5.9. STUDY CARD AND LETTER FOR GENERAL PRACTITIONER(S)

The patient will receive from the Investigating Centre at Visit 1 - Selection Visit:

- a personal card to be kept all along the study duration and providing the following information: patient's name, sponsor's name, study code, EUDRACT number, start date and expected end date of the study, complete address of the Investigating Centre with the name and phone number of the Investigator and a sponsor 24H/24 phone contact number in case of emergency (French and English languages): 33 (0)5 63 35 25 83. For Italy, this card will be in Italian only, without any English mention.
- in Italy, a letter to be given to his/her general practitioner. This letter intends to inform the general practitioner(s) (and any other doctors who take care of the patient) that the patient participates to the clinical study. It describes the study treatment and includes some information on the forbidden treatment during the study.

Final version 1122/1185

## 6. STUDY TREATMENT

The Clinical Pharmacy Department of the Institut de Recherche Pierre Fabre (IRPF) will supply the investigational centres with the treatment necessary for the conduct of the trial.


F373280 and placebo will be prepared in Soft Capsules similar presentation.

#### • F373280

Formulation of F373280, 1 g, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: Panthenyl ester of DHA, gelatine, glycerol, titanium, dioxide, purified water.

#### Placebo

Formulation of placebo matching tested product, Soft Capsules: oral administration, oblong size 20, off-white, Soft Capsules containing: paraffin liquid, fish flavour, gelatine, glycerol, titanium, dioxide, purified water.

Placebo and F373280 capsules will be packaged in opaque blisters.

## 6.2. PACKAGING AND LABELLING

The treatment units will be packed and labelled by the Clinical Pharmacy Department of the IRPF according to European Directive and local requirements.

## 6.2.1. Packaging

Each treatment unit will be composed of 3 cases for a 12-week treatment period.

Two 12-week treatment units will contain 3 cases, each case of 4-week treatment containing: 10 blister packs of four 1 g F373280 soft capsules or 1 g placebo soft capsules each.

## 6.2.2. Labelling

Investigational Products will be labelled according to the following rules:

Labelling should comply with the local requirements for Investigational Medicinal Products.

Final version 1123/1185

On the treatment units and cases, the labels will bear the following indications:

- a) name and address of the sponsor
- b) protocol number
- c) packaging batch number
- d) treatment number
- e) storage conditions
- f) expiry date
- g) pharmaceutical dose form
- h) route of administration
- i) quantity of dosage units
- j) direction for use
- k) legal statements:
- -"for clinical trial only", "keep out of the reach and the sight of children", "please return to your doctor any unused product", respect the prescribed dose"

On the treatment unit, another label will be affixed with the mention of the Investigator's name and patient's code (completed by the Investigator).

In addition, on each case will be mentioned the case number and a detachable label will bear the following indications:

- Protocol number
- Packaging batch number
- Expiry date
- Case number
- Treatment number

On the blister pack, the label will mention the protocol number, the packaging batch number, the case number and the treatment number.

## 6.3. DISTRIBUTION TO CENTRE AND STORAGE

The Clinical Pharmacy Department of the IRPF will supply the Investigational Centre with the treatment units along the study according to the need, upon request triggered by the patient's selection

Final version 1124/1185

As soon as the Pharmacist or the Investigator receives the trial medication, he/she will check the contents and immediately acknowledges the receipt in the IVRS/IWRS. The copy of the acknowledgement will be kept in the Investigator's or the Pharmacist's file. The same procedure will be applied to all further supplies during the course of the trial.

At the time of the delivery to the Centre, the following information will be provided:

- Details of storage conditions that should be respected
- And, upon request and for the 1<sup>st</sup> delivery only, a letter of release for the Investigational Medicinal Product from the Sponsor's Qualified Person

The CRA will ensure during the monitoring visits that trial medications have been received in good conditions and the acknowledgment of receipt has been performed adequately.

Treatment units should remain intact until dispensation to the patients. They should be kept at temperature below 30°C in an appropriate lockable room only accessible to the person authorised to dispense them, under the responsibility of the Pharmacist or the Investigator.

In the case of undue delay in study execution, the Pharmacist or the Investigator should ensure that the expiry date has not been exceeded.

## 6.4. ALLOCATION OF TREATMENTS AND DISPENSATION TO PATIENT

A randomisation list will be established by the Clinical Pharmacy Department of the IRPF. This list will be computer-generated with internal software. The randomisation methodology is validated by the Biometry Department before generation.

Treatments F373280 or placebo will be balanced in a 1:1 ratio.

As the treatment units are prepared for 12-week treatment periods, the Investigator will have to allocate a treatment number at inclusion visit (V2) and another one at visit 6.

For each patient, the treatment number given at visit 6 will not be the same that the one given at inclusion visit (V2).

The treatment numbers will be given through the IVRS/IWRS.

At selection visit (V1), practically, once patient's eligibility is confirmed:

- The Investigator:
- Contacts the IVRS/IWRS

Final version 1125/1185

- Answers the questions related to the patient
- The IVRS/IWRS company:
- Confirms this information by fax/email to the Investigator
- Fills the "Request for Delivery of Investigational Product" form and sends it by email and/or fax to the Clinical Pharmacy Department of the *IRPF*.
- The Clinical Pharmacy Department of the *IRPF* sends the corresponding treatment unit to the Investigator within 5 days from reception of the email request form.

At inclusion visit (V2), the treatment number to be allocated for the first 12-week period to the patient is given by the IVRS/IWRS.

At visit 6, the Investigator will contact again the IVRS/IWRS to obtain the treatment number for the last 12-week period of treatment.

The Investigator will dispense to the patient the 4-week treatment cases (one or two according to the visit) which label indicates the treatment number and the administration period.

## 6.5. DRUG ADMINISTRATION

#### **6.5.1.** Duration of Treatment

For a patient completing the study, the theoretical study treatment exposure to F373280 or placebo will be 24 weeks.

If the ECV is postponed by 1 week to allow INR stabilization, the treatment duration will be 25 weeks.

## 6.5.2. Dose Schedule

One soft capsule of 1g of F373280 or placebo to be taken each day during 24 weeks.

## 6.5.3. Route and Conditions of Administration

The soft capsules are to be taken orally. One soft capsule is to be taken each evening with the dinner during 24 weeks.

Final version 1126/1185


The Investigator should maintain accurate written records of drug received, dispensed, returned and any remaining treatment units, on the drug accountability form. These records should be made available for Clinical Research Associate (CRA) monitoring. The packaging of the medication should remain intact until just before the dispensation.

At each visit, the Investigator will record the number of soft capsules returned by each patient using the appropriate page of the e-CRF.

At the end of the study, all used and unused treatments including packaging should be noted, and return is organised by the CRA to the Clinical Pharmacy Department of the IRPF for destruction. A copy of the drug accountability form should be provided by the Investigator to the CRA.

#### 6.7. RECALL OF INVESTIGATIONAL PRODUCTS

In case of recall of investigational products (decided by the Competent Authorities or the Sponsor), the Investigator will immediately be informed by the Sponsor.

The Investigator in collaboration with the Sponsor's representatives (Study Manager, CRA) must urgently:

- Stop the delivery of the concerned investigational products to the patients.
- Inform the concerned patients that they must immediately stop taking these investigational products and bring them back.

The Study Manager/CRA organises the return of the recalled products to the Clinical Pharmacy Department of the IRPF according to the Sponsor's procedures.

## 7. CONCOMITANT TREATMENTS

Any existing concomitant treatment (at selection visit), any new concomitant treatment or change in the dosage of an existing concomitant treatment during the course of the study must be noted on the electronic Case Report Forms (e-CRF). All treatments should be evaluated by the Investigator at patient's selection, and treatment prolongation or stop during the study should be considered.

Final version 1127/1185

For all concomitant treatments taken during the study, the following information must be noted in the relevant section(s) of the e-CRF:

- The name of the treatment and its form
- The reason for prescription
- The route of administration
- The daily dose
- The duration of treatment.

#### 7.1. VITAMIN K ANTAGONIST TREATMENT

VKA should be given for at least 3 weeks before ECV and continued for the whole study duration. However, VKA should be stopped in case of occurrence of VKA intolerance during the study and the patient should be withdrawn from the study. The VKA used will be left to the decision of each Investigator according to his/her local practice.

#### 7.2. PROHIBITED TREATMENTS

- Class I and class III antiarrhythmic treatments:
  - Class I:
    - o Class IA: Disopyramide, Procainamide, Quinidine
    - o Class IB: Lidocaine, Mexiletine
    - o Class IC: Flecainide, Propafenone
  - Class III: Dofetilide, Ibutilide, Sotalol, Amiodarone, Dronedarone.
- Ranolazine
- Any PUFA
- Any oral anticoagulant treatment other than VKA: new oral anticoagulants (dabigatran, rivaroxaban, apixaban), or irreversible antiplatelet agents P2Y12 inhibitors such as ticlopidine, clopidogrel or prasugrel
- Dietary supplement with Omega 3 or Omega 6

Final version 1128/1185

Prohibited treatments at selection must not be prescribed for the duration of the study except in case of occurrence of an adverse event or AF episode that requires a corrective treatment in the interest of the patient's health.

## 7.3. AUTHORISED TREATMENTS

Other treatments will be authorised during the study duration.

However, if medication other than study drugs is administered at any time from the start of the study, details must be recorded in the e-CRF. During the study, patients must be asked whether they have been on a course of prescribed drug treatment or have taken any OTC or herbal drugs since the visit.

## 8. EVALUATION CRITERIA

## 8.1. PRIMARY EFFICACY CRITERION

## 8.1.1. Time to the first Atrial Fibrillation Recurrence or Atrial Flutter Emergence

## 8.1.1.1. Definition

Time to first AF recurrence or atrial flutter emergence is defined by the time to first episode of AF or atrial flutter (symptomatic or not) lasting for at least 10 minutes.

#### 8.1.1.2. Schedule

The heart rhythm follow up will be performed from the end of ECV visit (visit 3) to the final study visit (visit 9).

For randomised patients with spontaneous cardioversion before ECV, the recurrence of AF or the emergence of atrial flutter will be assessed after visit 3 (from week 5).

## 8.1.1.3. Evaluation Methods

• 7-day holter monitor:

Final version 1129/1185

The heart rhythm monitoring will be carried out from visit 3 to visit 4 using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) fixed after ECV visit.

Following holter monitoring, the heart rhythm will be documented using Trans Telephonic ECG Monitoring (TTEM).

## • Trans Telephonic ECG Monitoring:

The ECG follow up will be documented using the TTEM: one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). The patient will be requested to contact the Central Reading Laboratory for transmission of each stored TTEM.

Moreover, if patient experiences AF or atrial flutter symptoms during this TTEM period, it should be documented using the TTEM.

In case of AF recurrence or atrial flutter emergence and provided that the patient does not require a cardioversion or an introduction of an anti-arrhythmic at Investigator's judgement, the patient could be maintained in the study with the treatment in order to assess a spontaneous cardioversion. For that purpose the patient will continue to transmit a TTEM once a week.

## • Process of centralisation of ECG (Holter and TTEM)

ECG (Holter and TTEM) will be centralized by the Central Reading Laboratory. The ECG will be validated by a trained technician, then analysed by a cardiologist. The cardiologist interpretation will be emailed to the site (or per fax on request of the site). The investigator will be asked to review and sign these documents.

The Holter and TTEM process will be fully described in separate documents.

## 8.2. SECONDARY EFFICACY CRITERIA

## 8.2.1. Numbers of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.1.1. Definition

Number of AF episodes will consist in the assessment of AF episodes with duration at least 10 minutes ( $N_{Sup10}$ ) and of less than 10 minutes ( $N_{Inf10}$ ), respectively.

Final version 1130/1185

#### 8.2.1.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the study visit 4.

#### 8.2.1.3. Evaluation Methods

• 7-day holter monitor:

The heart rhythm monitoring will start using a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) after ECV visit from visit 3 to visit 4.

## 8.2.2. Duration of AF episodes in the first week following visit 3 (ECV visit)

## 8.2.2.1. Definition

Duration of AF episodes will consist in the sum of duration of each AF episode.

## 8.2.2.2. Schedule

The heart rhythm follow up will be performed from the end of successful ECV visit (visit 3) to the follow up study visit (visit 4).

## 8.2.2.3. Evaluation Methods

Duration of AF episodes will be assessed using the 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording.

## 8.2.3. Clinical parameters evaluation

#### 8.2.3.1. EHRA score assessment

## 8.2.3.1.1. *Definition*

AF related symptoms will be evaluated by the EHRA (European Heart Rhythm Association) score [20]. The following items "during presumed arrhythmia episodes" are checked to determine the score: palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety.

Classification of AF-related symptoms (EHRA score) are as follows:

Final version 1131/1185

- EHRA I 'No symptoms'
- EHRA II 'Mild symptoms'; normal daily activity not affected
- EHRA III 'Severe symptoms'; normal daily activity affected
- EHRA IV 'Disabling symptoms'; normal daily activity discontinued

This classification relates exclusively to the patient-reported symptoms.

In addition to this score, the frequency will be classified in three groups, namely occasionally (less than once per month), intermediate (1/month to almost daily) and frequent at least daily.

#### 8.2.3.1.2. Schedule

EHRA evaluation will be performed in case of evocative symptoms of arrhythmia.

## 8.2.3.1.3. Evaluation Methods

EHRA evaluation will be collected by Central Reading Laboratory during TTEM period.

## 8.2.3.2. Time to first AF recurrence less than 10 minutes

Time to first AF recurrence less than 10 minutes will be assessed during TTEM period.

## 8.2.3.3. Recurrence of symptomatic AF

Recurrence of symptomatic AF will be assessed during TTEM period.

The number of recurrences of symptomatic AF consists of the number of AF recurrences associated with a symptom (palpitation, fatigue, dizziness, dyspnea, chest pain and anxiety) and confirmed by an ECG.

The time to first symptomatic AF recurrence is defined by the time to first episode of symptomatic AF.

## 8.2.3.4. Number and duration of hospitalizations

- Number and duration of hospitalizations for cardiovascular events
- Hospitalization for AF treatment

Final version 1132/1185

- Hospitalization for worsening of heart failure
- Hospitalization for myocardial infarction
- All cause of hospitalization
- Number and duration of hospitalizations for thromboembolic stroke

## 8.2.4. Cardioversion assessment

- Assessment of spontaneous cardioversion before visit 3
- Assessment of successful cardioversion at visit 3 (i.e. return to sinus rhythm)
- Shocks distribution (1, 2 or 3 shocks)
- Number of patients needing another cardioversion after initial ECV

## 8.2.5. Evolution of echocardiographic parameters

## 8.2.5.1. **Definition**

The following echocardiographic parameters will be assessed: Left atrial diameter (mm), LAA (cm²), Left atrial volume (ml), Left atrial volume/BSA (ml/m²), LVEF (%), Left ventricular end diastolic volume/BSA (ml/m²), Left ventricular end systolic volume/BSA (ml/m²), Left ventricular end diastolic volume (ml), Left ventricular end systolic volume (ml), Left ventricular end systolic diameter (mm) and Left ventricular end systolic volume (ml).

## 8.2.5.2. Schedule

Measurements will be performed at visit 1 and visit 2 to check the eligibility of the patient.

Measurements performed at visit 4, visit 6 and visit 9 are done to follow the echocardiographic evolution of the patients in sinus rhythm.

#### 8.2.5.3. Evaluation method

The echography evaluations will be carried out according to the recommendations for chamber quantification drawn up by the American Society of Echocardiography and the European

Final version 1133/1185

Association of Echocardiography [23]. So, the recommended method for volume measurements is to use the biplane method of discs (modified Simpson's rule) from 2-D measurement.

## 8.3. BIOMARKER ASSESSMENT: RED BLOOD CELL CONCENTRATIONS OF DHA

#### 8.3.1. Definition

Because of the limited human tissue accessibility for biopsy, red blood cell DHA contents is a marker of tissue DHA concentration [13], [14].

## 8.3.2. Blood samples

#### 8.3.2.1. Collection schedule

Blood samples will be collected to determine the red blood cells (RBC) concentrations of DHA.

Blood samples will be performed at visit 2 before treatment, visit 3, visit 6 and visit 9.

Actual sampling times will be individually reported in the e-CRFs.

## 8.3.2.2. Technical handling

Two blood samples (2 x 4 ml) will be collected in EDTA tubes. They will be homogenized slowly by inverting the tube without shaking, stored between  $+2^{\circ}\text{C}/+8^{\circ}\text{C}$  in a fridge (no freezing will be allowed) and sent to Analytical Centre in refrigerated conditions (between  $+2^{\circ}\text{C}$  and  $+8^{\circ}\text{C}$ ). Analysis will be performed within 2 weeks following reception at the Analytical Centre.

#### 8.3.3. DHA concentration measurement

Analytical determination of RBC concentrations of DHA will be carried out by the Analytical Centre.

Lipids will be extracted from red blood cells samples with a mixture of hexane/isopropanol after acidification [17]. Total lipid extracts will be saponified and methylated. The fatty acid methyl esters (FAME) will be extracted and analyzed by Gas Chromatography.

Identification of FAME will be based on retention times obtained for FAME prepared from fatty acid standards. The area under peaks will be determined using ChemStation Software (Agilent)

Final version 1134/1185

and results will be expressed as % of total fatty acids. DHA concentration will be calculated using the internal standard and expressed as  $\mu g/g$  for red blood cells samples. Thus, omega-3 index will be assessed. The omega-3 index represents the content of EPA plus DHA in red blood cells (expressed as a percent of total fatty acids). It is a biomarker considered as a new marker of risk for death from coronary disease [18].

Results of this analytical determination will be kept confidential by the dosing centre until the end of the study, and will be provided only at the end of the study (after database lock) in a separate file.

## **8.4. SAFETY ASSESSMENT**

#### **8.4.1.** Adverse Events

At selection, any concomitant disease will be reported on the e-CRF. At each further visit, the occurrence of AEs since the last visit will be based on the patient's spontaneous reporting, the Investigator's non-leading questioning and his/her clinical evaluation. All AEs will be reported on the e-CRF (see section 10).

## **8.4.2.** Laboratory Investigations

#### 8.4.2.1. Schedule

Laboratory investigations will be performed at visit 1 (before treatment) and visit 9 (end of treatment) or End of Treatment visit.

At visit 3 and 6, only a standard haematologic dosage will be performed.

Furthermore the kalemia will be checked before electrical cardioversion at visit 3.

The total volume of blood samples taken for haematology and biochemistry analysis should not exceed 30 ml.

#### 8.4.2.2. Technical Procedures and Parameters

The following tests will be performed:

Final version 1135/1185

<u>Haematology</u>: haematocrit, haemoglobin, RBC count, white blood cells (WBC) count, WBC

differential counts (% and/or absolute), reticulocytes, platelets.

<u>Biochemistry</u>: sodium, potassium, bicarbonate, chloride, alkaline phosphatase, gamma GT,

albumin, total bilirubin, conjugated bilirubin, creatinine, aspartate

aminotransferase (AST), alanine aminotransferase (ALT), fasting glucose,

total cholesterol, cholesterol (HDL, LDL), triglycerides, creatine

phosphokinase (CPK), fibrinogen.

Blood samples will be taken in the morning in fasting conditions.

The estimation of GFR at selection relies on the measurement of serum creatinine and the Cockcroft-Gault formula:

Cockcroft-Gault formula

- with serum creatinine expressed as mg/L:

in men:

GFR (ml/min) = [(140-age) x weight / (7.2 x serum creatinine in mg/L)]

in women:

GFR (ml/min) =  $[(140\text{-age}) \times \text{weight} / (7.2 \times \text{serum creatinine in mg/L})] \times 0.85$ 

- with serum creatinine expressed as µmol/l:

GFR (ml/min) = [(140-age) x weight / serum creatinine in  $\mu$ mol/l] x k,where k = 1.23 for men, 1.04 for women.

(weight in kg, age in years)

Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

## 8.4.3. Global Physical Examination

A global physical examination including the measurement of body weight will be carried out on each body system at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

Final version 1136/1185

The Body surface area (BSA) will be calculated at the same visits using Mostellers' formula:

 $BSA = [(Weight x Height)/3600]^{1/2}$ 

(Weight in kg, height in cm)

The physical examination will be globally evaluated as "normal/abnormal". Further target inspection will be undertaken for any abnormal finding.

## 8.4.4. Vital Signs

Vital signs will consist in blood pressure and heart rate at rest.

#### 8.4.4.1. Schedule

Vital signs will be measured at each visit.

## 8.4.4.2. Technical Procedure and Parameters

Systolic blood pressure (SBP) and diastolic blood pressure (DBP), expressed in mmHg, will be measured after at least 5 minutes in supine position and after 2 minutes in standing position.

The heart rate (HR), expressed in beats per minute (bpm), will be measured by auscultation by counting the beats for at least 30 seconds, after at least 5 minutes in supine position and after 2 minutes in standing position.

Bodyweight will be measured with patient in underwear and with the same balance at each visit.

## 8.4.5. Electrocardiogram (ECG)

#### 8.4.5.1. Schedule

An ECG will be recorded after at least 10 minutes of rest at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9 using a usual standardised 12-lead cardiograph.

## 8.4.5.2. Technical Procedure and Parameters

## • Electrocardiogram:

The global interpretation from manual reading (normality, clinical relevance) and HR (bpm), PR (ms), QRS (ms), QT (ms), QTcB (ms), QTcF (ms), repolarisation patterns will be reported in the

Final version 1137/1185

e-CRF. Each print-out will include the patient's code, date, time, technician's initials and investigator's signature.

In case of thermic paper ECG print out, a photocopy will be made by the centre to ensure safe filing.

24 hour-Holter - ECG

An ambulatory continuous 24-hour ECG (5-leads/2 or 3 channels) will be recorded at selection visit using a holter ECG, in order to confirm persistent AF.

## **8.4.6.** Coagulation parameters

Coagulation assessment will be evaluated by the following parameters:

- Prothrombin Time/INR (PT/INR)
- Activated Partial Thromboplastin Time (aPTT)
- Thrombin Clotting Time (TCT)

The recommendations for the controls of INR are the following [25, 26]:

- 1) During the pre-cardioversion period, if the anticoagulation by VKA has to be initiated, the treatment must be initiated at least 3 weeks prior to cardioversion then the INR will be monitored as follow:
  - The adjustment of the dosage of VKA should be performed stepwise by controlling INR 2
     to 3 times a week until stabilization within the target range (2 3) on 2 successive tests.
  - When the INR is within the target range (2 3) on 2 successive tests, the dose of VKA should be maintained. Then the controls of INR will be progressively spaced within a few weeks.
  - When INR is stabilized, at least one test should be performed each week.
  - In all cases, an INR control must be performed within 24 h before ECV.
- 2) During the pre-cardioversion period, if the anticoagulation by VKA was already initiated, the INR will be monitored as follow:
  - One INR per week up to ECV
  - An INR control must be performed within 24 h before ECV
- 3) After cardioversion : one INR every 4 weeks
- 4) Throughout the duration of the study if INR > 3 the advocated actions are:

Final version 1138/1185

- No transesophageal echocardiography before cardioversion
- For asymptomatic patients:
  - 3 < INR < 4: no omission of VKA (dose adjustment if required), no vitamin K
  - $4 \le INR < 6$ : omit one dose of VKA, no vitamin K
  - $6 \le INR < 10$ : interrupt VKA, vitamin K 2 mg orally
  - INR ≥ 10: interrupt VKA, vitamin K 5 mg orally
     For INR ≥ 6, an adverse event has to be reported (asymptomatic overdose).

Anti-coagulation by VKA should be given at least 3 weeks before ECV and continued for the whole study duration.

aPTT and TCT will be performed at visit 1, visit 2, visit 3, visit 6, visit 7, and visit 9.

The quantity of blood samples collected at each time for coagulation parameters will be 2 ml. Additional tests may be done at the Investigator's discretion, in the patient's interest. In case of any abnormal and/or clinically significant results, the Investigator should order laboratory control tests.

#### 8.5. CONCOMITANT TREATMENTS

Concomitant treatments will be evaluated at each study visit.

Requirements related to patient's concomitant treatments started before selection visit and continued throughout the trial, or started during the trial, can be found in section 7.

#### 8.6. COMPLIANCE

The patient will be reminded at each visit to bring back at the following visit any used or unused remaining soft capsule, blister and case.

At each visit (except at visit 4), the Investigator will record the number of supplied and remaining soft capsules in the e-CRF.

## 9. STUDY PROCEDURES

Visit 1 - Selection Visit (Week - 4 to Week -1):

Final version 1139/1185

The patient considered eligible for selection by the Investigator will be informed of the characteristics and the consequences of the trial both verbally and by reviewing the patient's information sheet and consent form (see section 14.3). If the patient accepts to participate in the study, he/she will sign the informed consent form and will keep a copy.

The patient will be assessed for the following:

- Demographic characteristics (gender, age, height, body surface area)
- Personal and medico-surgical history
- Habits (Tobacco, alcohol consumption, dietary habits including fish consumption...)
- Cardiovascular diseases, mainly detailed history of Heart Failure and AF characteristics
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Concomitant diseases, adverse signs or symptoms (able to be used for treatment emergent AE determination)
- Concomitant treatments (authorised, disallowed)
- Global physical examination/bodyweight
- Vital signs
- Biology: haematology, biochemistry, assessment of coagulation parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Biology assessment of renal function: creatinine or estimated glomerular filtration rate If the results of the above assessments are compatible with the selection criteria:
  - A 24-hour continuous ECG ambulatory recording (Holter ECG) device will be installed on the patient to monitor the patient heart rhythm. The patient will be requested to bring back the device after the termination of 24 hours recording. The recording will be transmitted from the Investigational site to the Central Reading Laboratory. The Central Reading Laboratory will send his/her assessment regarding the confirmation of persistent AF within 2 working days to the Investigator.

Final version 1140/1185

• The patient will enter the selection and pre-cardioversion periods in which anticoagulant (VKA) will be adjusted to achieve ideally an International Normalized Ratio (INR) in the range of 2 to 3 before ECV.

At the end of the visit, the Investigator will contact the IVRS/IWRS to confirm the patient selection (which will automatically order the treatment delivery) and organise the appointment for the next visit.

The patient will receive from the investigational centre the participant card to be kept for all the duration of the study.

## **Visit 2 - Inclusion Visit (Day 1):**

If the patient's behaviour during the selection period and/or the result of complementary examinations, particularly the confirmation of the presence of persistent AF by the Central Reading Laboratory during this period and the laboratory tests, are compatible with the inclusion criteria, the patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: red blood cell concentrations of DHA and coagulation parameters Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination/bodyweight
- Vital signs
- Echocardiography using a two-dimensional echocardiography
- 12-lead ECG
- Urine pregnancy test for women of child bearing potential

If the results of the above assessments are compatible with the inclusion criteria, the patient will be included and the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 2 for the first 12-week period.

Between this Inclusion visit and the next visit (V3), the INR will be closely monitored (refer to paragraph 8.4.6) in order to fulfil the ECV conditions (refer to paragraph 3).

Final version 1141/1185

At the end of the visit, the Investigator will organise the appointment for the next visit and will give the treatment for the next 4-week period (one case of treatment).

## Visit 3 (Week 4: D28 -2/+7 days) cardioversion:

Patient will be assessed for the following criteria:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Haematology, RBC concentrations of DHA, Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT)
- Global Physical examination /bodyweight
- Vital signs
- 12-lead ECG
- Electrocardioversion (ECV): ECV has to be performed 4 weeks after randomization in patients with AF. ECV will be performed in the morning, with the patient in the fasting state and without dyskalemia. An INR value control must be performed within 24h before ECV. INR values ≥ 2 on the 3 last tests performed before ECV are required. However, if only 2 INR values are ≥ 2 among those 3 last tests, an ECV can be performed if the presence of atrial thrombosis can be excluded with an ECHO–TE (transesophageal echocardiography) performed on the same day (before ECV) and the patient can continue the study. Anesthesia will be induced and patients will be cardioverted with administration of a synchronized, biphasic current. The initial shock will be set at 100 J if the body weight is less than 70 kg and at 150 J for higher body weights. Successful cardioversion will be defined as recovery of sinus rhythm lasting at least 1 minute after the shock. If unsuccessful, a second 200-J shock, and eventually a third 200-J shock, will be administered. Failure of ECV is defined as the persistence of AF after the third attempt at cardioversion. After the procedure, patients will be monitored on telemetry for at least 6 hours before discharge.

Final version 1142/1185

Patients who will not revert to sinus rhythm or with early AF relapse or early atrial flutter emergence within the observation period after ECV will be withdrawn from the study and will be considered to have finished their follow-up.

At the end of the visit, a 7-day continuous ECG (5-leads/2 or 3 channels) ambulatory recording (holter ECG) will be installed on the patient in order to monitor the patient heart rhythm after ECV.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

At the end of the visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next 8-week period (two cases of treatment).

## Visit 4 (Week 5: D35 -2/+7 days):

After removal of the continuous ECG ambulatory device, the patient will be assessed for the following criteria:

- Assessment of AE
- Concomitant treatments (authorised, disallowed)
- Bodyweight (bodyweight measured at V3 to be used)
- Vitals Signs
- Echocardiography using a two-dimensional echocardiography

At the end of the visit, the patient will be given the TTEM device for cardiac monitoring. The patient will be clearly instructed on the frequency and modalities of transmission. The patient will be requested to perform one transmission per week from this visit (initial call to perform with the patient) to the visit 9 (week 24 – end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

## Visit 6\* (Week 12: D84 $\pm$ 7 days) - Visit 7 (Week 16: D112 $\pm$ 7 days) :

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following criteria:

Adverse events

Final version 1143/1185

- Concomitant treatments (authorised, disallowed)
- Laboratory examination: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time (aPTT), Thrombin Clotting Time (TCT). However, in case of discontinuation of anticoagulation after ECV due to occurrence of VKA intolerance, the monitoring of INR, aPTT and TCT should be stopped.
- Global Physical examination/bodyweight
- Vital signs
- 12-lead ECG
- The cardiac monitoring will be continued using the TTEM device through one transmission per week from the day of visit 4 (end of week 5) to visit 9 (week 24, end of study). Moreover, in case of AF or atrial flutter symptoms, additional transmissions may be performed.

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused capsules for each 4-week treatment period.

In addition, at visit 6:

- the investigator will contact the IVRS/IWRS to obtain the treatment unit number to be dispensed at visit 6 for the last 12-week period.
- an echocardiography will be performed, an haematology examination will be done and the RBC concentration of DHA will be measured.

At the end of each visit, the Investigator will organise the appointment for the next visit and give the treatment to be taken during the next treatment period: one case at visit 6 and two cases at visit 7.

## Visit 9\* - End-of-Study Visit (Week 24: D168 $\pm$ 7 days):

\*see amendment PA05 dated 22OCT2014

Patient will be assessed for the following:

- Adverse events
- Concomitant treatments (authorised, disallowed)
- Global Physical examination/bodyweight

Final version 1144/1185

Vital signs

• 12-lead ECG

• Laboratory examination: haematology, biochemistry, assessment of coagulation

parameters: Prothrombin Time/INR (PT/INR), Activated Partial Thromboplastin Time

(aPTT), Thrombin Clotting Time (TCT), Red blood cell concentration of DHA.

• Urine pregnancy test for women of childbearing potential

• Echocardiography using a two-dimensional echocardiography

The Investigator will collect all unused cases, blisters and soft capsules, and will count the unused

soft capsules.

The total volume of blood collected should be about 90 ml for the study duration (30 ml for the

total volume of haematology and biochemistry, 2 ml for each blood samples for coagulations

parameters and 4 ml for each blood samples of DHA).

10. ADVERSE EVENTS: DEFINITION AND REPORTING

10.1. ADVERSE EVENTS

**10.1.1.** Definition of Adverse Events

An AE is any adverse change from the patient's baseline condition, i.e. any subjective signs and

symptoms or change in a concomitant disease present at the Selection Visit considered or not

related to the treatment.

AE includes intercurrent signs, symptoms, illnesses and significant deviations from baseline for

vital signs and laboratory values which may occur during the course of the clinical study.

All laboratory tests for which abnormal results are collected after study treatment initiation should

be repeated until the values return to normal or to a stable status. Abnormal results are defined as

those falling out of the laboratory normal ranges and that are clinically significant. The frequency

of such checks should be defined by the Investigator according to the degree of abnormality.

Final version 1145/1185

In all cases, the aetiology should, as much as possible, be identified and *Pierre Fabre Médicament* notified.

## 10.1.2. Grading of Adverse Events

Adverse or intercurrent events are graded as follows:

- Mild: awareness of signs or symptoms, but easily tolerated
- Moderate: uncomfortable enough to cause interference with usual activity
- Severe: incapacity with inability to work or do usual activity

## 10.1.3. Reporting of Adverse Events

The records of AE in the e-CRF describe the nature (diagnosis, signs and symptoms), severity, onset date, stop date, outcome and actions taken, and relationship to study treatment (in the Investigator's opinion). It must be specified whether the event is serious or not.

## 10.2. SERIOUS ADVERSE EVENTS (SAE)

#### 10.2.1. Definition

A SAE includes, but is not necessarily restricted to, any event which:

- Results in death (whatever may be the cause)
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Requires the patient's hospitalisation or prolongation of current hospitalisation \*
- Is a congenital anomaly or birth defect

Other events such as cancer and any additional adverse experience or abnormal laboratory values occurring during the study period, defined by the protocol as serious or which the Investigator considers significant enough or that suggest a significant hazard, contra-indications, side effect or precaution, must be handled as serious adverse events.

Any overdosage meeting a seriousness criteria should be reported as a SAE (see section 10.3).

Final version 1146/1185

Any pregnancy occurring during/after exposure to the study drug(s) should be reported on the SAE notification form (see section 10.4).

- \* any hospitalisation, or prolongation of hospitalisation due to the circumstances listed below:
  - planned (as per protocol) medical/surgical procedure
  - preparation for routine health assessment/procedure (e.g. routine colonoscopy)
  - planned medical/surgical admission (planned prior to entry into study trial, appropriate documentation required)
  - administrative or social reasons (e.g. lack of housing, economic inadequacy, care-giver respite, family circumstances)

will not be reported as a SAE.

## 10.2.2. Reporting of SAE

All Serious Adverse Events, according to the above-mentioned definitions and regardless of treatment or relationship to study drug, and occurring once the informed consent form has been signed, must be reported by the Investigator as soon as he/she is informed of the event.

The Investigator must notify the Sponsor of this event by sending, within 24 hours, the "Notification of serious adverse event" form ("first notification") with all the available information about the event (see appendix 17.2), to the Sponsor's Corporate Vigilances e-mail dedicated box:

## HQ.pharmacovigilance@pierre-fabre.com

In case it is not possible to send the report by e-mail it can be sent by FAX at the following number:

+ 33 1 49 10 80 90

In case of non-inclusion, the reporting period ends when the non-inclusion is documented.

## 10.2.3. Follow-up of SAE

The Investigator must draw-up a specific clinical report and use the "Notification of serious adverse event" form ("follow-up") (see appendix 17.2) and collect the results of the carried out examinations and the reports of hospitalisation.

Final version 1147/1185

The serious adverse events must be followed up until resolution or stabilisation.

## 10.2.4. SAE Occurring After the Study

Any SAE occurring during 30 days following the end of the study for the patient should be notified to the Sponsor.

Must also be notified to the Sponsor any event occurring at any time after the end of the study for the patient which may be related to the study treatment in the Investigator's opinion.

#### 10.3. REPORTING OF OVERDOSAGE TO THE SPONSOR

For the purpose of this trial, an overdosage will be defined as any dose exceeding the planned prescribed dose of the study drug or the administration of any dose of an associated product that is considered both excessive and medically important.

In the absence of seriousness criteria, the overdosage and associated adverse event if any, are reported only on the Adverse Event page of the e-CRF. <u>If the definition</u> of seriousness criteria <u>is</u> <u>met</u>, the SAE notification form must also be transmitted to the Sponsor.

## 10.4. REPORTING OF PREGNANCY TO THE SPONSOR

Pregnancies discovered in the period in between the informed consent form signed but before any study drug exposure are not to be reported to the Sponsor unless associated to a seriousness criteria (e.g. serious adverse event study-protocol related procedure). If pregnancy is confirmed, the women must not be administered the study drug and must be withdrawn immediately from the study.

If pregnancy is suspected while the patient is receiving study treatment, the study drug should be discontinued immediately until the result of the pregnancy testing is known. If pregnancy is confirmed, then the study treatment is permanently discontinued in an appropriate manner and the patient is withdrawn from the study.

The Investigator must report to the Sponsor any pregnancy which occurs during or after the patient has been exposed to the study drug and until 30 days after the last study drug administration. The Investigator must immediately notify the Sponsor using the SAE notification form and also report the pregnancy on the AE page of the e-CRF.

Final version 1148/1185

Women who become pregnant after exposure to the study drug must be followed by the Investigator until the completion/termination of the pregnancy. If the pregnancy goes to term, the outcome will have to be reported to the Sponsor (baby's healthy status).

# 10.5. SPONSOR'S RESPONSIBILITIES FOR SAFETY REPORTING PURPOSES

Sponsor will submit expedited and periodic reports to both Competent Authorities and Ethics Committees per corporate standard operating procedures as regards to the EU directive 2001/20/EC taking into account local specific requirements.

## 11. DATA COLLECTION AND STUDY MONITORING

#### 11.1. DATA COLLECTION

## 11.1.1. Case Report Form

An e-CRF will be used to record all patient data required by the protocol except the central ECG (Holter ECG, TTEM) and DHA data which will be transferred from vendors to the subcontractor as electronic data files that will be loaded into the study database.

The e-CRF should be fully validated, compliant with ICH-GCP requirements and European regulations and should include a traceability system for data corrections and deletions (audit trail).

Prior to the start of the study, the Investigator will complete a "Delegation of significant study-related duties" form. The signature and initials of all personal in charge of e-CRF completion should be recorded on this form. Each person involved in e-CRF completion, review, correction and / or validation will be trained and will have an individual login and access code to the e-CRF. Training sessions will be held by the subcontractor for all participants using this tool. An e-CRF user manual will be available for investigators and CRAs.

All the information included into the e-CRF will be recorded from source documents onto the e-CRF by an authorised person.

Final version 1149/1185

The Investigator is responsible for the management and accuracy of the information on the e-CRF. At each monitoring visit, the e-CRF(s) should be at the CRA's disposition for review and validation

At the end of the study, a CD-ROM containing the pdf version of all e-CRFs (including audit-trail) will be sent by the subcontractor to the Sponsor and to the investigational sites for archiving. The subcontractor must store all study data for at least 15 years after the end of the study and ensure their legibility and accessibility during all the storage period.

#### 11.1.2. Source Documents

A source document is an original record or certified copy of an original record of clinical findings, observations or any other medical or paramedical activities performed during the clinical trial, necessary for the transcription and the verification of the collected data.

Source documents along with all other trial-related documents (copies of all "informed consent" forms, e-CRFs CD-ROM, drug inventories and any correspondence related to the study) must be kept in the investigator's file throughout the study, and then, must be stored in the study centre's archives for a period of at least 15 years or as per local legal requirements, whatever is the longest.

For further details see section 15.2.

#### 11.2. STUDY MONITORING

## 11.2.1. Monitoring visits

On-site visits will be carried out by a representative of the Sponsor's staff (Study Manager or CRA) prior to study initiation and at regular intervals (every 4 to 6 weeks) throughout the study. Additional visits and communication by telephone fax or meeting may be performed if necessary. Any site visit performed by the Sponsor's representatives will be recorded in the Investigator's study file.

Final version 1150/1185

#### 11.2.1.1. Site Preselection Visit

Before selecting a centre for the study, a visit will be carried out by the CRA and/or the Study Manager to ensure that the Investigator has the necessary capacities (availability, patient's recruitment, environment), technical means and staff to carry out the study.

#### 11.2.1.2. Initiation Visit

Before the start of the study at all investigational sites, an initiation visit will be carried out by the CRA to check at the latest that:

- The Investigator:
- has received the technical protocol, administrative and financial agreement signed by all parties
- has received the written statement of the Ethics Committee approval and the list of its members and their functions
- The original dated and signed *curriculum vitae* of the investigator(s) has been collected
- Laboratory normal ranges have been collected
- All study materials are available on the study site
- All participants agree with the monitoring procedures and know the study procedures
- All participants are aware of a possible audit or inspection

The CRA has also to provide training on the study protocol requirements and study specific procedures.

## 11.2.1.3. Follow-up Visits

Throughout the study, regular follow-up visits will be carried out by the CRA to check compliance with GCP, patient's informed consents, strict application of the protocol, conformity of the data entered on the e-CRF with the source documents and ensure its correct completion, adverse events reporting, proper retention, storage and management of the study medication, as well as the source and other trial-related documents.

Final version 1151/1185

## 11.2.1.4. Closing Visit

At the end of the study, a final visit will be carried out by the CRA to:

- Verify that the e-CRFs CD-ROM with pdf files are correctly stored
- Control the accountability of intact and used treatment units and return them to the Clinical Pharmacy Department of the *IRPF* for destruction
- Obtain the last data clarifications and/or solutions if any
- Collect the patient's consent forms in sealed envelopes (except in case of specific country requirements),
- Make an on-site review of all study documentation and complete it if necessary
- And finally, remind the Investigator of his regulatory obligations, study document archiving process and duration.

#### 11.2.2. Direct Access to Source Documents

In accordance to the requirements of the GCP, all Sponsor representatives (Study Manager, CRA and Auditors) have to be given a direct access to all source and study data to perform quality monitoring/audit, thus ensuring accuracy and completeness of data).

Investigators are reminded that all Sponsor representatives keep professional confidentiality with regards to the patient data.

## 11.3. INDEPENDENT DATA MONITORING COMMITTEE

An Independent Data Monitoring Committee (IDMC) will be established to assess at intervals the progress of the clinical trial, the compliance with the inclusion criteria, the quality of follow up, the quality of primary end point measures, the safety data. The IDMC will thereafter recommend to the Sponsor whether to continue, modify, or stop the study.

The IDMC operating procedures will be described in an independent document.

Final version 1152/1185
## 12. DATA MANAGEMENT

All clinical data related to the study will be collected and saved in a computerised database by the Data Management Department of the subcontractor and under the supervision of the Data Manager of Pierre Fabre Biometry (PFB) according to the following procedures.

## 12.1. DATA ENTRY

All required data will be collected by the Investigator or authorised designee (duly identified into the delegation task list) on the e-CRFs.

The e-CRFs used for this study will be developed and maintained by the Data Management Department of the subcontractor and approved by the Sponsor.

Electronic data (Holter ECG, TTEM and DHA) will be transferred by the 3<sup>rd</sup> party vendor according to the specifications given by the Data Manager of the subcontractor. These data will be captured and handled in accordance with the European GCP ICH E6 guideline.

## 12.2. DATA CLEANING

The subcontractor will define in the Data Validation Plan for reviewing and querying data, descriptions of both manual and electronic edit checks. Upon Sponsor approval, the subcontractor will program the checks.

The subcontractor will review the data over the course of the study, working with the Sponsor to identify data inconsistencies. The Investigator will be asked to resolve queries by making changes directly into the e-CRF.

## 12.3. DATA CODING

Adverse events, concomitant diseases, medical/surgical histories will be coded by the subcontractor using the MedDRA dictionary (latest version in use).

Concomitant medication will be coded by the subcontractor using the WHO-DRUG dictionary (latest version in use).

The Sponsor Clinical Development Physician will validate the coding.

Final version 1153/1185

## 12.4. DATA STORAGE

Computer data files as well as their modifications will be archived by the subcontractor and kept available upon request of the Sponsor.

## 12.5. DATABASE LOCK

The validated database will be locked by the subcontractor upon request of the Data Manager of PFB following the completion of all steps required, i.e. data entry and check of all data, resolution of all queries, validation of the coding, Clinical and Products Safety databases reconciliation and validation committee.

Then, the subcontractor will transfer the locked database in SAS format to the Data Manager of PFB who assume storage on the PFB secured server.

## 13. STATISTICAL ANALYSIS

After the database lock and the randomisation code release, the statistical analysis will be performed by PFB or under the supervision of the statistician of PFB using SAS® software, according to the Statistical Analysis Plan approved by the Validation Committee.

## 13.1. GENERAL CONSIDERATIONS

The main objective of the study is to assess the efficacy of F373280 versus placebo on the maintenance of sinus rhythm after direct ECV in patients with persistent AF and chronic heart failure.

Only the primary analysis of the primary efficacy criterion, on which is based the sample size justification, may lead to a causal interpretation. All other statistical results are to be regarded within a descriptive perspective.

The statistical significance level of the various two sided tests of all analyses will be 5 %.

## 13.2. SAMPLE SIZE

Assuming an AF recurrence or atrial flutter emergence rate of 85% under placebo and 65% under active group, i.e. a clinically relevant difference  $\Delta$  of 20%, a sample size of 64 assessable patients

Final version 1154/1185

per group is required, using a log-rank test of survival curves with a 80 % power and a 5 % two-sided significance level.

According to the previous assumptions and assuming a rate of not assessable patients of 15%, a minimum of 76 patients will have to be randomised per group.

Due to the premature stop of the recruitment 135 patients were finally randomised.

## 13.3. PROTOCOL DEVIATIONS

Prior to the database lock and the randomisation code release, the Validation Committee members will review the protocol deviations and will classify them as either minor or major. A protocol deviation will be considered major when it is likely to bias significantly the treatment effect estimate based on the primary efficacy criterion.

Patients with major deviation(s) will be excluded from the Per Protocol data set (see section 13.4).

A listing of all protocol deviations will be provided for all randomised patients, including the type (major/minor) of protocol deviations according to the decisions made by the members of the Validation Committee.

The number and percentage of patients with major protocol deviations will be tabulated by treatment group and type of major protocol deviations on the Full Analysis Set defined in section 13.4.

## 13.4. DATA SETS ANALYSED

The following 3 data sets will be analysed (as defined by the Validation Committee):

- The Safety Set composed of all randomised patients having received at least one dose of the study treatment. This data set will be used to perform analyses of Safety.
- The Full Analysis Set (FAS) composed of all randomised patients having received at least one dose of the study treatment and with a successful cardioversion observed at visit 3. This data set will be used to perform analyses of Efficacy.
- The Per Protocol Set (PP) which is the subset of the Full Analysis Set composed of all patients with a primary efficacy criteria available and without any major protocol

Final version 1155/1185

deviation or other source of bias for primary criteria analyses. This data set will be used to perform the supportive analysis of the primary efficacy criterion.

## 13.5. HANDLING OF DROPOUTS AND MISSING DATA

## **13.5.1. Dropouts**

The number of patients who withdraw from the study after their randomisation will be provided by treatment group for all treated patients (Safety Set). All withdrawn patients will be further described regarding their time to dropout and reasons for withdrawal.

## 13.5.2. Repositioning of Visits

No repositioning of visits will be done.

## 13.5.3. Missing Data

Missing values will not be substituted by estimated values, but considered as missing in statistical analysis.

## 13.6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Before the first trial drug intake, patient's background, medical and surgical history, demographic data and disease characteristics will be described by treatment group on the Safety Set.

- <u>Quantitative parameters</u> will be described by treatment group and overall using the following: number of patients, number of missing data, mean, standard deviation, minimum, median and maximum values.
- Qualitative parameters will be described by treatment group and overall using frequencies.

Concomitant diseases, as well as medical and surgical histories will be tabulated descriptively by treatment group and overall using the MedDRA codes of System Organ Classes and preferred terms.

Final version 1156/1185

If more than 10% of patients are excluded from the FAS and PP set, the description of patients by treatment group at selection and inclusion will be repeated on the FAS and PP set for all parameters.

No statistical test of comparability of treatment groups at baseline will be performed.

## 13.7. EFFICACY ANALYSIS

## 13.7.1. Primary Criterion

## 13.7.1.1. Primary Analysis

The primary criteria, time to first recurrence of AF or atrial flutter emergence, will be analysed using the Kaplan Meier method and compared with the Log rank test. Hazard ratios and 95% confidence intervals will be estimated with the Cox regression model.

The primary analysis will be performed on the FAS.

## 13.7.1.2. Supportive Analysis

The primary analysis will be repeated on the PP set.

## 13.7.1.3. Additional Analysis

To take into consideration the sample size reduction, the **predictive probability of success** with the expected sample size based on observed data, the **predictive power** and the **conditional power** will be provided to support the statistical decision.

## 13.7.2. Secondary Criteria

All secondary analyses will be performed on the FAS. If more than 10% of patients are excluded from the PP set, the secondary analyses will be repeated on the PP set.

## 13.7.2.1. Numbers of Atrial Fibrillation Episodes in the first week following V3

Both the numbers of AF episodes (symptomatic or not) lasting for at least 10 minutes and with duration less than 10 minutes ( $N_{Sup10}$  and  $N_{Inf10}$ ) will be described by treatment group and compared by the chi-square test (or CMH test adjusted for centre) or Fisher's exact Test.

Final version 1157/1185

## 13.7.2.2. Duration of Atrial Fibrillation Episodes in the first week following V3

The duration of all AF Episodes will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centres effects) or Wilcoxon test.

## 13.7.2.3. Time to first AF recurrence less than 10 minutes or symtomatic

The time to the first AF recurrence less than 10 minutes and the time to the first symptomatic AF recurrence will be analysed as the primary analysis.

## 13.7.2.4. Clinical parameters evaluation

The EHRA score will be described by treatment group and analysed using a chi-squared test (or CMH test adjusted for centre) or Fisher's exact Test.

The frequency of presumed arrhythmia will be described by treatment group.

The number of recurrence of symptomatic AF, of hospitalizations (for cardiovascular events, for thromboembolic stroke and for all causes), of spontaneous cardioversion, of successful cardioversion (including number of shocks distribution) and the number of patients needing cardioversion after initial ECV will be described by treatment group and compared using a chi-square test or a Fisher Test (if the numbers are relevant).

The duration of hospitalizations for cardiovascular events, for thromboembolic stroke and for any cause will be described by treatment group and compared using the Student t (or using an ANOVA with treatment and centre effects) or Wilcoxon test.

The echocardiographic parameters values will be described at each time (V1, V2, V4, V6 and V9) and changes described from V4 to V9 and from V2 to V9.

## 13.7.2.5. Biomarker analysis: red blood cell concentrations of DHA

Values and changes from baseline for red blood cell concentration of DHA will be performed by treatment group and assessment time.

## 13.8. SAFETY ANALYSIS

The Safety Set will be used to perform all analyses of the safety criteria.

Final version 1158/1185

#### 13.8.1. Adverse Events

Any adverse event having been reported during the study for a given patient will be classified by preferred term and corresponding system organ class using the MedDRA terminology.

Adverse events will be classified as:

- Treatment emergent adverse events, *i.e.*, any adverse event which occurs or worsens on study treatment during the randomised period.
- Or non treatment emergent adverse events, *i.e.*, any adverse event which occurs during the run-in period (before V2) or is reported as concomitant disease with the same intensity.

For each study period, any patient with at least one reported adverse event will be classified as a patient:

- With at least one adverse event
- With at least one treatment emergent adverse event
- With one TEAE
- With two TEAEs
- With at least three TEAEs
- With at least one related TEAE
- With an adverse event leading to the study treatment discontinuation (definitive or temporary)
- With an adverse event leading to withdrawal
- With at least one serious adverse event.

Numbers and percentages of patient with at least one reported treatment emergent adverse event will be tabulated by treatment group:

- By system organ class
- By system organ class and preferred term
- By system organ class and preferred term, taking into consideration its most severe intensity

Final version 1159/1185

• And by system organ class and preferred term, taking into consideration the most severe relationship to the study treatment.

Recurring adverse events (*i.e.*, adverse events classified with the same preferred term) for a given patient will only be counted once and only their most severe intensity or most severe relationship to the study treatment will be tabulated.

The number and percentage of patient with at least one most common (<u>reported in 1% patients in any group</u>) drug related TEAE ("not excluded or unassessable") will be tabulated by Preferred Term and Treatment group in decreasing order for the treatment group (<u>for all patients</u>).

The number and percentage of patients with at least one reported most common treatment emergent adverse event will also be plotted by treatment group. This graphical representation will highlight the frequencies of the most severe intensities reported by system organ class and preferred term.

SAE will also be described on an individual basis: treatment group, patient's code, sex and age, Investigator's reported term, preferred term, time of onset according to the time of the first study treatment administration, duration, action taken regarding the study treatment administration, use of a corrective treatment, outcome and relationship to the study treatment in the Investigator's opinion.

## 13.8.2. Clinical Laboratory Evaluation

For each laboratory parameter, data will be tabulated by treatment group and assessment time.

The absolute changes post-trial drug administration - baseline (the baseline value being the value measured on the last blood sample collected before the first trial drug administration) will be calculated and tabulated by parameter, treatment group and post-trial drug administration assessment time. Results of retests performed post-trial drug administration will not be analysed and tabulated. They will only be displayed in individual data listings.

For all biochemistry parameters, scatter plots highlighting individual results will display the baseline and week 24 of the laboratory measurements for each patient by locating the point defined by the baseline value on the abscissa and respectively week 24 value in the ordinate.

For all haematology parameters, scatter plots highlighting individual results will display the baseline and week 4, week 12 and week 24 of the laboratory measurements for each patient by

Final version 1160/1185

locating the point defined by the baseline value on the abscissa and respectively week 4, week 12 and week 24 value in the ordinate.

Each treatment group will be differently identified. The first bisecting line (45° line), the lines of lower and upper normal range, the lines of Potentially Clinically Significant Change (PSC) range and Clinically noteworthy abnormal laboratory value (CNALV) range added on the plots (see Appendix 17.3).

For all blood laboratory parameters, shift tables will be provided to depict the numbers of patients with post-trial drug administration variations at each assessment time as compared to the baseline values (measured on the last blood sample collected before the first trial drug administration) by treatment group. A 3-point scale (low, normal, high) will be used as defined by the normal ranges in use in the laboratory in charge of the assays.

CNALV (see in Appendix 17.3) will be identified and described on an individual basis. If relevant, five separate individual data listings by treatment group will be provided:

- CNALV for haemoglobin (including corresponding individual results of erythrocytes and haematocrit)
- CNALV for neutrophils or leucocytes (including corresponding individual results of basophils, eosinophils, lymphocytes and monocytes)
- CNALV for platelets (including corresponding individual results of erythrocytes and leucocytes)
- CNALV for liver function parameters (including corresponding individual results of gamma-GT)
- CNALV for serum creatinine

## 13.8.3. Global Physical Examination

Recorded data of the global physical examination performed will not be tabulated as any abnormal findings post-randomisation should be reported as AEs (if clinically significant).

Physical examination assessments will be provided in the listings of individual data.

Final version 1161/1185

## 13.8.4. Vital Signs, Physical Findings and Other Observations Related to Safety

## 13.8.4.1. Vital Sign Measurements Over Time

For each parameter (systolic blood pressure, diastolic blood pressure and HR in supine and standing positions), descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.2. Body weight

Descriptive statistics over time of values and changes from baseline will be tabulated by treatment group and assessment time.

## 13.8.4.3. Individual Patient Changes

The number and percentage of patient with at least one Predefined Potentially Clinically Significant Change (PSC) and with at least one PSC Leading to Clinically Significant Value (PSCV) will be tabulated by treatment group (see Table 1 in Appendix 17.3).

According to the pharmacological drug profile mentioned previously in this Protocol, the changes from baseline to the maximum and/or minimum post-baseline value could be categorized and tabulated by treatment group with frequencies and decreasing cumulative percentages.

If there is a signal of a drug effect toward one direction rather than the other, additionally shift tables of variations from baseline to the maximum or minimum post-baseline value could be also provided (see Table 2 to 4 in Appendix 17.3).

An individual data listing of patients with symptomatic or asymptomatic orthostatic hypotension will be provided by treatment group (see Table 5 in Appendix 17.3).

## 13.8.5. ECG

Frequencies on the clinical interpretation (normal, abnormal CS or NCS) will be presented by treatment group and assessment time. Individual tabulated data for ECG abnormalities will be also displayed.

Final version 1162/1185

## 13.8.6. Coagulation parameters

Scatter plots highlighting individual results for coagulation parameters (prothrombin time/INR, activated partial thromboplastin time and thrombin clotting time) before and after study treatment administration will be produced.

## 13.9. CONCOMITANT TREATMENTS

Concomitant treatments will be tabulated by treatment group within a descriptive perspective. They will be classified by therapeutic area according to the WHO-DRUG dictionary using the "anatomical therapeutic chemical" classification on the safety set.

## 13.10. COMPLIANCE

The percentage of compliance will be described by treatment group using the quantity

$$Compliance(\%) = \frac{Estimated\_actual\_consumption}{Theoretical\_consumption} \times 100$$

with: Estimated actual consumption = number of tablets provided at the start of study (Visit 2) minus number of tablets returned at the end of study (Visit 9)

Theoretical consumption = number of days of treatment intake planned between the start and the end of study (168 days  $\pm$  7days)

## 13.11. INTERIM ANALYSIS AND DATA MONITORING

No analyses of efficacy data are planned for IDMC that ensures that the overall probability of type I error is controlled. No Type I error and sample size adjustments are necessary. Any recommendations of the IDMC to alter study conduct will be based on safety, so IDMC monitoring of the study will not affect the statistical operating characteristics of the final analysis.

Final version 1163/1185

The IDMC will review, two times during the study period (after the first 30 subjects will have been randomized and when the first 80 subjects will have terminated their study participation), safety data results across treatment groups and judges whether the overall safety and feasibility (not futility) of the trial remain acceptable.

## 14. GENERAL ETHICAL CONSIDERATIONS

## 14.1. ETHICAL CONDITIONS

This study is performed in accordance with the principles stated in the Declaration of Helsinki (1964) and subsequent amendments and in accordance with the Good Clinical Practice Guideline (CPMP/ICH/135/95).

## 14.2. ETHICS COMMITTEE AND LEGAL REQUIREMENTS

All the documents required by National Regulations and any other informative documents that may be requested are submitted for review to an Ethics Committee whose procedures and operations meet the GCP and National Legal Requirements.

Depending on National Regulations, the application is submitted to the Ethics Committee by the Sponsor (or representative) or by the Investigator.

A copy of the formal written approval from the Ethics Committee is provided to the Sponsor (directly by the Ethics Committee or via the Investigator) with a list of names and qualifications of its members.

The request for authorisation by the Competent Authority or its notification if required (depending on National Regulations) is carried out by the Sponsor.

The screening of patients does not start before the approval of the Ethics Committee has been obtained and the study authorised by the Competent Authority or notified to the Competent Authority (depending on National Regulations).

Final version 1164/1185

# 14.3. PATIENT'S INFORMATION LEAFLET AND INFORMED CONSENT FORM

An information must be given to the patients before their decision to participate or abstain from participation.

This information is based on the elements set out in the Declaration of Helsinki and the ICH GCP Guidelines. It must also describe the measures taken to safeguard patient's privacy and protection of personal data, according to European Directive 95/46 EC or other local regulation.

Restraints and risks must be explained, as well as the right to discontinue participation in the study at any stage, without affecting their further relationship with the Investigator and/or their future care.

The written information and consent form must be submitted to the patient with an oral explanation. It must be agreed and signed by the patient before any study-related procedure starts.

This information and consent procedure is under the Investigator's responsibility.

The information and consent document are made in triplicate: the original copy is kept by the Investigator, one copy is given to the patient and the last copy is kept by the Clinical Quality Assurance Unit of the Sponsor in a sealed envelope at the end of study (except in case of specific country requirement).

Specific areas of the Sponsor's copy are not triplicated to avoid the reading of the patient's surname (except the first 3 letters), first name, address and signature.

If any information becomes available during the trial that may be relevant to the patient's willingness to keep on participating in the trial, an updated written informed consent must be submitted to the patient to confirm agreement to continue participating.

## 14.4. PERSONAL DATA PROTECTION

All information from this study (excluding data from the informed consent) is entered into a computer under the Sponsor's responsibility in accordance with the French law, "Loi Informatique et Libertés" (January 6, 1978, and subsequent amendments) and with the European Directive 95/46/CE.

Final version 1165/1185

## 14.5. INSURANCE POLICY

In accordance with the provisions of the law and the GCP, the Sponsor Pierre Fabre Médicament, has an insurance policy intended to guarantee against possible damage resulting from the research.

The studies and/or experiments performed on behalf of the Sponsor Pierre Fabre Médicament are specifically and expressly guaranteed.

It is advisable to underline that non compliance with the Research Legal Conditions is a cause for guarantee exclusion.

## 15. ADMINISTRATIVE PROCEDURES

## 15.1. PROTOCOL AMENDMENT

Neither the Investigator nor the Sponsor may alter the protocol without the authorisation of the other party.

All changes to the protocol are subject to an amendment which must be dated and signed by both parties and must appear as an amendment to the protocol.

Substantial amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities.

Urgent amendments are submitted for approval / authorisation to the Ethics Committees and Competent Authorities, but could be implemented immediately under specific conditions defined with the Sponsor.

## 15.2. SOURCE DOCUMENTS, INVESTIGATOR'S FILE STORAGE

The Investigator:

- Keeps all trial-related documents in appropriate file folders. Records of patient, original
  informed consent forms, source documents, a CD Rom containing a pdf copy of e-CRF,
  drug inventory, Ethics Committees and Sponsor correspondence pertaining to the study
  must be kept on file.
- Retains all documents relating to the screening (consent and investigation results) of all
  patients included in the trial or not.

Final version 1166/1185

- Retains a list of the patient's names, addresses (and/or number of medical file), code
   numbers to allow checking of data reported on e-CRFs with those from source documents.
- Authorises direct access to source documents for monitoring, audits and inspections.
- The trial-related documents must be retained as strictly confidential at the Investigator's site for at least 15 years or according to local requirements, whatever is the longest after the completion or discontinuation of the trial (European Directive 2003/63/EC).

#### 15.3. END OF THE STUDY

## 15.3.1. Definition of the End of Study

The end of study is the last visit of the last patient undergoing the trial.

Any change to this definition during the study, for whatever reason, must be notified as a substantial amendment.

## 15.3.2. Early Study Termination

## 15.3.2.1. Early Study Termination Decided by the Sponsor

The Sponsor may discontinue the study at any time for any of the following reasons:

- Lack of recruitment
- Deviations from good clinical practice and/or regulations
- Poor product safety
- New information that could jeopardise the patient's safety
- Stopping of the development ...

## 15.3.2.2. Early Study Termination Decided by the Competent Authorities

The Competent Authorities may suspend or prohibit a study if they consider that either the conditions of authorisation are not being met or has doubt about the safety or scientific validity of the study.

Final version 1167/1185

## **15.4. AUDIT**

The Sponsor is responsible for making sure that both its representatives (Study Manager, CRA...) and the Investigator fulfil the requirements as specified by the GCP Guideline.

An audit can be organised internally at Pierre Fabre Médicament and at the investigational site where the e-CRFs are matched against source documents.

All study documentation must be directly accessible to auditors.

The practical conditions for the audit are discussed between the Investigator and the Clinical Quality Assurance Department.

Oral information about the audit results are given to the Investigator.

## 15.5. INSPECTION

The Health Authorities may inspect any investigation site or the Sponsor in the course of the study or after its completion, to verify the conduct of the study and quality of the data. The Investigator must provide to the inspectors direct access to study documents.

## 15.6. CONFIDENTIALITY

The present materials (protocol and related documentation, e-CRF, Investigator's Brochure) contain confidential information.

Except if agreed in writing with the Study Manager, the Investigators must hold such information confidential, and must not disclose it to others (except where required by Applicable Law).

## 15.7. CLINICAL STUDY REPORT

Data analysis and clinical study report writing are under the Sponsor's responsibility.

Upon data analysis completion, a final report including a review of the objectives and methods, a presentation and a discussion of the results is drawn up according to ICH Guidelines (Structure and Content of Clinical Study Reports, ICH-E3, CPMP/ICH/137/95).

The report is a clinical and statistical integrated report. It must be signed by the Sponsor's representative(s) and the Coordinating Investigator.

Final version 1168/1185

## 15.8. STUDY RESULTS COMMUNICATION

Upon completion of the study, the global results of the Research are communicated to the Investigator. According to the Local Regulation, the patient can ask the Investigator for the results.

## 15.9. STUDY RESULTS PUBLICATION

The information and data collected during the conduct of this clinical study are considered confidential and are used by the Sponsor in connection with the development of the study drug. This information may be disclosed if deemed necessary by the Sponsor.

To allow the use of the information derived from this clinical study and to insure compliance with Current Regulations, the Investigator must provide the Sponsor with complete test results and all data collected during the study.

Only the Sponsor may make study information available to physicians and to Regulatory Agencies, except as required by Current Regulations.

All the results of this study including data, reports, discoveries and inventions resulting from the study, are the property of the Sponsor.

In the event the Sponsor chooses to publish study data, the manuscript must be provided to the author(s) at least 30 days prior to the expected date of submission to the intended publisher.

The Investigator(s) can reserve the right to publish or present study data; if so, the manuscript or abstract must be provided to the Sponsor for review at least 30 days prior to the expected date of submission to the intended publisher or of planned presentation.

In addition, if necessary, (the) Investigator(s) shall withhold publication for an additional 60 days, to allow the filing of a patent application, or to allow the Sponsor to take any measures he deems appropriate to establish and preserve his proprietary rights.

It is agreed that publication of study results by each site shall be made only as part of a publication of the study results obtained by all sites performing the protocol, once the study is completed and finalised.

Final version 1169/1185

The authors list is agreed by all Investigators prior to publication. The names of the authors are provided according to their participation in the design of the protocol as well as their recruitment of eligible and analysable patients.

Final version 1170/1185

## 16. REFERENCES

- [1]. F373280 INVESTIGATOR'S BROCHURE, version October 2013
- [2]. NODARI S., TRIGGIONAI M., CAMPIA U., MANERBA A., MILESI G., CESANA M.B., GHEORGHIADE M., DEI CAS L. n-3 Polyunsaturated Fatty Acids in the prevention of atrial Fibrillation Recurrences after electrical cardioversion. A prospective, Randomised study *Circulation*, 2011; 124:1100-1106
- [3]. NODARI S., TRIGGIANI M., CAMPIA U., MANERBA A., MILESI G., CESANA M B., GHEORGHIADE M., DEI CAS L. Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy *J. Am. Coll. Cardiol.* 2011;57;870-879
- [4]. MOERTL D., HAMMER A., STEINER S., HUTULEAC R., VONBANK K., BERGER R.

  Dose-dependant effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of non ischemic origin: A double-blind, placebo-controlled, 3-arm study *American Heart Journal 2011; 161:915.e1-915.e9 volume 161, number 5*
- [5]. GISSI-HF INVESTIGATORS
  Effects of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GSSI-HF Trial): a randomised, double-blind, placebo-controlled trial

  The lancet on line August 2008
- [6]. CAMM A.J., KIRCHHOF P., LIP G.Y., SCHOTTEN U., SAVELIEVA I., ERNST S., VAN GELDER I.C., AL-ATTAR N., HINDRICKS G., PRENDERGAST B., HEIDBUCHEL H., ALFIERI O., ANGELINI A., ATAR D., COLONNA P., DE CATERINA R., DE SUTTER J., GOETTE A., GORENEK B., HELDAL M., HOHLOSER S.H., KOLH P., LE HEUZEY J.Y., PONIKOWSKI P., RUTTEN F.H. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery, Eur Heart J. 2010 Oct;31(19):2369-429
- [7]. KOWEY PR, REIFFEL JA, ELLENBOGEN KA, NACCARELLI GV, PRATT CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomised controlled trial. *JAMA*. 2010;304:2363–2372.

Final version 1171/1185

[8]. BIANCONI L., CALO L., MENNUNI M., SANTINI L., MOROSETTI P., AZZOLINI P., BARBATO G., BISCIONE F., ROMANO P., SANTINI M. N-3 polyunsaturated fatty acids for the prevention of arrhythmia recurrence after electrical cardioversion of chronic persistent atrial fibrillation: a randomised, double-blind, multicentre study *Europace (2011) 13, 174-181* 

- [9]. OMACOR® SUMMARY PRODUCT CARACTERISTICS (SPC) dated 17/02/2012
- [10]. BEPANTHENE ® SUMMARY PRODUCT CARACTERISTICS (SPC)
- [11]. TOUBOUL P, BRUGADA J, CAPUCCI A, CRIJNS HJ, EDVARDSSON N, HOHNLOSER SH.

Dronedarone for prevention of atrial fibrillation: a dose-ranging study. *Eur Heart J 2003;24(16):1481-7*.

[12]. LE HEUZEY JY AND ALL.

A Short-Term, Randomised, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Dronedarone versus Amiodarone in Patients with Persistent Atrial Fibrillation: The DIONYSOS Study.

J Cardiovasc Electrophysiol.

[13]. METCALF G.R., JAMES J.M., GIBSON A.R., EDWARDS J., STUBBERFIELD J., STUKLIS R., YOUNG D.G., ROBERTS-THOMSON K. & CLELAND G.L.M.L. & OKEN H.

Effects of fish-oil supplementation on myocardial fatty acids in humans. *Am J Clin Nutr (2007); 85 : 1225.* 

[14]. ARTERBURN M.L. & OKEN H.

Distribution, interconversion and dose response of n-3 fatty acids in humans. *Am J Clin Nutr* (2006);83: 1469-1473S.

[15]. TIELEMAN RG, VAN GELDER IC, CRIJNS HJ, DE KAM PJ, VAN DEN BERG MP, HAAKSMA J, VAN DER WOUDE HJ, AND ALLESSIE MA.

Early recurrences of atrial fibrillation after electrical cardioversion: a result of fibrillation-induced electrical remodelling of the atria? J. Am. Coll. Cardiol. 1998;31;167-173

[16]. SALM P, TAYLOR PJ, KOSTNER K

Simultaneous quantification of total eicosapentaenoic acid, docosahexaenoic acid and arachidonic acid in plasma by high-performance liquid chromatography-tandem mass spectrometry.

Biomed Chromatogr 2011 Jun; 25(6):652-9.

[17]. LEGRAND P., SCHMITT B., MOUROT J., CATHELINE D., CHESNEAU G., MIREAUX M., KERHOAS N., WEILL P.

Final version 1172/1185

The consumption of food products from linseed-fed animals maintains erythrocyte omega-3 fatty acids in obese human. *Lipids*, 2010, 45, 11-19.

[18]. HARRIS WS, VON SCHACKY C.

The Omega-3 Index: a new risk factor for death from coronary heart disease? *Prev Med. 2004 Jul; 39(1):212-20* 

[19]. ABSTRACT: P5161.

NODARI S, MANERBA A., MADURERI A., BERLINGHIERI N., PULCINI E., FRATTINI S., METRA M, DEI CAS L.

Effects of Polyunsaturated Fatty Acids n-3 (PUFA n-3) in the prophylaxis of atrial fibrillation relapses after external electric cardioversion

World Congress of Cardiology 2006, 2-6 September, Barcelona – Spain

[20]. KIRCHHOF P., AURICCHIO A., BAX J., CRIJNS H., CAMM J., DIENER HC., GOETTE A., HINDRICKS G., HOHNLOSER S., KAPPENBERGER L., KUCK KH., LIP HYG., OLSSON B., MEINERTZ T., PRIORI S., RAVENS U., STEINBECK G., SVERHAGE E., TIJSSEN J., VINCENT A., BREITHARDT G.

Outcome parameters from a consensus conference organized by the German Atrial Fibrillation Competence NETwork and the European Heart Rhythm Association.

Europace 2007, 9, 1006-1023

## [21]. EUROPEAN MEDICINES AGENCY

Addendum to the guideline on antiarrhythmics on atrial fibrillation and atrial flutter.

EMA/CHMA/EWP/213056/2010

## [22]. OWEN AJ, PETER-PRZYBOROWSKA BA, HOY AJ, MCLENNAN PL.

Dietary fish oil dose- and time-response effects on cardiac phospholipid fatty acid composition.

Lipids. 2004;39:955–961

[23]. ROBERTO M. LANG, MICHELLE BIERIG, RICHARD B. DEVEREUX, FRANK A. FLACHSKAMPF\*, ELYSE FOSTER, PATRICIA A. PELLIKKA, MICHAEL H. PICARD, MARY J. ROMAN, JAMES SEWARD, JACK SHANEWISE, SCOTT SOLOMON, KIRK T. SPENCER, MARTIN ST. JOHN SUTTON, WILLIAM STEWART.

Recommendations for chamber quantification Eur J Echocardiography (2006) 7, 79-108

[24]. JOHN J.V. McMURRAY, STAMATIS ADAMOPOULOS, STEFAN D. ANKER, ANGELO AURICCHIO, MICHAEL BÖHM, KENNETH DICKSTEIN, VOLKMAR FALK, GERASIMOS FILIPPATOS, CÂNDIDA FONSECA, MIGUEL ANGEL GOMEZ-SANCHEZ, TINY JAARSMA, LARS KØBER, GREGORY Y.H. LIP, ALDO PIETRO MAGGIONI, ALEXANDER PARKHOMENKO, BURKERT

Final version 1173/1185

# M. PIESKE, BOGDAN A. POPESCU, PER K. RØNNEVIK, FRANS H. RUTTEN, JUERG SCHWITTER, PETAR SEFEROVIC, JANINA STEPINSKA, PEDRO T. TRINDADE, ADRIAAN A. VOORS, FAIEZ ZANNAD, ANDREAS ZEIHER

ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012 European Heart Journal (2012) 33, 1787–1847

[25]. AGENCE NATIONALE DE SECURITE DU MEDICAMENT ET DES PRODUITS DE SANTE (ANSM).

Bon usage des médicaments antivitamine K (AVK) Actualisation – Juillet 2012

[26]. GILLES PERNOD, ANNE GODIER, CLAIRE GOZALO, BENJAMIN TREMEY, PIERRE SIE

French clinical practice guidelines on the management of patients on vitamin K antagonists in at-risk situations (overdose, risk of bleeding, and active bleeding) *Thrombosis Research 126 (2010) e167–e174* 

Final version 1174/1185

## 17. APPENDICES

Final version 1175/1185

## 17.1. DECLARATION OF HELSINKI

## WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the: 29th WMA General Assembly, Tokyo, Japan, October 1975 35th WMA General Assembly, Venice, Italy, October 1983 41st WMA General Assembly, Hong Kong, September 1989 48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996 52nd WMA General Assembly, Edinburgh, Scotland, October 2000 53th WMA General Assembly, Washington 2002 (Note of Clarification on paragraph 29 added) 55th WMA General Assembly, Tokyo 2004 (Note of Clarification on Paragraph 30 added) 59th WMA General Assembly, Seoul, October 2008

#### A. INTRODUCTION

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data. The Declaration is intended to be read as a whole and each of its constituent paragraphs should not be applied without consideration of all other relevant paragraphs.
- 2. Although the Declaration is addressed primarily to physicians, the WMA encourages other participants in medical research involving human subjects to adopt these principles.
- 3. It is the duty of the physician to promote and safeguard the health of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 4. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 5. Medical progress is based on research that ultimately must include studies involving human subjects. Populations that are underrepresented in medical research should be provided appropriate access to participation in research.
- 6. In medical research involving human subjects, the well-being of the individual research subject must take precedence over all other interests.
- 7. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best current interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 8. In medical practice and in medical research, most interventions involve risks and burdens.
- 9. Medical research is subject to ethical standards that promote respect for all human subjects and protect their health and rights. Some research populations are particularly vulnerable and need special protection. These include those who cannot give or refuse consent for themselves and those who may be vulnerable to coercion or undue influence.
- 10. Physicians should consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.

## B. PRINCIPLES FOR ALL MEDICAL RESEARCH

11. It is the duty of physicians who participate in medical research to protect the life, health, dignity,

Final version 1176/1185

- integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects.
- 12. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 13. Appropriate caution must be exercised in the conduct of medical research that may harm the environment.
- 14. The design and performance of each research study involving human subjects must be clearly described in a research protocol. The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, other potential conflicts of interest, incentives for subjects and provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study. The protocol should describe arrangements for post-study access by study subjects to interventions identified as beneficial in the study or access to other appropriate care or benefits.
- 15. The research protocol must be submitted for consideration, comment, guidance and approval to a research ethics committee before the study begins. This committee must be independent of the researcher, the sponsor and any other undue influence. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration. The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No change to the protocol may be made without consideration and approval by the committee.
- 16. Medical research involving human subjects must be conducted only by individuals with the appropriate scientific training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional. The responsibility for the protection of research subjects must always rest with the physician or other health care professional and never the research subjects, even though they have given consent.
- 17. Medical research involving a disadvantaged or vulnerable population or community is only justified if the research is responsive to the health needs and priorities of this population or community and if there is a reasonable likelihood that this population or community stands to benefit from the results of the research
- 18. Every medical research study involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and communities involved in the research in comparison with foreseeable benefits to them and to other individuals or communities affected by the condition under investigation.
- 19. Every clinical trial must be registered in a publicly accessible database before recruitment of the first subject.
- 20. Physicians may not participate in a research study involving human subjects unless they are confident that the risks involved have been adequately assessed and can be satisfactorily managed. Physicians must immediately stop a study when the risks are found to outweigh the potential benefits or when there is conclusive proof of positive and beneficial results.
- 21. Medical research involving human subjects may only be conducted if the importance of the objective outweighs the inherent risks and burdens to the research subjects.
- 22. Participation by competent individuals as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no competent individual may be

Final version 1177/1185

- enrolled in a research study unless he or she freely agrees.
- 23. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information and to minimize the impact of the study on their physical, mental and social integrity.
- 24. In medical research involving competent human subjects, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information. After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.
- 25. For medical research using identifiable human material or data, physicians must normally seek consent for the collection, analysis, storage and/or reuse. There may be situations where consent would be impossible or impractical to obtain for such research or would pose a threat to the validity of the research. In such situations the research may be done only after consideration and approval of a research ethics committee.
- 26. When seeking informed consent for participation in a research study the physician should be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent should be sought by an appropriately qualified individual who is completely independent of this relationship.
- 27. For a potential research subject who is incompetent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the population represented by the potential subject, the research cannot instead be performed with competent persons, and the research entails only minimal risk and minimal burden.
- 28. When a potential research subject who is deemed incompetent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 29. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research population. In such circumstances the physician should seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research should be obtained as soon as possible from the subject or a legally authorized representative.
- 30. Authors, editors and publishers all have ethical obligations with regard to the publication of the results of research. Authors have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. They should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results should be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest should be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

Final version 1178/1185

## C. ADDITIONAL PRINCIPLES FOR MEDICAL RESEARCH COMBINED WITH MEDICAL CARE

- 31. The physician may combine medical research with medical care only to the extent that the research is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 32. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best current proven intervention, except in the following circumstances:
  - The use of placebo, or no treatment, is acceptable in studies where no current proven intervention exists; or
  - Where for compelling and scientifically sound methodological reasons the use of placebo is necessary to determine the efficacy or safety of an intervention and the patients who receive placebo or no treatment will not be subject to any risk of serious or irreversible harm. Extreme care must be taken to avoid abuse of this option.
- 33. At the conclusion of the study, patients entered into the study are entitled to be informed about the outcome of the study and to share any benefits that result from it, for example, access to interventions identified as beneficial in the study or to other appropriate care or benefits.
- 34. The physician must fully inform the patient which aspects of the care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never interfere with the patient-physician relationship.
- 35. In the treatment of a patient, where proven interventions do not exist or have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. Where possible, this intervention should be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information should be recorded and, where appropriate, made publicly available.

Final version 1179/1185

## 17.2. SAE REPORT FORM

Final version 1180/1185

Final version 1181/1185

| Transmission date | | | (ddmmyyyy) | Country: | | |
|---|---|---|---|---|---|---|
| SAE N° | | FI | RST NOTIFICATION | FOLLOW-U | UP N° | |
| > CONCOMITANT M<br>(EXCEPT THE TREA | EDICATION SING<br>ATMENTS GIVEN | CE TRIAL INITIATIO<br>FOR THE SAE) | N and UP UNTIL TH | E OCCURRENCE O | F THE SAE | |
| Trade name<br>(or INN) | Daily dose | Start date (dd/mm/yy) | Ongoing at occurence of the event | Stop date<br>(dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ➤ MEASURES TAKEN | FOLLOWING T | HE SAE | l l | | | |
| • Study treatment | TOLLOWING II | HE SAE | | | | |
| ☐ No change | | | | | | |
| C | ication, specify : | | Modification D | ate: | //_ | |
| ☐ Temporarily d | | | Readministration date | e: | //_ | |
| ☐ Withdrawn | | | End date | : | / / | |
| ☐ Not applicable | e | | | | | |
| • The event led to: | | | | | | |
| | f corrective or symp | tomatic treatments: | | | | |
| <b>r</b> | T | I | Ongoing at | | Route of | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | occurence of the event | Stop date<br>(dd/mm/yy) | admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Discontinuation | on of concomitant tre | eatments: | | 1 | l | |
| Trade name<br>(or INN) | Daily dose | Start date<br>(dd/mm/yy) | Ongoing at occurence of the event | Stop date (dd/mm/yy) | Route of admin. | Indication |
| | | // | | // | | |
| | | // | | // | | |
| | | // | | // | | |
| ☐ Others, specif | y : | • | | • | | |
| > OUTCOME | | | | | | |
| ☐ Not recovered/No ☐ Recovered/Resolv In case of death | | ☐ Recovering/Resolvir☐ Fatal | ☐ Unknown | l/Resolved | | |
| ➤ INVESTIGATOR CA | AUSALITY ASSES | SMENT (investigator) | s assessment to be don | e as soon as nossible) | | |
| Study drug: | 1001111110010 | | tudy protocol: | c as soon as possible) | | |
| □ Not Suspected Comments: | □ Suspected | □ Not Susp | | Suspected | | |

Final version 1182/1185

Enclose in the notification the results of carried out examinations, reports of hospitalisation, etc...

# 17.3. PREDEFINED LIMITS OF LABORATORY AND VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CHANGES AND VALUES

List of Predefined Potentially Clinically Significant Change For Laboratory Values<sup>(\mathrice{m})</sup>

| PARAMETERS | | UNIT | PSC | |
|--------------|------------------------|--------|----------|-------------|
| | | | Decrease | Increase |
| MUSCLE | Creatine Phosphokinase | U/1 | - | 236 |
| KIDNEY | Creatinine | μmol/l | - | 35 |
| | Urea | mmol/l | - | 3.2 |
| | Uric acid | μmol/l | _ | 119 |
| | Phosphate | mmol/l | 0.39 | 0.39 |
| | Calcium | mmol/l | 0.30 | 0.30 |
| ELECTROLYTES | Sodium | mmol/l | 8 | 8 |
| | Potassium | mmol/l | 1.1 | 1.1 |
| | Chloride | mmol/l | 8 | 7 |
| | Bicarbonate | mmol/l | 7 | 8 |
| METABOLISM/ | Glucose (random) | mmol/l | 3 | 3.7 |
| NUTRITIONAL | Albumin | g/l | 6 | 6 |
| No IMIIONAL | Protein | g/l | 11 | 10 |
| | Cholesterol | mmol/l | _ | 1.97 |
| | HDL cholesterol | mmol/l | 0.91 | 0.85 |
| | LDL cholesterol | mmol/l | 2.17 | 2.04 |
| | Triglycerides | mmol/l | - | 2.91 |
| ERYTHROCYTES | Erythrocyte count | T/1 | 0.7 | 0.7 |
| | Haemoglobin | g/l | 20 | - |
| | Haematocrit | 1 | 0.06 | 0.06 |
| | MCV | fl | 7 | 7 |
| | MCH (Fe) | fmol | 0.19 | 0.19 |
| | MCHC (Fe) | mmol/l | 2 | 2 |
| LEUKOCYTES | Leukocyte count | G/l | 4.2 | 3.8 |
| DIFFERENTIAL | Neutrophils | G/l | 3.47 | 3.19 |
| COUNT | Lymphocytes | G/l | 1.76 | 1.63 |
| | Monocytes | G/l | - | 0.49 |
| | Eosinophils | G/l | - | 0.41 |
| | Basophils | G/l | - | 0.14 |
| URINE | Specific gravity | - | 0.017 | 0.015 |
| | рН | - | 2 | 2 |
| LIVER | Total bilirubin | μmol/l | - | 10 |
| | ASAT (SGOT) | U/1 | - | N x (23/36) |
| | ALAT (SGPT) | U/l | - | N x (28/45) |
| | Gamma GT | U/l | - | N x (25/38) |
| | Alkaline phosphatase | U/l | | N x (30/95) |

N = upper limit of normal range

Final version 1183/1185

<sup>(¤)</sup> Delta-limits from « Routine Laboratory Tests in Clinical Trials » W. Leigh Thompson, Rocco L. Brunelle, Gregory G. Enas, Patrick J. Simpson and Randy L. Walker Lilly Research Laboratories, Lilly Corporate Centre, Indianapolis, Indiana in « Clinical Trials and Tribulations » 1988.

## **Definition of Clinically Noteworthy Abnormal Laboratory Values (CNALV)**

| | PARAMETERS | CNALV |
|---|---|---|
| HAEMOGLOBIN | | <ul> <li>Decrease of at least 2g/dl and value &lt; 10 g/dl whatever the baseline value</li> <li>If missing baseline: value &lt;10g/dl</li> </ul> |
| NEUTROPHILS | | • < 1 500/mm <sup>3</sup> whatever the baseline value |
| WBC (if missing | g value for neutrophils) | $\bullet$ < 3 000/mm <sup>3</sup> whatever the baseline value |
| PLATEL | ETS | $\bullet$ < 100 000/mm <sup>3</sup> whatever the baseline value |
| SERUM ( | CREATININE | <ul> <li>Increase of at least 30 % as compared to baseline value and value &gt; 150 μmol/l whatever the baseline value</li> <li>If missing baseline: value &gt; 150 μmol/l</li> </ul> |
| LIVER F | UNCTION TESTS | |
| | ALAT | <ul> <li>If normal baseline: <ul> <li>ALAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N :</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N : <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | ASAT | <ul> <li>If normal baseline: <ul> <li>ASAT &gt; 2 N</li> </ul> </li> <li>If abnormal baseline: <ul> <li>if baseline value ≤ 2.5 N:</li> <li>increase of at least 100 % as compared to baseline value</li> </ul> </li> <li>if baseline value &gt; 2.5 N: <ul> <li>value &gt; 5 N</li> </ul> </li> </ul> |
| and/or | Alkaline phosphatase (AP) | <ul> <li>If normal baseline:</li> <li>AP &gt; 1.25 N</li> <li>If abnormal baseline:</li> <li>AP &gt; 2 N</li> </ul> |
| and/or | Total bilirubin (TB) | <ul> <li>If normal baseline:</li> <li>TB &gt; 1.5 N</li> <li>If abnormal baseline:</li> <li>TB &gt; 2 N</li> </ul> |

## N=upper limit of normal range

International consensus Meeting. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1990;28:317-322 Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced liver disorders: report of an Standardisation of definitions and criteria of causality assessment of adverse drug reactions: drugs-induced cytopenia. International Journal of Clinical Pharmacology, Therapy and Toxicology, 1991;29:75-81

Final version 1184/1185

Table 1: Predefined Limits for Potentially Clinically Significant Changes (PSC) and PSC Leading to Clinically Significant Values (PSCV)

| Parameter | PSC | PSCV |
|---|---|---|
| SBP | Increase ≥ 20 mmHg | $SBP \ge 160 \text{ mmHg and increase} \ge 20 \text{ mmHg}$ |
| | Decrease ≥ 20 mmHg | $SBP \le 90 \text{ mmHg}$ and decrease $\ge 20 \text{ mmHg}$ |
| DBP | Increase ≥ 10 mmHg | DBP ≥ 100 mmHg and increase ≥ 10 mmHg |
| | Decrease ≥ 10 mmHg | $DBP \leq 50$ mmHg and decrease $\geq 10$ mmHg |
| HR | Increase ≥ 10 bpm | $HR \ge 110$ bpm and increase $\ge 10$ bpm |
| | Decrease ≥ 10 bpm | $HR \le 50$ bpm and decrease $\ge 10$ bpm |

Table 2: Predefined Classes for changes from Baseline to the Maximum (and/ or Minimum) Post-baseline Value

| Classes of Change from Baseline to the Maximum<br>Post-baseline Value | | | Classes of Chan<br>Minimum Post-b | ge from Baseline<br>oaseline Value | to the |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| All | All | All | All | All | All |
| ≥ 0 | ≥ 0 | ≥ 0 | ≤ 0 | ≤ 0 | ≤ 0 |
| > 0 | > 0 | > 0 | < 0 | < 0 | < 0 |
| ≥ 10 | ≥ 5 | ≥ 10 | ≤ -10 | ≤ - 5 | ≤ -10 |
| ≥ 20 | ≥ 10 | ≥ 20 | ≤ -20 | ≤ -10 | ≤ -20 |
| ≥ 30 | ≥ 15 | ≥ 30 | ≤ -30 | ≤ -15 | ≤ -30 |
| ≥ 40 | ≥ 20 | | ≤ -40 | ≤ -20 | |
| | ≥ 25 | | | ≤ -25 | |
| | ≥ 30 | | | ≤ -30 | |

Table 3: Classes for Vital Signs Maximum or Minimum Values

| Classes for the Maximum Post-baseline Value for each parameter | | Classes for the Minimum Post-baseline Value for each parameter | | | |
|---|---|---|---|---|---|
| SBP mmHg | DBP mmHg | HR bpm | SBP mmHg | DBP mmHg | HR bpm |
| < 120 | < 80 | ≤50 | ≤90 | ≤50 | ≤50 |
| [120;140] | [80;90[ | <i>[50;75]</i> | [90 ;120] | [50;80] | <i>[50 ;75]</i> |
| [140;160] | [90;100] | [75;100] | [120;140] | [80;90] | [75;100] |
| ≥ 160 | ≥ 100 | ≥ 100 | ≥ 140 | ≥ 90 | ≥ 100 |

Table 4: Classes for Maximum or Minimum of BP in its entirety

| Classification of Maximum Values for Blood | Classification of Minimum Values Blood |
|---|---|
| Pressure (mmHg) | Pressure (mmHg) |
| SBP < 140 and DBP < 90 | SBP > 90 and DBP > 50 |
| SBP [140;160[ and DBP < 100 | $SBP \le 90 \text{ or } DBP \le 50$ |
| or DBP [90;100[ and SBP < 160 | 3B1 ≥ 90 01 DB1 ≥ 30 |
| $SBP \ge 160 \text{ or } DBP \ge 100$ | |

**Table 5: Definition of orthostatic hypotension** 

| Orthostatic Hypotension * |
|---|
| SBP Decrease $\geq 20$ mmHg or DBP Decrease $\geq 10$ mmHg between supine and standing positions |

<sup>\*</sup> Consensus Committee of the American Autonomic Society and the American Academy of Neurolog: Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Neurology 1996;46:1470-3.

Final version 1185/1185